

# **PARTNER 3:**

A Prospective, Randomized, Controlled, Multi-Center Study to Establish the Safety and Effectiveness of the SAPIEN 3 Transcatheter Heart Valve in Low Risk Patients who have Severe, Calcific, Aortic Stenosis Requiring Aortic Valve Replacement

NCT02675114

**Dec 2018** 

### **PARTNER 3 - Low Risk**

A Prospective, Randomized, Controlled, Multi-Center Study to Establish the Safety and Effectiveness of the SAPIEN 3 Transcatheter Heart Valve in Low Risk Patients who have Severe, Calcific, Aortic Stenosis Requiring Aortic Valve Replacement

# **Clinical Protocol Study Number - 2015-08**

Version 5.0

**DEC 2018** 

Study Sponsor: Edwards Lifesciences LLC One Edwards Way Irvine, CA 92614

PROPRIETARY DATA: This document and the information contained herein may not be reproduced, used or disclosed without written permission from Edwards Lifesciences LLC.

Edwards, Edwards Lifesciences, the stylized E logo, Certitude, Edwards Commander, Edwards SAPIEN, Edwards SAPIEN 3, SAPIEN, and SAPIEN 3 are trademarks of Edwards Lifesciences Corporation.

# **TABLE OF CONTENTS**

| PROTOCOL | SYNOPSIS | 4 |
|---|---|---|
| 1.0 | INTRODUCTION | 12 |
| 2.0 | STUDY OBJECTIVE | 22 |
| 3.0 | STUDY DESIGN | 22 |
| 4.0 | ENROLLMENT | 22 |
| 5.0 | STUDY DEVICE | 22 |
| 6.0 | STUDY ENDPOINTS | 26 |
| 7.0 | STUDY POPULATION | 28 |
| 8.0 | STUDY PROCEDURES | 31 |
| 9.0 | ADVERSE EVENTS | 50 |
| 10.0 | RISKS AND BENEFIT ANALYSIS | 54 |
| 11.0 | STATISTICAL ANALYSIS | 56 |
| 12.0 | STUDY ADMINISTRATION | 67 |
| 13.0 | ETHICAL AND REGULATORY CONSIDERATIONS | 72 |
| Appendix A | Abbreviations | 76 |
| Appendix B | Definitions | 78 |
| Appendix C | Instructions For Use (IFU) | 97 |
| Appendix D | Physician and Support Staff Training | 98 |
| Appendix E | Six Minute Walk Test | 101 |
| Appendix F | Frailty Index | 108 |
| Appendix G | Mini Mental State Examination (MMSE) | 110 |
| Appendix H | NIH Stroke Scale (NIHSS) | 111 |
| Appendix I | Modified Rankin Scale (mRS) | 122 |
| Appendix J | Echocardiogram | 124 |
| Appendix K- | 1 Computed Tomography (CT) | 163 |
| Appendix K- | 2 Sub-Study CT | 216 |
| Appendix L | Histopathology | 234 |
| Appendix M | EQ-5D-5L | 238 |
| Appendix N | Kansas City Cardiomyopathy Questionnaire (KCCQ) | 241 |
| Appendix O | SF-36 | 245 |
| Appendix P | References | 251 |
| Appendix Q | Actigraphy/QOL Sub-Study QOL measures [Enrollment Closed] | 254 |

## **Tables**

| Table 1.1-1: Criteria for Determining Severity of Aortic Stenosis | 12 |
|---|---|
| Table 1.2.1-1: Primary Endpoint Analysis – Non Inferiority Test SAPIEN 3 vs. SAPIEN | 16 |
| Table 1.2.1-2: Death and Stroke at 30 Days (SAPIEN 3 vs. SAPIEN VI Population) | 17 |
| Table 1.2.1-3: Aortic Insufficiency at 30 Days (SAPIEN 3 vs. SAPIEN VI Population) | 17 |
| Table 1.2.1-4: Major Vascular Complications at 30 Days (SAPIEN 3 vs. SAPIEN VI Population) | 17 |
| Table 1.2.1-5: PIIS3 – Clinical Outcomes at 30 Days and 1 Year in Combined S3HR/INOP Cohort (AT | Population) 18 |
| Table 1.2.2-1: PIIS3 - 30-Day Clinical Events in S3i (AT Population) | 19 |
| Table 5.1.1-1: Device Sizing | 24 |
| Table 8.3.2-1: Recommended anticoagulation/antithrombotic regimen | 36 |
| Figures | |
| Figure 1.1.3-1 Edwards TAVR Technology | 14 |
| Figure 1.1.3-2: SAPIEN 3 THV | |
| Figure 1.2.2-1: Moderate/Severe PVL at 30 Days of SAPIEN Valves | 20 |
| Figure 5.1.1-1 Edwards SAPIEN 3 Model 9600TEX | 23 |

#### **PROTOCOL SYNOPSIS**

**Title** A prospective, randomized, controlled, multi-center study to

establish the safety and effectiveness of the SAPIEN 3 transcatheter heart valve in low risk patients who have severe, calcific, aortic stenosis requiring aortic valve

replacement.

**Purpose** To establish the safety and effectiveness of the Edwards

SAPIEN 3 (Edwards Lifesciences, Irvine, California) Transcatheter Heart Valve (THV) in patients with severe, calcific aortic stenosis who are at low operative risk for

standard aortic valve replacement (AVR).

Study Device Edwards SAPIEN 3 THV system Model 9600 TFX (20, 23,

26 and 29 mm) with the associated delivery systems.

**Control** Commercially available surgical bioprosthetic aortic valve

replacement

**Study Design** Prospective, randomized, controlled, multi-center.

Patients will be randomized 1:1 to receive either transcatheter heart valve replacement (TAVR) with the Edwards SAPIEN 3 or aortic valve replacement with a commercially available surgical bioprosthetic valve. A subset of eligible patients from each study arm will be enrolled in a computed tomography (CT) sub-study and/or an Actigraphy/QOL sub-study [enrollment closed] at select

sites.

Patient Population Patients with severe, calcific, aortic stenosis requiring aortic

valve replacement who are at low operative risk

Sample Size PARTNER 3 Randomized Trial:

Up to 1182 patients will be enrolled.

**PARTNER 3 Sub-studies:** 

Of the 1182 patients, a subset of patients will be enrolled in the following sub-studies:

- CT Sub-study (up to 440)
- Actigraphy/QOL Sub-study (up to 400) [Enrollment Closed]

### **PARTNER 3 Single-Arm Registries:**

Additional patients will be enrolled in the following singlearm registries:

Alternative Access Registry (100) [Enrollment Closed]

- Bicuspid Registry (up to 75)
- Underrepresented Populations Registry (up to 100)

### **Study Sites**

Up to 85 actively enrolling sites will participate.

Selected sites will participate in a CT sub-study, an Actigraphy/QOL sub-study [enrollment closed], or the

Underrepresented Populations Registry.

#### Visit Schedule

Screening, Procedure, Post Procedure, Discharge, 30 day, 6 month, and annually through 10 years.

### **Primary Endpoint**

### Safety and Effectiveness:

Composite endpoint of all-cause mortality, all stroke, and rehospitalization (valve-related or procedure-related and including heart failure) at 1 year post procedure.

### Secondary Endpoints for Labeling

- 1. New onset atrial fibrillation at 30 Days
- 2. Length of index hospitalization
- 3. Death, KCCQ < 45 or KCCQ decrease ≥ 10 points at 30 days
- 4. Death or All Stroke at 30 days
- 5. All Stroke at 30 days

### **Additional Safety and Effectiveness Endpoints**

- Mortality (all cause & cardiovascular) at 30 days and 1 year
- Stroke (disabling and nondisabling) at 30 days and 1 year
- 3. Death or stroke at 1 year
- 4. Death or disabling stroke at 30 days and 1 year
- 5. Vascular complications (major) at 30 days and 1 year
- 6. Bleeding complications (life-threatening, disabling, or major) at 30 days and 1 year
- 7. Myocardial infarction at 30 days and 1 year
- 8. Acute kidney injury at 30 days

- 9. Renal replacement therapy at 1 year
- New permanent pacemaker implantation resulting from new or worsened conduction disturbances at 30 days and 1 year
- 11. Coronary obstruction requiring intervention at 30 days and 1 year
- 12. New York Heart Association class at 30 days and 1 year
- 13. Hemodynamic valve performance evaluation by echocardiography for aortic valve stenosis and aortic valve regurgitation (paravalvular & central) at 30 days, and years 1, 2, 3, 4, 5, 7, and 10
- Rehospitalization (valve- or procedure-related including heart failure) at 30 days, 1 year and annually (up to year 10)
- 15. New onset atrial fibrillation at 1 year
- 16. ICU days and discharge location
- 17. Structural valve deterioration at years 1-5, 7 and 10
- 18. Days alive and out of hospital at 1 year
- 19. Six-minute walk test at 30 days and 1 year
- 20. Health status as evaluated by Quality of Life questionnaires
  - KCCQ at 30 days and 1 year
  - EQ-5D-5L at 30 days and 1 year
  - SF-36 at 30 days and 1 year

#### **Inclusion Criteria**

Candidates for this study must meet all of the following inclusion criteria:

- 1. Severe, calcific aortic stenosis as follows:
- AVA  $\leq 1.0 \text{ cm}^2 \text{ or AVA index } \leq 0.6 \text{ cm}^2/\text{m}^2$
- Jet velocity ≥ 4.0 m/s or mean gradient ≥ 40 mmHg AND
- 1) NYHA Functional Class ≥ 2 OR 2) exercise test that demonstrates a limited exercise capacity, abnormal BP response, or arrhythmia OR 3)

asymptomatic with LVEF <50%

Note: Qualifying echo must be within the 90 days prior to randomization.

- 2. Heart team agrees the patient has low risk of operative mortality and has an STS < 4.
- The study patient has been informed of the nature of the study, agrees
  to its provisions and has provided written informed consent as
  approved by the Institutional Review Board (IRB)/Ethics Committee
  (EC) of the respective clinical site.

#### **Exclusion Criteria**

Candidates will be excluded from the study if any of the following conditions are present:

- 1. Native aortic annulus size unsuitable for sizes 20, 23, 26, or 29 mm THV based on 3D imaging analysis
- 2. Iliofemoral vessel characteristics that would preclude safe placement of the introducer sheath.
- 3. Evidence of an acute myocardial infarction ≤ 1 month (30 days) before randomization
- 4. Aortic valve is unicuspid, bicuspid, or is non-calcified
- 5. Severe aortic regurgitation (>3+)
- 6. Severe mitral regurgitation (>3+) or ≥ moderate stenosis
- 7. Pre-existing mechanical or bioprosthetic valve in any position. (of note, mitral ring is not an exclusion).
- 8. Complex coronary artery disease:
  - Unprotected left main coronary artery
  - Syntax score > 32 (in the absence of prior revascularization)
  - Heart Team assessment that optimal revascularization cannot be performed.
- 9. Symptomatic carotid or vertebral artery disease or successful treatment of carotid stenosis within 30 days of randomization
- Leukopenia (WBC < 3000 cell/mL), anemia (Hgb < 9 g/dL), Thrombocytopenia (Plt < 50,000 cell/mL), history of bleeding diathesis or coagulopathy, or hypercoagulable states.

- Hemodynamic or respiratory instability requiring inotropic support, mechanical ventilation or mechanical heart assistance within 30 days of randomization
- 12. Hypertrophic cardiomyopathy with obstruction (HOCM)
- 13. Ventricular dysfunction with LVEF < 30%
- 14. Cardiac imaging (echo, CT, and/or MRI) evidence of intracardiac mass, thrombus or vegetation
- 15. Inability to tolerate or condition precluding treatment with antithrombotic/anticoagulation therapy during or after the valve implant procedure
- 16. Stroke or transient ischemic attack (TIA) within 90 days of randomization
- 17. Renal insufficiency (eGFR < 30 ml/min per the Cockcroft-Gault formula) and/or renal replacement therapy
- 18. Active bacterial endocarditis within 180 days of randomization
- Severe lung disease (FEV1 < 50% predicted) or currently on home oxygen
- 20. Severe pulmonary hypertension (e.g., PA systolic pressure ≥ 2/3 systemic pressure)
- 21. History of cirrhosis or any active liver disease
- 22. Significant frailty as determined by the Heart Team (after objective assessment of frailty parameters).
- 23. Significant abdominal or thoracic aortic disease (such as porcelain aorta, aneurysm, severe calcification, aortic coarctation, etc.) that would preclude safe passage of the delivery system or cannulation and aortotomy for surgical AVR.
- 24. Hostile chest or conditions or complications from prior surgery that preclude safe reoperation (e.g., mediastinitis, radiation damage, abnormal chest wall, adhesion of aorta or IMA to sternum, etc.)
- 25. Patient refuses blood products
- 26. BMI >  $50 \text{ kg/m}^2$
- 27. Estimated life expectancy < 24 months
- 28. Absolute contraindications or allergy to iodinated contrast that cannot be adequately treated with pre-medication

- 29. Immobility that would prevent completion of study procedures (e.g. six-minute walk tests, etc.)
- 30. Patient is not a candidate for both arms of the study (not applicable to single-arm registries)
- 31. Currently participating in an investigational drug or another device study.

Note: Trials requiring extended follow-up for products that were investigational, but have since become commercially available, are not considered investigational trials. Observational studies are not considered exclusionary.

### CT Imaging Sub-Study Inclusion Criteria

Sites with the ability to perform high quality multi-phasic, ECG-gated CT scans (i.e., 4D) will be selected to participate in a CT sub-study

All CT sub-study participants must meet inclusion criteria 1-3 above

### CT Imaging Sub-Study Exclusion Criteria

In addition to the exclusion criteria noted above, patients will be excluded from the sub- study if the following is present:

- 1. Condition requiring or planned use of anticoagulants following the valve implant procedure
- 2. GFR < 50
- 3. Inability to perform high-quality MDCT study for any reason (e.g., atrial fibrillation with rapid ventricular response)

### Actigraphy/QOL Sub-Study Eligibility Criteria [Enrollment Closed]

Select sites will be invited to participate in an Actigraphy/QOL sub-study. Patients must meet all the eligibility criteria of the PARTNER 3 study. In addition, they must demonstrate a basic working knowledge of and ability to use the devices specified in the sub-study. Patients who are non-ambulatory (i.e., wheelchair bound) will not be eligible.

#### Alternative Access Registry Eligibility Criteria [Enrollment Closed]

Patients who do not have appropriate iliofemoral access as defined in exclusion criterion number 2 but meet all other inclusion and exclusion criteria should be considered for enrollment in the alternative access registry.

#### **Bicuspid Registry Eligibility Criteria**

Patients with a bicuspid valve as determined by the CT core lab (e.g., exclusion criterion 4) should be considered for enrollment in this registry if they meet all other eligibility criteria and none of the following additional exclusion criteria:

- 1. Aneurysmal ascending aorta (i.e., >4.0 cm)
- 2. Severe or bulky calcification of the left ventricular outflow tract (LVOT) or raphe that

would increase the risk of annular injury or significant paravalvular leak (PVL) post TAVR

- 3. Coronary anatomy that increases the risk of coronary artery obstruction post TAVR
- 4. Positive urine or serum pregnancy test in female subjects of childbearing potential

### **Underrepresented Populations Registry Eligibility Criteria**

Up to ten (10) sites from underrepresented geographical locations will be selected to enroll patients in a single-arm registry for underrepresented populations. Patients at these sites are eligible for this registry if they meet all eligibility criteria above for the randomized cohort.

### **Principal Investigators**

Martin B. Leon, M.D., FACC New York Presbyterian Hospital/Columbia University Medical Center New York, NY

Michael J. Mack, M.D., FACC Baylor University Medical Center/The Heart Hospital Baylor Plano Plano, TX

**Sponsor** Edwards Lifesciences LLC

One Edwards Way Irvine, CA 92614

### **INVESTIGATOR SIGNATURE PAGE**

A Prospective, Randomized, Controlled, Multi-Center Study to Establish the Safety and Effectiveness of the SAPIEN 3 Transcatheter Heart Valve in <u>Low Risk</u> Patients who have Severe, Calcific, Aortic Stenosis Requiring Aortic Valve Replacement

| study is conducted in compliance with the protocol, Good Clinical Practice applicable regulatory requirements. | e and all |
|---|---|
| Investigative Site Name | |
| Site Principal Investigator Name (print) | |
| Site Principal Investigator Signature Date | |

I have read this protocol and agree to adhere to its requirements. I will ensure that the

#### 1.0 INTRODUCTION

### 1.1 Background

Prolonged average life expectancy has resulted in an aging population and consequently an increase in the number of patients with acquired, calcific, severe, symptomatic aortic stenosis (AS). Surgical aortic valve replacement (SAVR) has been the standard of care therapy for patients suffering from severe AS. In the aged population, many patients are too sick to undergo AVR, or have extensive comorbidities that preclude the option for surgery [1].

AS is a progressive, debilitating and life-threatening disease if left untreated. Affected individuals are typically > 65 years of age. Bicuspid aortic valve morphology is a common congenital valvular abnormality, occurring in 0.5% to 2% of the general population [2]. AS is also a frequent complication in this population and may occur at a younger age in patients with a bicuspid valves, when compared with patients with a tricuspid aortic valve morphology [3, 4]. The pathology involves progressive calcification of the leaflet bodies which limits normal cusp opening during systole.

The pathophysiology of AS includes an increase in afterload, progressive hypertrophy of the left ventricle, valve obstruction, and a subsequent decrease in systemic and coronary blood flow. Cellular aging and degeneration have been implicated in this form of the disease; diabetes mellitus and hypercholesterolemia are risk factors.

Typically, patients with AS are free from cardiovascular symptoms (e.g. angina, syncope, and/or heart failure) until late in the course of the disease. However, once symptoms manifest, the prognosis is poor without intervention. Survival analyses have demonstrated that the interval from onset of symptoms to time of death is approximately two years in patients with heart failure, three years in those with syncope, and five years in those with angina [5]. Gardin [6] reported that among symptomatic patients with moderate-to- severe AS treated medically, mortality rates after the onset of symptoms were approximately 25% at 1 year, and 50% at 2 years. More than 50% of the reported deaths were sudden.

Grading the severity of AS is based on a variety of hemodynamic and natural history data. According to the ACC/AHA guidelines, AS is best described as a continuum. Relief of aortic valve obstruction typically results in a reduction of symptoms and improvements in hemodynamic parameters, global left ventricle systolic function, as well as a reversal of left ventricular hypertrophy [7].

Echocardiographic criteria for determining the severity of AS, as defined by the 2006 published practice guidelines of the joint ACC/AHA Task Force are described below in Table 1.1-1.

Table 1.1-1 Criteria for Determining Severity of Aortic Stenosis

| Indicator | Mild | Moderate | Severe |
|--------------------|-------|-----------|--------|
| Jet velocity (m/s) | < 3.0 | 3.0 - 4.0 | > 4.0 |

| Mean Gradient (mmHg) | < 25 | 25 - 40 | > 40 |
|---------------------------|-------|-----------|-------|
| Valve area (cm²) | > 1.5 | 1.0 - 1.5 | < 1.0 |
| Valve area index (cm²/m²) | | | < 0.6 |

# 1.1.1 Treatment options prior to introduction of transcatheter aortic valve replacement (TAVR)

Treatment options for patients suffering from symptomatic aortic stenosis, prior to the introduction of transcatheter aortic valve replacement (TAVR), included palliation of symptoms without valve replacement (non-surgical standard therapy), or surgical aortic valve replacement (AVR). Treatment options were determined by patient risk for morbidity or mortality after surgery and patient choice. Non-surgical treatment options, including balloon aortic valvuloplasty, did not provide sustained hemodynamic improvement and have led to poor quality of life and shortened life expectancies [8-10]. Patients considered poor candidates for AVR typically present with significant multiple morbidities or anatomical limitations [11].

Patient frailty may also contribute to the decision to forego surgery. Surgical AVR has demonstrated excellent long term outcomes for patients with aortic valve stenosis, even in high risk populations (STS PROM > 10) [8-10,12-14].

### 1.1.2 Transcatheter aortic valve replacement (TAVR)

Transcatheter aortic valve replacement (TAVR) was first performed in man in 2002 [15], followed by clinical trials and approval for commercialization in Europe in 2007 [16, 17]. It is currently estimated that approximately 300,000 patients have undergone TAVR worldwide. The Edwards THV global clinical research program includes more than 30,000 patients enrolled in 18 clinical studies that include first-inman, feasibility, and pivotal studies as well as randomized controlled trials and post market registries. Results and outcomes from these trials have been publically reported at medical congresses and in peer-reviewed scientific journals. References are provided in [18-25]. The randomized PARTNER I Trial produced the most conclusive evidence of safety and effectiveness of the Edwards SAPIEN THV in high surgical risk (Cohort A) and inoperable (Cohort B) patients with severe, symptomatic aortic stenosis [cite Cohort A and B papers]. The PARTNER II trial has shown safety and effectiveness of the next generation SAPIEN XT THV in high risk and inoperable patients (Cohort B). More recently results of the SAPIEN 3 THV have also demonstrated safety and effectiveness in high risk or greater risk patients with symptomatic heart disease due to severe native calcific aortic stenosis. Early results in intermediate risk patients treated with SAPIEN 3 THV have been presented and longer term intermediate risk results with the SAPIEN XT THV and SAPIEN 3 THV are pending.

### 1.1.3 General Overview of the Study Valve Technology

Edwards Lifesciences has pioneered three variations of heart valve implantation devices over the past 50 years, starting with the first mechanical heart valve in 1960,

followed by the introduction of bioprosthetic tissue valves in 1976 and the advancement of bovine pericardial bioprostheses in the 1980's. The evolution of valve replacement therapy was again expanded in 2004, with the acquisition of transcatheter heart valve technologies from percutaneous valve technologies (PVT). Edwards's research and development expertise in bioprosthetic heart valves was applied to the development of the first generation SAPIEN™ transcatheter heart valve (THV) in 2006 and the introduction of the second generation Edwards SAPIEN XT™ THV in 2008. The current generation Edwards SAPIEN 3 THV was approved by the FDA in June 2015 for patients with aortic valve stenosis who are inoperable or high risk.

Figure 1.1.3-1 Edwards TAVR Technology



The original Edwards SAPIEN THV was comprised of a radiopaque, stainless steel expandable support structure (stent), with an integrated unidirectional trileaflet tissue valve, and a polyethylene terephthalate (PET) fabric cuff. The SAPIEN XT THV has incorporated a cobalt chromium alloy stent and a proprietary valve leaflet shape. The valve tissue is fabricated from three equal sections of bovine pericardium that have been preserved in low concentration solutions of buffered glutaraldehyde to fully crosslink the tissue, while preserving its flexibility and strength. All SAPIEN family THV valves are treated with the Edwards ThermaFix™ process.

The SAPIEN 3 system was designed to improve the rates of procedure related adverse events such as paravalvular leak, major vascular complications and major bleeding. The SAPIEN 3 system also improves ease of use over previous

generations by improving coaxial valve alignment with a greater degree of distal flex in the transfemoral Commander delivery system, with a flex indicator on the handle that shows the degree of articulation in the delivery system, and smaller expandable sheaths with minimum access vessel diameter requirements as low as 5.5 mm.

The inflow aspect of the SAPIEN 3 THV contains an external layer of polyethylene terephthalate (PET) with integral scalloped geometry that is intended to acutely fill the voids between the valve frame and native annulus caused by eccentric calcium deposits and enhances the chronic re-endothelialization process to create a tissue bridge across these voids.



Figure 1.1.3-2: SAPIEN 3 THV

As with the previous generation valve (SAPIEN XT THV), the SAPIEN 3 THV leaflets are designed to be in the semi-closed configuration at the first heartbeat. The SAPIEN 3 THV leaflets, however, were given a small "cap" at the leaflet tips to accommodate proper coaptation under all deployment configurations (i.e., nominal, under, over, and oval). The commissure attachments of the SAPIEN 3 THV also differ slightly from the SAPIEN XT THV; the leaflets are attached via a soft integral tissue tab that is inserted into slots on the frame (rather than attached to a metal bar, as is the SAPIEN XT THV).

Delivery of the SAPIEN 3 THV may be preceded by dilation of the stenotic native aortic valve by means of balloon aortic valvuloplasty (BAV). Predilation tests the expansion capacity of the native valve and prepares the annulus for implantation of the THV. For the Commander delivery system, the THV is carefully mounted and crimped proximal to the balloon. The delivery system is then inserted into the femoral artery (retrograde approach), through the Edwards Expandable Introducer Sheath Set (eSheath), and into a straight section of the descending aorta. The balloon catheter is then brought underneath the valve, in the correct location for valve delivery. The steerable delivery system is then advanced over the aortic arch and delivered to the site of the native stenotic aortic valve.

### 1.2 SAPIEN 3 Clinical History

There were two cohorts, in the PARTNER II (PII) Trial assessing the latest SAPIEN 3 (S3) THV in patients with symptomatic severe aortic stenosis: the high risk operable/inoperable cohort (PIIS3 HR), with nested registry (NR7 – size 20mm) and the intermediate risk cohort (PIIS3i). All patients receiving the S3 THV presented with severe symptomatic calcific aortic stenosis requiring aortic valve replacement (AVR) and due to co-morbidities were at intermediate or higher risk for open chest surgery.

#### 1.2.1 PIIS3HR Cohort of the PARTNER II Trial Results

The PIIS3HR Cohort of the PARTNER II trial was a single arm, non-randomized, historical- controlled study to compare the third generation Edwards SAPIEN 3 THV system with the first generation Edwards SAPIEN THV system in patients who either have high risk for surgery or cannot undergo surgery (inoperable). The 20 mm valve size was introduced into the trial after enrollment was completed with the three larger sizes (23, 26, and 29 mm), thus a separate nested registry, NR7, with identical inclusion/exclusion criteria as the PIIS3HR Cohort except for the aortic annulus diameter, was created to collect data for the 20 mm valve.

Data was collected on 583 eligible patients enrolled at 29 investigational sites in the United States, who were successfully implanted with a SAPIEN 3 THV, which constitutes the Valve Implant (VI) population. Among the VI population, 491 patients were implanted via the transfemoral (TF) access route, and 92 patients via the transapical (TA) or transaortic (TAo) access route. The overall (N=583) average patient age was  $82.6 \pm 8.1$  years, and the average STS score was  $8.6 \pm 3.7$ .

The primary endpoint; composite rate of all-cause mortality, all stroke, and Al ≥ moderate at 30 days was 6.7% in the SAPIEN 3 cohort and 15.6% in the SAPIEN cohort, as shown in Table 1.2.1-1. The resulting proportion difference in the average treatment effect on the treated (ATT) was -6.9% (90% CI: [-13.3%, -0.5%]). Since the upper limit of the CI was < 7.5%, the non–inferiority was met.

Table 1.2.1-1: Primary Endpoint Analysis – Non Inferiority Test SAPIEN 3 vs. SAPIEN

| (PIIS3HR VI<br>Population) Event<br>at 30 days | SAPIEN 3 (N=583) | SAPIEN (N=326) | Weighted Proportion Difference in Average Treatment Effect on the Treated (ATT) |
|---|---|---|---|
| Composite of Death,<br>Stroke and Al ≥<br>Moderate | 6.7% [5.1%, 8.6%] <sup>1</sup> | 15.6% [12.6%, 19.5%] <sup>1</sup> | -6.90% [-13.3%, -0.5%] |
| 90% stratified Wilson confidence interval | | | |

<sup>2.</sup> Wald-type two-sided 90% confidence interval using weighted mean and SD

The Kaplan-Meier (K-M) estimates for all-cause mortality, cardiac mortality, and all stroke at 30 days for the SAPIEN 3 cohort and the SAPIEN cohort are provided in Table 1.2.1-2.

Table 1.2.1-2: Death and Stroke at 30 Days (SAPIEN 3 vs. SAPIEN VI Population)

| | SAPIEN 3<br>(N= 583) | | | SAPIEN<br>(N= 326) | | |
|---|---|---|---|---|---|---|
| Events at 30<br>Days | No.<br>Events | No. Pts<br>with<br>Events | K-M Estimated<br>Event Rate <sup>1</sup><br>(95% CI) | No.<br>Events | No. Pts<br>with<br>Events | K-M Estimated<br>Event Rate<br>(95% CI) |
| Death | 13 | 13 | 2.2%<br>([1.3%, 3.8%]) | 15 | 15 | 4.6%<br>([2.8%, 7.5%]) |
| Cardiac Death | 8 | 8 | 1.4%<br>([0.7%, 2.7%]) | 10 | 10 | 3.1%<br>([1.7%, 5.7%]) |
| All Stroke | 9 | 9 | 1.6%<br>([0.8%, 3.0%]) | 14 | 14 | 4.3%<br>([2.6%, 7.2%]) |

<sup>1</sup>Kaplan-Meier (K-M) estimates at 30 days used time to first event for each patient. Events occurring after 30 days were not included in this analysis.

The proportion of patients with AI  $\geq$  moderate at 30 days was 3.0% in the SAPIEN 3 cohort and 14.3% in the SAPIEN cohort, which were found to be statistically significantly different (p=0.0051;Table 1.2.1-3).

Table 1.2.1-3: Aortic Insufficiency at 30 Days (SAPIEN 3 vs. SAPIEN VI Population)

| Event at 30<br>Days | SAPIEN 3<br>(N = 583) | SAPIEN<br>(N = 326) | Weighted Proportion Difference in Average Treatment Effect on the Treated (ATT) | P-value |
|---|---|---|---|---|
| AI ≥Moderate,<br>n/Total no. (%)<br>[95% CI] | 16/532<br>(3.0%)<br>[1.7%, 4.8%] <sup>1</sup> | 40/280<br>(14.3%)<br>[10.4%, 18.9%] <sup>1</sup> | -13.1%<br>[-22.2%, -3.9%] <sup>2</sup> | 0.0051 |

<sup>1. 95%</sup> Clopper-Pearson Exact confidence interval.

The rate of major vascular complications at 30 days post implantation is shown in Table 1.2.1-4. The rate was 5.0% for the SAPIEN 3 cohort and 10.1% for the SAPIEN cohort, which were found to be not statistically significantly different (p=0.0578).

Table 1.2.1-4: Major Vascular Complications at 30 Days (SAPIEN 3 vs. SAPIEN VI Population)

| Event at 30 Day | SAPIEN 3<br>(N=583) | SAPIEN<br>(N=326) | Weighted Proportion Difference in Average Treatment Effect on the Treated (ATT) | P-value |
|---|---|---|---|---|
| Major Vascular<br>Complications, n/Total<br>no. (%) [95% CI] | 29/583<br>(5.0%)<br>[3.4%, 7.1%] | 33/326<br>(10.1%)<br>[7.1% , 13.9%] <sup>1</sup> | -8.0%<br>[-16.2%, 0.3%] <sup>2</sup> | 0.0578 |

<sup>1. 95%</sup> Clopper-Pearson Exact confidence interval.

<sup>2.</sup> The Wald-type two-sided 90% confidence interval using weighted mean and SD.

<sup>2.</sup> The Wald-type two-sided 90% confidence interval using weighted mean and SD.

Professor Howard Hermann presented the 1-year results from the PIIS3HR cohort at the TCT annual meeting (15 October 2015, San Francisco, California, USA). There were 384 high surgical risk patients (HR) (66.0%) and 199 inoperable patients (INOP) (34%) in this cohort. Between the 30-day and 1-year follow-up there were 71 additional deaths and 5 patients withdrew their participation in the study.

| Table 1.2.1-5: PIIS3 – Clinical Outcomes at 30 Days and 1 Year | in |
|----------------------------------------------------------------|----|
| Combined S3HR/INOP Cohort (AT Population) | |

| Clinical Outcomes (%) | 30 Days | 1 Year |
|---|---|---|
| All-Cause Mortality | 2.2 | 14.4 |
| Cardiac Mortality | 1.4 | 8.1 |
| All Strokes | 1.4 | 4.3 |
| Disabling Stroke* | 0.9 | 2.4 |
| Rehospitalization | 8.0 | 17.1 |
| New Permanent Pacemaker | 13.3 | 16.9 |
| Surgical AVR | 0.2 | 0.6 |
| Structural Valve Deterioration | 0 | 0 |
| Valve Thrombosis | 0 | 0 |
| *No differences between TF and TA/TAo or between HR and INOP subgroup defined as modified Rankin Score ≥ 2 – CEC adjudicated. | | |

A paired analysis of paravalvular regurgitation (PVL) confirmed a sustained change in the none/trace measurement of 64.3% at 30 days and 68.1% at 1 year (Figure 2). No severe PVL was reported and only 2.5% and 2.7% moderate PVL at 30 days or 1 year. A Kaplan- Meier survival analysis by 30 day PVL demonstrated no difference in survival between patients with none/trace and mild PVL (88.0% and 85.9%) but a significant difference in survival between moderate/severe PVL (61.9%) and none/trace PVL (log rank p=0.0015) and mild PVL (log rank p=0.0058).

#### 1.2.2 PIIS3i Cohort of the PARTNER II Trial Results

The PIIS3i Cohort consists of intermediate operable risk patients, who received the Edwards SAPIEN 3 THV. To assure that patients were of "intermediate" risk, an STS score of 4-8% was selected as the inclusion criteria.

The PIIS3i Cohort is a single arm non-randomized, historical-controlled study to compare the transcatheter heart valve therapy with the third generation SAPIEN 3 THV system, to surgical AVR in patients who have an intermediate risk for surgery (control arm patients from PARTNER II Cohort A). The S3 THV was available in 20, 23, 26, and 29 mm sizes. The primary endpoint for the PIIS3i Cohort is a non-hierarchical composite endpoint of death, all stroke, and Al ≥ moderate at 1 year. The primary analysis is a non-inferiority analysis.

A total of 1078 patients were enrolled in S3i, across 51 different sites. The majority of patients were male (62%) and the average patient age was reported as 81.9 years. The average STS score was 5.3% (median 5.2%). The transfemoral access approach was used for valve delivery in 89.0%, transapical approach in 7% and

transaortic approach in 4.0%.

Treatment was conducted with the implantation of a size 26mm valve in 43.7% of patients, followed by size 23mm in 32.2%, size 29mm in 20.0% and size 20mm in 4.1% of patients.

Functional improvement was observed in the AT population of the S3i Cohort, as the number of patients with NYHA classification III/IV decreased from baseline to 30 days from 90% to 13% and 73% to 6%, respectively.

At ACC in 2015, Dr. Susheel Kodali presented 30-day data for S3i, as seen in Table 1.2.2-1 below. S3i clinical events and historical SAPIEN family moderate/severe paravalvular leak at 30 days are described below in Table and Figure 1.2.2- 1 respectively.

Table 1.2.2-1: PIIS3 - 30-Day Clinical Events in S3i (AT Population)

| Event (%) | S3i<br>Overall<br>(n=1076) | \$3i<br>TF<br>(n= 951) | S3i<br>TA/TAo<br>(n=125) |
|---|---|---|---|
| All-Cause Death | 1.1 | 1.1 | 1.6 |
| Cardiovascular Death | 0.9 | 0.9 | 8.0 |
| All Strokes | 2.60 | 2.42 | 4.00 |
| Disabling* | 1.02 | 0.95 | 1.60 |
| Non-Disabling | 1.58 | 1.47 | 2.40 |
| TIA | 0.37 | 0.42 | 0 |
| Major Vascular Complication | 5.6 | 5.9 | 3.2 |
| Life-Threatening Bleeding | 5.4 | 4.4 | 12.9 |
| Annular Rupture | 0.2 | 0.2 | 0 |
| Myocardial Infarction | 0.3 | 0.3 | 0 |
| Coronary Obstruction | 0.4 | 0.4 | 0 |
| Acute Kidney Injury | 0.5 | 0.3 | 1.6 |
| New Permanent Pacemaker | 10.1 | 10.4 | 7.2 |
| Aortic Valve Reintervention | 0.7 | 0.8 | 0 |
| Endocarditis | 0.1 | 0.1 | 0 |



Figure 1.2.2-1: Moderate/Severe PVL at 30 Days of SAPIEN Valves

Although patients with bicuspid valve morphology have historically been excluded from TAVR studies and are not included in the data summaries above, recent reports on the use of S3 in these patients is feasible and effective with favorable valve performance [38].

### 1.3 Design Rationale for the Expanded Indication Trial

Earlier TAVR studies, such as those evaluating the SAPIEN (2006) and SAPIEN XT (2009) THVs, had very selective inclusion criteria that required that the patient populations be high risk for surgery (STS>8) and non-operable, due to concerns of procedural complications including stroke, vascular complications, paravalvular leak (PVL), and conduction disturbances.

As TAVR technology has evolved (Figure 1.1.3-1), such as with the introduction of the S3 enhanced frame geometry, lower frame height, outer skirt to reduce PVL, and improved delivery system utilizing reduced access-vessel diameter requirements, and new studies demonstrate procedural complication rates similar to AVR, there has been a natural progression towards indications including operable patients with decreasing risk profiles.

The tenacious pursuit of technological advances in THV, in combination with over a decade of clinical outcomes, operator experience and input has yielded favorable and steadily improving safety and efficacy. Ongoing studies of the latest generation valve (S3) demonstrate very low rates of significant paravalvular regurgitation, major vascular complications, and bleeding complications; and in intermediate-risk patients - markedly low mortality and stroke at 30 days.

### 1.3.1 Rationale for CT Sub-Study

There have been recent reports of abnormal imaging findings as assessed by multiphasic, ECG-gated CT (i.e., 4D CT) in some patients in the absence of clinical symptoms or echocardiographic abnormalities following TAVR [29, 30]. The abnormal imaging has been described as "leaflet thickening" and "reduced leaflet mobility". This imaging phenomenon has not been definitely linked with clinical valve thrombosis which occurs in 1% or less of TAVR and SAVR bioprostheses. The purpose of the CT sub-study is to further investigate this phenomenon with the following specific objectives:

- 1. Establish the prevalence of the imaging abnormality.
- 2. Establish the relationship between the imaging abnormality and patient, procedural and pharmacology factors.
- 3. Establish the relationship between imaging abnormalities and clinical events.

### 1.3.2 Rationale for Actigraphy/QOL [Enrollment Closed]

Traditional, face-to-face methods for measuring quality of life (QOL) and functional status at defined time points can lack the precision needed to detect changes on a more frequent or even day to day basis. Advances in mobile health (mHealth) technology may enable more regular, convenient and accurate tracking of QOL and physical activity information through applications and wearable devices. These technologies have the potential to help gather more and better data on patients' response to therapy and progression of disease.

The purpose of this sub-study is to investigate the feasibility of assessing change in QOL and activity levels using electronic patient-reported outcome (ePRO) applications and wearable activity trackers. The end goal is to publish study results and explore new and innovative ways of assessing QOL and functional status of aortic stenosis patients with low surgical risks.

### 1.3.3 Rationale for Underrepresented Registry

With the growing use of TAVR for heart valve repair, some US centers are considered "high-volume" due to the number of TAVR procedures performed each year. Results from past TAVR trials have shown that these centers enroll predominately Caucasian patients. Many patients that would benefit from TAVR are not enrolled into trials due to their inability to travel to the larger TAVR centers, due to cultural/socio-economic pressure to remain within their own community, or because there is no referral base for reaching these patients and increasing awareness of TAVR. In order to expand the study of TAVR to a broader group of patients, Edwards is reaching-out to these underrepresented patients by selecting ten additional sites with a predominantly diverse ethnic, cultural, non-Caucasian patient base that perform a more limited number of TAVR procedures per year.

#### 2.0 STUDY OBJECTIVE

The purpose of this trial is to establish the safety and efficacy of the Edwards SAPIEN 3 THV device in patients with severe, calcific, aortic stenosis who are at low operative risk for SAVR.

### 3.0 STUDY DESIGN

This is a prospective, randomized, controlled, multi-center study. Qualified study patients will be randomized 1:1 to receive either the Edwards SAPIEN 3 transcatheter heart valve through iliofemoral access, or SAVR with a commercially available bioprosthetic valve. Selected sites will enroll qualified patients into a CT sub-study. Selected sites may also enroll patients in an Actigraphy/QOL sub-study [Enrollment Closed].

Additional patients will be enrolled in the following single-arm registries:

- Alternative Access Registry (100) [Enrollment Closed]
- Bicuspid Registry (up to 75)
- Underrepresented Populations Registry (up to 100)

#### 4.0 ENROLLMENT

Up to 1182 qualified patients will be randomized at up to 65 actively enrolling sites in the US. It is anticipated that approximately 5-10 sites may be selected outside of the US. Further, up to ten (10) separate US sites from targeted geographic areas will be selected to enroll patients in a single-arm registry for underrepresented populations. No site will be allowed to enroll more than 15% of patients. Edwards will notify investigative sites of enrollment closure.

### **Sub-studies**

Of the 1182 patients, a subset of patients will also be enrolled in the following randomized substudies:

- CT sub-study (up to 440)
- Actigraphy/QOL sub-study (up to 400) [Enrollment Closed]

### Registries

Additional patients will be enrolled in the following single-arm registries:

- Alternative Access Registry (100) [Enrollment Closed]
- Bicuspid Registry (up to 75)
- Underrepresented Populations Registry (up to 100)

### 5.0 STUDY DEVICE

The commercially available Edwards SAPIEN 3 THV and Commander Delivery System will be provided for use in this study for transfemoral delivery of the SAPIEN 3 THV.

### Alternative Access Registry [Enrollment Closed]

The Edwards Commander Delivery System will be provided for subclavian delivery and the Edwards Certitude Delivery System will be provided for transapical and transaortic delivery of the SAPIEN 3 THV as part of Alternative Access Registry.

### **Edwards SAPIEN 3 System**

- Edwards SAPIEN 3 Transcatheter Heart Valve [Model 9600TFX (in 20 mm, 23 mm, 26 mm and 29 mm sizes)]
- Edwards Commander Delivery System (Models 9600LDS20, 9600LDS23, 9600LDS26 and 9600LDS29)
- Edwards Certitude Delivery System (Models 9620TA20, 9620TA23, 9620TA26 and 9620TA29, 9600SDS20, 9600SDS23, 9600SDS26 and 9600SDS29)
- Edwards Certitude Introducer Sheath Set [Models 9620IS18 (18F) and 9620IS21 (21F), 9600IS18 and 9600IS21]
- Edwards Crimper (Model 9600CR)

#### 5.1 Device Descriptions

### 5.1.1 Edwards SAPIEN 3 THV

The SAPIEN 3 THV (Figure 5.1.1-1) is a catheter-delivered heart valve that combines a balloon expandable stent and bioprosthetic valve technology.

The device is comprised of a balloon-expandable, radiopaque, cobalt-chromium alloy frame, a trileaflet bovine pericardial tissue valve, a polyethylene terephthalate (PET) internal fabric skirt, and a PET external sealing ring. The valve tissue is treated with Edwards ThermaFix process, packaged and terminally liquid sterilized in a buffered glutaraldehyde solution.

Figure 5.1.1-1 Edwards SAPIEN 3 Model 9600TFX



The device leaflets are designed to be in the semi-closed configuration at the first heartbeat. The leaflets have a small "cap" at the leaflet tips to accommodate proper coaptation under all deployment configurations (i.e., nominal, under, over and oval). The leaflets are attached via a soft integral tissue tab that is inserted into slots on the frame.

The SAPIEN 3 is available in 4 sizes (Table 5.1.1-1).

| <b>Table 5.1.1-1</b> | Device Sizing |
|----------------------|---------------|
| \ / I A | . 0: |

| Native Valve<br>Annulus Size | Native Valve Annulus Size (CT) | | THV Size | Valve |
|---|---|---|---|---|
| (TEE) | Area | Area Derived<br>Diameter | THV SIZE | Height |
| 16-19 mm | 273 – 345 mm2 | 18.6-21 mm | 20 mm | 15.5 mm |
| 18-22 mm | 338 – 430 mm2 | 20.7-23.4 mm | 23 mm | 18 mm |
| 21-25 mm | 430 – 546 mm2 | 23.4-26.4 mm | 26 mm | 20 mm |
| 24-28 mm | 540 – 683 mm2 | 26.2-29.5 mm | 29 mm | 22.5 mm |

THV size recommendations are based on native valve annulus size, as measured by transesophageal echocardiography (TEE) or computed tomography (CT). Patient anatomical factors and multiple imaging modalities should be considered during THV size selection.

### 5.1.2 Edwards Commander Delivery System

The Commander Delivery System includes:

- Loader
- Qualcrimp Accessory
- 2-piece Crimp Stopper

### **Commander Delivery System**

The Edwards Commander Delivery System consists of a balloon catheter for deployment of the THV and a Flex Catheter to aid in valve alignment to the balloon, tracking and positioning of the THV. The delivery system includes a tapered tip to facilitate crossing of the aortic valve. The handle contains a Flex Wheel to control flexing of the Flex Catheter, and a Balloon Lock and Fine Adjustment Wheel to facilitate valve alignment and positioning of the valve within the aortic annulus. A stylet is included within the guidewire lumen of the delivery system. The Balloon Catheter has radiopaque Valve Alignment Markers defining the working length of the balloon. A radiopaque Center Marker in the balloon is provided to help with valve positioning. A radiopaque Triple Marker proximal to the balloon indicates the Flex Catheter position during deployment.

### **Certitude Delivery System**

The Edwards Certitude Delivery System includes a handle with a Flex Wheel for articulation of the Ballon Catheter and a Loader. The loader allows for the delivery of the crimped THV through the hemostasis valves of the sheath. Three radiopaque indicators on the catheter shaft define the position on the ballon where the THV should be crimped and also provide visualization of the balloon. The THV is crimped between the two radiopaque shoulders on the distal and proximal ends of the balloon. A radiopaque Center Marker in the balloon is provided to help with valve positioning. An inflation and guidewire hub is housed in the handle assembly. A 2-piece crimp stopper and the Qualcrimp crimping accessory are packaged with the delivery system for use during crimping of the THV.

#### Loader

The loader is used to aid insertion of the delivery system into the sheath, and may be removed to utilize the full working length of the inserted device.

#### **Qualcrimp Accessory**

The Qualcrimp accessory is a foam tube composed of polyurethane sponge covered in an outer layer of PET. The SAPIEN 3 THV is placed within the Qualcrimp accessory prior to placing it in crimper. The Qualcrimp accessory is intended to protect the leaflets of the SAPIEN 3 THV during crimping.

### 2-piece Crimp Stopper

This component is discussed in section 5.1.4.

### 5.1.3 Certitude Delivery System

The Certitude Delivery System includes:

- Loader (see 5.1.2)
- Qualcrimp Accessory (see 5.1.2)
- 2-piece Crimp Stopper (see 5.1.4)

The Edwards Certitude Delivery System includes a handle with a Flex Wheel for articulation of the Balloon Catheter and a Loader. The loader allows for the delivery of the crimped THV through the hemostasis valves of the sheath. Three radiopaque indicators on the catheter shaft define the position on the balloon where the THV should be crimped and also provide visualization of the balloon. The THV is crimped between the two radiopaque shoulders on the distal and proximal ends of the balloon. A radiopaque Center Marker in the balloon is provided to help with valve positioning. An inflation and guidewire hub is housed in the handle assembly. A 2-piece crimp stopper and the Qualcrimp crimping accessory are packaged with the delivery system for use during crimping of the THV.

### 5.1.4 Edwards Crimper

The Crimper reduces the diameter of the SAPIEN 3 THV to mount it to the delivery system. The Crimper is comprised of a compression mechanism that is closed with a handle located on the housing. The Crimper is used with a 2-piece Crimp Stopper (packaged with the delivery system) to correctly crimp the THV to the appropriate size.

The SAPIEN 3 THV, the associated Delivery Systems and components will be used per the Instructions for Use (IFU) and after sufficient training of physicians/site personnel has been achieved as determined by the study sponsor. Further descriptions of these devices are provided in the respective IFUs (Appendix C).

#### 6.0 STUDY ENDPOINTS

### 6.1 Primary Endpoint Safety and Effectiveness:

Composite endpoint of all-cause mortality, all stroke, and rehospitalization (valve-related or procedure-related and including heart failure) at 1 year post procedure.

### 6.2 Secondary Endpoints for Labeling

- 1. New onset atrial fibrillation at 30 Days
- 2. Length of index hospitalization
- 3. Death, KCCQ < 45 or KCCQ decrease ≥ 10 points at 30 days
- 4. Death/All Stroke composite at 30 days
- 5. All Stroke at 30 days

### 6.3 Additional Safety and Effectiveness Endpoints

- 1. Mortality (all cause & cardiovascular) at 30 days and 1 year
- 2. Stroke (disabling and nondisabling) at 30 days and 1 year
- 3. Death or stroke at 1 year
- Death or disabling stroke at 30 days and 1 year
- 5. Vascular complications (major) at 30 days and 1 year
- 6. Bleeding complications (life threatening, disabling, or major) at 30 days and 1 year
- 7. Myocardial infarction at 30 days and 1 year
- 8. Acute kidney injury at 30 days
- 9. Renal replacement therapy at 1 year
- 10. New permanent pacemaker implantation resulting from new or worsened conduction disturbances at 30 days and 1 year
- 11. Coronary obstruction requiring intervention at 30 days and 1 year
- 12. New York Heart Association class at 30 days and 1 year
- 13. Hemodynamic valve performance evaluation by echocardiography for aortic valve stenosis and aortic valve regurgitation (paravalvular & central) at 30 days, and years 1, 2, 3, 4, 5, 7, and 10.

- 14. Rehospitalization (valve-related or procedure-related and including heart failure) at 30 days, 1 year, and annually (up to 10 years).
- 15. New onset atrial fibrillation at 1 year
- 16. ICU days, and discharge location
- 17. Structural valve deterioration at years 1-5, 7 and 10
- 18. Days alive and out of hospital at 1 year
- 19. 6-minute walk test at 30 days and 1 year
- 20. Health status as evaluated by Quality of Life questionnaires
  - a. KCCQ at 30 days and 1 year
  - b. EQ-5D-5L at 30 days and 1 year
  - c. SF-36 at 30 days and 1 year

### 6.4 Actigraphy/QOL Substudy Outcome Measures [Enrollment Closed]

### **Primary Outcome Measures:**

- 1. Quality of life as assessed by visual analog scale for pain (VAS Pain) through 30 days.
- 2. Activity during daytime hours (6 am to 10 pm) as assessed by mean daily steps walked through 30 days.

### **Secondary Outcome Measures:**

- 1. Quality of life as assessed by
  - a. VAS Pain 31-44 days
  - b. Kansas City Cardiomyopathy Questionnaire (KCCQ-12) through 44 days
  - c. PF-10 Physical Component Summary through 44 days
- 2. Activity during daytime hours (6 am to 10 pm) through 44 days
  - a. Mean daily steps walked
  - b. Number of minutes active
  - c. Number of minutes sedentary
  - d. Total activity count of the most active 10 hours in the day (which need not be 10 consecutive hours)

#### 7.0 STUDY POPULATION

The study population will be comprised of patients with severe, calcific, aortic stenosis who are at low operative risk for SAVR.

#### 7.1 Inclusion Criteria

All study participants must meet the following inclusion criteria.

- 1. Severe, calcific aortic stenosis meeting the following criteria:
  - AVA  $\leq 1.0 \text{ cm}^2 \text{ or AVA index } \leq 0.6 \text{ cm}^2/\text{m}^2$
  - Jet velocity ≥ 4.0 m/s or mean gradient ≥ 40 mmHg <u>AND</u>
  - 1) NYHA Functional Class ≥ 2 OR 2) exercise tolerance test that demonstrates a limited exercise capacity, abnormal BP response, or arrhythmia OR 3) asymptomatic with LVEF <50%

Note: Qualifying echo must be within the 90 days prior to randomization.

- 2. Heart team agrees the patient has a low risk of operative mortality and an STS < 4.
- The study patient has been informed of the nature of the study, agrees to its
  provisions and has provided written informed consent as approved by the
  Institutional Review Board (IRB)/Ethics Committee (EC) of the respective
  clinical site.

#### 7.2 Exclusion Criteria

Candidates will be excluded from the study if any of the following conditions are present:

- 1. Native aortic annulus size unsuitable for sizes 20, 23, 26, or 29mm THV based on 3D imaging analysis
- 2. Iliofemoral vessel characteristics that would preclude safe passage of the introducer sheath
- Evidence of an acute myocardial infarction ≤ 1 month (30 days) before randomization
- Aortic valve is unicuspid, bicuspid, or non-calcified
- 5. Severe aortic regurgitation (>3+)
- 6. Severe mitral regurgitation (>3+) ≥ moderate stenosis
- 7. Pre-existing mechanical or bioprosthetic valve in any position. (of note, mitral ring is not an exclusion).
- 8. Complex coronary artery disease:

- a. Unprotected left main coronary artery
- b. Syntax score > 32 (in the absence of prior revascularization)
- c. Heart Team assessment that optimal revascularization cannot be performed
- 9. Symptomatic carotid or vertebral artery disease or successful treatment of carotid stenosis within 30 days of randomization
- Leukopenia (WBC < 3000 cell/mL), anemia (Hgb < 9 g/dL), Thrombocytopenia (Plt < 50,000 cell/mL), history of bleeding diathesis or coagulopathy, or hypercoagulable states
- 11. Hemodynamic or respiratory instability requiring inotropic support, mechanical ventilation or mechanical heart assistance within 30 days of randomization
- 12. Hypertrophic cardiomyopathy with obstruction (HOCM)
- 13. Ventricular dysfunction with LVEF < 30%
- 14. Cardiac imaging (echo, CT, and/or MRI) evidence of intracardiac mass, thrombus or vegetation
- 15. Inability to tolerate or condition precluding treatment with antithrombotic/anticoagulation therapy during or after the valve implant procedure
- 16. Stroke or transient ischemic attack (TIA) within 90 days of randomization
- 17. Renal insufficiency (eGFR < 30 ml/min per the Cockcroft-Gault formula) and/or renal replacement therapy at the time of screening.
- 18. Active bacterial endocarditis within 180 days of randomization
- 19. Severe lung disease (FEV1 < 50% predicted) or currently on home oxygen
- 20. Severe pulmonary hypertension (e.g., PA systolic pressure ≥ 2/3 systemic pressure)
- 21. History of cirrhosis or any active liver disease
- 22. Significant frailty as determined by the Heart Team (after objective assessment of frailty parameters).
- Significant abdominal or thoracic aortic disease (such as porcelain aorta, aneurysm, severe clacification, aortic coarctation, etc.) that would preclude safe passage of the delivery system or cannulation and aortotomy for surgical AVR
- 24. Hostile chest or conditions or complications from prior surgery that would preclude safe reoperation (i.e., mediastinitis, radiation damage, abnormal chest wall, adhesion of aorta or IMA to sternum, etc.)

- 25. Patient refuses blood products
- 26. BMI >  $50 \text{ kg/m}^2$
- 27. Estimated life expectancy < 24 months
- 28. Absolute contraindications or allergy to iodinated contrast that cannot be adequately treated with pre-medication
- 29. Immobility that would prevent completion of study procedures (e.g. six-minute walk tests, etc.)
- 30. Patient is not a candidate for both arms of the study (not applicable to single-arm registries)
- 31. Currently participating in an investigational drug or another device study. Note: Trials requiring extended follow-up for products that were investigational, but have since become commercially available, are not considered investigational trials. Observational studies are not considered exclusionary.

### 7.3 CT Imaging Sub-Study

Sites with the ability to perform high quality 4D scans will be selected to participate in a CT sub-study.

### 7.3.1 Inclusion Criteria

All CT sub-study participants must meet inclusion criteria listed in Section 7.1.

#### 7.3.2 Exclusion Criteria

In addition to the exclusion criteria in section 7.2, candidates will be excluded from the sub- study if the following is present:

- 1. Condition requiring or planned use of anticoagulants following the valve implant procedure.
- 2. GFR <50
- 3. Inability to perform high-quality MDCT study for any reason (e.g., atrial fibrillation with rapid ventricular response)

### 7.4 Actigraphy/QOL Sub-Study Eligibility Criteria [Enrollment Closed]

Select sites will be invited to participate in an Actigraphy/QOL sub-study. Patients must meet all the eligibility criteria of the PARTNER 3 study in sections 7.1 and 7.2. In addition, they must demonstrate a basic working knowledge of and ability to use the devices specified in the sub-study. Patients who are non-ambulatory (i.e, wheelchair bound) will not be eligible.

### 7.5 Alternative Access Registry Eligibility Criteria [Enrollment Closed]

Patients who do not have appropriate iliofemoral access as defined in exclusion criterion 2 in Section 7.2 but meet all other inclusion and exclusion criteria should be considered for enrollment in the alternative access registry.

### 7.6 Bicuspid Registry Eligibility Criteria

Patients who have a bicuspid valve as determined by the CT core lab (e.g., exclusion criterion 4) should be considered for enrollment in this registry if they meet all other eligibility criteria in Sections 7.1 and 7.2 and none of the following additional exclusion criteria:

- 1. Aneurysmal ascending aorta (i.e., >4.0 cm)
- Severe or bulky calcification of the left ventricular outflow tract (LVOT) or raphe that would increase the risk of annular injury or significant paravalvular leak (PVL) post TAVR
- 3. Coronary anatomy that increases the risk of coronary artery obstruction post TAVR
- 4. Positive urine or serum pregnancy test in female subjects of childbearing potential

### 7.7 Underrepresented Populations Registry Eligibility Criteria

Up to ten (10) sites from underrepresented geographical locations will be selected to enroll patients in a single-arm registry for underrepresented populations. Patients at these sites are eligible for this registry if they meet all eligibility criteria in Sections 7.1 and 7.2.

#### 8.0 STUDY PROCEDURES

### 8.1 Screening Period

The screening period is designed to obtain patient consent, determine patient eligibility for the study, and to submit the presentation for case review. The Screening Visit procedures will occur within the 30 days prior to the valve implant procedure, unless otherwise noted below. All patients that sign an informed consent will be entered into the electronic database (EDC) and be assigned a Subject ID. All assessments performed will be entered into EDC.

Patients that have signed the informed consent and do not meet the inclusion/exclusion criteria in Section 7.1 and 7.2 will be considered a Screen Failure (SF). All assessments performed and the inclusion or exclusion criteria that was not met will be entered into EDC.

The patient status will be considered 'Discontinued' if the following occur during the screening period:

- The patient withdraws consent or expires prior to or after the Case Review.
- The patient completes all of the screening procedures, including Case Review call, and the Case Review is not approved.

All assessments performed and the reason for discontinuation will be entered into EDC and the Exit form will be completed.

The following information will be collected during the screening period:

### Consent:

Patient informed consent completion, (section 8.1.1)

### Operability:

STS Risk Score

#### Other Assessments:

- Logistic EuroSCORE
- EuroSCORE II

### Systems:

- Medical history and physical assessment (including height, weight, blood pressure, and heart rate).
- Medications including all antithrombotics/anticoagulants and HMG coA reductase inhibitors.

### **Cardiopulmonary:**

- Canadian Cardiovascular Society (CCS) status of angina
- 12-lead ECG
- New York Heart Association Class (NYHA Classification)
- Comprehensive transthoracic (TTE) echocardiogram, including assessment
  of aortic valve gradients (mean and peak), areas, indices, degree of
  regurgitation, left ventricle systolic function (global and segmental).
   Qualifying echo must be performed within 90 days prior to randomization.
- Cardiac imaging (TEE, CT, or cardiac MRI) with 3D reconstruction to determine aortic valve annulus area. Qualifying cardiac imaging must be performed within 1 year prior to randomization, unless clinically indicated.
- CT Angiography, including thoracic and abdomen scan with visualization of iliac and femoral arteries. Qualifying iliofemoral CT must be performed within 1 year prior to randomization.
- Left heart catheterization to assess the severity of aortic stenosis and severity of coronary artery disease, if applicable. Qualifying catheterization must be performed within 1 year prior to randomization, unless clinically indicated.
- SYNTAX Score for significant native coronary artery disease (CAD)
- Pulmonary Function Test for patients with a history of lung disease

### **Neurological Assessments:**

- Mini Mental State Examination (MMSE), (Appendix G)
- National Institutes of Health Stroke Scale (NIHSS), (Appendix H)
- Modified Rankin Scale (mRS), (Appendix I)

Every effort should be made to have a neurologist (or neurology fellow) perform the NIHSS and mRS assessments. If it is not possible to have the neurologist/fellow perform the assessments within the protocol-specified visit window, a certified study team member may perform the assessments.

#### **Functional Assessments:**

- Six Minute Walk Test (6MWT), (Appendix E)
- Frailty Index (5 Meter Walk Test (5MWT), grip strength, Activities of Daily Living (ADL), and Albumin laboratory) (Appendix F)
- Quality of Life Assessments
  - KCCQ (Appendix N)
  - EQ-5D-5L (Appendix M)
  - SF-36 (Appendix O)

### **Clinical Laboratory Tests:**

- WBC, Hgb, and platelet count
- PT or INR
- CK/CKMB and/or troponins ≤ 72 hours before the valve implant procedure
- Creatinine
- eGFR
- Albumin (as part of Frailty Index)
- Total Bilirubin
- AST/ALT (required for patients with chronic liver disease)
- B-type natriuretic peptide (BNP)

### 8.1.1 Informed Consent

The study investigator(s) and support staff will approach patients with severe, aortic stenosis to assess their interest in participating in the study by providing them an overview of the study including the background, risks, benefits and study procedures. If patients are interested in participating in the study, the study patient will sign the Institutional Review Board (IRB) approved informed consent form prior to any study specific procedures are performed. All patients consented should be entered into the study's electronic database (EDC).

#### 8.1.2 Case Review

The Case Review Board is a select review committee comprised of Investigators who are participating in the trial. The role of the Case Review Board is to review submitted cases to determine if the patient is an appropriate candidate for the trial, with a focus on confirming patient operative risk, valve sizing, appropriate vascular

access, valve morphology and any relevant clinical factors impacting enrollment eligibility. In addition, the Heart Team's strategy for treatment of concomitant coronary artery disease will be reviewed, as applicable. Before a case is submitted for review, the site Principal Investigator and Heart Team will screen the patient for operative risk and fundamental enrollment criteria. It is required that at least one site surgeon Investigator personally examine the patient to determine operative risk. Once fully screened and deemed an appropriate candidate, the site will submit the case for review and approval consideration by the Case Review Board. The Sponsor will maintain a record of the case presentation and case approval notes.

### 8.2 Randomization and Enrollment

Once all screening procedures have been completed, all inclusion/exclusion criteria have been confirmed and the Case Review has been completed and approved, the patient is eligible to be randomized or enrolled into one of the single-arm registries.

Randomization will occur centrally. To randomize a patient, the investigative site will enter the subject into the designated electronic system and obtain the treatment assignment (TAVR or SAVR). Once the assignment has been made, the subject will be considered randomized and enrolled into the study.

All randomized patients will be considered part of the Intent to Treat (ITT) population. Randomized patients are considered enrolled in the study; for the randomized patients, the terms "randomized" and "enrolled" have the same meaning.

If the patient has been enrolled and the patient withdraws consent prior to the valve implant procedure start, the patient will be considered discontinued. All assessments performed and the reason for withdrawal will be entered into EDC and the Exit form will be completed.

### 8.3 Procedure (Day 0)

The valve implant procedure should occur within 14 days of randomization and no later than 30 days after informed consent is obtained. The date of the valve implant procedure is considered Day 0. The valve implant procedure will be considered to have started when:

- The first interventional access related puncture (venous or arterial) is established for TAVR.
- The first skin incision is performed for SAVR.

Performance of TEE does not by itself constitute start of procedure.

For those patients receiving TAVR, the commercially available SAPIEN 3 THV with the Commander Delivery System, or the Certitude Delivery system if treated with a transapical or transaortic approach as part of the Alternative Access registry [enrollment closed], and components will be used per the most current Instructions for Use (IFU) at all times for device sizing, preparation, and recommended implant

procedure. Refer to Appendix C for the IFUs to be used in this study.

For those patients receiving SAVR, a commercially available bioprosthetic surgical valve and associated components will be used according to institution standard of care.

Day 0 will be used to schedule all subsequent visits and calculate visit windows. Patients who receive the assigned TAVR or SAVR implant will continue in the study and complete the study through year 10 according to the visits and events described in section 8.0 and Schedule of Procedures.

Day 0 valve implant procedure assessments will include the following:

### Systems:

- Medications including all antithrombotics/anticoagulants and HMG coA reductase inhibitors.
- Adverse event assessment

### Cardiopulmonary:

- Comprehensive transthoracic (TTE) or transesophageal (TEE) echocardiogram
- Supra-aortic angiogram or TEE

If the valve implant is aborted (prior to or after the start of the valve implant procedure), the Day 0 visit may be re-scheduled if the patient continues to meet all inclusion/exclusion criteria.

### 8.3.1 Device Preparation

A detailed description of device preparation and required equipment is supplied in the Instructions for Use (Appendix C).

#### 8.3.2 Procedure Recommendations

Table 8.3.2-1 outlines the recommended anticoagulation/antithrombotic regimen. The categories were developed by The PARTNER II Trial Patient and Procedure Management

Steering Committee. There are no current validated guidelines in this specific study population, however, the literature was surveyed and used as guidance for the following proposed guidelines [26].

NOTE: The CHAD score only applied to patients in Atrial Fibrillation (AF) and had not been validated in non-AF patient populations; therefore the CHAD score reference was used as one among many guidelines to establish the risk stratification for intensity of anticoagulation regimen.
Table 8.3.2-1 Recommended anticoagulation/antithrombotic regimen

| AVR | TAVR |
|---|---|
| Pre valve impl | ant procedure |
| Aspirin 81-100 mg QD | Aspirin 81-100 mg QD |
| <ul> <li>Patients with BMS within one month or drug eluting stent (DES) within 12 months should be continued on Clopidogrel/prasugrel prior to their implant procedure</li> <li>Patients in atrial fibrillation on warfarin should be bridged with LMW or UF heparin prior to the implant procedure</li> <li>Patients with persistent or paroxysmal atrial fibrillation, not on anticoagulation, will not be required to have a TEE to rule out LA thrombus prior to the implant procedure. If intraprocedural TEE during AVR reveals thrombus, implant procedure will be aborted and delayed until patient has been on warfarin or dabigatran for 30 days. In patients in the surgical group with LA clot seen on intraoperative TEE, implant procedure can proceed per surgical standard of care</li> </ul> | <ul> <li>Patients with BMS within one month or DES within 12 months should be continued on Clopidogrel/prasugrel prior to their implant procedure</li> <li>Patients in atrial fibrillation on warfarin should be bridged with LMW or UF heparin prior to the implant procedure</li> <li>Patients with persistent or paroxysmal atrial fibrillation, not on anticoagulation, will not be required to have a TEE to rule out LA thrombus prior to implant procedure. If intraprocedural TEE during TAVR reveals thrombus, implant procedure will be aborted and delayed until patient has been on warfarin or dabigatran for 30 days. Note: thrombus must be eliminated in order to proceed with TAVR.</li> <li>In patients undergoing concomitant TAVR/PCI, clopidogrel loading with either 300mg or 600mg prior to the implant procedure is recommended in addition to ASA</li> </ul> |
| Intrapro | |
| Heparin will be given to achieve/ maintain ACT≥250 | Heparin will be given to achieve/ maintain ACT <u>&gt;</u> 250 sec. |

| | AVR | TAVR |
|---|---|---|
| | Post valve imp | lant procedure |
| Category I for Stroke Risk No atrial fibrillation, No recent stents | <ul> <li>ASA 81mg qd</li> <li>Clopidogrel 75qd started 24<br/>hours post-surgery for at least<br/>one month if clinically safe and<br/>at the discretion of the surgical<br/>team. In centers that use<br/>warfarin post-surgical AVR,<br/>Clopidogrel will not be started</li> </ul> | <ul> <li>ASA 81mg qd</li> <li>Clopidogrel 300mg load within 6 hours of the implant procedure (either pre or post)</li> <li>Clopidogrel 75mg qd for at least one month post implant procedure</li> </ul> |
| Category II for Stroke Risk No atrial fibrillation, recent stents | <ul> <li>ASA 81mg qd</li> <li>Clopidogrel should not be discontinued prior to surgery if patient had BMS within one month or DES in 12 months</li> <li>Clopidogrel 75qd started 24 hours post-surgery if clinically safe and continued for at least one month post-surgical AVR in those with BMS and a total</li> </ul> | <ul> <li>ASA 81mg qd</li> <li>Clopidogrel 75mg qd should be continued prior to the implant procedure and after the implant procedure without interruption for at least one month after BMS and 12 months after DES</li> </ul> |
| Category III for Stroke Risk Atrial fibrillation, no recent stents | <ul> <li>ASA 81mg qd</li> <li>Patients should be started on warfarin or dabigatran 24 hours post AVR if clinically safe and this should be continued for at least one month or indefinitely if possible. If clinically safe, patient's being started on warfarin should be bridged with unfractionated or low molecular weight heparin until INR therapeutic.</li> <li>If patients are not a candidate for warfarin or dagibatran, Clopidogrel 75mg qd (in addition to ASA 81 mg) can be</li> </ul> | <ul> <li>ASA 81mg qd</li> <li>Patients should be started on warfarin or dabigatran 24 hours post TAVR if clinically safe and this should be continued for at least one month or indefinitely if possible. If clinically safe, patients started on warfarin should be bridged with unfractionated or low molecular weight heparin until INR therapeutic.</li> <li>If patients are not a candidate for warfarin or dagibatran, Clopidogrel 75mg qd can be considered as an alternative</li> </ul> |

| | AVR | TAVR |
|---|---|---|
| Category IV<br>for Stroke<br>Risk<br>Atrial<br>fibrillation,<br>recent<br>stents | <ul> <li>ASA 81mg qd</li> <li>Clopidogrel 75mg qd for at least one month post BMS or 12 months post DES</li> <li>Patients should be started on warfarin or dabigatran 24 hours post AVR if clinically safe and continued indefinitely. If clinically safe, patients being started on warfarin should be bridged with UF or LMW heparin until INR therapeutic.</li> </ul> | <ul> <li>ASA 81mg qd</li> <li>Clopidogrel 75mg qd for at least one month post BMS or 12 months post DES</li> <li>Patients should be started on warfarin or dabigatran 24 hours post TAVR if clinically safe and continued indefinitely. If clinically safe, patient's being started on warfarin should be bridged with UF or LMW heparin until INR therapeutic.</li> </ul> |

Note: Any changes to antithrombotic/anticoagulation regimen from study visit to study visit will be noted on the Case Report Form (CRF) including reason for change.

# 8.3.3 Antibiotic Prophylaxis

Study patients should be prophylactically treated for endocarditis per the recommendations of the American Heart Association.

#### 8.3.4 Contrast Media

Careful management of contrast media is required. Accurate measurement of the contrast used will be captured in the case report form.

# 8.3.5 Radiation Precautions

Radiation precautions will be adhered to per institutional standards. Total procedural radiation exposure will be documented on the case report forms in accordance with institutional measures (i.e. total procedural fluoroscopy time, dosage, etc.).

Radiation exposure of 6-15 mSv is estimated for the Screening CT and each Sub-study CT [27]. If a radiation induced skin injury is suspected, the Investigator should see the patient at an office visit, and should arrange for appropriate follow-up care.

#### 8.4 Post Procedure

The post implant procedure time period is defined as the 48 hours after the patient exits the cath lab/ operating room. Study patients will be continuously monitored clinically, hemodynamically, and electrocardiographically during catheterization for all local, systemic side effects and complications. After completion of the implant procedure, all study patients will be monitored per institution standard of care. Subsequent monitoring will also be continued according to institutional standard of care.

The following information will be collected during the Post Procedure time period:

## Systems:

- Medications including all antithrombotics/anticoagulants and HMG coA reductase inhibitors.
- Adverse event assessment

# Cardiopulmonary:

12-lead ECG

## **Clinical Laboratory Tests:**

- WBC, Hgb, and platelet count
- PT or INR
- CK/CKMB and/or Troponins will be performed to monitor the patient's cardiac enzymes at 3 different time intervals. Of note, patients discharged prior to the completion of 24 hour series of lab tests will not be issued deviations.
  - The first lab draw post implant procedure (within 8 hours of exit from the cath lab
    - / operating room)
  - The second lab draw, (6 8 hours after the first lab draw)
  - The third lab draw, (6 8 hours after the second lab draw)
- Creatinine

## Neurological assessments:

NIHSS

All patients should be assessed post-procedure to determine if there is evidence of neurological impairment. If symptoms of stroke are suspected, the NIHSS should be performed. For all patients diagnosed with stroke after procedure, a follow-up mRS assessment 90 days after the diagnosis should be performed (on site or phone calls). Evaluation of stroke by mRS between 30 and 90 days is acceptable if 90-day follow-up not available. Every effort should be made to have a neurologist (or neurology fellow) perform the assessment. If it is not possible to have the neurologist/fellow complete this within the protocol-specified visit window, a certified study team member may perform the assessments.

# 8.5 Discharge

Discharge is the actual date and time the patient is discharged. For patients discharged within 48 hours of exiting the cath lab / operating room, it is not required to repeat tests collected during the Post Procedure period that are also required for the discharge visit. If the patient was discharged over a weekend or holiday, the discharge assessments may be completed on the last weekday prior to discharge.

The following information will be collected for study patients within 24 hours of the date and time of discharge.

## Systems:

- Physical assessment including weight, blood pressure, and heart rate
- Medications including all antithrombotics/anticoagulants and HMG coA reductase inhibitors.
- Adverse event assessment

# Cardiopulmonary:

- NYHA classification
- Comprehensive transthoracic echocardiogram (TTE)

# **Clinical Laboratory Tests:**

- WBC, Hgb, and platelet count
- PT or INR
- Creatinine
- BNP

# **Neurological Assessments:**

NIHSS

All patients should be assessed at Discharge to determine if there is evidence of neurological impairment. If symptoms of stroke are suspected, the NIHSS should be performed. For all patients diagnosed with stroke after procedure, a follow-up mRS assessment 90 days after the diagnosis should be performed (on site or phone calls). Evaluation of stroke by mRS between 30 and 90 days is acceptable if 90-day follow-up not available. Every effort should be made to have a neurologist (or neurology fellow) perform the assessment. If it is not possible to have the neurologist/fellow complete this within the protocol-specified visit window, a certified study team member may perform the assessments.

## 8.6 Post Procedure Follow Up Visits

## 8.6.1 30 Day Post Procedure Visit

The 30 day post procedure visit window will be calculated from the Day 0 valve implant date. The visit window is +7 days.

The following data will be collected for all study patients 30 days post implant procedure.

## Systems:

- Physical assessment including weight, blood pressure, and heart rate
- Medications including all antithrombotics/anticoagulants and HMG coA reductase inhibitors.
- Adverse event assessment

## Cardiopulmonary:

- 12-lead ECG
- NYHA classification
- Comprehensive transthoracic echocardiogram (TTE)
- CT Scan (only for those patients in the CT sub-study) (section 12.5.2.1)

## **Neurological Assessments:**

- MMSE
- NIHSS
- Modified Rankin Scale

For all patients diagnosed with stroke between discharge and 30 days post-procedure, a follow-up mRS assessment 90 days after the diagnosis should be performed (on site or phone calls). Evaluation of stroke by mRS between 30 and 90 days is acceptable if 90-day follow-up not available. Every effort should be made to have a neurologist (or neurology fellow) complete the NIHSS and mRS assessment. If it is not possible to have the neurologist/fellow complete this within the protocol-specified visit window, a certified study team member may perform the assessments.

#### **Functional Assessments:**

- 6MWT
- Quality of Life Questionnaires
  - KCCQ
  - EQ-5D-5L
  - SF-36

## **Clinical Laboratory Tests:**

- WBC, Hgb, and platelet count
- Creatinine
- BNP

## 8.6.2 6 Month Post Procedure Visit

The 6 month post implant procedure visit window will be calculated from the Day 0 visit date. The visit window is +14 days.

The following data will be collected for all study patients 6 months post valve implant procedure.

#### Systems:

- Physical assessment including weight, blood pressure, and heart rate
- Medications including all antithrombotics/anticoagulants and HMG-CoA reductase inhibitors.
- Adverse Event assessment

## Cardiopulmonary:

NYHA classification

## **Neurological Assessments:**

The following assessments should be completed for all patients diagnosed with stroke after the procedure:

- NIHSS
- Modified Rankin Scale

For all patients diagnosed with stroke between 30 days and 6 months post-procedure, a follow-up mRS assessment 90 days after the diagnosis should be performed (on site or phone calls). Evaluation of stroke by mRS between 30 and 90 days is acceptable if 90-day follow-up not available. Every effort should be made to have a neurologist (or neurology fellow) perform the assessment. If it is not possible to have the neurologist/fellow complete this within the protocol-specified visit window, a certified study team member may perform the assessments.

#### **Functional Assessments:**

- Quality of Life Questionnaires
  - KCCQ
  - EQ-5D-5L
  - SF-36

## 8.6.3 12 Month Post Procedure Visit

The 12 month post implant procedure visit window will be calculated from the Day 0 valve implant date. The visit window is +30 days.

The following data will be collected for all study patients 12 month post implant procedure.

#### Systems:

- Physical assessment, (including weight and blood pressure)
- Medications including all antithrombotics/anticoagulants and HMG-CoA reductase inhibitors.
- Adverse Event assessment

## Cardiopulmonary:

- 12 lead ECG
- NYHA classification
- Comprehensive transthoracic echocardiogram (TTE)
- CT Scan (only for those patients in the CT sub-study)

## **Neurological Assessments:**

MMSE

The following assessments should be completed for all patients diagnosed with stroke after the procedure:

- NIHSS
- Modified Rankin Scale

For all patients diagnosed with stroke between 6 months and 12 months post-procedure, a follow-up mRS assessment 90 days after the diagnosis should be performed (on site or phone calls). Evaluation of stroke by mRS between 30 and 90 days is acceptable if 90-day follow-up not available. Every effort should be made to have a neurologist (or neurology fellow) perform the assessment. If it is not possible to have the neurologist/fellow complete this within the protocol-specified visit window, a certified study team member may perform the assessments.

#### **Functional Assessments:**

- 6MWT
- Quality of Life Questionnaires
  - KCCQ
  - EQ-5D-5L
  - SF-36

# 8.6.4 Years 2 through 10 Annual Post Procedure Visit

The yearly post implant procedure visit window will be calculated from the Day 0 valve implant date. The visit window is +45 days.

The following data will be collected for all study patient's years 2 through 10 annually post implant procedure visit.

## Systems:

- Physical assessment including weight, blood pressure and heart rate
- Medications including all antithrombotics/anticoagulants and HMG coA reductase inhibitors.
- · Adverse event assessment

# Cardiopulmonary:

- NYHA classification
- Comprehensive transthoracic echocardiogram (TTE) [years 2, 3, 4, 5, 7, and 10 only]

#### **Functional Assessments:**

- Quality of Life Questionnaire
  - KCCQ
  - SF-36

## **Neurological Assessment (2 Year Post Procedure Visit only):**

For all patients diagnosed with stroke between 1 year and up to 2 years post-procedure, a follow-up mRS assessment 90 days after the diagnosis should be performed (on site or phone calls). Evaluation of stroke by mRS between 30 and 90 days is acceptable if 90-day follow-up not available. Every effort should be made to have a neurologist (or neurology fellow) perform the assessment. If it is not possible to have the neurologist/fellow complete this within the protocol-specified visit window, a certified study team member may perform the assessments.

#### 8.7 Missed Visits

Site personnel should make all reasonable efforts to locate and communicate with the subject at each visit time point. For each missed visit, a minimum of 3 attempts to contact the subject should be recorded in source documentation, including date, time and name of site personnel trying to make contact.

# 8.8 Lost to Follow-Up

If the patient has missed multiple visits (with multiple attempts to contact as noted in section 8.9) and no record of death is found, the patient may be considered a lost to follow up. All assessments performed and the reason for discontinuation will be entered into EDC and Exit form completed.

## 8.9 Discontinuation after entering procedure room

Every patient should be encouraged to remain in the study until they have completed the protocol required follow-up period. If the patient discontinues prematurely from the study, the reason for discontinuation must be documented. All attempts should be made to have the patient come into the clinic for an Exit visit.

If the following situations occur, the patient status will be considered 'Discontinued':

- The patient has entered the cath lab or operating room (procedure room) and an inclusion or exclusion criteria failure has been found.
- The patient has entered the procedure room and expires prior to the start of the valve implant procedure.
- The patient expires after the procedure has started.
- The patient withdraws consent after the valve implant procedure and prior to the final study visit.
- The patient expires after the valve implant procedure and prior to the final study visit.

If the patient is randomized to TAVR but has a THV other than the SAPIEN 3 implanted, the patient status will be considered discontinued and the patient will be monitored through Day 30 or until any AEs occurring are resolved.

All assessments performed and the reason for discontinuation will be entered into EDC and Exit form completed.

# 8.10 Randomized TAVR patient receives SAVR

Patients who are randomized to TAVR but undergo SAVR will continue in the study and complete all remaining study visits. The reason for conversion from TAVR to SAVR will be entered into EDC.

# 8.11 Death Registries

In the event of a patient lost to follow-up or early withdrawal, Edwards may opt to search the Social Security Death Index and/or other death registries. If the patient is confirmed to be expired, Edwards may opt to obtain the death certificate.

# **Schedule of Procedures**

| | Screening | Procedure<br>(Valve Implant) | Post<br>Procedure | Discharge | 30D | 6M | 12M | 2-10Y |
|---|---|---|---|---|---|---|---|---|
| Visit Window | Day -30 <sup>d</sup> | Day 0 | | | +7 days | +14 days | +30 days | +45 days |
| Physical Assessment | | | | | | | | |
| Informed Consent | Х | | | | | | | |
| Medical History | Х | | | | | | | |
| Physical Assessment | Х | | | Х | Х | Х | Х | Х |
| CCS Angina | X | | | | | | | |
| NYHA Classification | X | | | Х | Х | Х | Х | Х |
| MMSE | Х | | | | Х | | Х | |
| STS Risk Score | Х | | | | | | | |
| Logistic EuroSCORE | Х | | | | | | | |
| EuroSCORE II | Х | | | | | | | |
| SYNTAX Score | X | | | | | | | |
| Medications | X | Х | Х | Х | Х | Х | Х | Х |
| Adverse Event Assessment | | Х | Х | Х | Х | Х | Х | Х |
| NIHSSa | Х | | Хa | Хa | Х | Хa | Χa | |
| Modified Rankin Scale <sup>a</sup> | Х | | | | Х | Хa | Χa | |
| 6 Minute Walk Test | X | | | | Х | | Х | |
| Frailty Index <sup>k</sup> | Х | | | | | | | |
| Laboratory Measurements | | | | | | | | |
| WBC, Hgb, Platelet Count | Х | | Х | Х | Х | | | |
| PT or INR | X | | Х | Х | | | | |
| CK/CKMB and/or Troponins | <b>X</b> b | | Χc | | | | | |
| eGFR | Х | | | | | | | |
| Creatinine | Х | | Х | X | Х | | | |
| Albumin, Total Bilirubin | Х | | | | | | | |
| AST/ALT <sup>m</sup> | Х | | | | | | | |
| BNP | Х | | | Х | Х | | | |

| | Screening | Procedure (Valve Implant) | Post Procedure | Discharge | 30D | 6M | 12M | 2-10Y |
|---|---|---|---|---|---|---|---|---|
| Visit Window | Day -30 <sup>d</sup> | Day 0 | | | +7 days | +14 days | +30 days | +45 days |
| Non-Invasive Tests | | | | | | | | |
| Pulmonary Function Test (PFT) | Χı | | | | | | | |
| ECG | Х | | Х | | Х | | Х | |
| Echocardiogram (TTE) | Xe | <b>X</b> j | | Х | Х | | Х | Xe |
| Final Eligibility Review | | | | | | | | |
| Case Review <sup>i</sup> | Х | | | | | | | |
| Invasive Tests | | | | | | | | |
| Sub-study CTf | | | | | Х | | Х | |
| 3D Cardiac imaging (CT, TEE, or<br>cardiac MRI) հ | Х | | | | | | | |
| Iliofemoral CT Angiography <sup>g</sup> | Х | | | | | | | |
| Valve implant procedure (TAVR or SAVR) | | Х | | | | | | |
| Cardiac Catheterization | Х | | | | | | | |
| Supra-aortic angiogram or TEE | | <b>X</b> <sup>j</sup> | | | | | | |
| Quality-of-Life Assessments | | | | | | | | |
| KCCQ | Х | | | | Х | Х | Х | Х |
| EQ-5D-5L | Х | | | | Х | Х | Х | |
| SF-36 | Х | | | | Х | Х | Х | Х |

- a All patients should be assessed post-procedure to determine if there is evidence of neurological impairment. If symptoms of a stroke are suspected, the NIHSS should be performed. Every effort should be made to have a neurologist or neurology fellow perform the neurological assessments. 6M and 1Y assessments to be performed only for patients diagnosed with a stroke after the procedure.
- b CK/CKMB and/or Troponins are required ≤ 72 hours before the valve implant procedure.
- c Post Procedure CK/CKMB and/or Troponins are required at 3 different time intervals: 1.) At the first lab draw post valve implant procedure (within 8 hours of exiting the cath lab or operating room) 2.) At the second lab draw 6 8 hours after the first lab draw 3.) At the third lab draw 6 8 hours after the second lab draw.
- d Screening procedures will be completed within 30 days prior to the valve implant procedure unless otherwise noted.
- e Qualifying echocardiogram must have been performed within the 90 days prior to randomization. Echocardiograms to be obtained years 2, 3, 4, 5, 7, and 10.
- f Only for those patients participating in the CT sub-study (section 12.5.2.1). Additionally, if the patient presents with symptoms, an unscheduled CT scan should be performed,
- g Includes thoracic and abdomen scan with visualization of iliac and femoral arteries.
- h All patients will have cardiac imaging at the screening visit regardless of participation in the CT sub-study.
- i Case Review will be completed when all screening procedures have been completed, all inclusion/exclusion criteria have been fundamentally confirmed and the site is ready to present a case.
- j TTE or TEE on date of valve implant procedure.
- k Frailty Index includes activities of daily living (ADLs), 5 meter walk test (5MWT), grip strength, and albumin laboratory.
- I Only for patients with a history of lung disease.
- m Only required for patients with chronic liver disease.

# 8.12 Procedures for Actigraphy/QOL Sub-study [Enrollment Closed]

Patients will receive a tablet and wearable activity tracker during the screening process and prior to randomization. A trained research assistant at each site will instruct patients on how to wear and use the devices. Baseline QOL and activity will be established during a pre-procedure phase (between screening and the procedure date). A preprogrammed algorithm will send alarm prompts to complete the VAS Pain assessment on the tablet every other day beginning at screening and ending on day 44 post procedure. The KCCQ-12 and PF-10 Physical will be completed via the tablet at 1, 2, 3, 5 and 6 week time points following the procedure. Activity data will be tracked continuously in 15-minute increments from screening through 44 days post procedure. Quality of life data will be captured via Medidata's Patient Cloud ePRO system, which allows patients to enter questionnaire data into commercially available smartphones and tablets that automatically synchronize with the Medidata platform. Activity data will be captured via Medidata's mobile health offering, which involves direct integration with wearable devices (i.e., Garmin Vivofit2). Activity data is authenticated and securely ingested by the Medidata Clinical Cloud, where it is then audited, processed and integrated with the rest of the clinical record.

# Schedule of Procedures Actigraphy/QOL Sub-Study [Enrollment Closed]

| | Screening | | | Post-Procedure | | | | | | | | | | | | | | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | | | Time window: + 12 hours | | | | | | | | | | | | | | | | | | | | | | |
| | | | + 2 | + 4 | 6 | +<br>8 | + 10 | + 12 | + 13 | + 14 | +<br>16 | + 18 | + 20 | + 22 | + 24 | + 26 | + 28 | + 30 | + 32 | + 34 | + 36 | + 37 | + 38 | +<br>40 | + 42 | + 44 |
| VAS Pain | Х | dure Day | Х | Х | Х | Х | Х | Х | | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | | Х | Х | Х | Х |
| | | roce | | | L | | L | | | | L | | Time | wind | ow: + | 1 day | 7 | I | | L | | L | | ı | | |
| KCCQ-12 | X | Pr | | | Х | | | | Х | | | | X | | | | | | | | | Х | | | | Х |
| PF-10 | Х | | | | Х | | | | Х | | | | Х | | | | | | | | | Х | | | | Х |

#### Notes:

- ePRO based VAS pain assessment will be completed every other day. A 12 hour time window will be allowed for patients to complete each assessment
- ePRO based KCCQ-12 and PF-10 assessments will be completed at 1-week, 2-weeks, 3-weeks, 5-weeks and 6-weeks post procedure. A one day time window will be allowed for patients to complete each assessment. Note: to lessen patient burden, ePRO based KCCQ-12 and PF-10 assessments will not be completed at baseline and 30-day follow-up as paper based assessments are already administered at those time points
- Paper based KCCQ, EQ-5D-5L and SF-36 will be administered at screening, 30-days, 6 months, 12 months. Note: KCCQ-12 and PF-10 scores can be derived from the longer KCCQ and SF-36 instruments
- Daily activity data is defined based on the subject's time zone and day

#### 9.0 ADVERSE EVENTS

#### 9.1 Adverse Event

An Adverse Event (AE) is any untoward medical occurrence, unintended disease or injury or untoward clinical signs (including abnormal laboratory findings) in patients, users or other persons, whether or not related to the investigational medical device.

Adverse events may be volunteered by patients, elicited by the Investigator or designee, the CEC, safety team, monitoring team, or collected via observation by the Investigator. All AEs will be assessed by the Investigator who will determine whether or not the event is related to the device and/or implant procedure, and whether or not the event meets serious criteria. If it is determined that an AE has occurred, the investigator should obtain all the information required to complete the AE Form of the CRF.

In addition, patients will be instructed to contact the investigator, and/or study coordinator if any significant adverse events occurs between study visits.

All clinically significant AEs will be reported by the Investigator and reviewed by the Sponsor in compliance with applicable regulations as indicated below section 9.5.

## 9.2 Serious Adverse Event

An Adverse Event is considered serious if the event:

- Leads to death;
- Leads to a serious deterioration in the health of the study patient that:
  - Results in life-threatening illness or injury;
  - Results in a permanent impairment of a body structure or a body function;
  - Requires inpatient hospitalization or prolongation of existing hospitalization:
  - Results in medical or surgical intervention to prevent permanent impairment to body structure or a body function;
- Led to fetal distress, fetal death or congenital abnormality or birth defect;
- Significant medical event.

Important medical events that do not meet the above criteria may still be considered an SAE if they seriously jeopardize the patient and require immediate medical or surgical intervention to prevent one of the aforementioned outcomes.

Death should not be recorded as an adverse event, but should only be reflected as an outcome to another specific AE.

# 9.3 Anticipated Adverse Events

Anticipated adverse events are AEs that have been identified as possible adverse events related to the investigational device or implant procedure.

# 9.4 Unanticipated Adverse Device Effect

An Unanticipated Adverse Device Effect (UADE) is any serious adverse effect on health or safety or any life-threatening problem or death caused by, or associated with a device, if that effect, problem, or death was not previously identified in nature, severity, or degree of incidence in the investigational plan or application (including a supplementary plan or application), or any other unanticipated serious problem associated with a device that relates to the rights, safety or welfare of patients.

The Investigator shall submit to the Sponsor and the reviewing EC/IRB a report of any UADE occurring during an investigation as soon as possible, but no later than 10 working days of awareness.

All UADE adverse events must be followed until resolution or until a stable clinical endpoint is reached. All required treatments and outcomes of the UADE adverse event must be recorded.

Edwards will notify FDA as well as all participating clinical investigators and IRBs of all UADEs that occur during this study within 10 working days after becoming aware of the event. Investigators are responsible for reviewing information received about UADEs.

## 9.5 AE Reporting Requirements

All relevant AEs will be captured from the time of randomization/enrollment until the study patient's participation has ended (i.e. completion of study or withdrawal of consent).

Adverse events must be followed until resolution, stabilization or study completion. The AE and/or SAE should be reported, and CRF Forms completed **as soon as possible but no later than 10 working days of awareness**.

In the event that the EDC system is not in service, a paper copy of the AE Case Report Form (CRF) must be faxed or emailed to Sponsor THV Medical Safety at (949) 809-2933 or emailed to THV\_Safety@edwards.com within 10 business days of becoming aware of the event. At the time of initial notification, the following minimal information must be provided:

- Study site
- Patient ID
- Adverse event description
- Causal relationship to device and implant procedure
- Aware date

The site will provide a copy of supporting documentation (example: admission H&P, implant procedure reports, anesthesia records, discharge summary, echocardiogram and ECG reports, laboratory results, etc.) for all endpoint-related and device or procedure-related events and UADEs to Edwards Lifesciences (or designee). Source documentation may be requested by the Edwards Medical Safety Officer for other AEs in order to verify that events are being assessed appropriately.

Enrolling sites must provide to the Sponsor at a minimum an admission history and physical, index procedure report and discharge from index hospitalization along with relevant echocardiographic reports. This will be done irrespective of subject having any AE/SAE.

All AEs must be reported over the 12 month period following the initial valve implant procedure. Reportable AEs after year 1 through year 10 or study exit include only the following events:

- All AEs that are assessed or suspected to be device or implant procedure related
- All AEs that meet the criteria for serious adverse event irrespective of device or implant procedure relationship
- All AEs considered to be an Unanticipated Adverse Device Effect

The site Principal Investigator is responsible for informing the Institutional Review Board (IRB) of SAEs, UADE and/or AEs as required. A copy of this report should be provided to the Sponsor (or designee).

## **Events that do not Require Reporting to the Sponsor:**

For purposes of this study, the following events will not be required to be reported as adverse events to the Sponsor, because they are normally expected to occur in conjunction with transcatheter valve implantation and surgical valve replacement or are associated with customary, standard care of patients undergoing THV implantation or surgical AVR:

- Post-operative pain.
- Post-anesthesia emesis, nausea, or headache (within 24 hours of procedure).
- Electrolyte imbalance without clinical sequelae following procedure, even if requiring correction.
- Pre-planned future surgical procedures not associated with the study procedure or device.
- Low grade temperature increase (≤ 101°F or 38.5°C).
- Dizziness: Imprecise term commonly used to describe various symptoms such as faintness, giddiness, imbalance, lightheadedness, unsteadiness or vertigo without signs of TIA or stroke.
- Elevated white blood count, outside the standard laboratory normal value, without signs and symptoms of infection.

- Minor, localized tenderness, swelling, induration, oozing, etc. at incision / delivery system insertion site.
- Systolic or diastolic blood pressure changes that do not require treatment or intervention.
- Thrombocytopenia: does not become an AE until treatment is administered;
   Suspected heparin-induced thrombocytopenia (HIT) should be reported
- Hyperglycemia The use of insulin in the post-operative period does not constitute hyperglycemia if during the index hospitalization. An elevated blood sugar of less than 250 mg/dl during the first 48 hours post-operative does not constitute hyperglycemia.
- Expected, non-clinically significant events such as non-significant lab variances.

# 9.6 Pre-existing Condition

Pre-existing medical conditions or symptoms reported prior to subject enrollment will not be recorded as an AE. In the event there is a worsening in the pre-existing medical condition or symptoms due to the device, implant procedure, or study related procedures, then an AE must be recorded.

Death should not be recorded as an adverse event, but should only be reflected as an outcome to another specific AE.

# 9.7 Causality of AEs

For each AE, the Investigator will determine whether the event is related to the device and/or the implant procedure, and whether the event meets the definition of a SAE as outlined in section 9.2.

The causal relationship of the event to the device and the implant procedure will be categorized as follows:

- **None:** The event is not associated with the device or implant procedure. There is no relation between the event and the device or implant procedure.
- Possibly Related: The temporal sequence between the device or implant
  procedure and the event is such that the relationship is not unlikely or there is no
  contradicting evidence that can reasonably explain the study patient's condition.
  There is a possibility of any relation between the event and the device or implant
  procedure.
- Definitely Related: The temporal sequence is relevant or the event abates upon device application completion/removal or the event cannot be reasonably explained by the patient's condition or comorbidities. The event is related or most likely associated with the device or implant procedure.

# 9.8 Sponsor Assessment of AEs

All AEs will be reviewed by the Medical Safety Officer. Each AE will be assessed as to its relationship to the study device and/or implant procedure, whether it was

anticipated or not anticipated, (based on the list of potential risks provided in section 10.2), and whether it qualifies as an SAE.

## 9.9 Device Malfunctions

A device malfunction is defined as the failure of a device to meet its performance specifications or otherwise perform as intended. Performance specifications include all claims made in the labeling for the device. The intended performance of a device refers to the intended use for which the device is labeled or marketed.

All device malfunctions with or without adverse events should be reported to Edwards Lifesciences as soon as possible (preferably within 24 hours) but no later than 10 working days of awareness.

#### 10.0 RISKS AND BENEFIT ANALYSIS

There are potential risks associated with transcatheter valve replacement. There are risks related to the overall procedures (complications associated with standard cardiac catheterization, balloon valvuloplasty, local and/or general anesthesia) as well as additional possible risks uniquely associated with the use of the study valve and its delivery systems.

## 10.1 Potential Benefits

There are no guaranteed benefits from participation in this study. Information gained from this study may be of benefit to other people with the same medical condition in the future. The long-term results of using the SAPIEN 3 THV are not known at the present time. Alternative treatments include surgical AVR and BAV.

Implantation of the transcatheter heart valve may result in improved valvular function, acute alleviation of symptoms related to aortic stenosis, and improved quality of life in patients with low operative risk of mortality.

#### 10.2 Potential Risks

There are potential risks associated with transcatheter valve replacement. There are risks related to the overall procedures (complications associated with standard cardiac catheterization, balloon valvuloplasty, local and/or general anesthesia) as well as additional possible risks uniquely associated with the use of the study valve and its delivery systems.

Potential risks associated with anesthesia and interventional procedures include but are not limited to:

- Abnormal lab values (including electrolyte imbalance)
- Allergic reaction to anesthesia, contrast media or device materials
- Anemia

- Angina
- Arrhythmia
- Bleeding
- Cardiovascular injury including perforation or dissection of vessels, ventricle, myocardium or valvular structures that may require intervention
- Conduction system injury (defect) which may require a permanent pacemaker
- Death
- Embolization including air, calcific/thrombotic valve material, or thrombus
- Exercise intolerance or weakness
- Femoral AV fistula or pseudoaneurysm
- Fever
- Heart failure
- Heart murmur
- Hematoma
- Hemorrhage requiring transfusion or intervention
- Hypertension or hypotension
- Infection including septicemia and endocarditis
- Inflammation
- Myocardial infarction
- Pain or changes at the access site
- Paralysis
- Pericardial effusion or cardiac tamponade
- Peripheral ischemia or nerve injury
- Permanent disability
- Pleural effusion
- Pulmonary edema
- Renal insufficiency or renal failure
- Reoperation
- Respiratory insufficiency or respiratory failure
- Restenosis
- Retroperitoneal bleed
- Stroke/transient ischemic attack, clusters or neurological deficit
- Syncope

In addition to the risks listed above, additional potential risks specifically associated with the use of the SAPIEN 3 THV, the delivery systems and/or accessories include, but may not be limited to, the following:

- Cardiac arrest
- Cardiac failure or low cardiac output
- Cardiogenic shock
- Coronary flow obstruction/transvalvular flow disturbance
- Device degeneration
- Device embolization
- Device explants
- Device migration or malposition requiring intervention
- Device thrombosis requiring intervention

- Emergency cardiac surgery
- Hemolysis
- Injury to mitral valve
- Mechanical failure of delivery system, and/or accessories
- Non-emergent reoperation
- Nonstructural dysfunction
- Paravalvular or transvalvular leak
- Structural valve deterioration (wear, fracture, calcification, leaflet tear/tearing from the stent posts, leaflet retraction, suture line disruption of components of a prosthetic valve, thickening, stenosis)
- Valve deployment in unintended location
- Valve regurgitation
- Valve stenosis
- Valve thrombosis

## 10.2.1 Risk Minimization

Product handling and implant procedure guidance are provided in the IFU and training manual, which will be used for device training to minimize risks associated with device use.

Additionally, efforts will be made to minimize risks through site/investigator selection and management. First, site and investigator selection criteria are established to ensure that the study personnel and their institutions are qualified to screen, perform and manage the study procedures as well as support the associated requirements for research. Second, the trial management structure is designed to provide disciplined oversight of the trial activities including close monitoring of site and personnel performance and also support opportunities for investigators and study personnel to share best practices through investigator meetings, ongoing education and case reviews.

The SAPIEN 3 THV represents a third generation THV for Edwards Lifesciences and was developed with the experience from the first and second generation SAPIEN THVs. The SAPIEN 3 System has undergone extensive clinical testing in the aortic position and is commercially available for TAVR in the US and countries that honor the CE mark.

#### 11.0 STATISTICAL ANALYSIS

## 11.1 Sample Size Calculations

The sample size for the trial is based on obtaining at least 90% power to pass the 1-year safety and effectiveness endpoint.

Event rate estimates for the primary safety and effectiveness endpoint were based on data from prior studies. Since the current study patients are a lower risk

population, and to account for procedural refinement over time in both arms as well as changes in definitions for components of the endpoint, the rates have been lowered.

The sample size is based on the composite primary endpoint which assumes an event rate of 16.6% in the SAVR arm and 14.6% in the TAVR arm. A randomized sample size of 864 patients with 1-year data would produce 90% power for passing the endpoint. The test statistic used for this computation is the one-sided Z test (Unpooled), at alpha = 0.025, using the specified non-inferiority margin of 6.0%. The sample size was computed in PASS.

The sample size determination was based on a pure frequency analysis, whereas the endpoint analysis will use the Kaplan-Meier estimates. Since the two methods are equivalent in the absence of censoring, and a sufficient number of uncensored patients is anticipated, the sample size should be adequate.

Because the feasibility assumptions are uncertain in this previously unstudied population, an actual sample size of 1000 has been chosen, which is higher than the minimum statistically justified size to allow for trial contingencies, such as withdrawals and lost to follow-up.

# 11.2 Analysis Populations

- The Intent to Treat (ITT) population consists of all randomized patients.
- The As Treated (AT) population is the subset of the ITT population consisting of all patients for whom the index procedure is begun, whether or not the index procedure is completed. If multiple procedures were attempted, the last procedure with the study valve deployed will be considered the index procedure and used for determining the As Treated trial arm assignment and the date of the index procedure will be used for determining all follow-up visits and related assessment. A randomized TAVR patient for whom the TAVR procedure is never started will not be part of the AT population, even if that patient should receive a SAVR implant.
- The Valve Implant (VI) population is the subset of the AT population consisting of all patients who receive and retain the intended valve during the index procedure. Patients who receive a valve in valve implant will be part of the VI population. Patients who are converted from TAVR to SAVR during the procedure will not be part of the VI population.

The AT population will be the primary population for trial endpoint analysis. The VI population will be used for analysis of echo data and related endpoints. Selected sensitivity analyses will be performed using the ITT population.

## 11.3 Timing

- The index procedure date is defined as Day 0. For randomized patients who do
  not have the procedure attempted, the randomization date will be used as Day
  0.
- Time intervals for events will be computed by subtracting the event date minus day 0. For example, if the procedure occurs on January 1, and the patient dies on January 31, the death will be considered a 30 day death for analysis.
- The timing for all visits will be based on the index procedure date. If the patient never receives the procedure the 30-day visit will never be due; later visits for such patients will be based on the randomization date.
- In analysis of time-dependent variables, one year is defined as 365.25 days, and one month as 30.4375 (= 365.25/12) days.

For information depending on follow-up windows any visit within the specified window will be used, without regard to the actual timing of the visit.

- Analysis close date:
  - The analysis close date for the initial analysis will be the earlier of the following two dates: One year past the last index procedure
  - One year plus 60 days past the last randomization. This condition is in order to account for a potential patient with a severely delayed procedure.
- The analysis close date for later reports will be determined prior to the report.
   Unless otherwise specified such dates will be at annual intervals past the initial analysis close date.
- All database information will be used to determine patient survival as of the analysis close date.
- Adverse events occurring after the relevant analysis close date will not be included in adverse event analysis.
- Information dependent on a visit window, such as echo or NYHA, will be included in analysis as long as the window starts on or before the analysis close date.

# 11.4 Primary endpoint analysis (Non-inferiority)

The primary safety and effectiveness endpoint is the composite of all-cause mortality, all stroke, and rehospitalization (valve-related or procedure-related and including heart failure) at 1 year post procedure. The endpoint will be evaluated as a non-inferiority analysis based on a non-inferiority margin of 6.0%. The components of

the composite endpoint will be evaluated by the CEC.

To precisely formulate the test, let  $r_T$  denote the true event proportion in the test arm at 1 year, and  $r_C$  denote the true event proportion in the Control arm at 1 year. The hypotheses are:

$$H_0: r_T - r_C \ge \Delta$$
  
 $H_A: r_T - r_C < \Delta$ 

The value  $\Delta$  is the non-inferiority margin, and is taken to be 0.06. The test will be performed as a one-sided test at alpha = 0.025.

A 95% confidence interval for the difference  $r_T$  -  $r_C$  will be computed using the Kaplan-Meier algorithm with the standard errors being computed using Greenwood's formula. The null hypothesis shall be rejected at alpha = 0.025 if the upper confidence limit is less than 0.06.

Covariates will not be included in analysis of the primary endpoint.

# 11.5 Primary Endpoint (Superiority) and Secondary endpoints for labeling

The analysis for the superiority in the primary endpoint and secondary endpoints for labeling will be performed only if the primary endpoint passes the non-inferiority test.

The superiority in the primary endpoint and secondary endpoints will be evaluated for labeling purposes in the order shown below. Each endpoint will be tested between the treatment arms by a two-sided test at alpha = 0.05. If any of the endpoints does not achieve statistical significance at alpha = 0.05, the lower endpoints in the list will not be considered for this purpose. The analyses will be performed in the As Treated population.

# 1. New onset atrial fibrillation, as a superiority analysis comparing trial arms (Secondary endpoint for labeling)

Let rT and rC be the true new onset atrial fibrillation rate at 30 days for test and control arms respectively. The hypotheses for the superiority test are:

$$H_0$$
:  $r_T = r_C$   
 $H_A$ :  $r_T \neq r_C$ 

The endpoint will be evaluated as a binary endpoint. The trial arms will be compared using the Fisher's exact test. The null hypothesis shall be rejected and the superiority will be established if the p-value of test is less than 0.05 and the point estimates  $\hat{r_T} < \hat{r_C}$ .

The counts and percentages of the new onset atrial fibrillation at 30 days will be presented for TAVR and SAVR arms, the p-value of trial arm comparison will

also be presented. The subjects with pre-procedural atrial fibrillation or those undergoing concomitant ablation will be excluded from the analysis unless CEC adjudicated the event as "new onset" or "both".

# 2. Length of index hospitalization, as a superiority analysis comparing trial arms (Secondary endpoint for labeling)

Let  $d_T$  and  $d_C$  be the distribution of the true lengths of index hospitalization for test and control arms, respectively. For this analysis, patients who die before discharge will be considered to have been discharged on the death date. The hypotheses for the superiority test are:

$$H_0$$
:  $d_T = d_C$   
 $H_A$ :  $d_T \neq d_C$ 

Length of index hospitalization will be treated as a continuous variable, with trial arms compared using the Wilcoxon rank-sum test. The null hypothesis shall be rejected and the superiority will be established if the p-value of test is less than 0.05 and the point estimates of the median lengths  $\hat{d}_T < \hat{d}_C$ .

The mean, standard deviation, median, minimum and maximum of Length of index hospitalization will be presented for TAVR and SAVR arms, the p-value of trial arm comparison will also be presented.

# 3. Primary endpoint as a superiority analysis comparing trial arms

The superiority test for the primary endpoint will be performed as a one-sided test at 0.025, where  $\alpha$  is the amount of Type I error passed, The hypotheses for the superiority test are:

H<sub>0</sub>: 
$$r_T \ge r_C$$
 or equivalently H<sub>0</sub>:  $r_T - r_C \ge 0$   
H<sub>A</sub>:  $r_T < r_C$  H<sub>A</sub>:  $r_T - r_C < 0$ 

The following Z statistic will be used for the superiority test.

$$Z = \frac{\hat{r}_T - \hat{r}_C}{\sqrt{s_T^2 + s_C^2}}$$

The null hypothesis shall be rejected and the superiority will be established if the p-value of the one-sided Z test is less than 0.025.

# 4. KCCQ and death composite at the 30 day visit, as a superiority analysis comparing trial arms (Secondary endpoint for labeling)

Let  $r_T$  and  $r_C$  be the true rate of the composite events at 30 days for test and control arms respectively. The hypotheses for the superiority test are:

$$H_0$$
:  $r_T = r_C$   
 $H_A$ :  $r_T \neq r_C$ 

The endpoint will be evaluated as a binary endpoint. The trial arms will be compared using Fisher's exact test. The null hypothesis shall be rejected and the superiority will be established if the p-value of test is less than 0.05 and the point estimates  $\hat{r}_T < \hat{r}_C$ .

A patient will be counted as meeting this endpoint if one or more of the following three conditions hold.

- a) The patient dies on day 30 or earlier, whether or not a KCCQ score has been collected within the follow-up window.
- b) The KCCQ score at the 30 day visit is < 45.
- c) The KCCQ score at 30 days is ≥ 10 points decreased from the baseline score.

Missing data will be handled as described in section 11.8.5.

# 5. Death/All Stroke composite at 30 days, as a superiority analysis comparing trial arms (Secondary endpoint for labeling)

Let  $r_T$  and  $r_C$  be the true rate of the death/all stroke composite events at 30 days for test and control arms, respectively. The hypotheses for the superiority test are:

$$H_0$$
:  $r_T = r_C$   
 $H_A$ :  $r_T \neq r_C$ 

The endpoint will be evaluated as a binary endpoint. The trial arms will be compared using the Fisher's exact test. The null hypothesis shall be rejected and the superiority will be established if the p-value of test is less than  $\alpha$  and the point estimates  $\hat{r}_T < \hat{r}_C$ .

The counts and percentages of the composite event at 30 days will be presented for TAVR and SAVR arms, the p-value of trial arm comparison will also be presented.

# 6. All Stroke at 30 days, as a superiority analysis comparing trial arms (Secondary endpoint for labeling)

Let  $r_T$  and  $r_C$  be the true stroke rate at 30 day for test and control arms, respectively. The hypotheses for the superiority test are:

$$H_0$$
:  $r_T = r_C$   
 $H_A$ :  $r_T \neq r_C$ 

Stroke will be evaluated as a binary endpoint. The trial arms will be compared using the Fisher's exact test. The null hypothesis shall be rejected and the superiority will be established if the p-value of test is less than  $\alpha$  and the point estimates  $\hat{r}_T < \hat{r}_C$ .

The number of events, number of patients with event and Kaplan-Meier estimates of stroke rate at 30 day will be presented for TAVR and SAVR arms, the p-value of trial arm comparison will also be presented.

# 11.6 Additional Safety and Effectiveness Endpoints

The endpoints in this section will be evaluated according to the general statistical methods described in section 11.8. These endpoints will not be subject to the formal multiple comparisons correction; they are presented as part of the totality of information. All the statistical tests between the treatment arms will be two-sided tests at alpha=0.05.

- Mortality (all cause & cardiovascular) at 30 days and 1 year
- Stroke (disabling and nondisabling) at 30 days and 1 year
- Death or stroke at 1 year
- Death or disabling stroke at 30 days and 1 year
- Vascular complications (major) at 30 days and 1 year
- Bleeding complications (life threatening, disabling or major) at 30 days and 1 year
- Myocardial infarction at 30 days and 1 year
- Acute kidney injury at 30 days
- Requirement for renal replacement therapy at 1 year
- New permanent pacemaker implantation resulting from new or worsened conduction disturbances at 30 days and 1 year.
- Coronary obstruction requiring intervention at 30 days and 1 year

- New York Heart Association class at 30 days and 1 year
- Hemodynamic valve performance evaluation by echocardiography for aortic
  valve stenosis and aortic valve regurgitation at 30 days and years 1, 2, 3, 4, 5,
  7, and 10. Echo readings to be evaluated include aortic valve area, mean
  gradient, peak gradient, perivalvular aortic regurgitation, total aortic
  regurgitation, and mitral regurgitation.
- Rehospitalization (valve-related or procedure-related and including heart failure) at 30 days, 1 year and annually (up to 10 years)
- Days alive and out of hospital at 1 year
- Six-minute walk test at 30 days and 1 year
- Health status as evaluated by Quality of Life questionnaires at 30 days and 1 year
- New onset atrial fibrillation at 1 year
- ICU days and discharge location
- Structural valve deterioration at years 1-5,7 and 10

# 11.7 Additional analyses

- Baseline data will be reported by summary statistics, separately by trial arm with p- values.
- The various procedural variables will be reported by summary statistics, separately by trial arm with *p*-values.
- Visit compliance data will be presented.
- Analysis of echo and procedural variables will be presented by valve size, at the various echo collection time points.
- Analyses past one year will be the same as the analyses for 1 year, but limited to those variables collected after the 1 year visit.

# 11.8 General Statistical Methodology

## 11.8.1 Time Dependent Variables

Time-dependent variables will be analyzed using the Kaplan-Meier algorithm, with standard errors computed by Greenwood's formula. The number of patients-at-risk will be computed at exact time points, without reference to any nominal follow-up windows. The log-rank statistic will be used for any comparison among groups.

Thirty day analysis will present both pure frequency and Kaplan-Meier rates; for later analyses only Kaplan-Meier rates will be presented. Kaplan-Meier rates will be presented at 30 days and 1 year as well as other time points as appropriate.

#### 11.8.2 Continuous and ordinal variables

- For continuous variables, summary statistics will include means, standard
  deviations, medians and quartiles. Confidence limits will be computed using the
  t-distribution. Groups will be compared using t-tests or analysis of variance.
   Where severe departures from normality are observed, comparisons will also be
  performed using the Wilcoxon rank-sum test.
- For ordinal variables, summary statistics will include medians and quartiles; means will also be presented when appropriate. Group comparisons will be performed using the Wilcoxon rank-sum test.
- NYHA and regurgitation will be considered as ordinal variables. Group counts and means will be presented for these variables.

## 11.8.3 Categorical Variables

- For categorical variables, summary statistics will include counts and percentages.
   Confidence limits for binary variables will be computed using the exact binomial distribution.
- Categorical variables will be compared by Fisher's exact test.

# 11.8.4 Non-Inferiority Analyses

- Non-inferiority tests at a point in time are based on the rate difference approach.
- The test is performed at a point in time T, using the Kaplan-Meier estimates for freedom from the endpoint being evaluated, and the Greenwood standard errors for these estimates. The test will be performed by computing the two-sided 95% confidence limit for the event rate difference (TAVR SAVR). The acceptance criterion is that the upper confidence limit is less than Delta, where Delta is the predetermined non-inferiority margin of 6.0%.
- In analysis of the primary endpoint, there will be little or no censored data. The only censoring would be due to lost to follow-up or withdrawal from the trial.
- It is conceivable that there will be no censored data at all in evaluating the
  primary endpoint. In such a case the Kaplan-Meier estimators are pure
  proportions, and the Greenwood variance is the standard variance for an
  estimated proportion. The confidence limits would agree with those produced by

standard frequency analysis.

• For the primary endpoint in this trial the non-inferiority margin of 6.0% has been chosen.

## 11.8.5 Missing Data

- Missing variables will not be imputed for planned analyses, except where otherwise specified.
- The primary safety and effectiveness endpoint will be based on Kaplan-Meier estimates, which automatically account for censored data.
- For sensitivity purposes, tipping point analyses for the primary endpoints are defined in the SAP.
- Tipping point analysis will also be presented for the secondary endpoint involving KCCQ.

## 11.8.6 Multiple comparisons

A formal multiple comparisons analysis is presented in section 11.5 for the named secondary endpoints for labeling purposes. In all other cases p-values will be presented as computed, without any adjustments for the comparisons.

## 11.8.7 Adverse event analysis

- Adverse event analysis will involve both site and CEC reporting.
  - Where events have been adjudicated by the CEC, those adjudications will be used in preference to site reports.
  - Where site events are analyzed, the MedDRA coding will be used. The underlying site evaluations will not be used for analysis, but may appear in listings as appropriate.
- Adverse events to be analyzed include the composites involved in the primary and secondary endpoints, as well as all events contained in these composites. All events adjudicated by the CEC will also be analyzed.
- Adverse event tables will present data at 30 days, 6 months, and 1 year. The
  tables will include counts of events, patients with event, and Kaplan-Meier event
  rates at the specific time point. The trial arms will be compared by the log-rank
  test
- Late adverse events (> 30 days) will be analyzed by a constant hazard model, and upper one-sided confidence limits will be given for the rates.

 Adverse event data past 1 year will be presented as counts of events and patients with event. No formal analyses will be performed for such data.

## 11.8.8 Periodic analyses

Periodic analyses will be performed during the trial to the extent required by the appropriate regulatory authorities and the DSMB. The sample size and endpoint timing for this trial is fixed in advance, and not based on these periodic analyses. Accordingly, there is no adjustment to alpha.

Other than the required reports mentioned in the previous paragraph, there will be no reporting of trial outcome data prior to the 1-year analysis close date.

It is anticipated that reporting will continue throughout the trial, with formal reports based on analysis close dates at annual intervals.

# 11.8.9 Quality of life questionnaires

Quality of life questionnaires will be scored according to algorithms provided by the vendor. The various summary scores produced by the algorithms will be analyzed as continuous variables.

# 11.8.10 General Specifications

- Trial arm comparisons will be presented wherever meaningful. *P*-values will be computed using a null hypothesis of no difference.
- Unless otherwise specified, Wald *p*-values will be presented.
- Unless otherwise specified, confidence limits and hypotheses tests will be two sided, using alpha = 0.05.
- Unless otherwise specified, the precise form of each algorithm will be the default of SAS, using the latest release installed at Edwards at the time of analysis. This will be version
   9.3 or later.
- Various CRFs will contain comment fields. Data in these fields will not be analyzed, but listings will be provided for internal use on request.

## 11.9 CT Sub-Study

The purposes of the study are to:

1. Investigate the prevalence of the imaging abnormality.

The prevalence data come in two forms. A Yes/No value, which will be analyzed as a binary variable. A grading, which will be analyzed as an ordinal variable.

2. Investigate the relationship between the imaging abnormality and patient, procedural and pharmacology factors.

The Yes/No value will be the dependent variable in logistic regression models, with the independent variables chosen based on potential clinical relevance.

Multivariable models will be developed if the univariate analyses so suggest.

3. Investigate the relationship between imaging abnormalities and clinical events.

The clinical events to be considered will include stroke, TIA, and death. These will be modeled as time-dependent variables using proportional hazards regression, with the Yes/No value of the imaging abnormality as an independent variable.

Key echo parameters (valve area, mean gradient, and AR) will be modeled, with the Yes/No value of the imaging abnormality as an independent variable.

This sub-study analysis is unpowered.

The choice of variables for items 2 and 3 will be based on the tables presented in the papers of Makkar [26] and Pache [27].

It should be noted that the prior studies found few statistically significant baseline predictors of the imaging abnormality, and they found only minor clinical impact resulting from the abnormality. There is no reason to expect any different results in this sub-study.

## 12.0 STUDY ADMINISTRATION

# 12.1 General Study Organization

Edwards Lifesciences is the Study Sponsor and has the overall responsibility for the conduct of the study, including assurance that the study meets the regulatory requirements of the appropriate regulatory bodies.

Edwards Lifesciences will be responsible for obtaining IDE approval for the study, selecting investigators, ensuring that sites have IRB/EC approval prior to investigational device shipment, and conducting clinical site monitoring to ensure that patients are being properly consented and the study is being conducted according to the protocol.

As appropriate, Edwards Lifesciences will submit changes in the Investigational Plan to the FDA and Investigators to obtain IRB/EC re-approval.

Edwards Lifesciences will maintain copies of correspondence, data, shipment of devices, adverse device effects and other records related to the clinical trial as appropriate.

Edwards Lifesciences will submit all reports required by the FDA as identified in 21 Code of Federal Regulations (CFR) 812.150(B). This includes UADEs, withdrawal of IRB/EC approval, current investigators list, annual progress reports, recall information, final reports and protocol violations.

# 12.2 Data Safety Monitoring Board (DSMB)

A Data Safety Monitoring Board (DSMB) will monitor all AEs and SAEs to provide safety oversight. DSMB members will not be involved in the study and have no conflict of interest. At least one member will be a cardiothoracic surgeon with specific expertise in aortic stenosis. DSMB activities, including stopping rules for early termination, will be defined in the DSMB Charter.

# 12.3 Clinical Event Adjudication Committee (CEC)

The Clinical Events Committee (CEC) will adjudicate endpoint events and provide assessment of SAEs and device/procedure relatedness from enrollment through the primary endpoint. The CEC will include cardiologists and cardiothoracic surgeons with experience in the field of aortic stenosis who are not involved in the study and have no conflict of interest. CEC activities will be defined in the CEC Charter.

## 12.4 Study Procedures

### 12.4.1 Echocardiogram

Study patients will receive an echocardiogram at the visits specified in section 8.0. A central imaging core lab will be established to independently review and analyze echocardiographic images. A standardized protocol for acquiring images will be developed by the core lab and be provided to the clinical sites prior to study initiation. Sites will be trained on acquiring images prior to study initiation. Appendix J includes the echocardiogram manual of operations.

#### 12.4.2 Computed Tomography (CT)

All study patients will have a screening CT as referenced in section 8.0. Sites will be trained on acquiring images prior to study initiation. In addition, all Screening CTs will be independently analyzed with regards to annular measurements by a CT/angiographic core lab. Appendix K-1 includes CT acquisition information.

# 12.4.2.1 CT Sub-Study

Study patients enrolled in the CT sub-study will have a 4D CT at visits specified in section

8.1. A central imaging core lab will independently review sub-study CTs. Appendix K-2 includes the sub-study CT acquisition information.

Investigational sites will be blinded to the resulting images unless specific clinical or echo abnormalities are present.

If any of the following events occur, a repeat 4D CT will be mandated unless the event occurs within 24 hrs of the 30 day CT; in which case the CT will be unblinded.

- Any neurological event
- Any potential embolic event
- Myocardial infarction
- A change in echo parameters including an increase in mean gradient of 10-20 mm Hg or a change in DVI of 0.05 - 0.1

Patients whose initial imaging data are determined to be unevaluable will not undergo subsequent imaging.

# 12.4.3 Quality of Life Questionnaires

Investigational sites will be provided with paper QoL questionnaires (KCCQ, EQ-5D-5L, and the SF-36). Patient questionnaires will be IRB approved prior to patient administration.

Investigational staff will administer patient questionnaires to study patients. Patients will be instructed to complete each questionnaire at visits specified in section 8.0. The patient will be instructed by the investigational staff to sign and date the paper questionnaire once the questionnaire is completed. Patients will be instructed by the investigational staff not to change questionnaire answers once the questionnaire has been completed. Investigational sites should retain the completed questionnaire in the patients' source documents. Site staff will enter data collected from the completed patient questionnaire into the EDC.

The patient level summary scores will be computed by the Edwards Biostatistics group, and these scores will be used in evaluating protocol endpoints. A QoL core lab may prepare reports of additional analyses.

Quality of life will be measured through standard surveys:

- The Kansas City Cardiomyopathy Questionnaire (KCCQ) is an assessment of disability and quality of life impairment due to congestive heart failure.
- 2) EQ-5D-5L is a standardized questionnaire for describing and valuing patients' health- related quality of life for clinical and economic appraisal.

3) The SF- 36 is a generic health status instrument and rating scale that allows mapping of health status to population-level utility weights. This is an important metric for cost- effectiveness analysis.

## 12.4.4 Image Management

A central image management lab will be established to receive, maintain, and provide cardiac images (echocardiogram and CT) to the appropriate core lab for analyzing.

Instructions for image upload will be provided to investigative staff prior to study initiation. Investigative staff should upload all images to the image management core lab within 5 business days of data collection.

### 12.4.5 Histopathology

Histopathology studies of explanted valves will be performed. Explants will be appropriately prepared and preserved and sent to the independent histopathology laboratory for macroscopic and microscopic analysis. Investigational valves that are removed at any time with an allegation of device malfunction should be returned to the Sponsor for evaluation. All other explants (those not with an allegation of device malfunction) should be sent to the Histopathology Core Lab. Appendix L contains a complete explant protocol which includes detailed procedures for the histopathology studies.

Gross pathological examination of the entire valve and the support structure (i.e., and shape, if occurrence of intravascular trauma, tissue abrasion, uniformity of the frame, position the natural valve cusps) will be assessed.

The valves will be assessed for cusp excursion and the presence of leaflet fenestrations, rigidity tears, hematoma, thrombi and calcified nodules, cell proliferation tissue overgrowth.

fibrous sheath, and local inflammatory reaction. (One half of each leaflet must be used for the quantitative determination of inorganic calcium and phosphate).

# 12.5 Training

To ensure proper device usage, uniform data collection, and protocol compliance, training is required for relevant study site personnel in accordance to roles outlined in the Delegation of Authority (DoA).

At the beginning of the study, Edwards Lifesciences will provide training to site personnel. Training will include review of the instructions for use of the device, study protocol, case review process, identification of eligible patients, instructions on inhospital data collection, standardized data collection for core laboratory analysis,

methods for soliciting data from alternative sources, and regulatory requirements.

Documentation of site personnel qualification and training should be maintained in the site's clinical trial files and copies collected and forwarded for the Sponsor site file.

Ongoing training may be provided in one of the following formats by the Sponsor or its designee: live training sessions, teleconference, WebEx, online, or read and review. The Sponsor reserves the right to enforce retraining for sites who have demonstrated study or implant procedure compliance issues.

# 12.6 Device Management

# 12.6.1 Study Device

All SAPIEN 3 products will be supplied by Edwards Lifesciences. Each SAPIEN 3 THV will have a unique identifier which should be recorded in the patient's medical file as well as on the implant card that is given to the patient.

Refer to Appendix C for the IFUs to be used in this study. The IFUs will also be available electronically.

### 12.6.2 Device Storage

All SAPIEN 3 System components provided for the study should be stored in a secure location where only study personnel can access the device for use. Only physicians identified in the Investigator's Delegation of Authority Log on file at Edwards Lifesciences may implant this device in study patients.

#### 12.6.3 Device Accountability

The study site will maintain detailed records of the receipt and disposition of all investigational devices on the Device Accountability Log (DAL). Device disposition will be verified by the clinical monitor periodically throughout the study. The Investigator will return unused devices to Edwards along with the completed device disposition log at completion of the investigation. Use of the SAPIEN 3 THV and accessories provided for use in the study is prohibited outside of this protocol.

# 12.7 Data Management

Edwards Lifesciences will provide data management through a secure, password protected Electronic Data Capture (EDC) system accessible via the Internet. A unique Patient ID will be assigned for each patient enrolled in the study. All pertinent data will be entered by the study site and core lab personnel into the electronic Case Report Forms (eCRFs).

Every reasonable effort should be made to complete data entry within 5 business
days of data collection. Data review by Edwards Lifesciences personnel will occur remotely as well as during on site monitoring. Data discrepancies will be queried and resolved through the EDC system.

The site Principal Investigator or designee must ensure the accuracy and completeness of the recorded data and then provide his/her electronic signature on the appropriate eCRFs. Changes to data previously submitted to the Sponsor will require a new electronic signature to acknowledge/approve the changes.

# 12.8 Monitoring Procedures

All clinical sites will be monitored periodically by Edwards Lifesciences or designee to ensure compliance with the protocol and the Investigator's Agreement and that all study patients have been properly consented. The monitor will ensure that the completed eCRFs match the source documents and work with the site to resolve differences through electronically generated queries or formal action items.

Edwards Lifesciences will evaluate circumstances where an investigator deviates from the clinical protocol and will retain the right to remove either the investigator or the investigational site from the study.

# 12.9 Auditing

The study may be subject to a quality assurance audit by Edwards Lifesciences or a designee, as well as inspection by appropriate regulatory authorities. It is important that the Investigator and relevant study personnel are available during any audits and that sufficient time is devoted to the process. In the event of an audit by regulatory authorities, the Investigator should contact Edwards Lifesciences as soon as possible.

### 12.10 Record Retention

All clinical sites will maintain study records for a minimum of two years after marketing for this patient population approval is obtained or after the site is notified by Edwards

Lifesciences that the study has been terminated. Record retention dates will be provided to all parties concerned by Edwards Lifesciences.

# 13.0 ETHICAL AND REGULATORY CONSIDERATIONS

# 13.1 Compliance with Good Clinical Practices

The Investigator will ensure that this study is conducted in accordance with Good Clinical Practice (GCP) and applicable regulatory (local) requirements.

## 13.2 Institutional Review Board/Ethics Committee

This protocol, the proposed Informed Consent Form (ICF), other written patient information and any proposed advertising material must be submitted to the IRB for written approval. A copy of the written IRB approval of the protocol and ICF must be received by Edwards Lifesciences before recruitment of patients into the study and shipment of investigational product.

The Investigator must submit and, where necessary, obtain approval from the IRB for all subsequent protocol amendments and changes to the ICF.

The Investigator is responsible for obtaining annual IRB approval and renewal throughout the duration of the study. Copies of the Investigator's reports and the IRB continuance of approval must be sent to Edwards Lifesciences.

## 13.3 Patient Informed Consent

Edwards Lifesciences will provide a sample ICF to the Investigator to prepare for use at his/her site. The site-specific ICF must be in agreement with current GCP guidelines.

Edwards Lifesciences must approve the site-specific ICF prior to submission to the IRB. The reviewing IRB must approve the ICF before use at that site.

Before participating in the clinical trial, each patient must give written Informed Consent after the context of the study has been fully explained in a language that is easily understood by the patient. The subject must also be given the opportunity to ask questions and have those questions answered to his/her satisfaction.

A copy of each patient's signed and dated consent form must be maintained by each Investigator in a designated clinical trial administrative file. A signed copy of the consent form must be given to each subject. The consent process must be documented in the subject's medical chart.

Any modifications to the site-specific ICF must be approved by Edwards Lifesciences and the IRB.

## 13.4 Confidentiality

All data used in the analysis and reporting of this evaluation will be without identifiable reference to the patient. Authorized personnel assigned by Edwards Lifesciences will have access to the confidential files and will have the right to inspect and copy all records pertinent to this trial. All data used in the analysis and reporting of this evaluation will be without identifiable reference to the subject.

# 13.5 Investigator Records

Records to be maintained by the Investigator include, but are not limited to, the following:

- Clinical trial protocol and all amendments
- Signed Clinical Trial Agreement and any amendments
- IRB approval letters, including continuing reviews and all amendments/changes
- IRB approved informed consent documents

The following records must be maintained for each subject enrolled in the trial:

- Signed patient informed consent
- All relevant source documentation for study visits and study-related procedures
- Supporting documentation of any adverse events

# 13.6 Investigator Reports

Adverse event reporting requirements are discussed in section 9.0.

<u>Withdrawal of IRB Approval</u>. Within 5 working days, the Principal Investigator will report to Edwards Lifesciences a withdrawal of approval by the reviewing IRB of the investigator's part of an investigation.

<u>Informed Consent</u>. If an investigator uses a device without obtaining informed consent, the investigator shall report such use to Edwards Lifesciences and the reviewing IRB within 5 working days after the use occurs.

<u>Progress Reports</u>. The Principal Investigator will submit progress reports on the investigation to Edwards Lifesciences and the IRB at least yearly.

<u>Final Report</u>. Upon completion or termination of this Trial, the Principal Investigator must submit a final written report to Edwards Lifesciences and the IRB as required by the regulations. The report must be submitted within 3 months of completion or termination of the trial.

# 13.7 Amending the Protocol

This protocol must be followed exactly. It can be altered only by written amendments made by Edwards Lifesciences. Following appropriate approval by Edwards Lifesciences, the amended protocol will be submitted to the required regulatory agencies before being distributed to all enrolling sites. Each site must obtain IRB/EC approval, complete required training (if any, and as required by DoA role), and receive written approval from Edwards Lifesciences before implementing the revised protocol.

## 13.8 Protocol Deviations

An investigator must not make any changes or deviate from this protocol, except to protect the life and physical well-being of a subject in an emergency. Emergency changes to protect the life of the patient do not require prior approval, but must be reported to Edwards Lifesciences and the reviewing IRB within 5 days of the incident.

Each deviation from the protocol must be documented with the date and reason for the deviation and reported to Edwards Lifesciences as soon as possible, and to the IRB per local guidelines and government regulations.

# 13.9 Publication Policy

Publication or presentation of the overall clinical study results and/or site-specific results requires prior written approval of Edwards Lifesciences. If Edwards Lifesciences approves the publication or presentation of the overall clinical study results and/or site-specific results, then Institutions and Investigators will comply with the Publications and Public Disclosure section of the Clinical Trial Agreement. Edwards Lifesciences will provide statistical support for the publication process.

# Appendix A Abbreviations

| Abbreviation | Full Term |
|--------------|------------------------------------------------|
| ACT | Activated Clotting Time |
| AE | Adverse Event |
| AR | Aortic Regurgitation |
| ASD | Atrial Septal Defect |
| AT | As Treated |
| AV | Atrioventricular |
| AV | Aortic Valve |
| BARC | Bleeding Academic Research Consortium |
| BAV | Balloon Aortic Valvuloplasty |
| CBC | Complete Blood Count |
| CEC | Clinical Events Committee |
| CFR | Code of Federal Regulations |
| CHD | Congenital Heart Defects |
| CHF | Congestive Heart Failure |
| CK-MB | Creatine Kinase MB |
| СРВ | Cardiopulmonary Bypass |
| СТ | Computed Tomography |
| CTA | Computed Tomography Angiography |
| CV | Curriculum Vitae |
| DAL | Device Accountability Log |
| DOA | Delegation of Authority |
| DSMB | Data Safety Monitoring Board |
| EC | Ethics Committee |
| ECG | Electrocardiogram |
| Echo | Echocardiogram |
| eCRF | Electronic Case Report Form |
| EDC | Electronic Data Capture |
| EMEA | Europe, Middle East, Africa |
| ePRO | Electronic Patient-Reported Outcome |
| FDA | Food and Drug Administration |
| GCP | Good Clinical Practice |
| Hct | Hematocrit |
| Hgb | Hemoglobin |
| ICF | Informed Consent Form |
| IDE | Investigational Device Exemption |
| IFU | Instructions For Use |
| INR | International Normalized Ratio |
| IRB | Institutional Review Board |
| ISO | International Organization for Standardization |

| Abbreviation | Full Term |
|--------------|-------------------------------------------------|
| KM | Kaplan Meier |
| LAR | Legally Authorized Representative |
| LBBB | Left Bundle Branch Block |
| LVOT | Left Ventricular Outflow Tract |
| MI | Myocardial Infarction |
| MR/MRI | Magnetic Resonance / Magnetic Resonance Imaging |
| NYHA | New York Heart Association |
| PA | Pulmonary Artery |
| PCWP | Pulmonary Capillary Wedge Pressure |
| PET | Polyethylene Terephthalate |
| PLT | Platelets |
| QOL | Quality of Life |
| RA | Right Atrium |
| RBC | Red Blood Cell |
| RV | Right Ventricle |
| SAE | Serious Adverse Event |
| SAVR | Surgical Aortic Valve Replacement |
| STS | Society of Thoracic Surgeons |
| TAVR | Transcatheter Aortic Valve Replacement |
| THV | Transcatheter Heart Valve |
| TIA | Transient Ischemic Attack |
| TTE | Transthoracic Echocardiogram |
| UADE | Unanticipated Adverse Device Effect |
| VARC | Valve Academic Research Consortium |
| VAS | Visual Analogue Scale |
| VI | Valve Implant |
| WBC | White Blood Cell |

# Appendix B Definitions

| Term | Definition | Reference/<br>Justification |
|---|---|---|
| Adverse Event (AE) | Any untoward medical occurrence, unintended disease or injury, or untoward clinical signs (including abnormal laboratory findings) in subjects, users or other persons, whether or not related to the investigational medical device | ISO 14155-1:2011<br>GCP |
| Access Site | Any location (arterial or venous) traversed by a guidewire, a catheter or a sheath for TAVR or skin incision for SAVR | VARC 1 |
| Access site related complication | Any adverse clinical consequence possibly associated with any of the access sites used during the procedure | VARC 1 |
| Acute kidney injury | An abrupt loss of kidney function, resulting in the retention of urea and other nitrogenous waste products The increase in creatinine meeting at least Stage 1 must | Sponsor/VARC 2 |
| | occur within 48 hours. Staging will be based on the worse stage that occurs within 7 days of the index procedure. | |
| | Stage 1 • Increase in serum creatinine to 150-199% (1.5-1.99 × increase compared with baseline) OR increase of ≥0.3 mg/dL (≥26.4 mmol/L) OR • Urine output <0.5 ml/kg per hour for >6 but <12 hours | |
| | Stage 2 • Increase in serum creatinine to 200-299% (2.0-2.99 × increase compared with baseline) OR • Urine output <0.5 ml/kg per hour for >12 but <24 hours | |
| | Stage 3 • Increase in serum creatinine to ≥300% (>3 × increase compared with baseline) OR serum creatinine of ≥4.0 mg/dL (≥354 mmol/L) with an acute increase of at least 0.5 mg/dL (44 mmol/L) OR • Urine output <0.3 ml/kg per hour for ≥24 hours OR • Anuria for ≥12 hours | |
| | Patients receiving renal replacement therapy (dialysis, hemodialysis, peritoneal dialysis, hemofiltration, transplant) are considered to meet Stage 3 criteria irrespective of other criteria irrespective | |
| Anemia | A condition in which the blood is deficient in red blood cells, in hemoglobin, or in total volume, without clear evidence of overt bleeding, that is actionable (e.g. requires medications, transfusion etc) | Sponsor |

| Term | Definition | Reference/<br>Justification | |
|---|---|---|---|
| Angina / Cardiac<br>chest pain | Chest pain due to a heart muscle | in inadequate supply of oxygen to the | Sponsor |
| Angina, grading | Grade | Description | Canadian |
| scale | Grade I | Ordinary physical activity, such as walking and climbing stairs, does not cause angina. Angina occurs with strenuous, rapid, or prolonged exertion at work or during recreation | Cardiovascular<br>Society |
| | Grade II | Slight limitation of ordinary activity. Angina occurs with walking or climbing stairs rapidly, walking uphill, walking or stair climbing after meals, walking in the cold, into the wind, while under emotional stress, or during the first hours after awakening. Walking more than two blocks on the level and climbing more than one flight of ordinary stairs at a normal pace and in normal conditions, does not cause angina | |
| | Grade III | Marked limitation of ordinary physical activity. Angina occurs with walking one to two blocks on the level and climbing one flight of stairs in normal conditions and at a normal pace | |
| | Grade IV | Inability to carry on any physical activity without discomfort. Angina syndrome may be present at rest | |
| Aortic coarctation | A narrowing of the a ligamentum arterios | aorta usually in the area of the sum | Groenemeijer BE,<br>Bakker A, Slis HW,<br>Waalewijn RA,<br>Heijmen RH. An<br>unexpected finding<br>late after repair of<br>coarctation of the<br>aorta. Netherlands<br>Heart Journal.<br>2008;16(7-8):260-<br>263. |

| Term | Definition | Reference/<br>Justification |
|---|---|---|
| Aortic dissection | Aortic dissection is a separation of an intimal of wall that may or may not require intervention | Sponsor |
| Aortic stenosis, native | Aortic stenosis is classified as "severe" when the following are present: • Jet velocity > 4.0 m/s • Mean gradient > 40mmHg • Valve area < 1.0 cm <sup>2</sup> • Valve area index < 0.6cm <sup>2</sup> /m <sup>2</sup> | 2014 AHA/ACC |
| Arrhythmia /<br>Conduction<br>System Injury<br>(Defect) | Arrhythmia: an irregular heart rate or abnormal rhythm resulting in symptoms or requiring medical intervention. Conduction system defect: an impairment of the electrical pathways and specialized muscular fibers that conduct impulses through the heart (ex. bundle branch block, heart block, etc.). | Sponsor |
| Bicuspid aortic<br>valve | Congenital malformation resulting in 2 functioning leaflets as defined by Sievers and Schmidtke | A classification<br>system for the<br>bicuspid aortic valve<br>from 304 surgical<br>specimens. Sievers<br>HH, Schmidtke C. J<br>Thorac Cardiovasc<br>Surg. 2007<br>May;133(5):1226-33. |
| Bioprosthetic valve dysfunction | Bioprosthetic valve dysfunction can be structural (ex. leaflet tears, leaflet mobility restriction, etc.) or non-structural (ex. paravalvular leak or endocarditis) or hemodynamic(aortic regurgitation or aortic stenosis) or a combination of these dysfunctions. Patients with BVD maybe asymptomatic or symptomatic requiring medical therapy (ex. addition of anticoagulation), hospitalization, or require intervention and/or valve explant. | Sponsor |
| Bleeding | Bleeding, including, but not limited to fatal bleed, bleeding associated with transfusion, drop in Hgb or visible sign of blood loss For the purposes of this trial, an overt source of bleeding for subjects undergoing TF-TAVR is > 100 mL blood loss during the procedure. For subjects undergoing SAVR and for subjects undergoing TAVR using an alternative approach (i.e. TAo, TA), an overt source of bleeding is considered to be > 600 mL bloody chest tube output (as captured on Intake and Output Chart, I/O) within 24 hours of leaving the OR/cath lab or bleeding requiring a transfusion of RBCs | Sponsor |
| CABG | Coronary artery bypass surgery | Sponsor |

| Term | Definition | Reference/<br>Justification |
|---|---|---|
| Cardiac arrest | Cardiopulmonary arrest or circulatory arrest, is a sudden stop in effective blood circulation due to the failure of the heart to contract effectively or at all | Sponosor / STS |
| Cardiogenic<br>shock | Sustained (>30 min) episode of systolic BP <90 mmHg and/or cardiac index <2.2 L/min/m2 determined to be secondary to cardiac dysfunction, and/or the requirement for parenteral inotropic or vasopressor agents or mechanical support (e.g., intra-aortic balloon pump, extracorporeal circulatory support, ventricular assist device) to maintain BP and cardiac index above those specified levels | 2014 ACC/AHA Key Data Elements and Definitions for Cardiovascular Endpoint Events in Clinical Trials |
| Cardiac<br>tamponade | Evidence of a new pericardial effusion associated with hemodynamic instability evident by: 1. Echo showing pericardial fluid and signs of tamponade such as right heart compromise, or 2. Systemic hypotension due to pericardial fluid compromising cardiac function | VARC 2 / STS |
| Hypertrophic Cardiomyopathy | Cardiomyopathy is a term applied to a wide spectrum of cardiac diseases in which the predominant feature is poor myocardial function in the absence of any anatomic abnormalities. Idiopathic hypertrophic subaortic stenosis (IHSS) is also know as hypertrophic obstructive cardiomyopathy (HOCM), and is characterized by a primary hypertrophy of the myocardium. The obstructive forms involve different degrees of dynamic subvalvar aortic obstruction from a thickened ventricular wall and anterior motion of the mitral valve. Cardiomyopathies are into three entities: 1. Dilated, characterized by ventricular dilatation and systolic dysfunction 2. Hypertrophic, characterized by physiologically inappropriate hypertrophy of the left ventricle 3. Restrictive, characterized by diastolic dysfunction, with a presentation often identical to constrictive pericarditis. | STS Congenital Heart Surgery Database Data Specifications |

| Term | Definition | | | Reference/<br>Justification |
|---|---|---|---|---|
| Cerebrovascular<br>disease | Cerebrovascular di<br>an area of the brair<br>by ischemia or blee<br>blood vessels are in | STS | | |
| | It includes: | | | |
| | Stroke TIA Noninvasive demonstrate major extrate brain Previous concervascularity intervention This does not included is eases or other a metabolic and another services. | | | |
| CHADS <sub>2</sub> Score<br>(Annual Stroke<br>Risk) | The CHADS2 score risk in patients with determine which ar appropriate. The CHADS2 score schema that can be ischemic stroke in a valvular AF. | Gage BF, Waterman AD, Shannon W, Boechler M, Rich MW, Radford MJ. Validation of Clinical Classification Schemes for Predicting Stroke: Results From the National Registry of | | |
| | | Annual Stroke ris | sk | Atrial Fibrillation. |
| | CHADS₂ Score | Stroke Risk % | 95% <u>CI</u> | <i>JAMA.</i><br>2001;285(22):2864- |
| | 0 | 1.9 | 1.2–3.0 | 2870. |
| | 1 | 2.8 | 2.0–3.8 | doi:10.1001/jama.285<br>.22.2864 |
| | 2 | 4.0 | 3.1–5.1 | .22.2004 |
| | 3 | | | |
| | 4 | | | |
| | 5 | | | |
| | 6 | 18.2 | 10.5–27 | |
| Chest deformity<br>(see also "Hostile<br>chest)" | Chest deformities the procedure and inclusive integrals at the procedure and inclusive integrals. | Sponsor | | |

| Term | Definition | | | | | | | Reference/<br>Justification |
|---|---|---|---|---|---|---|---|---|
| Child-Pugh<br>Classification | The Child-Pugh score consists of five clinical features and is used to assess the prognosis of chronic liver disease and cirrhosis: | | | | | | | CHOLONGITAS, E., |
| | Measu | re | 1 pc | int | 2 poin | ts | 3 points | M., TERRENI, N.,<br>PATCH, D. and<br>BURROUGHS, A. K. |
| | Total biliri<br>µmol/l (m | | <34 ( | (<2) | 34-50 (2 | -3) | >50 (>3) | (2005), Systematic review: the model for end-stage liver |
| | Serum alb<br>g/dl<br>Prothron | Í | >3. | .5 | 2.8-3.5 | 5 | <2.8 | disease – should it replace Child-Pugh's |
| | time,<br>prolonga<br>(secs | tion | <4. | .0 | 4.0-6.0 | ) | > 6.0 | classification for assessing prognosis in cirrhosis. |
| | Ascite | s | Nor | ne | Mild | | Moderate to<br>Severe | Alimentary Pharmacology & Therapeutics, 22: |
| | Hepatic<br>encephalopati | | Nor | ne | Grade I-II<br>suppress<br>with<br>medication | sed | Grade III-IV (or refractory) | 1079–1089. doi:<br>10.1111/j.1365-<br>2036.2005.02691. |
| | Chronic liver disease is classified into Child-Pugh class A to C, employing the added score from above: | | | | | | | |
| | Points | Cla | ss | | ne year<br>urvival | Τv | vo year survival | |
| | 5-6 | A | | | 100% | | 85% | |
| | 7-9 | В | | | 81% | | 57% | |
| 10-15 C 45% 35 | | | | | 35% | | | |
| Coagulopathy | A pathologic condition that affects the ability of the blood to coagulate. Examples include | | | | | | | |

| Term | Definition | Reference/<br>Justification |
|---|---|---|
| Congestive Heart<br>Failure (CHF) | Diagnosis requires physician documentation or report of any of the following: | STS |
| Cardiopulmonary bypass (CPB) | Bypass of the heart and lungs as in open heart surgery | Sponsor |
| Conversion to open surgery | Any conversion to complete TAVR procedure secondary to any procedure-related complications | Sponsor |
| Coronary artery disease (CAD) | Coronary artery disease is characterized by a narrowing or "stenosis" of the blood vessels to the heart resulting in inadequate blood flow to the heart muscle itself. | STS |
| Coronary obstruction | Angiographic or echocardiographic evidence of a new, partial or complete, obstruction of a coronary ostium, either by the valve prosthesis itself, the native leaflets, calcifications, or dissection, occurring during or after the TAVR or SAVR procedure. Mechanical coronary artery obstruction following TAVR or index SAVR includes: • impingement of the coronary ostia by the valve support structure in the setting of suboptimal valve positioning and/or 'small aortic root' anatomy; OR • displacement of native aortic valve leaflets towards the coronary ostia during TAVR; OR • suture-related kinking or obstruction or cannulation-related obstruction of the coronary ostia associated with SAVR. | VARC 2/STS |
| Device | For the determination of device relationship, the study device consists of: • The Edwards SAPIEN 3 valve • The Edwards Valve Delivery System • The Edwards Expandable Sheath • Any surgical valve used implanted during index procedure | Sponsor |
| Device (Valve)<br>fracture | The separation of any portion of the frame into two or more parts; as may be determined by radiography, computed tomography,magnetic resonance imaging or by direct examination. | Sponsor |

| Term | Definition | Reference/ |
|---|---|---|
| Device<br>malfunction | The failure of a device to meet any of its performance specifications or otherwise perform as intended. Performance specifications include all claims made in the labeling of the device. | FDA., 21 CFR<br>803.3(m) |
| Device (Valve)<br>thrombosis | Any thrombus attached to or near an implanted valve that occludes part of the blood flow path, interferes with valve function, or is sufficiently large to warrant treatment. Note that valve-associated thrombus identified at autopsy in a patient whose cause of death was not valve-related should not be reported as valve thrombosis | VARC 2 |
| Endocarditis | Endocarditis must meet at least 1 of the following criteria: 1. Patient has organisms cultured from valve or vegetation 2. Patient has 2 or more of the following signs or symptoms: • Fever (>38°C) • New or changing murmur • Embolic phenomena • Skin manifestations (i.e., petechiae, splinter hemorrhages, painful subcutaneous nodules) • CHF • Cardiac conduction abnormality With no other recognized cause and at least 1 of the following: a. organisms cultured from 2 or more blood cultures b. organisms seen on Gram's stain of valve when culture is negative or not done c. valvular vegetation seen during an invasive procedure or autopsy d. positive laboratory test on blood or urine (e.g., antigen tests for H influenzae, S pneumoniae, N meningitidis, or Group B Streptococcus) e. evidence of new vegetation seen on echocardiogram and if diagnosis is made antemortem, physician institutes appropriate antimicrobial therapy. Infection of the endocardial surface of the heart which may include one or more heart valves, the mural endocardium, or a septal | STS |
| EuroSCORE II | defect http://www.euroscore.org/calc.html | European System for<br>Cardiac Operative<br>Risk Evaluation |
| EuroSCORE,<br>logistic | http://www.euroscore.org/calcold.html | European System for<br>Cardiac Operative<br>Risk Evaluation |
| Explant | Removal of the investigational valve implant for any reason | Sponsor |

| Term | Definition | Reference/<br>Justification |
|---|---|---|
| Hemolysis | Evidence of RBC destruction best explained by hemolysis (LDH >350 u/L and decreased haptoglobin based on site lab normals) and no other explanation for the findings. Microscopic evidence may be considered supportive. | Sponsor |
| Hospitalization<br>(repeat) | Any <i>unplanned</i> admission to the hospital (including an emergency department visit) for either a diagnostic or therapeutic purpose (e.g. diuretics, inotropes, chronotropes, oral or intra-venous therapy) following discharge from the index hospitalization | Sponsor |
| Hospitalization for CHF | An event where the patient is admitted to the hospital with a primary diagnosis of CHF where the length of stay is at least 24 h (or extends over a calendar date if the hospital admission and discharge times are unavailable), and the patient exhibits new or worsening symptoms of CHF on presentation, has objective evidence of new or worsening CHF, and receives initiation or intensification of treatment specifically for CHF. | 2014 ACC/AHA Key<br>Data Elements and<br>Definitions for<br>CardiovascularEndpo<br>int Events in Clinical<br>Trials/VARC 2 |
| | Clinical symptoms of CHF include, but not limited to a pulmonary edema, hypoperfusion, or documented volume overload AND administration of IV diuresis or inotropic therapy, performance of aortic valvuloplasty, institution of mechanical support (IABP or ventilation for pulmonary oedema) or haemodialysis for volume overload. | |
| Hypertension | Systolic pressure > 140 or a diastolic pressure > 90 mmHg | Sponsor |
| Hypotension | Systolic pressure < 90 or a diastolic pressure < 60 mmHg | Sponsor |
| Index<br>hospitalization | The beginning of the Index Hospitalization is defined as the day the patient is admitted for valve implant procedure and continues until the patient is discharged from the hospital. | Sponsor |
| Infection | Known infection requiring intravenous antibiotics for other than prophylaxis, and/or extended hospitalization | Sponsor |
| Lung disease,<br>severe | FEV1 < 50% predicted or currently on home oxygen | Sponsor |
| Liver disease, chronic | MELD Score ≥ 10 or Child-Pugh Class B or C | Sponsor |

| Term | Definition | Reference/<br>Justification |
|---|---|---|
| Mini-mental state examination (MMSE) | A questionnaire that is used extensively in clinical and research settings to measure cognitive impairment. | Pangman, VC; Sloan, J; Guse, L. (2000). "An Examination of Psychometric Properties of the Mini-Mental State Examination and the Standardized Mini-Mental State Examination: Implications for Clinical Practice". Applied Nursing Research 13 (4): 209–213. |
| MELD (Model<br>For End-Stage<br>Liver Disease)<br>Score | A scoring system for assessing the severity and quantification of chronic liver disease. It is preferable to using the calculator (http://www.mdcalc.com/meld-score-model-for-end-stage-liver-disease-12-and-older/) to calculate the MELD as there are several caveats relating to minimum and maximum values assigned in the MELD Values should be no more than 48 hours old In interpreting the MELD Score in hospitalized patients, the 3 month mortality is: 40 or more — 71.3% mortality 30–39 — 52.6% mortality 20–29 — 19.6% mortality 10–19 — 6.0% mortality | Wiesner et al. Model<br>for end-stage liver<br>disease (MELD) and<br>allocation of donor<br>livers.<br>Gastroenterology<br>(2003) vol. 124 (1) pp.<br>91-6 |
| Modified Rankin<br>Scale (mRS) | <ul> <li>&lt;9 — 1.9% mortality</li> <li>A commonly used scale for measuring the degree of disability or dependence in the daily activities of people who have suffered a stroke, as follows:</li> <li>0 No symptoms at all</li> <li>1 No significant disability despite symptoms; able to carry out all usual duties and activities</li> <li>2 Slight disability; unable to carry out all previous activities, but able to look after own affairs without assistance</li> <li>3 Moderate disability; requiring some help, but able to walk without assistance</li> <li>4 Moderately severe disability; unable to walk without assistance and unable to attend to own bodily needs without assistance</li> <li>5 Severe disability; bedridden, incontinent and requiring constant nursing care and attention</li> <li>6 Dead</li> </ul> | Van Swieten, J. C., et al. "Interobserver agreement for the assessment of handicap in stroke patients." Stroke 19.5 (1988): 604-607. |

| Term | Definition | Reference/<br>Justification |
|---|---|---|
| Mortality, all- | Cardiovascular mortality | VARC 2 |
| cause | _ | |
| | Any of the following criteria: | |
| | Death due to proximate cardiac cause (e.g. myocardial infarction, cardiac tamponade, worsening heart failure) | |
| | Death caused by non-coronary vascular conditions<br>such as neurological events, pulmonary embolism,<br>ruptured aortic aneurysm, dissecting aneurysm, or<br>other vascular disease | |
| | All procedure-related deaths, including those related<br>to a complication of the procedure or treatment for a<br>complication of the procedure | |
| | <ul> <li>All valve-related deaths including structural or<br/>nonstructural valve dysfunction or other valve-<br/>related adverse events</li> </ul> | |
| | <ul><li>Sudden or unwitnessed death</li><li>Death of unknown cause</li></ul> | |
| | Non-cardiovascular mortality Any death in which the primary cause of death is clearly related to another condition (e.g. trauma, cancer, suicide). | |
| Myocardial<br>Infarction | An acute ischemic event that is associated with documented and clinically significant myocardial necrosis Any one of the following criteria meets the diagnosis for MI: | STS |
| | Detection of a rise and/or fall of cardiac biomarker values [preferably cardiac troponin (cTn)] with at least one value above the 99th percentile upper reference limit (URL) and with at least one of the following: | |
| | - Symptoms of ischemia | |
| | <ul> <li>New or presumed new significant ST-segment—<br/>T wave (ST-T) changes or new left bundle<br/>branch block (LBBB)</li> </ul> | |
| | - Development of pathological Q waves in the ECG | |
| | <ul> <li>Imaging evidence of new loss of viable<br/>myocardium or new regional wall motion<br/>abnormality</li> </ul> | |
| | Identification of an intracoronary thrombus by angiography | |

| Term | Definition | Reference/<br>Justification |
|---|---|---|
| National<br>Institutes of<br>Health Stroke<br>Scale (NIHSS) | The NIHSS can help physicians determine the severity of a stroke, predict clinical outcomes and can help guide management. | NIHSS |
| New York Heart<br>Association<br>Classification<br>(NYHA) | NYHA Class Functional Capacity Patients with cardiac disease but without resulting limitation of physical activity. Ordinary physical activity does not cause undue fatigue, palpitation, dyspnea, or anginal pain. Patients with cardiac disease resulting in slight limitation of physical activity. They are comfortable at rest. Ordinary physical activity results in fatigue, palpitation, II dyspnea, or anginal pain. Patients with cardiac disease resulting in marked limitation of physical activity. They are comfortable at rest. Less than ordinary activity causes fatigue, palpitation, III dyspnea, or anginal pain. Patients with cardiac disease resulting in inability to carry on any physical activity without discomfort. Symptoms of heart failure or the anginal syndrome may be present even at rest. If any physical activity is undertaken, discomfort is increased. | The Criteria Committee of the New York Heart Association. (1994). Nomenclature and Criteria for Diagnosis of Diseases of the Heart and Great Vessels. (9th ed.). Boston: Little, Brown & Co. pp. 253–256. |
| Paravalvular<br>Leak | Paravalvular or paraprosthetic leak (PVL) is a complication associated with the implantation of a prosthetic heart valve whether traditional (surgical) or a transcatheter (TAVR) approach. PVL refers to blood flowing through a channel between the structure of the implanted valve and cardiac tissue as a result of a lack of appropriate sealing | ESC |

| Term | Definition | Reference/<br>Justification |
|---|---|---|
| Peripheral<br>vascular disease<br>(PVD) | Includes peripheral arterial disease of upper and lower extremity, renal, mesenteric, and abdominal aortic systems, as follows: Claudication, either with exertion or at rest Amputation for arterial vascular insufficiency Vascular reconstruction, bypass surgery, or percutaneous intervention to the extremities (excluding dialysis fistulas and vein stripping) Documented abdominal aortic aneurysm with or without repair Positive noninvasive test (e.g., ankle brachial index =< 0.9, ultrasound, magnetic resonance or computed tomography imaging of > 50% diameter stenosis in any peripheral artery, i.e., renal, subclavian, femoral, iliac) or angiographic imaging Peripheral arterial disease excludes disease in the carotid, cerebrovascular arteries or thoracic aorta. PVD does not include DVT. | STS |
| Porcelain aorta<br>or severely<br>atherosclerotic<br>aorta | Heavy circumferential calcification or severe atheromatous plaques of the entire ascending aorta extending to the arch such that aortic cross-clamping is not feasible. | VARC 2 |
| Pulmonary<br>hypertension | A mean pulmonary artery pressure >or equal 25 mm Hg in presence of LAP/wedge <= 15 mm Hg | ACC |
| Pre-existing condition | A pre-existing condition is one that is present at the start of study treatment. A preexisting condition is not an adverse event unless it worsens as a result of the study treatment. | Sponsor |

| Term | Definition | | | | Reference/<br>Justification |
|---|---|---|---|---|---|
| Prosthetic aortic valve stenosis | | Normal | Mild | Moderate/severe | VARC-2 |
| criteria <sup>a</sup> | | | | | |
| Ontona | Quantita | tive Paramet | ters (flow-c | dependent) <sup>b</sup> | |
| | Peak velocity<br>(m/s) | <3 m/s | 3-4 m/s | >4m/s | |
| | Mean gradient<br>(mmHg) | <20 mmHg | 20-40<br>mmHg | >40 mmHg | |
| | Quantitat | tive paramet | ers (flow-ir | ndependent) | |
| | Doppler velocity index <sup>c</sup> | >0.35 | 0.35-0.25 | <0.25 | |
| | Effective orifice aread | >1.1 cm <sup>2</sup> | >1.1-0.8<br>cm <sup>2</sup> | <0.8 cm <sup>2</sup> | |
| | Effective orifice areae | >0.9 cm <sup>2</sup> | >0.9-0.6<br>cm <sup>2</sup> | <0.6 cm <sup>2</sup> | |
| | (50–70 mL).<br><sup>b</sup> These parame<br>concomitant ao<br><sup>c</sup> For LVOT >2.5 | ters are mor<br>rtic regurgita<br>cm, signific<br>of BSA ≥1.6<br>e and the siz | re affected<br>ation.<br>cant stenos<br>cm² (note<br>ze of the n | al stroke volume by flow, including sis criteria is <0.20. : dependent on the ative annulus). | |

| Term | Definition | | | | Reference/<br>Justification |
|---|---|---|---|---|---|
| Prosthetic aortic valve | | Normal | Mild | Moderate/severe | VARC 2 |
| regurgitation<br>criteria | | Semi-quant | l<br>titative Parame | ters | |
| | Diastolic flow<br>reversal in the<br>descending<br>aorta—PW | Absent or brief early diastolic | Intermediate | Prominent,<br>holodiastolic | |
| | Circumferential extent of prosthetic valve paravalvular regurgitation (%) <sup>a</sup> | <10% | 10-29% | ≥30% | |
| | | Overetites | 45 | .h | |
| | Regurgitant | Quantita | tive parameters | 30 | |
| | volume<br>(mL/beat) | <30 mL | 30-59 mL | ≥60 mL | |
| | Regurgitant | | | | |
| | fraction (%) EROA (cm²) | <30%<br>0.10 cm <sup>2</sup> | 30-49%<br>0.10-0.29<br>cm <sup>2</sup> | ≥50%<br>≥0.30 cm² | |
| | compared with | n the quant | titative Doppl | mate the severity<br>er.<br>sis criteria is <0.20. | |
| Reintervention | after the comp | olanted or o | operated val<br>ne valve impl | r replaces a<br>ve, which occurrs<br>ant procedure and<br>hese interventions | STS/AATS |
| | <ul><li>Surgio</li><li>Valve</li></ul> | | alvuloplasty<br>alve replacer<br>k closure | ment | |

| Term | Definition | Reference/<br>Justification |
|---|---|---|
| Serious Adverse<br>Event (SAE) | Adverse Event that: • Leads to death; | ISO 14155-1:2011<br>FDA (21 CFR 312.32<br>(a) |
| | <ul> <li>Leads to a serious deterioration in the health of<br/>the study patient that:</li> </ul> | |
| | o Results in life-threatening illness or injury; | |
| | <ul> <li>Results in a permanent impairment of a<br/>body structure or a body function;</li> </ul> | |
| | <ul> <li>Requires inpatient hospitalization or<br/>prolongation of existing hospitalization;</li> </ul> | |
| | <ul> <li>Results in medical or surgical intervention<br/>to prevent permanent impairment to body<br/>structure or a body function;</li> </ul> | |
| | <ul> <li>Led to fetal distress, fetal death or congenital<br/>abnormality or birth defect;</li> <li>Significant medical event</li> </ul> | |
| | Important medical events that do not meet the above criteria may still be considered an SAE if they seriously jeopardize the patient and require immediate medical or surgical intervention to prevent one of the aforementioned outcomes. | |
| Sternal wound dehiscence | Opening of sternal with negative cultures and no signs of infection requiring a procedure or operation for treatment | Sponsor |
| Valve implant procedure | Placement of study device and/or additional procedures occurring in the cath lab and/or operating room which are completed prior to subject transfer to a post-procedure recovery unit (e.g. Recovery Room, ICU/CCU, etc. The valve implant procedure will be considered to have started when: | Sponsor |
| | <ul> <li>The first interventional access related puncture<br/>(venous or arterial) is established for TAVR.</li> <li>The first skin incision is performed for SAVR.</li> </ul> | |
| | Performance of TEE does not by itself constitute start of procedure | |
| Valve<br>Thrombosis | Valve thrombosis is any thrombus not caused by infection attached to or near an operated valve that occludes part of the blood flow path, interferes with valve function, or is sufficiently large to warrant treatment. | VARC2 |
| Stroke /<br>Transient<br>Ischemic Attack | Diagnostic Criteria | VARC 2 |

| Term | Definition | Reference/<br>Justification |
|---|---|---|
| (TIA) | Acute episode of a focal or global neurological deficit with at least one of the following: | |
| | <ul> <li>□ change in level of consciousness</li> <li>□ hemiplegia</li> <li>□ hemiparesis</li> <li>□ numbness or sensory loss affecting one side of the body</li> <li>□ dysphasia or aphasia</li> <li>□ hemianopia</li> <li>□ amaurosis fugax</li> <li>□ or other neurological signs or symptoms consistent with stroke</li> </ul> | |
| | Duration of a focal or global neurological deficit >24 h; <b>OR</b> <24 h, if available neuroimaging documents a new hemorrhage or infarct; <b>OR</b> the neurological deficit results in death | |
| | No other readily identifiable nonstroke cause for the clinical presentation (e.g., brain tumor, trauma, infection, hypoglycemia, peripheral lesion, pharmacological influences)to be determined by or in conjunction with designated neurologist* | |
| | Confirmation of the diagnosis by at least one of the following#: | |
| | <ul> <li>□ Neurology or neurosurgical specialist</li> <li>□ Neuroimaging procedure (MR or CT scan)</li> <li>□ Clinical presentation alone</li> </ul> | |
| | Stroke definitions†: | |
| | □ Non-disabling: a mRS score of less than 2 at 90 days or the last available clinical visit with evaluable data or one that does not result in an increase of at least one mRS category from an individual's pre-stroke baseline | |
| | □ Disabling: a mRS score of 2 or more at 90 days or the last available clinical visit with evaluable data and an increase of at least one mRS category from an individual's pre-stroke baseline | |
| | Stroke classification: | |
| | ☐ Hemorrhagic: an acute episode of focal or global cerebral or spinal dysfunction caused by intraparenchymal, intraventricular, or subarachnoid hemorrhage. | |

| Term | Definition | Reference/<br>Justification |
|---|---|---|
| | ☐ <i>Ischemic:</i> an acute symptomatic episode of focal cerebral, spinal, or retinal dysfunction caused by an infarction of the central nervous system tissue | |
| | ☐ <i>Undetermined:</i> stroke with insufficient information to allow categorization as ischemic or hemorrhagic. | |
| | Transient Ischemic Attack (TIA) | |
| | Duration of focal or global neurological deficit <24 h, any variable neuroimaging does not demonstrate a new hemorrhage or infarct | |
| | *Patients with non-focal global encephalopathy will not be reported as a stroke without unequivocal evidence based upon neuroimaging studies. #If a stroke is reported without evidence of confirmation of the diagnosis by one of these methods, the event may still be considered a stroke on the basis of the clinical presentation alone. †Modified Rankin score assessments should be made by qualified individuals according to a certification process. | |
| Structural performance | Evaluation of migration, embolization, fracture, or thrombosis | FDA |
| Structural<br>Valvular<br>Deterioration<br>(SVD) | Structural valve deterioration includes dysfunction or deterioration exclusive of infection or thrombosis as determined by reoperation, autopsy or clinical investigation. The term structural deterioration refers to changes intrinsic to the valve, such as wear, fracture, calcification, leaflet tear, leaflet retraction, suture line disruption of components a prothetic valve, thickening, stenosis | Akins, Cary W., et al. "Guidelines for reporting mortality and morbidity after cardiac valve interventions." European Journal of Cardio-Thoracic Surgery 33.4 (2008): 523-528. |
| STS Adult<br>Cardiac Surgery<br>Risk Calculator | The Society of Thoracic Surgeons' risk models predict the risk of operative mortality and morbidity after adult cardiac surgery on the basis of patient demographic and clinical variables. | STS |
| Syncope | http://riskcalc.sts.org/stswebriskcalc/#/ A fainting spell or loss of consciousness | STS |
| SYNTAX Score | An angiographic grading tool to determine the complexity of coronary artery disease. <a href="http://www.syntaxscore.com/">http://www.syntaxscore.com/</a> <a href="http://ir-nwr.ru/calculators/syntaxscore/frameset.htm">http://ir-nwr.ru/calculators/syntaxscore/frameset.htm</a> | |

| Term | Definition | Reference/<br>Justification |
|---|---|---|
| 6 Minute Walk<br>Test | A performance-based measure of functional exercise capacity. The test measures the distance an individual is able to walk over a total of six minutes on a hard, flat surface. See more at: http://www.rheumatology.org/I-Am-A/Rheumatologist/Research/Clinician-Researchers/Six-Minute-Walk-Test-SMWT#sthash.cFCDWfkn.dpuf | ATS |
| THV-in-THV | An additional valve prosthesis is implanted within a previously implanted prosthesis because of suboptimal device position and/or function, during or after the valve implant procedure | VARC 2 |
| Transient<br>Ischemic Attack<br>(TIA) | See "Stroke / Transient Ischemic Attack (TIA)" | |
| Unanticipated<br>Adverse Device<br>Effect (UADE) | Any serious adverse effect on health or safety or any life-threatening problem or death caused by, or associated with, a device, if that effect, problem, or death was not previously identified in nature, severity, or degree of incidence in the investigational plan or application (including a supplementary plan or application), or any other unanticipated serious problems associated with a device that relates to the rights, safety, or welfare of patients. | FDA |
| Vascular injury | Injury that may be caused by a guidewire, vascular sheath, delivery catheter, or any balloon used for aortic valve predilatation and can include arterial dissection, perforation, arteriovenous fistula, pseudoaneurysm formation, retroperitoneal hemorrhage, or incomplete arteriotomy closure. Venous injuries can include perforation, tears and thromboembolism. Cardiac vascular injury can include perforation or tearing of the major cardiac structures that require repair. | Sponsor |
| Valve<br>malpositioning | Valve migration After initial correct positioning, the valve prosthesis moves upward or downward, within the aortic annulus from its initial position, with or without consequences | VARC 2 |
| | Valve embolization The valve prosthesis moves during or after deployment such that it loses contact with the aortic annulus | |
| | Ectopic valve deployment Permanent deployment of the valve prosthesis in a location other than the aortic root | |

# Appendix C Instructions For Use (IFU)

Refer to device package label to access electronic IFU or contact an Edwards Clinical Affairs representative.

# Appendix D Physician and Support Staff Training

Title: Edwards Lifesciences Physician Training and Procedural Case Support Plan

Date: October 2017

**Purpose**: The purpose of this plan is to document and standardize the requirements for physician training for transcatheter heart valve (THV) implantation. It further describes the procedural case support provided by an Edwards Lifesciences representative (e.g., Clinical Specialist).

Scope: This plan applies to the implanting physician Investigators (Interventional Cardiologists/Surgeon for the PARTNER 3 trial. This plan addresses training for current users who have previously completed training under prior Edwards's trials and newly designated implanting physicians.

# I. Current User Physician Training Plan

## 1. Didactic Presentation and Device Demonstration

A didactic presentation including room set-up and patient preparation, sizing, device description and usage, procedural steps, complications and technical tips is given to the implanting physicians. In addition, a hands-on device demonstration is given. Both the didactic presentation and device demonstration are provided by an Edwards Lifesciences representative (e.g., Edwards Clinical Specialist).

## 2. Documentation

Training for the implanting physicians will be documented on the appropriate Training Forms (i.e., checked-off, dated and signed) by an Edwards Lifesciences representative as training is completed. Training records are maintained by Edwards Lifesciences in addition to being filed in the site study files.

# **II.** New User Physician Training Plan includes:

# 1. THV Fundamentals Training Program

All new implanting physicians must attend the Edwards THV Fundamentals Training Program, which consists of the following:

- a) Didactic training/review of training manual: Focuses of key aspects of patient evaluation, device overview, procedural and technical tips, potential complications and troubleshooting tips.
- b) Device demonstration
- c) Simulation: Not required. Used as an enhancement to device demonstration and procedure training when available or applicable.
- d) Case observation or Case Review: 1 case observation or case review prior to first THV case.
- e) Certain requirements may be waived for physicians with applicable prior experience including but not limited to: prior involvement in THV or procedural development, or prior clinical experience in the aortic position. Any requirements waived to be indicated by a letter to file summarizing the reason for waiver and applicable prior experience.

## 2. Proctoring

The implanting physician must be proctored by an experienced physician for a minimum of two successful valve implantation procedures and deemed ready for independence by both the proctor and Clinical Specialist. These are to be performed at the Investigator's institution with his staff. If the proctor is not satisfied that these two procedures provide sufficient preparation, then subsequent proctoring sessions may be added as needed. Proctor requirements may be waived for physicians with applicable prior experience including but not limited to: prior involvement in THV or procedural development, or prior clinical experience in the aortic position. Any requirements waived to be indicated by a letter to file summarizing the reason for waiver and applicable prior experience.

## 3. Proctor Requirements

An implanting physician is considered a proctor only after having completed a minimum of eight procedures. Proctors should have extensive experience in recognition and management of intraprocedural complications and advanced troubleshooting skills.

# 4. Refresher THV Fundamentals Training

Required for implanting physicians if greater than 3 months from THV Fundamentals completion to first case or 5 months in between THV cases.

## 5. Didactic Presentation and Device Demonstration

Once THV Fundamentals Training and Proctoring have been complete, the implanting physicians required to be trained by an Edwards Representative (e.g., Clinical Specialist) on the study specific didactic presentation and receive a hands-on device demonstration (if different from training received for commercial device).

# 6. Documentation

Training for the implanting physicians will be documented on the appropriate Training Forms (i.e., checked-off, dated and signed) by an Edwards Lifesciences representative as training is completed.

Training records are maintained by Edwards Lifesciences and copies will be filed in the site study files.

# **III. Procedural Case Support**

An Edwards Lifesciences representative (e.g., Clinical Specialist) will attend all procedures to answer device and procedural questions, and is responsible for ensuring that all Edwards THV devices are prepared in accordance to the Instructions for Use Throughout the PARTNER 3 trial in no instance will any site perform a THV procedure without an Edwards's representative (e.g., Clinical Specialist) present.

# Appendix E Six Minute Walk Test

# **American Thoracic Society**

# ATS Statement: Guidelines for the Six-Minute Walk Test

THIS OFFICIAL STATEMENT OF THE AMERICAN THORACIC SOCIETY WAS APPROVED BY THE ATS BOARD OF DIRECTORS MARCH 2002

### CONTENTS

Purpose and Scope
Background
Indications and Limitations
Contraindications
Safety Issues
Technical Aspects of the 6-Minute Walk Test
Required Equipment
Patient Preparation
Measurements
Quality Assurance
Interpretation
References

### PURPOSE AND SCOPE

This statement provides practical guidelines for the 6-minute walk test (6MWT). Specifically, it reviews indications, details factors that influence results, presents a brief step-by-step protocol, outlines safety measures, describes proper patient preparation and procedures, and offers guidelines for clinical interpretation of results. These recommendations are not intended to limit the use of alternative protocols for research studies. We do not discuss the general topic of clinical exercise testing.

As with other American Thoracic Society statements on pulmonary function testing, these guidelines come out of a consensus conference. Drafts were prepared by two members (P.L.E. and R.J.Z.) and were based on a comprehensive Medline literature search from 1970 through 2001, augmented by suggestions from other committee members. Each draft responded to comments from the working committee. The guidelines follow previously published methods as closely as possible and provide a rationale for each specific recommendation. The final recommendations represent a consensus of the committee. The committee reviewed in five years and in the meantime encourages further research in areas of controversy.

### BACKGROUND

There are several modalities available for the objective evaluation of functional exercise capacity. Some provide a very complete assessment of all systems involved in exercise performance (high tech), whereas others provide basic information but are low tech and are simpler to perform. The modality used should be chosen based on the clinical question to be addressed and on available resources. The most popular clinical exercise tests in order of increasing complexity are stair climbing, a 6MWT, a shuttle-walk test, detection of exercise-induced asthma, a cardiac stress test (e.g., Bruce protocol), and a cardio-

Am J Respir Crit Care Med Vol 166. pp 111–117, 2002 DOI: 10.1164/rccm.166/1/111 Internet address: www.atsjournals.org pulmonary exercise test (1, 2). Other professional organizations have published standards for cardiac stress testing (3, 4).

Assessment of functional capacity has traditionally been done by merely asking patients the following: "How many flights of stairs can you climb or how many blocks can you walk?" However, patients vary in their recollection and may report overestimations or underestimations of their true functional capacity. Objective measurements are usually better than self-reports. In the carly 1960s, Balke developed a simple test to evaluate the functional capacity by measuring the distance walked during a defined period of time (5). A 12-minute field performance test was then developed to evaluate the level of physical fitness of healthy individuals (6). The walking test was also adapted to assess disability in patients with chronic bronchitis (7). In an attempt to accommodate patients with respiratory disease for whom walking 12 minutes was too exhausting, a 6-minute walk was found to perform as well as the 12-minute walk (8). A recent review of functional walking tests concluded that "the 6MWT is easy to administer, better tolerated, and more reflective of activities of daily living than the other walk tests" (9).

The 6MWT is a practical simple test that requires a 100-ft hallway but no exercise equipment or advanced training for technicians. Walking is an activity performed daily by all but the most severely impaired patients. This test measures the distance that a patient can quickly walk on a flat, hard surface in a period of 6 minutes (the 6MWD). It evaluates the global and integrated responses of all the systems involved during exercise, including the pulmonary and cardiovascular systems, systemic circulation, peripheral circulation, blood, neuromuscular units, and muscle metabolism. It does not provide specific information on the function of each of the different organs and systems involved in exercise or the mechanism of exercise limitation, as is possible with maximal cardiopulmonary exercise testing. The self-paced 6MWT assesses the submaximal level of functional capacity. Most patients do not achieve maximal exercise capacity during the 6MWT; instead, they choose their own intensity of exercise and are allowed to stop and rest during the test. However, because most activities of daily living are performed at submaximal levels of exertion, the 6MWD may better reflect the functional exercise level for daily physical activities.

## INDICATIONS AND LIMITATIONS

The strongest indication for the 6MWT is for measuring the response to medical interventions in patients with moderate to severe heart or lung disease. The 6MWT has also been used as a one-time measure of functional status of patients, as well as a predictor of morbidity and mortality (see Table 1 for a list of these indications). The fact that investigators have used the 6MWT in these settings does not prove that the test is clinically useful (or the best test) for determining functional capacity or changes in functional capacity due to an intervention in patients with these diseases. Further studies are necessary to determine the utility of the 6MWT in various clinical situations.

Formal cardiopulmonary exercise testing provides a global assessment of the exercise response, an objective determination of functional capacity and impairment, determination of the appropriate intensity needed to perform prolonged exercise, quantification of factors limiting exercise, and a definition of the underlying pathophysiologic mechanisms such as the contribution of different organ systems involved in exercise. The 6MWT does not determine peak oxygen uptake, diagnose the cause of dyspnea on exertion, or evaluate the causes or mechanisms of exercise limitation (1, 2). The information provided by a 6MWT should be considered complementary to cardiopulmonary exercise testing, not a replacement for it. Despite the difference between these two functional tests, some good correlations between them have been reported. For example, a significant correlation (r = 0.73) between 6MWD and peak oxygen uptake has been reported for patients with end-stage lung diseases (36, 37).

patients with end-stage lung diseases (36, 37).

In some clinical situations, the 6MWT provides information that may be a better index of the patient's ability to perform daily activities than is peak oxygen uptake; for example, 6MWD correlates better with formal measures of quality of life (38). Changes in 6MWD after therapeutic interventions correlate with subjective improvement in dyspnea (39, 40). The reproducibility of the 6MWD (with a coefficient of variation of approximately 8%) appears to be better than the reproducibility of 1-second forced expiratory volume in patients with chronic obstructive pulmonary disease (COPD) (8, 41-43). Questionnaire indices of functional status have a larger hard-term variability (22-33%) than does the 6MWD (37).

short-term variability (22-33%) than does the 6MWD (37). The shuttle-walking test is similar to the 6MWT, but it uses an audio signal from a tape cassette to direct the walking pace of the patient back and forth on a 10-m course (44-47). The walking speed is increased every minute, and the test ends when the patient cannot reach the turnaround point within the required time. The exercise performed is similar to a symptom-limited, maximal, incremental treadmill test. An advantage of the shuttle walking test is that it has a better correlation with peak oxygen uptake than the 6MWD. Disadvantages include less validation, less widespread use, and more potential for cardiovascular problems.

### CONTRAINDICATIONS

Absolute contraindications for the 6MWT include the following: unstable angina during the previous month and myocar-

# TABLE 1. INDICATIONS FOR THE SIX-MINUTE WALK TEST

Pretrestment and positivaliment comparisons Lung transplantation (9, 10) Lung resection (11) Lung volume reduction surgery (12, 13) Pulmonary rehabilisation (14, 15) COPD (16-18) Pulmonary hypertension Heart failure (19, 20) Functional status (single measurement) COPD (21, 22) Cystic fitnessis (23, 24) Heart failure (25-27) Poripheral varcular disease (28, 29) Fibromyelyla (30) Older patients (31) Predictor of most (31) Predictor of most (31) Predictor of most (31) Predictor of (22, 33) COPD (34, 35) COPD (34, 35) Primary pulmonary hypertension (10, 36)

Definition of abbreviation: COPD = chronic obstructive pulmonary disease.

dial infarction during the previous month. Relative contraindications include a resting heart rate of more than 120, a systolic blood pressure of more than 180 mm Hg, and a diastolic blood pressure of more than 100 mm Hg.

Patients with any of these findings should be referred to the physician ordering or supervising the test for individual clinical assessment and a decision about the conduct of the test. The results from a resting electrocardiogram done during the previous 6 months should also be reviewed before testing. Stable exertional angina is not an absolute contraindication for a 6MWT, but patients with these symptoms should perform the test after using their antiangina medication, and rescue nitrate medication should be readily available.

#### Pationale

Patients with the previously mentioned risk factors may be at increased risk for arrhythmias or cardiovascular collapse during testing. However, each patient determines the intensity of their exercise, and the test (without electrocardiogram monitoring) has been performed in thousands of older persons (31, 48–50) and thousands of patients with heart failure or cardiomyopathy (32, 51, 52) without serious adverse events. The contraindications listed previously here were used by study investigators based on their impressions of the general safety of the 6MWT and their desire to be prudent, but it is unknown whether adverse events would occur if such patients performed a 6MWT; they are, therefore, listed as relative contraindications.

### SAFETY ISSUES

- Testing should be performed in a location where a rapid, appropriate response to an emergency is possible. The appropriate location of a crash cart should be determined by the physician supervising the facility.
- the physician supervising the facility.

  2. Supplies that must be available include oxygen, sublingual nitroglycerine, aspirin, and albuterol (metered dose inhalor or nebulizer). A telephone or other means should be in place to enable a call for help.
- 3. The technician should be certified in cardiopulmonary resuscitation with a minimum of Basic Life Support by an American Health Association-approved cardiopulmonary resuscitation course. Advanced cardiac life support certification is desirable. Training, experience, and certification in related health care fields (registered nurse, registered respiratory therapist, certified pulmonary function technician, etc.) are also desirable. A certified individual should be readily available to respond if needed.
- Physicians are not required to be present during all tests.
   The physician ordering the test or a supervising laboratory physician may decide whether physician attendance at a specific test is required.
- If a patient is on chronic oxygen therapy, oxygen should be given at their standard rate or as directed by a physician or a protocol

Reasons for immediately stopping a 6MWT include the following: (1) chest pain, (2) intolerable dyspnea, (3) leg cramps, (4) staggering, (5) diaphoresis, and (6) pale or ashen appearance.

Technicians must be trained to recognize these problems and the appropriate responses. If a test is stopped for any of these reasons, the patient should sit or lie supine as appropriate depending on the severity or the event and the technician's assessment of the severity of the event and the risk of syncope. The following should be obtained based on the judgment of the technician: blood pressure, pulse rate, oxygen saturation, and a physician evaluation. Oxygen should be administered as appropriate.

American Thoracic Society

### TECHNICAL ASPECTS OF THE 6MWT

The 6MWT should be performed indoors, along a long, flat, straight, enclosed corridor with a hard surface that is seldom traveled. If the weather is comfortable, the test may be performed outdoors. The walking course must be 30 m in length. A 100-ft hallway is, therefore, required. The length of the corridor should be marked every 3 m. The turnaround points should be marked with a cone (such as an orange traffic cone). A starting line, which marks the beginning and end of each 60-m lap, should be marked on the floor using brightly colored tape.

Rationale. A shorter corridor requires patients to take mo

time to reverse directions more often, reducing the 6MWD. Most studies have used a 30-m corridor, but some have used 20- or 50-m corridors (52-55). A recent multicenter study found no significant effect of the length of straight courses ranging from 50 to 164 ft, but patients walked farther on con-

tinuous (oval) tracks (mean 92 ft farther) (54).

The use of a treadmill to determine the 6MWD might save space and allow constant monitoring during the exercise, but the use of a treadmill for 6-minute walk testing is not recommended. Patients are unable to pace themselves on a treadmill. In one study of patients with severe lung disease, the mean distance walked on the treadmill during 6 minutes (with the speed adjusted by the patients) was shorter by a mean of 14% when compared with the standard 6MWD using a 100-ft hallway (57). The range of differences was wide, with patients walking between 400-1,300 ft on the treadmill who walked 1,200 ft in the hallway. Treadmill test results, therefore, are not interchangeable with corridor tests.

### REQUIRED EQUIPMENT

- 1. Countdown timer (or stopwatch)
- Mechanical lap counter
- 3. Two small cones to mark the turnaround points
- A chair that can be easily moved along the walking course Worksheets on a clipboard 4.
- A source of oxygen
- Sphygmomanometer
- 8. Telephone
- 9. Automated electronic defibrillator

### PATIENT PREPARATION

- 1. Comfortable clothing should be worn.
- Appropriate shoes for walking should be worn.
- Patients should use their usual walking aids during the test (canc, walker, etc.).
- The patient's usual medical regimen should be continued.
- 5. A light meal is acceptable before early morning or early af-
- Patients should not have exercised vigorously within 2 hours of beginning the test.

### MEASUREMENTS

- Repeat testing should be performed about the same time of day to minimize intraday variability.
- A "warm-up" period before the test should not be performed. The patient should sit at rest in a chair, located near the starting position, for at least 10 minutes before the test starts. During this time, check for contraindications, measure pulse and blood pressure, and make sure that clothing and shoes are appropriate. Compete the first portion of the worksheet (see the APPENDIX).

4. Pulse oximetry is optional. If it is performed, measure and record baseline heart rate and oxygen saturation (SpO2) and follow manufacturer's instructions to maximize the sig-nal and to minimize motion artifact (56, 57). Make sure the readings are stable before recording. Note pulse regularity

and whether the oximeter signal quality is acceptable

whether the oximeter signal quality is acceptable.

The rationale for measuring oxygen saturation is that although the distance is the primary outcome measure, improvement during serial evaluations may be manifest either by an increased distance or by reduced symptoms with the same distance walked (39). The SPO<sub>2</sub> should not be used for constant monitoring during the exercise. The technician must not walk with the patient to observe the SPO<sub>2</sub> if worn during the walk, the pulse oximeter must be lightweight (less than 2 pounds), battery powered, and held in place (perhaps by a "fanny pack") so that the patient does not have to hold or stabilize it and so that stride is not affected. Many pulse oximeters have considerable motion artifact that prevents oximeters have considerable motion artifact that prevents accurate readings during the walk. (57)

- 5. Have the patient stand and rate their baseline dyspnea and overall fatigue using the Borg scale (see Table 2 for the Borg scale and instructions [58]).
  Set the lap counter to zero and the timer to 6 minutes. As-
- semble all necessary equipment (lap counter, timer, clipboard, Borg Scale, worksheet) and move to the starting
- 7. Instruct the patient as follows:

"The object of this test is to walk as far as possible for 6 minutes. You will walk back and forth in this hallway. Six minutes is a long time to walk, so you will be exerting your-self. You will probably get out of breath or become exhausted. You are permitted to slow down, to stop, and to rest as necessary. You may lean against the wall while resting, but resume walking as soon as you are able.

You will be walking back and forth around the cones. You should pivot briskly around the cones and continue back the other way without hesitation. Now I'm going to show you. Please watch the way I turn without hesitation."

Demonstrate by walking one lap yourself, Walk and pivot around a cone briskly.

"Are you ready to do that? I am going to use this counter to keep track of the number of laps you complete. I will click it each time you turn around at this starting line. Remember that the object is to walk AS FAR AS POSSIBLE for 6 minutes, but don't run or jog.

Start now, or whenever you are ready."

### TABLE 2. THE BORG SCALE

| 0 | Nothing at all | |
|-----|-------------------|-------------------|
| 0.5 | Yery, very slight | (just noticeable) |
| | Maria Babe | |

Slight (light)

Moderate Somewhat severe Severe (heavy)

Very severe

10 Very, very severe (maximal)

This Borg scale should be printed on heavy paper (11 inches high and perhaps laminated) in 20-point type size. At the beginning of the 6-minute exercise, show the scale to the patient and eak the patient this: "Please grade your level of shortness of breash using this scale." Then sak this: "Please grade your level of staligue using this scale." At the end of the exercise, remind the patient of the breathing number that they choice before the exercise and ask the patient to grade their breathing fevel again. Then ask the patient to grade their level of fatigue, after reminding them of their grade before the exercise.

113

114

- 8. Position the patient at the starting line. You should also stand near the starting line during the test. Do not walk with the patient. As soon as the patient starts to walk, start the timer.
- 9. Do not talk to anyone during the walk. Use an even tone of voice when using the standard phrases of encouragement. Watch the patient. Do not get distracted and lose count of the laps. Each time the participant returns to the starting line, click the lap counter once (or mark the lap on the worksheet). Let the participant see you do it. Exaggerate the click using body language, like using a stopwatch at a race.

After the first minute, tell the patient the following (in even tones): "You are doing well. You have 5 minutes to go.

When the timer shows 4 minutes remaining, tell the pa-tient the following: "Keep up the good work. You have 4 minutes to go."

When the timer shows 3 minutes remaining, tell the patient the following: "You are doing well. You are halfway

When the timer shows 2 minutes remaining, tell the patient the following: "Keep up the good work. You have only 2 minutes left."

When the timer shows only 1 minute remaining, tell the patient: "You are doing well. You have only I minute to

Do not use other words of encouragement (or body language to speed up).

If the patient stops walking during the test and needs a rest, say this: "You can lean against the wall if you would like; then continue walking whenever you feel able." Do not stop the timer. If the patient stops before the 6 minutes are up and refuses to continue (or you decide that they should not continue), wheel the chair over for the patient to sit on, discontinue the walk, and note on the worksheet the distance, the time stopped, and the reason for stopping prematurely

When the timer is 15 seconds from completion, say this:
"In a moment I'm going to tell you to stop. When I do, just stop right where you are and I will come to you."

When the timer rings (or buzzes), say this: "Stop!" Walk over to the patient. Consider taking the chair if they look exhausted. Mark the spot where they stopped by placing a bean bag or a piece of tape on the floor.

- Post-test: Record the postwalk Borg dyspnea and fatigue levels and ask this: "What, if anything, kept you from walking farther?"
- 11. If using a pulse oximeter, measure SpO2 and pulse rate from the oximeter and then remove the sensor
- 12. Record the number of laps from the counter (or tick marks on the worksheet).
- 13. Record the additional distance covered (the number of meters in the final partial lap) using the markers on the wall as dis-tance guides. Calculate the total distance walked, rounding to the nearest meter, and record it on the worksheet.
- 14. Congratulate the patient on good effort and offer a drink

### **OUALITY ASSURANCE**

### Sources of Variability

There are many sources of 6MWD variability (see Table 3) The sources of variability caused by the test procedure itself should be controlled as much as possible. This is done by fol-

lowing the standards found in this document and by using a quality-assurance program.

### **Practice Tests**

A practice test is not needed in most clinical settings but should be considered. If a practice test is done, wait for at least I hour before the second test and report the highest 6MWD as the patient's 6MWD baseline.

Rationale. The 6MWD is only slightly higher for a second 6MWT performed a day later. The mean reported increase ranges from 0 to 17% (23, 27, 40, 41, 54, 59). A multicenter study of 470 highly motivated patients with severe COPD performed two 6MWTs 1 day apart, and on average, the 6MWD was only 66 ft (5.8%) higher on the second day (54).

Performance (without an intervention) usually reaches a plateau after two tests done within a week (8, 60). The training effect may be due to improved coordination, finding optimal stride length, and overcoming anxiety. The possibility of a practice or training effect from tests repeated after more than a month has not been studied or reported; however, it is likely that the effect of training wears off (does not persist) after a

### Technician Training and Experience

Technicians who perform 6MWTs should be trained using the standard protocol and then supervised for several tests before performing them alone. They should also have completed cardiopulmonary resuscitation training.

Rationale. One multicenter study of older people found

that after correction for many other factors, two of the technicians had mean 6MWDs that were approximately 7% lower than the other two sites (31).

### Encouragement

Only the standardized phrases for encouragement (as speci-

fied previously here) must be used during the test.

Rationale. Encouragement significantly increases the distance walked (42). Reproducibility for tests with and without encouragement is similar. Some studies have used encouragement every 30 seconds, every minute, or every 2 minutes. We have chosen every minute and standard phrases. Some studies (53) have instructed patients to walk as fast as possible. Although larger mean 6MWDs may be obtained thereby, we recommend that such phrases not be used, as they emphasize ini-tial speed at the expense of earlier fatigue and possible excessive cardiac stress in some patients with heart disease.

# TABLE 3. 6MWD SOURCES OF VARIABILITY

Factors reducing the 6MWD

Older age

Higher body weight Female sex

Impaired cognition

impaired cognition
A shorter corridor (more turns)
Pulmonary disease (COPD, asthma, cystic fibrosis, interstitial lung disease)
Cardiovascular disease (angina, MI, CHF, stroke, TIA, PVD, AAI)
Musculosteletal disorders (arbitilis, anide, knee, or hip injuries, mascle weating, etc.)

Factors increasing the 6MWD Taller height (longer fogs)

Male sex High motivation

A patient who has previously performed the test

Medication for a disabiling disease taken just before the test. Oxygen supplementation in patients with exercise-induced hypoxemia

Dallation of abbreviations: COPD = chronic obstructive pulmonary disease; 6MWD = 6-minute waiting distance.

American Thoracic Society

# 115

### Supplemental Oxygen

If oxygen supplementation is needed during the walks and serial tests are planned (after an intervention other than oxygen therapy), then during all walks by that patient oxygen should be delivered in the same way with the same flow. If the flow must be increased during subsequent visits due to worsening gas exchange, this should be noted on the worksheet and considered during interpretation of the change noted in 6MWD. The type of oxygen delivery device should also be noted on the report: for instance, the patient carried liquid oxygen or pushed or pulled an oxygen tank, the delivery was pulsed or continuous, or a technician walked behind the patient with the oxygen source (not recommended). Measurements of pulse and SpO<sub>2</sub> should be made after waiting at least 10 minutes after any change in oxygen delivery.

ter any change in oxygen delivery.

Rationale. For patients with COPD or interstitial lung discase, oxygen supplementation increases the 6MWD (17, 59, 61, 63). Carrying a portable gas container (but not using it for supplemental oxygen) reduced the mean 6MWD by 14% in one study of patients with severe respiratory disability, but using the container to deliver supplemental oxygen during the exercise increased the mean 6MWD by 20-35% (59).

### Medications

The type of medication, dose, and number of hours taken before the test should be noted.

Rationale. Significant improvement in the distance walked, or the dyspnea scale, after administration of bronchodilators has been demonstrated in patients with COPD (62, 63), as well as cardiovascular medications in patients with heart failure (19).

### INTERPRETATION

Most 6MWTs will be done before and after intervention, and the primary question to be answered after both tests have been completed is whether the patient has experienced a clinically significant improvement. With a good quality-assurance program, with patients tested by the same technician, and after one or two practice tests, short-term reproducibility of the 6MWD is excellent (37). It is not known whether it is best for clinical purposes to express change in 6MWD as (1) an absolute value, (2) a percentage change, or (3) a change in the percentage of predicted value. Until further research is available, we recommend that change in 6MWD be expressed as an absolute value (e.g., the patient walked 50 m farther).

A statistically significant mean increase in 6MWD in a

A statistically significant mean increase in 6MWD in a group of study participants is often much less than a clinically significant increase in an individual patient. In one study of 112 patients (half of them women) with stable, severe COPD, the smallest difference in 6MWD that was associated with a noticeable clinical difference in the patients' perception of exercise performance was a mean of 54 m (95% confidence interval, 37-71 m) (64). This study suggests that for individual patients with COPD, an improvement of more than 70 m in the 6MWD after an intervention is necessary to be 95% confident that the improvement was significant. In an observational study of 45 older patients with heart failure, the smallest difference in 6MWD that was associated with a noticeable difference in their global rating of worsening was a mean of 43 m (20). The 6MWD was more responsive to deterioration than to improvement in heart failure symptoms.

### Reported Mean Changes in 6MWD After Interventions

Supplemental exygen (4 L/min) during exercise in patients with COPD or interstitial lung disease increased mean 6MWD by approximately 95 m (36%) in one study (59). Patients taking

an inhaled corticosteroid experienced a mean 33 m (8%) increase in 6MWD in an international COPD study (16). Patients with COPD in a study of the effects of exercise and diaphragmatic strength training experienced a mean increase in 6MWD of 50 m (20%) (65). Lung volume reduction surgery in patients with very severe COPD has been reported to increase 6MWD by a mean of 55 m (20%) (13).

Cardiac rehabilitation in patients referred with various heart diseases increased 6MWD by a mean of 170 m (15%) in a recent study (66). In 25 older patients with heart failure, an angiotensin-converting enzyme inhibitor medication (50 mg captopril per day) improved 6MWD a mean of 64 m (39%) compared with a mean increase of only 8% in those receiving a placebo (19).

### Interpreting Single Measurements of Functional Status

Optimal reference equations from healthy population-based samples using standardized 6MWT methods are not yet available. In one study, the median 6MWD was approximately 580 m for 117 healthy men and 500 m for 173 healthy women (50). A mean 6MWD of 630 m was reported by another study of 51 healthy dider adults (55). Differences in the population sampled, type and frequency of encouragement, corridor length, and number of practice tests may account for reported differences in mean 6MWD in healthy persons. Age, height, weight, and sex independently affect the 6MWD in healthy adults; therefore, these factors should be taken into consideration when interpreting the results of single measurements made to determine functional status. We encourage investigators to publish reference equations for healthy persons using the previously mentioned standardized procedures.

A low 6MWD is nonspecific and nondiagnostic. When the 6MWD is reduced, a thorough search for the cause of the impairment is warranted. The following tests may then be helpful: pulmonary function, cardiac function, ankle-arm index, muscle strength, nutritional status, orthopedic function, and cognitive function.

### Conclusions

The 6MWT is a useful measure of functional capacity targeted at people with at least moderately severe impairment. The test has been widely used for preoperative and postoperative evaluation and for measuring the response to therapeutic interventions for pulmonary and cardiac disease. These guidelines provide a standardized approach to performing the 6MWT. The committee hopes that these guidelines will encourage further research into the 6MWT and allow direct comparisons among different studies.

This statement was developed by the ATS Committee on Proficiency Standards for Clinical Pulmonary Function Laboratories.

Members of the committee are:

Members of the committee are:

ROINT O, CAMO, M.D., Chair\*

RICHIED CASALUR, PH.D., M.D.,

ALAN L. COLER, M.D.,

PAU, L. EWIELT, M.D.,

NE R. MECHATIR, M.D.,

ROY T, MCKAY, PH.D.,

DOUGLAS JOHNOON, M.D.,

AC S, WANARS, M.D.,

A HOC COmmittee members are:

VAN BITTHER, M.D.,

CAN MOTTHUR, R.T.T.

"Willing Committee Members

### References

 Wasserman K, Hansen JB, Sue DY, Casaburi R, Whipp BJ. Principles of exercise testing and interpretation, 3rd edition. Philadelphia: Lippincott, Williams & Wilkins; 1999.

- Weisman IM, Zeballoz RJ. An integrated approach to the interprotation of cardiopulmonnry exercise testing. Clin Chest Med 1994;15:421-445.
   Fletcher GF, Balady G, Frodelicher VF, Hartley LH, Haskell WL, Poliok ML. Exercise standards: a statement for healthcare professionals from the American Heart Association: writing group. Circulation 1995; 91:580-615.
- Pina IL, Balady GJ, Hanson P, Labovitz AJ, Medonna DW, Myers J. Gulde-lines for clinical exercise testing laboratories: a statement for healthcare professionals from the Committee on Exercise and Cardiac Rehabilita-tion, American Heart Association. Circulation 1995;91:912–921.
- 5. Balke B. A simple field test for the assessment of physical fitness. CARI Report 1963;63:18.
- Cooper KH. A means of assessing maximal oxygen intake: correlation between field and treadmill tosting. JAJAA 1968;203:201–204.
   McGavin CR, Gupta SP, McI ardy GJR. Twelve-minute walking test for assessing disability in chronic bronchitis. BAJ 1976;1:822–823.
- Bustand RJA, Pang J, Gross BR, Woodcock AA, Goddes DM. Two-six-, and 12-minute walking tests in respiratory disease. BMJ 1982; 284:1607-1608.
- Solway S, Brooks D, Lacasso Y, Thomas S. A qualitative systematic overview of the measurement properties of functional walk tests used
- in the cardiorespiratory donsain. Chest 2001;119:256-270.

  10. Kadikar A, Maurer J, Kesten S. The six-minute walk test: a guide sessment for lung transplantation. J Heart Lung Transplant 1997;16;
- 11. Holden DA, Rice TW, Stelmach K, Meeker DP. Exercise testing, 6 mi walk, and stair climb in the evaluation of patients at high risk for pul-
- walk, and stair climb in the evaluation of patients at high risk for pulmonary resection. Chest 1992;102:1774–1779.

  12. Sciurba FC, Rogers RM, Keenna RJ, Slivka WA, Goresan J 3rd, Ferson PF, Holbert JM, Brown ML, Landemena RJ. Improvement in pulmonary function and elastic recoil after lung-reduction surgery for differe emphysema. N Engl J Med 1996;334:1095–1059.

  13. Criner GJ, Cordova FC, Furukawa S, Kuzma AM, Travaline JM, Leyenson V, O'Brien GM. Prospective randomized trial comparing bilateral lung volume reduction surgery to pulmonary rehabilitation in severe COPD. Ann J Respir Crit Care Med 1999;160/2018–2027.

  14. Sinclair DJM, Ingazam CG. Controlled trial of supervised exercise training in chronic brouchitis. BMJ 1980;280:519–521.

  15. Roomi J, Johnson MM, Waters K, Yohannes A, Itelm A, Connolly MJ. Respiratory schabilitation, exercise capacity and quality of life in

- Roomi J, Johnson MM, Waters K, Yohannes A, Helm A, Connouly AH.
  Respiratory shabilitation, exercise capacity and quality of life in
  chronic nirways disease in old age. Age Ageing 1996;25:12-16.
   Paggino PL, Dahle R, Bakran I, Frith L, Hollingworth K, Etthimiou J,
  Multicentre randomised placebo-controlled trial of inhabed fluticasone propionate in patients with COPD. Lancet 1998;351:773-780.
   Leggett RJ, Frenley DC. Portable oxygen and exercise tolerance in patients with chronic hypoxic cor pulmonate. BMJ 1977;2:84-86.
   Spence DPS, Hay JG, Carter J, Pearson MG, Calverley PMA. Oxygen
- desaturation and breathlessness during corridor walking in COPD: effect of oxitroplum bromide. Thorax 1993;48:1145-1150.

  19. DeBock V, Mets T, Romsgnoll M, Derde MP, Captopril treatment of
- chronic heart finiture in the very old. J Gerantal 1994;49:M148-M152.

  20. O'Keeffe ST, Lye M, Donnnellan C, Carmichael DN. Reproducibilit and responsiveness of quality of life assessment and six minute with test in elderly heart failure patients. Heart 1998;80:377-382. 21. Bernstein ML, Despars JA, Singh NP, Avalos K, Sinnsbury DW, Light
- R.W. Re-analysis of the 12 minute walk in patients with COPD. Chen 1994;105:163–167.
- 22. Hajiro T, Nishimura K, Tsukino M, Ikeda A, Koyama H, Izumi T. Analysis of clinical methods used to evaluate dyspines in patients with COPD. Am J Respir Crit Care Med 1998;158:1185-1189.

  23. Gulmans VAM, vanVeldhoven NHMJ, dchleer K, Helders PJM. The
- six-minute walking test in children with cystle fibrosis: reliability and validity. Pediatr Pulmonol 1995;22:85-89.
- 24. Nixon PA, Joswiak ML, Fricker PJ, A six-minute walk test for assessing exercise tolerance in severely ill children. J Pediatr 1996;129:362-366.

  25. Bittner V. Six-minute walk test in patients with cardiac dysfunction. Cartille Management of the patients of the cardiac dysfunction. Cartille Management of the patients with cardiac dysfunction.
- diologia 1997;42:897-902.

  26. Pectors P, Mots T. The 6 minute walk as an appropriate exercise test in elderly patients with chronic heart failure. J Gerontol 1996;51A:
- M147-M151.

  27. Zugck C, Kruger C, Durr S, Gerber SH, Haunstetter A, Hornig K, Kubler W, Hanss M. Is the 6-minute welk test a reliable substitute for the department of the configuration of the details of the configuration. peak oxygon uptake in patients with dilated cardiomyopathy? Eur Heart J 2000;21:540-549.
- Montogomery PS, Gardner AW. The clinical utility of a six-minute walk test in peripheral arterial occlusive disease patients. J Am Geriatr Soc 1998;46:706-711.

- 29. Cahan MA, Montgomery P, Otis RB, Clancy R, Flinn W, Gardner A.
- Canan MA, Boongomery F, Ous Rds, Cannoy R, Fanni W, Ostonier The effect of cigarents smoking status on six-minute walk distance in patients with intermittent claudication. Anglology 1999;90:537–546.
   King S, Wessel J, Bhambhani Y, Maikala R, Sholter D, Maksymowych W, Valldiya and reliability of the 6 minute walk in persons with fibromyalgia. J Rhennatol 1999;26:2233–2237.
- mynlgia. J. Rhenuntof 1999;26:2233-2237.

  I. Enright PL, McBurale MA, Bittner V, Tracy RP, McNamara R, Newman AB, the Cardiovascular Health Study. The six minute walk test: a quick measure of functional status in elderly adults. Chest (in press)

  32. Bittner V, Weiner DH, Yusuf S, Rogers WJ, Mohryer KM, Bangdiwala SI, Kronenberg MW, Kostis JB, Kohn RM, Guillotte M, et al. Prediction of metablish and morbidity with 5. Sanipulse walk test in patients.
- tion of mortality and morbidity with a 6-minute walk test in patients with left ventricular dysfunction. JAMA 1993;270:1702-1707.

  33. Cahalla LP, Mathier MA, Semigran MJ, Dec GW, DiSalvo TG. The six-
- ntinute walk tost predicts peak oxygen uptake and survival in patients with advanced heart failure. Chest 1996;110:325-332.
- with envanced near inture. Crest 1590g110535-353.

  Cote CG, Celli BR. In patients with COPD, the distinct walking distance is a better predictor of health care utilization than FEV1, blood gases, and dyspine [abstract]. Eur Respir J 1986;383.

  Kessler R, Paller M, Fourgaut G, Mennecler B, Weltzenblum E. Predictive factors of hospitalization for acute exacerbation in a series of 64 patients with chronic obstructive pulmonary disease. Am J Respir Crit Care Med 1990;550; 52:154 Care Med 1999;159:158-164.
- Cahalin L, Pappagianopoulos P, Prevost S, Wain J, Ginns L. The relation ship of the 6-min welk test to nextmal oxygen consumption in trans
- ship of the 6-min welk test to maximal oxygen consumption an transplant candidates with end-stage lung disease. Chest 1995;108:432-459.

  37. Guyatt GH, Thompson PJ, Berman LB, Sullivan MJ, Townsend M, Jones NL, Pagsloy SO. How should we measure function in patients with chronic heart and lung disease? J Chronic Dis 1985;58:317-524.

  38. Guyatt GH, Townsend M, Keller J, Singer J, Nogradi S. Measuring func-
- tional status in chronic lung disease; conclusions from a random control trial. *Kespir Med* 1991;85(Suppl B):17-21.

  39. Niederman MS, Clemento PH, Fein AM, Feinsilver SH, Robinson DA,
- Howite JS, Bernstein MG. Benefits of a multidisciplinary pulmonary rehabilitation program: improvements are independent of lung func-tion. Chest 1991;99:798–804.

- Noseda A, Carpianu J, Prigogine T, Schmerber J. Lung function, maximum and submaximum exercise testing in COPD patients: reproducibility over a long interval. Lung 1989;167:247–257.
   Knox AJ, Morrison JF, Muers MF. Reproducibility of walking test results in chronic obstructive airways disease. Thorax 1988;43:383–392.
   Guyatt GH, Pugsley SO, Sullivan MJ, Thompson PJ, Berman LB, Jones NL, Fellen BL, Taylor DW. Effect of encouragement on walking test responses. Thorax 1984:39:318–322.

- NL, Falten EL, Taylor DW. Effect of encouragement on walking test performance. Thorax 1984;9:818-822.

  43. Leger LA. A maximal multistage 20-m shuttle run test to predict VO2 max. Eur J Appl Physiol 1982;49:1-12.

  44. Singh SJ, Morgan MDL, Scott S, Walters D, Hardman AE. Development of a shuttle walking test of disability in patients with chronic shrways obstruction. Thorax 1992;47:1019-1024.

  45. Revill SM, Morgan MDL, Singh SJ, Williams J, Hardman AE. The endurance shuttle walk: a new field test for the assessment of endurance capacity in chronic obstructive pulmonary disease. Thorax 1995;42:13-222.

  46. Singh SJ, Morgan MDL, Hardman AE, Rowe C, Bardsley PA. Comparison of oxygen uptake during a conventional treadmill test and the shuttle walking test in chronic airflow limitation. Eur Respir J 1994;7: 2016-2020. 2016-2020.
- Morales FF, Martinez A, Mendez M, Agnrrado A, Ortege F, Fernandez-Guerra J, Montemayor T, Burgos J. A shuttle walk test for assessment of functional capacity in chronic heart failure. Am Heart J 1999;138:292-298.
   Enright PL, Sherrill DL. Reference equations for the six-minute walk in healthy adults. Am J Respir Crit Care Med 1998;158:1384-1387.
   Barst RJ, Rubin LJ, McGoon MD, Caldwell EJ, Long WA, Levy PS.
- Surviva) in primary pulmonary hypertension with long-term cor-ous intravenous prostacyclin. Ann Intern Med 1994;121:409-415.
- Miyamoto S, Nagaya N, Satoh T, Kyotani S, Sakamaki F, Fujita M, Na-kanishi N, Miyatake K. Clinical correlates and prognostic aignificance of six-minute walk test in patients with primary pulmonary hyperten-
- sion. Am J Respir Crit Core Med 2000;161:487-492.

  51. Guyatt GH, Sullivan MJ, Thompson PJ, Fallen EL, Pugsley SO, Taylor DW, Bermen LB. The 6-minute walk: a new measure of exercise caocity in patients with chronic heart failure. Can Med Assac J 1985;
- 52. Lipkin DP, Scrivin AJ, Crake T, Poole-Wilson PA. Six minute walking test for assessing exercise capacity in chronic heart failure. BMJ 1986; 292:653-655.
- Troosters T, Gosselink R, Decramer M. Six minute walking distance in healthy elderly subjects. Eur Respir J 1999;14:270-274.

American Thoracic Society

117

- 54. Weiss RA, et al. Six minute walk test in severe COPD: reliability and effect of walking course layout and length. Paper presented at ACCP Conference; September 2000; Sun Francisco.

  55. Stevens D, Elpern E, Sharma K, Szidon P, Ankin M, Kesten S. Compar-
- Ison of hallway and treadmill sik-minute walk tests. Am J Respir Crit Care Med 1999;160:1540-1543.

  56. Jensen LA, Onyskiw PR. Prasnd NGN. Meta-analysis of arterial oxygen saturation monitoring by pulse oximetry in adults. Heart Lung 1998; 27:197-Los
- saturation monitoring by pulse oximetry in adults. Heart Lung 1998; 27:387-408.

  57. Barthelemy JC, Geyssant A, Riffat J, Antoniadis A, Berruyer J, La Cour JR. Accuracy of pulse oximetry during moderate exercise: a comparative study. Scand J Clin Lab Invest 1990;50:533-539.

  58. Borg GAV. Psycho-physical bases of perceived exertion. Med Scl Sports Exerc 1982;14:377-381.

  59. Leach RM, Davidson AC, Chinn S, Twort CHC, Cameron IR, Battemen NT. Portable liquid oxygen and exercise ability in source registeries.
- Losch Kel, Davidson AC, Chinn S, Twort CHC, Cameron IR, Batemon NT. Portable liquid oxygen and exercise ability in severe respiratory disability. Thorax 1992;47:781–789.
   Mungall IPF, Hainsworth R. Assessment of respiratory function in patients with chronic obstructive sirvays disease. Thorax 1979;34:254–258.
   Roberts CM, Bell J. Wedzichn JA. Comparison of the efficacy of a de-

- mand oxygen delivery system with continuous low flow oxygen in subjects with stable COPD and severe oxygen desaturation on walking. Thorax 1996;51:831-834.

  62. Hay JG, Stone P, Carter J, Church S, Eyre-Brook A, Pearson MG, Woodcock AA, Calverley PM. Bronchodilator reversibility, exercise performance and breathlessness in stable chronic obstructive pulmonary disease. Eur Respir J 1992;5:659-664.

  63. Grove A, Lipworth BJ, Reid P, Smith RP, Lanage L, Ingram CG, Jenkins RI, Winter JH, Dhillon DP. Effects of regular salmetered on lung function and exercise capacity in patients with COPD. Thorax 1996;51:689-693.

  64. Redelmeier DA, Bayoumi AM, Goldstein RS, Guyatt GH. Interpreting small differences in functional status: The six minute walk test in chronic lung disease patients. Ann J Respir Crit Care Med 1997;155:1278-1282.

  65. Weiner P, Magadle R, Berer-Yannay N, Davidovich A, Weiner M. The oumulative effect of long-acting bronchodilators, exercise, and inspiratory muscle training on the perception of dyspine in patients with advanced COPD. Client 2006;118:672-678.

  66. Bittner V, Sanderson B, Breland J, Adams C, Schuman C. Assessing functional capacity as an outcome in cardiac rehabilitation: role of the 6 minute walk test. Clinical Exercise Physiology 2000.

### APPENDIX

| The following | elements sho | uld be prese | nt on the 6h | WT W | orkshee | and report |
|---|---|---|---|---|---|---|
| Lap counter: | | | | - | 1000 | |
| Patient name: | | | Patient | ID#_ | · | |
| Walk # | Tech ID | : | Date: | | | |
| Gender: M F | Age: | Race: | Height: _ | _ft | _in, | meters |
| Weight: | lbs,k | g Bloo | od pressure: | / | | |
| Medications ta | ken before th | ne test (dose | and time): | 172 | | |
| Supplemental | oxygen durin | g the test: N | lo Yes, flo | w | _L/mii | n, type |
| | | Baseline | | End of | Test | |
| | Time | _:_ | | _:_ | _ | |
| | Heart Rate | | | _ | | |
| | Dyspnea | nemani. | | ( | Borg sca | le) |
| | Fatigue | | | () | Borg sca | ie) |
| | SpO <sub>2</sub> | % | | % | | |
| Stopped or pau | sed before 6 | minutes? N | o Yes, rea | son; _ | | |
| Other sympton | ns at end of e | xercise: ang | ina dizzine | ss hip | , leg, or | calf pain |
| Number of laps | :(×60) | meters) + fir | nal partial fo | p: | meters | = |
| Total distance v | walked in 6 n | inutes: | meters | | | |
| Predicted distar | nce: m | eters Per | rcent predict | ed: | _% | |
| Tech comments | s: | | | | | |
| Interpretatio | on (including | comparison | with a prein | tervent | ion 6M | WD): |
# Appendix F Frailty Index

The assessment should be administered by either an investigator or research coordinator. The study patient will first be given a series of questions related to their ability to perform activities of daily living and scored accordingly on their responses. The second portion of the assessment involves a series of three hand grip strength tests which are averaged. Study patients will then be given a score for frailty based on their average score. Finally, study patients will be asked to walk 5 meters. Based on the overall assessment, a score will be given for frailty.

#### **FRAILTY INDEX DATA**

| 1. Was Frailty Index Obtained? Yes No No |
|------------------------------------------|
| 2. Date Completed:/ |
| 3. Height (cm/in) |
| <b>4. Weight</b> (kg/lb) |
| 5. BMI |
| 6. Serum Albumin:g/dL |
| 7. Time (lab):: (24 Hr) |

# **Katz Activities of Daily Living**

| ACTIVITIES | INDEPENDENCE: | DEPENDENCE: |
|---|---|---|
| POINTS (1 OR 0) | (1 POINT) | (0 POINTS) |
| | NO supervision, direction or | WITH supervision, direction, |
| | personal assistance | personal assistance or total care |
| | (1 POINT) Bathes self completely or | (0 POINTS) Needs help with bathing |
| BATHING | needs help in bathing only a single | more than one part of the body, |
| POINTS: | part of the body such as the back, | getting in or out of the tub or |

| | genital area or disabled extremity. | shower. |
|---|---|---|
| | | Requires total bathing. |
| | (1 POINT) Gets clothes from closets | (0 POINTS) Needs help with |
| DRESSING | and drawers and puts on clothes | dressing self or needs to be |
| POINTS: | and outer garments complete with | completely dressed. |
| | fasteners. May have help tying | |
| | shoes. | |
| | (1 POINT) Goes to toilet, gets on and | (0 POINTS) Needs help transferring |
| TOILETING | off, arranges clothes, cleans genital | to the toilet, cleaning self or uses |
| POINTS: | area without help. | bedpan or commode. |
| | (1 POINT) Moves in and out of bed | (0 POINTS) Needs help in moving |
| TRANSFERRING | or chair unassisted. Mechanical | from bed to chair or requires a |
| POINTS: | transferring aides are acceptable. | complete transfer. |
| | (1 POINT) Exercises complete self | (0 POINTS) Is partially or totally |
| CONTINENCE | control over urination and | incontinent of bowel or bladder. |
| POINTS: | defecation. | |
| | (1 POINT) Gets food from plate into | (0 POINTS) Needs partial or total |
| FEEDING | mouth without help. Preparation of | help with feeding or requires |
| POINTS: | food may be done by another | parenteral feeding. |
| | person. | |
| TOTAL POINTS = | | |
| | 1 | <u> </u> |

| Grip S | Strength |
|--------|----------|
|--------|----------|

Note to the Examiner: Elbow should be at a 90 degree angle, with arm not resting on table or "pinned" against chest wall.

All tests should be completed with the dynamometer in the dominant hand.

\_\_\_\_\_ Grasp 1
\_\_\_\_\_ Grasp 2
\_\_\_\_\_ Grasp 3

\_\_\_\_\_ Average

Men Cutoff for grip strength (Kg) criterion for frailty

BMI  $\leq$  24 $\leq$  29BMI 24.1-26 $\leq$  30BMI 26.1-28 $\leq$  30BMI > 28 $\leq$  32

Women Cutoff for grip strength (Kg) criterion for frailty

BMI  $\leq 23$  $\leq 17$ BMI 23.1-26 $\leq 17.3$ BMI 26.1-29 $\leq 18$ BMI > 29 $\leq 21$ 

.....

# 5-Meter Walk \_\_\_\_\_ Seconds

Men Cutoff Time to walk 5 meters criterion for frailty

Height  $\leq$  173 cm  $\geq$  7 seconds Height > 173 cm  $\geq$  6 seconds

Women

Height  $\leq$  159 cm  $\geq$  7 seconds Height > 159 cm  $\geq$  6 seconds

# Appendix G Mini Mental State Examination (MMSE)

| | Date of Exa | mination/_/ | | Years of | |
|---|---|---|---|---|---|
| | Name | | Age | School Completed_ | |
| appear in pare | entheses. Administ | ration should be conducted | clearly and slowly to the ex<br>d privately and in the exami<br>correct. Begin by asking the | nee's primary languag | ge. |
| Do you ha | ave any trouble w | th your memory? | May I ask you some question | ons about your mem | ory? |
| ORIENTATIO | N TO TIME | | RESPONSE | | ORE |
| What is the | year? | _ | | 0 | 1 |
| | season? | _ | | 0 | 1 |
| | month of the ye | ar? | | 0 | 1 |
| | day of the week | | | 0 | 1 |
| | date? | - | 1000000 | 0 | 1 |
| ORIENTATIO | N TO PLACE* | | | | |
| Where are we | now? What is the. | | | | |
| | state (province)? | - | | | 1 |
| | county (or city/to | | | 0 | 1 |
| | city/town (or par | rt of city/neighborhood)? | | 0 | 1 |
| | building (name | or type)? | | 0 | 1 |
| | floor of the build<br>(room number or | - | | 0 | 1 |
| *Alternative place | A 100 C 100 C | | gly precise may be substituted an | noted. | |
| REGISTRATIO | ON* | | | | |
| | | av three words. You say | them back after I stop. Re | adv? | |
| Here they are | . APPLE (pause). I | PENNY (pause), TABLE (pa | use]. Now repeat those wor | ds back to me. | |
| | times, but score or | | | | |
| | APPLE | _ | | 0 | 1 |
| | PENNY | | | 0 | |
| | PENNY | _ | | | 1 |
| | TABLE | _ | | 0 | 1 |
| | TABLE<br>se words in mind. | | ay them again in a few min | utes. | |
| | TABLE<br>se words in mind. | | ay them again in a few min | utes. | |
| *Alternative word | TABLE<br>se words in mind.<br>sets (e.g., PONY, QUA | | | utes. | |
| *Alternative word ATTENTION | TABLE se words in mind. sets (e.g., PONY, QUA AND CALCULA | ARTER, ORANGE) may be substit<br>TION [Serial 7s]* | | utes. examinee. | |
| *Alternative word ATTENTION | TABLE se words in mind. sets (e.g., PONY, QUA AND CALCULA u to subtract 7 fro | ARTER, ORANGE) may be substit<br>TION [Serial 7s]* | tuted and noted when retesting an | utes. examinee. | |
| *Alternative word<br>ATTENTION<br>Now I'd like yo | TABLE se words in mind. sets (e.g., PONY, QUA AND CALCULA u to subtract 7 fro ke away 7? | ARTER, ORANGE) may be substituted to the substitute of the substit | tuted and noted when retesting an | utes. examince. till I tell you to stop. | 1 |
| *Alternative word<br>ATTENTION<br>Now I'd like yo<br>What is 100 tal | TABLE se words in mind. sets (e.g., PONY, QUA AND CALCULA u to subtract 7 fro ke away 7? Keep going. | ARTER, ORANGE) may be substitution [Serial 7s]* om 100. Then keep subtrac [93] | ting 7 from each answer ur | utes. examince. till I tell you to stop. | 1 |
| *Alternative word<br>ATTENTION<br>Now I'd like yo<br>What is 100 tal<br>If needed, say: | TABLE se words in mind. sets (c.g., PONY, QUA AND CALCULA u to subtract 7 fro ke away 7? Keep going. Keep going. | ARTER, ORANGE) may be substituted in the substitute of the substit | ting 7 from each answer ur | utes. examince. till I tell you to stop. 0 | 1 1 1 |
| *Alternative word<br>ATTENTION<br>Now I'd like yo<br>What is 100 tal<br>If needed, say:<br>If needed, say:<br>If needed, say: | TABLE se words in mind. sets (e.g., PONY, QUA AND CALCULA u to subtract 7 fro ke away 7? Keep going. Keep going. Keep going. | ARTER, ORANGE) may be substituted in the substitute of the substit | ting 7 from each answer ur | utes. examince. til I tell you to stop. 0 0 0 | 1 1 1 |
| *Alternative word<br>ATTENTION<br>Now I'd like yo<br>What is 100 tal<br>If needed, say:<br>If needed, say:<br>If needed, say:<br>If needed, say: | TABLE se words in mind. sets (e.g., PONY, QUA AND CALCULA u to subtract 7 fro ke away 7? Keep going. Keep going. Keep going. Keep going. Keep going. | ARTER, ORANGE) may be substituted in the substitute of the substit | tuted and noted when retesting an | utes. examince. till I tell you to stop. 0 0 0 0 0 | 1 1 1 1 |
| *Alternative word<br>ATTENTION<br>Now I'd like yo<br>What is 100 tal<br>If needed, say:<br>If needed, say:<br>If needed, say:<br>If needed, say: | TABLE se words in mind. sets (e.g., PONY, QUA AND CALCULA u to subtract 7 fro ke away 7? Keep going. Keep going. Keep going. Keep going. Keep going. | ARTER, ORANGE) may be substituted in the substitute of the substit | ting 7 from each answer ur | utes. examince. till I tell you to stop. 0 0 0 0 0 | 1 1 1 1 |
| *Alternative word<br>ATTENTION<br>Now I'd like yo<br>What is 100 tal<br>If needed, say:<br>If needed, say:<br>If needed, say:<br>If needed, say: | TABLE se words in mind. sets (e.g., PONY, QUA AND CALCULA u to subtract 7 fro ke away 7? Keep going. Keep going. Keep going. Keep going. Keep going. | ARTER, ORANGE) may be substituted in the substitute of the substit | tuted and noted when retesting an | utes. examince. till I tell you to stop. 0 0 0 0 0 | 1 1 1 1 |

MMSE Copyright © 1975, 1998, 2001 by MiniMental, LLC. All rights reserved. Published 2001 by PAR. May not be reproduced in whole or in part in any form or by any means without written permission of PAR. This form is printed in red and blue ink on white paper. Any other version is unauthorized.

9 8 7 Reorder #RO-4740 Printed in the U.S.A.

WARNING! PHOTOCOPYING OR DUPLICATION OF THIS FORM WITHOUT PERMISSION IS A VIOLATION OF COPYRIGHT LAWS.

| Substitute and score this item only if the examinee refuses to pe<br>Spell WORLD forward, then backward.<br>Correct forward spelling if misspelled,<br>but score only the backward spelling. | erform the | e Serial 7 | s task. | | | | |
|---|---|---|---|---|---|---|---|
| | (D = 1) | (L = 1) | (R=1) | (O = 1) | $(W \approx 1)$ | (0 | to 5) |
| RECALL | | R | ESPON: | SE | | | ORE |
| What were those three words I asked you to remember? | ? [Do not | offer any | hints. | | | Center | e ane) |
| APPLE | - | | | | | 0 | 1 |
| PENNY | | | | | | 0 | 1 |
| TABLE | | | | | | 0 | 1 |
| NAMING* | | 8 | | | | | |
| What is this? [Point to a pencil or pen.] | | - 33 | | | | 0 | 1 |
| What is this? [Point to a watch.] | | | | V-121-101111 | | 0 | 1 |
| *Alternative common objects (e.g., eyeglasses, chair, keys) may be sub | bstituted an | d noted. | | | | | |
| REPETITION | | | | | | | |
| Now I am going to ask you to repeat what I say. Ready? [Repeat up to 5 times, but score only the first trial.] | "NO IFS | , ANDS, | OR BUT | S." Now | you say th | at. | |
| NO IFS, ANDS, OR BUTS. | | | | | | 0 | 1 |
| COMPREHENSION Listen carefully because I am going to ask you to do so Take this paper in your right hand [pause], fold it in half | mething<br>[pause], | and put | it on the | e floor (d | or table). | | |
| TAKE IN RIGHT HAND | <u> </u> | | | | | 0 | 1 |
| FOLD IN HALF | | | | | | 0 | 1 |
| PUT ON FLOOR (or TABLE) | | | | | - | 0 | 1 |
| READING | | | | | | | |
| Please read this and do what it says. [Show examinee to | the words | on the s | timulus i | form.] | | | |
| CLOSE YOUR EYES | | | | | | 0 | 1 |
| WRITING | | | | | | | |
| Please write a sentence. [If examinee does not respond, Place the blank piece of paper (unfolded) in front of the examinethe sentence is comprehensible and contains a subject and a vertex. | nee and pr | rovide a p | en or per | ncil. Scor | e 1 point if<br>ing. | 0 | 1 |
| DRAWING | | | * | | | | |
| Please copy this design. [Display the intersecting pentage Score 1 point if the drawing consists of two 5-sided figures that in | | | | | | 0 | 1 |
| | | | | | | | - |
| Assessment of level of consciousness. | | | | 100 | Score =<br> l item scores.) | (30 pois | nts max.) |
| | natose/ | | | | | | |

# **CLOSE YOUR EYES**



# Appendix H NIH Stroke Scale (NIHSS)

| <u> </u> | 1 | | I | ŀ | 1 |
|----------|---|---|----|---|---|
| S | T | F | ₹C | K | E |
| S | ( | _ | A | L | E |

| Date of Exam:// | |
|-------------------------|------------------------|
| Print Name of Examiner: | Signature of Examiner: |

Administer stroke scale items in the order listed. Record performance in each category after each subscale exam. Do not go back and change scores. Follow directions provided for each exam technique. Scores should reflect what the patient does, not what the clinician thinks the patient can do. The clinician should record answers while administering the exam and work quickly. Except where indicated, the patient should not be coached (i.e., repeated requests to patient to make a special effort).

#### NOTE: Only a NIHSS certified team member may administer the test.

If there is an increase from the baseline stroke scale score, or evidence of a suspected stroke or TIA, capture the increase as an adverse neurological event and document the reason for the score increase. Administer the NIH Stroke Scale 30 days and 60 days after any neurological adverse event.

| Instructions | Scale Definitions | Score |
|---|---|---|
| Level of Coneclousness: The Investigator must choose a response if a full evaluation is prevented by such obstacles as an endotracheal tube, language barrier, orotracheal trauma/bandages. A 3 score is scored only if the patient makes no movement (other than reflexive posturing) in response to noxious stimulation. | O = Alert; keenly responsive. 1 = Not aiert; but arousable by minor stimulation to obey, answer, or respond. 2 = Not aiert; requires repeated stimulation to attend, or is obtunded and requires strong or painful stimulation to make movements (not stereotyped). 3 = Responds only with reflex motor or autonomic effects or totally unresponsive, flaccid, and flexic. | |
| 1b. LOC Questions: The patient is asked the month and his/her age. The answer must be correct – there is no partial credit for being close. Aphasic and stuporous patients who do not comprehend the questions will score 2. Patients unable to speak because of endotracheal intubation, cortracheal trauma, severe dysarthria from any cause, language barrier, or any other problem not secondary to aphasia are given a 1. It is important that only the initial answer be graded and that the examiner not "help" the patient with verbal or non-verbal cues. | Answers both questions correctly. Answers one question correctly. Answers neither question correctly. | |
| 1c. LOC Commands: The patient is asked to open and close the eyes and then to grip and release the non-paretic hand. Substitute another one step command if the hands cannot be used. Credit is given if an unequivocal attempt is made but not completed due to weakness. If the patient does not respond to command, the task should be demonstrated to him or her (pantomime), and the result scored (i.e., follows none, one or two commands). Patients with trauma, amputation, or other physical impediments should be given suitable one-step commands. Only the first attempt is scored. | Performs both tasks correctly. Performs one task correctly. Performs neither task correctly. | |
| Beef Gaze: Only horizontal eye movements will be tested. Voluntary or reflexive (oculocephalic) eye movements will be scored, but caloric testing is not done. If the patient has a conjugate deviation of the eyes that can be overcome by voluntary or reflexive activity, the score will be 1. If a patient has an isolated peripheral nerve paresis (CN III, IV or VI), score a 1. Gaze is testable in all aphasic patients. Patients with ocular trauma, bandages, pre-existing blindness, or other disorder of visual aculty or fields should be tested with reflexive movements, and a choice made by the investigator. Establishing eye contact and then moving about the patient from side to side will occasionally clarify the presence of a partial gaze palsy. | Normal. Partial gaze palsy; gaze is abnormal in one or both eyes, but forced deviation or total gaze paresis is not present. Forced deviation, or total gaze paresis not overcome by the oculocephalic maneuver. | |



| Instructions | Scale Definitions | Score |
|---|---|---|
| 3. Visual: Visual fields (upper and lower quadrants) are tested by confrontation, using finger counting or visual threat, as appropriate. Patients may be encouraged, but if they look at the side of the moving fingers appropriately, this can be scored as normal. If there is unilateral bilindness or enucleation, visual fields in the remaining eye are scored. Score 1 only if a clear-cut asymmetry, including quadrantanopta, is found. If patient is bilind from any cause, score 3. Double simultaneous stimulation is performed at this point. If there is extinction, patient receives a 1, and the results are used to respond to item 11. | 0 = No visual loss. 1 = Partial hemianopia. 2 = Complete hemianopia. 3 = Bilateral hemianopia (blind including cortical blindness). | _ |
| 4. Facial Palsy: Ask – or use pantomime to encourage – the patient to show teeth or raise eyebrows and close eyes. Score symmetry of grimace in response to noxious stimuli in the poorty responsive or non-comprehending patient. If facial trauma/bandages, orotracheal tube, tape or other physical barriers obscure the face, these should be removed to the extent possible. | Normal symmetrical movements. Minor paralysis (flattened nasolablal fold, asymmetry on smiling). Partial paralysis (total or near-total paralysis of lower face). Complete paralysis of one or both sides (absence of facial movement in the upper and lower face). | _ |
| Motor Arm: The limb is placed in the appropriate position: extend the arms (palms down) 90 degrees (if sitting) or 45 degrees (if supine). Drift is scored if the arm falls before 10 seconds. The aphasic patient is encouraged using urgency in the voice and pantomime, but not noxious stimulation. Each limb is tested in turn, beginning with the non-paretic arm. Only in the case of amputation or joint fusion at the shoulder, the examiner should record the score as untestable (UN), and clearly write the explanation for this choice. | O = No drift; limb holds 90 (or 45) degrees for full 10 seconds. 1 = Drift; limb holds 90 (or 45) degrees, but drifts down before full 10 seconds; does not hit bed or other support. 2 = Some effort against gravity; limb cannot get to or maintain (if cued) 90 (or 45) degrees, drifts down to bed, but has some effort against gravity. 3 = No effort against gravity; limb falls. 4 = No movement. UN = Amputation or joint fusion, explain: 5a. Left Arm 5b. Right Arm | _ |
| 6. Motor Leg: The limb is placed in the appropriate position: hold the leg at 30 degrees (always tested suplne). Drift is scored if the leg falls before 5 seconds. The aphasic patient is encouraged using urgency in the voice and pantomime, but not noxious stimulation. Each limb is tested in turn, beginning with the non-paretic leg. Only in the case of amputation or joint fusion at the hip, the examiner should record the store as untestable (UN), and clearly write the explanation for this choice. | 0 = No drift; leg holds 30-degree position for full 5 seconds. 1 = Drift; leg falls by the end of the 5-second period but does not hit bed. 2 = Some effort against gravity; leg falls to bed by 5 seconds, but has some effort against gravity. 3 = No effort against gravity; leg falls to bed immediately. 4 = No movement. UN = Amputation or joint fusion, explain: 6a. Left Leg 6b. Right Leg | |
| 7. Limb Ataxia: This Item is almed at finding evidence of a unilateral cerebellar lesion. Test with eyes open. In case of visual defect, ensure testing is done in intact visual field. The finger-nose-finger and heel-shin tests are performed on both sides, and ataxia is scored only if present out of proportion to weakness. Ataxia is absent in the patient who cannot understand or is paralyzed. Only in the case of amputation or joint fusion, the examiner should record the score as untestable (UN), and clearly write the explanation for this choice. In case of blindness, test by having the patient touch nose from extended arm position. | 0 = Absent. 1 = Present in one limb. 2 = Present in two limbs. UN = Amputation or joint fusion, explain: | |



Score Instructions Scale Definitions Sensory: Sensation or grimace to pinprick when tested, or withdrawal from noxious stimulus in the obtunded or aphasic Normal; no sensory loss. Mild-to-moderate sensory loss; patient feels pinprick is less sharp or is dull on the affected side; or there is a loss of patient. Only sensory loss attributed to stroke is scored as abnormal and the examiner should test as many body areas (arms superficial pain with pinprick, but patient is aware of being (not hands), legs, trunk, face) as needed to accurately check for hemisensory loss. A score of 2, "severe or total sensory loss," touched should only be given when a severe or total loss of sensation can Severe to total sensory loss; patient is not aware of being touched in the face, arm, and leg. be clearly demonstrated. Stuporous and aphasic patients will, therefore, probably score 1 or 0. The patient with brainstem stroke who has bilateral loss of sensation is scored 2. If the patient does not respond and is quadriplegic, score 2. Patients in a come (Item 1a=3) are automatically given a 2 on this item. Beet Language: A great deal of information about comprehension will be obtained during the preceding sections of No aphasia; normal. the examination. For this scale item, the patient is asked to Mild-to-moderate aphasia; some obvious loss of fluency or facility of comprehension, without significant limitation on describe what is happening in the attached picture, to name items ideas expressed or form of expression. Reduction of on the attached naming sheet and to read from the attached list of speech and/or comprehension, however, makes sentences. Comprehension is judged from responses here, as well conversation about provided materials difficult or as to all of the commands in the preceding general neurological impossible. For example, in conversation about provided exam. If visual loss interferes with the tests, ask the patient to identify objects placed in the hand, repeat, and produce speech. materials, examiner can identify picture or naming card content from patient's response. The intubated patient should be asked to write. The patient in a coma (Item 1a-3) will automatically score 3 on this Item. The examiner must choose a score for the patient with stupor or limited Severe aphasia; all communication is through fragmentary expression; great need for inference, questioning, and guessing by the listener. Range of information that can be cooperation, but a score of 3 should be used only if the patient is mute and follows no one-step commands. exchanged is limited; listener carries burden of communication. Examiner cannot identify materials provided from patient response. Mute, global aphasia; no usable speech or auditory comprehension. Dysarthria: If patient is thought to be normal, an adequate n = Normal sample of speech must be obtained by asking patient to read or Mild-to-moderate dysarthria; patient siurs at least some repeat words from the attached list. If the patient has severe words and, at worst, can be understood with some difficulty. aphasia, the clarity of articulation of spontaneous speech can be rated. Only if the patient is intubated or has other physical barriers Severe dysarthria; patient's speech is so siurred as to be to producing speech, the examiner should record the score as unintelligible in the absence of or out of proportion to any untestable (UN), and clearly write an explanation for this choice. dysphasia, or is mute/anarthric. Do not tell the patient why he or she is being tested. intubated or other physical barrier, UN = explain: Extinction and inattention (formerly Neglect): Sufficient No abnormality. information to identify neglect may be obtained during the prior Visual, tactile, auditory, spatial, or personal inattention or testing. If the patient has a severe visual loss preventing visual extinction to bilateral simultaneous stimulation in one of the double simultaneous stimulation, and the cutaneous stimuli are sensory modalities. normal, the score is normal. If the patient has aphasia but does appear to attend to both sides, the score is normal. The presence Profound hemi-inattention or extinction to more than one of visual spatial neglect or anosagnosia may also be taken as modality; does not recognize own hand or orients to only evidence of abnormality. Since the abnormality is scored only if present, the item is never untestable. one side of space.



You know how.

Down to earth.

I got home from work.

Near the table in the dining room.

They heard him speak on the radio last night.



# **MAMA**

TIP - TOP

FIFTY - FIFTY

**THANKS** 

**HUCKLEBERRY** 

**BASEBALL PLAYER** 

# Appendix I Modified Rankin Scale (mRS)

The Modified Rankin Scale (mRS) is a 6-point scale to determine if the patient is severely disabled (5), has a moderately severe disability (4), is moderately disabled (3), is slightly disabled (2), has no significant disability (1), or has no symptoms at all and is not limited (0).

# **Instructions**

The Modified Rankin Scale (mRS) will be administered to all study patients by a neurologist or neurology fellow. The mRS will be completed after the Mini Mental State Examination (MMSE) and the National Institutes of Health Stroke Scale (NIHSS).

Because subjects and family members may understate the severity of disability, it is important for the rating clinician to understand that the mRS is a clinical scale and not a patient-reported outcome. The clinician may ask questions but must assess the disability according to the 6-point scale whether or not in agreement with the subject, family, close friend, or caregiver.

The rater should use the best sources of information available. Information should be obtained from the patient and/or family, friends, nursing staff, physical and occupational therapists, any person who is familiar with the daily routine of the patient, and from medical records. The rater should interview both the patient and a close family member/friend or caregiver whenever possible. If the patient lacks insight into some difficulties, or responses are inconsistent, it is often helpful to interview a caregiver or relative independently.

#### **Modified Rankin Scale Interview**

**5\_Severe disability**; someone needs to be available at all times; care may be provided by either a trained or an untrained caregiver.

**Question**: Does the person require constant care?

**4\_Moderately severe disability**; need for assistance with some basic ADL, but not requiring constant care.

Question: Is assistance essential for eating, using the toilet, daily hygiene, or walking?

- **3\_Moderate disability**; need for assistance with some instrumental ADL but not basic ADL. <u>Question</u>: Is assistance essential for preparing a simple meal, doing household chores, looking after money, shopping, or traveling locally?
- **2\_Slight disability**; limitations in participation in usual social roles, but independent for ADL. <u>Questions:</u> Has there been a change in the person's ability to work or look after others if these were roles before stroke? Has there been a change in the person's ability to participate in previous social and leisure activities? Has the person had problems with relationships or become isolated? Do any of the following interfere with the subject's ability to perform all usual activities: difficulty reading or writing, difficulty speaking or finding the right word, problems with balance or coordination, visual problems, numbness (face, arms, legs, hands, feet), loss of movement (face, arms, legs, hands, feet), difficulty with swallowing, or other symptom resulting from stroke?
- **1\_No significant disability**; symptoms present but not other limitations. Question: Does the subject have any symptoms that do not interfere with the performance of all usual activities?
- **0\_No symptoms at all**; no limitations and no symptoms.

Note: The above questions are a modification of the questions from Wilson, et. al, Stroke. 2002:33:2243-2246 and are modified here for the use in Transcatheter heart valve trials for the FDA Division of CV Devices.

# Appendix J Echocardiogram



Title Echo Imaging Acquisition Manual-PARTNER3 Study -MOP # P3-001

ADDRESS
Locations Echo CoreLab

affected IUCPQ
2725 Chemin Ste-Foy

Québec, G1V-4G5

Edwards Lifesciences LLC One Edwards Way Irvine, CA 92614

Document Title: Echo Manual of Operations

Trial Sponsor: Edwards Lifesciences

Protocol Title: A Prospective, Randomized, Multi-Center, Controlled, Long-Term Study to

Establish the Safety and Effectiveness of the SAPIEN 3 Transcatheter Heart Valve (THV) in Patients with Symptomatic, Severe, Calcific Aortic

Phone: (418) 656-8711 ext. 5938

Stenosis Requiring Aortic Valve Replacement (AVR).

Protocol Identifier: US IDE Pivotal Trial #2015-08

#### Edwards Lifesciences LLC Protocol US IDE Pivotal Trial #2015-08

# TABLE OF CONTENTS 2. Study Overview 4 Purpose 4 Study Synopsis 4 Echo Qualification Submission Process 5 3.3 4.2 GE Vivid 7 System Specific Instructions for Archive Export (RAW Data DICOM 43 data) 27 4.4 Philips iE33 System Specific Instructions for Archive Export (NATIVE DICOM data) 33 5. Echo Quality Control Process 37 Echo Critique 37 6.1 6.2 6.3 6.4

Edwards Lifesciences LLC Protocol US IDE Pivotal Trial #2015-08

# 1. ABBREVIATIONS AND ACRONYMS

| 2D | two dimensional |
|---|---|
| AO | aorta |
| AS | aortic stenosis |
| ASE | American Society of Echocardiography |
| A2CH | apical 2-chamber |
| A4CH | apical 4-chamber |
| A5CH | apical 5-chamber Cleveland Clinic Coordinating Center for |
| C5R | Cleveland Clinic Coordinating Center for<br>Clinical |
| CD | compact disc |
| DCF | data clarification form |
| CW | Continuous wave |
| DICOM | Digital Imaging and Communications in Medicine |
| DOB | date of birth |
| EDTF | Echo Data Transmittal Form |
| DVD | digital video disc |
| EKG | electrocardiogram |
| ECHO | echocardiogram |
| FPS | frames per second |
| FR | frame rate |
| ICL | Imaging Core Lab |
| LA | Left atrium |
| LV | Left ventricle |
| MACE | Major Adverse Cardiac Events |
| NA | Not Applicable |
| NATIVE DICOM format | Philips proprietary format |
| PACS | Picture Archiving and Communication System |
| PLAX | parasternal long axis |
| PSAX | parasternal short axis |
| PVC | premature ventricular contraction |

Edwards Lifesciences LLC Protocol US IDE Pivotal Trial #2015-08

| PW | Pulsed wave |
|----------------|----------------------------------------|
| RAW Data DICOM | |
| format | GE proprietary format |
| SV | Sample volume |
| TAVR | Transcatheter Aortic Valve Replacement |
| THV | Transcatheter Heart Valve |

# 2. STUDY OVERVIEW

# 2.1 Purpose

The purpose of this Imaging Manual is to instruct sites in: 1) protocol-specific image acquisition requirements; 2) necessary documentation, image data submission instructions and data storage; and 3) the query resolution process for discrepancies and/or non-compliant data.

The goal of the echocardiographic imaging portion of this trial is to assist sites in obtaining high quality, reproducible, quantitative information about structure, function and hemodynamics of the Transcatheter Heart Valve (THV) in the aortic position. Echocardiographic measures of aortic valve area and function are used as markers for determination of success in this trial.

# 2.2 Study Synopsis

Refer to study protocol.

Version 1 - 26 MAY 2016


Edwards Lifesciences LLC Protocol US IDE Pivotal Trial #2015-08

#### 3. ECHO PROCESS

#### 3.1 Echo Qualification Submission Process

- 3.1.1 All sites new to the PARTNER trials will be asked to submit to the Imaging Core Lab, a de-identified sample of an echocardiogram performed for the Study protocol (Trial #2015-08) via Moving Pictures WebSend at <a href="https://www.mddximage.com">www.mddximage.com</a>. The purpose of the Site Echo Qualification Process is to ensure compatibility between site Echo acquisition and Core Lab analysis tools prior to subject recruitment and to ensure adherence to the imaging protocol.
- 3.1.2 A critique of the Echo qualification scan will be emailed to the site and study sponsor as notification of the qualification status
- 3.1.3 If the site does not qualify with the first submission, the Imaging Core Lab will use the critique to recommend changes for resubmission of another Echo study.

# 3.2 Echocardiographic Instrumentation

Complete echo-Doppler examinations are required at baseline, discharge, 30 days, 1 years, 2 years, 3 years, 4 years, 5 years, 7 years, 10 years.

Echocardiographic equipment manufacturer and model varies from site to site. Each site must maintain annual documentation by a third party ensuring the equipment has been validated and calibrated. Each enrolling site should strive to use the same echo instrument on all echo exams performed on an individual subject throughout the study. If more than one echo machine will be used in this trial, then the information above should be maintained for all of the machines that will be utilized. Each machine must have the capability to record proper date, time and subject identification (ID).

Digital Capture - Typically the transthoracic images are obtained with the subject in the left lateral decubitus position with head elevated 15 degrees during quiet respiration or end expiration. The two-dimensional images should be recorded on an ultrasound system that ALLOWS DIGITAL CAPTURE and has harmonic imaging capabilities using transducers in the range of 2.5 to 5.0 MHz. A qualified physician or sonographer must perform all ultrasound exams. Whenever possible, the same sonographer should perform all serial echoes on a given subject. At least three to five sinus cardiac cycles (depending on heart rate) of each view should be DIGITALLY CAPTURED during quiet respiration or at end expiration. At least three- to five-second capture should be recorded if the subject is in atrial fibrillation. For digital acquisition, obtain at least two sets of three complete cardiac cycles (normal sinus rhythm <90 beats per minute), and at least two sets of five complete cardiac cycles (normal sinus rhythm >90 beats per

Edwards Lifesciences LLC Protocol US IDE Pivotal Trial #2015-08

minute) for each required parameter. Cardiac cycles for assessment should not include PVCs or post-PVCs (compensatory pause). Imaging media provided should be labeled with protocol number, subject ID, study site, time and date of exam. The images MUST be exported in vendor specific proprietary (RAW Data / NATIVE) DICOM data format.

For each view, the gain, compression and image sector width should be optimized to ensure the best echocardiographic image of the endocardial borders.

Frame Rate - A minimum frame rate image acquisition of 40 frames per second (fps) is required for 2D imaging and 20 fps for Doppler imaging. Optimization of frame rate for 2D imaging is achieved by narrowing the sector width to include entire left ventricular (LV) (or right ventricular) myocardium without compromising LV walls and reduce depth to include 1/3 of left atrium (LA) to ensure full visualization of basal LV. Optimization of frame rate for Doppler imaging is achieved by reducing the color sector without cutting of important region of interest (ROI) segments.

ECG - All images should have a good quality ECG tracing on the screen and clear calibration markings on the imaging sector. ECG leads will be applied and the EKG control setting of the machine optimized to ensure a high quality EKG with adequate amplitude QRS complex for reliable digital capture (lead II equivalent preferred).

Doppler and M-Mode - For Doppler spectral and M-Mode tracings, the sweep speed should be at least 50 mm/sec and preferably 100 mm/sec and the scale and baseline should be adjusted to make sure that the entire Doppler and M-Mode signal is visualized. Time and velocity calibration markers must be present on the Doppler and M-Mode tracing. For spectral and color Doppler, the appropriate gain level should be selected that detects flow without extraneous noise or extension of signal into adjoining tissue.

Color Doppler - As defined in the ASE Guidelines for the Quantification of Native Valve Regurgitation, Nyquist settings for color Doppler assessment of the cardiac valves should be 50-60 cm/sec

Contrast - If visualization of the left ventricular endocardial border is inadequate, then an approved contrast agent can be administered following institutional standards. However, the contrast enhanced imaging should only be performed after all other images and parameters are obtained. Doppler signals should be repeated after 2D contrast images are acquired. When Doppler signals are obtained during the contrast phase of the study, the gain must be reduced to optimize the velocity signal.


J - 6

Edwards Lifesciences LLC Protocol US IDE Pivotal Trial #2015-08

#### Echo Visits Schedule -

| Visit | Submit to Core Lab | Range |
|-----------|--------------------|----------|
| Baseline | Yes | -90 days |
| Discharge | Yes | |
| 30 Day | Yes | +7 days |
| 1 Year | Yes | +30 days |
| 2–5 Year | Yes | +45 days |
| 7 Year | Yes | +45 days |
| 10 Year | Yes | +45 days |

Edwards Lifesciences LLC Protocol US IDE Pivotal Trial #2015-08

# 3.3 Echo Protocol Parameters and Imaging Guidelines

- 3.3.1 Begin with subject in the left lateral decubitus position. Echo bed cutout should be utilized to optimize apical views.
- Obtain PLAX views of the LV, LVOT, and aortic valve (see Figures 1 and
   2)

Figure 1



Figure 2




J-8

Edwards Lifesciences LLC Protocol US IDE Pivotal Trial #2015-08

3.3.3 Zoomed views of the LVOT and Aortic valve in both the PLAX and PSAX are acquired to identify the true LVOT dimension, AV annulus and stent diameter (see Figures 3 and 4).

Figure 3



Figure 4



Version 1 - 26 MAY 2016 CONFIDENTIAL

J-9

Edwards Lifesciences LLC Protocol US IDE Pivotal Trial #2015-08

- 3.3.4 2D, color, and CW Doppler imaging of the tricuspid valve and pulmonary valve in PSAX view (see Figure 5)
- 3.3.5 Color Doppler of zoomed Aortic valve must be obtained in the PLAX and PSAX to assess for paravalvular leaks: importance of multi-plane imaging (see Figures 5 and 6).

Figure 5



Figure 6




J - 10

Edwards Lifesciences LLC Protocol US IDE Pivotal Trial #2015-08

- 3.3.6 Color Doppler of the Mitral valve and Aortic valve should be obtained in multiple planes that can resolve the origins, maximum vena contracta width and maximum paths of the regurgitant jets.
- 3.3.7 Obtain a high PLAX view with transducer in second or third intercostal space to see ascending aorta (see Figure 7).

Figure 7



3.3.8 Obtain right ventricular inflow view: 2D on right atrium, tricuspid valve, pulmonary valve, Color Doppler and CW Doppler of tricuspid valve (see Figure 8)

Figure 8




Edwards Lifesciences LLC Protocol US IDE Pivotal Trial #2015-08

3.3.9 Obtain right ventricular outflow view: 2D of RVOT and main pulmonary artery, color and PW Doppler on pulmonary valve (see Figure 9).

Figure 9



3.3.10 Obtain apical 4-chamber view. It is imperative that all apical views be acquired on axis and not foreshortened. The apical myocardium should appear thin and pointed when in the correct plane. A foreshortened apex will appear rounded with thickened myocardium. If the image is foreshortened, apical contractility will appear to thicken towards the mitral valve rather than towards the contra lateral walls (see Figures 10 and 11).

Figure 10




Edwards Lifesciences LLC Protocol US IDE Pivotal Trial #2015-08

3.3.11 To ensure high frame rate image acquisition (frame rate of 40 to 90 FPS or 40% of heart rate), sector size should be narrowed to include entire LV myocardium; depth should be reduced to include 1/3 of left atrium to ensure full visualization of basal LV (see Figure 11).

Figure 11



3.3.12 Obtain PW and CW Doppler of mitral flow, tissue Doppler velocities at the lateral and medial aspects of the mitral annulus (see Figure 12)

Figure 12



Edwards Lifesciences LLC Protocol US IDE Pivotal Trial #2015-08

3.3.13 Obtain 4-chamber views of the right ventricle. Show a loop with focused view of the RV (see Figure 13)

Figure 13



3.3.14 Tissue Doppler imaging of the free-wall aspect of the tricuspid annulus (see Figure 14)

Figure 14



Edwards Lifesciences LLC Protocol US IDE Pivotal Trial #2015-08

3.3.15 In the apical 5-chamber view, obtain PW Doppler in LVOT and CW of the aortic valve. Obtain color Doppler of LVOT and aortic valve. (see Figure 15 for baseline study and Figure 16 for follow-up studies).

Figure 15



Figure 16



Edwards Lifesciences LLC Protocol US IDE Pivotal Trial #2015-08

3.3.16 For TAVR, obtain PW Doppler at 2 locations pre-stent and in-stent (see Figure 17). For SAVR, obtain PW Doppler pre-stent (see Figure 18).

Figure 17



Figure 18




Edwards Lifesciences LLC Protocol US IDE Pivotal Trial #2015-08

3.3.17 Obtain 2-chamber view: 2D of LV. Color Doppler of MR (see Figure 19)

Figure 19



3.3.18 Obtain 3-chamber view: 2D of aortic valve. PW Doppler of LVOT and CW Doppler of aortic valve. Color Doppler of LVOT and aortic valve. Color Doppler of MR (see Figure 20 for baseline study and Figure 21 for follow-up studies).

Figure 20




J - 17

Edwards Lifesciences LLC Protocol US IDE Pivotal Trial #2015-08

Figure 21



3.3.19 Obtain subcostal view: 2D, color Doppler of aortic valve, MR and TR, diastolic flow reversal of upper abdominal aorta (optional) (see Figure 22)

Figure 22



Edwards Lifesciences LLC Protocol US IDE Pivotal Trial #2015-08

3.3.20 Obtain right parasternal view: CW Doppler of aortic valve (in 40-50% of cases maximum aortic jet velocity is obtained at the right parasternal window (see Figure 23)

Figure 23



3.3.21 Obtain suprasternal notch view: If moderate or severe AR is suspected, then a PW spectral Doppler assessment of the proximal descending aorta should be performed to assess diastolic flow reversal. Place sample volume in the descending thoracic aorta below the take-off of the subclavian artery in the supra-sternal imaging plane. Set velocity scale between 60 and 80 cm/s above baseline (see Figure 24).

Figure 24



Edwards Lifesciences LLC Protocol US IDE Pivotal Trial #2015-08

3.3.22 The site is not required to perform any measurements for the study. The ICL will review each image make the required measurements and update the data into the study database.


Edwards Lifesciences LLC Protocol US IDE Pivotal Trial #2015-08

Table 2: Echo Protocol Imaging Acquisition

| | This table can be printed and used as a reference while performing the echo |
|---|---|
| | <ul> <li>Secure the study assigned Subject ID from the site coordinator. In the Echo ID field,<br/>type LASTNAME as EDWARD\$ Trial, FIRSTNAME subject initials, and Medical<br/>Record Number (MRN) 3-digit trial ID 4-digit site and 3-digit subject number</li> </ul> |
| | <ul> <li>Obtain 2 digital clips of 3 complete cardiac cycles (normal sinus rhythm) for each<br/>required parameter</li> </ul> |
| | <ul> <li>High 2D imaging frame rate: ≥40 FPS or 40% of heart rate</li> </ul> |
| | <ul> <li>Spectral Doppler (PW and CW) should be performed with the line of interrogation as<br/>parallel to flow as possible. Record Doppler at 100 mm/sec sweep speed.</li> </ul> |
| Acquisition<br>Requirements | <ul> <li>Pedoff (CW) aortic spectral display Doppler is required from; apical, suprasternal<br/>notch (SSN) and right parasternal (RPS) imaging windows. Please annotate on<br/>spectral display which view is being acquired.</li> </ul> |
| | <ul> <li>Per ASE guidelines, if 2 or more contiguous endocardial segments are not visible,<br/>echo contrast should be used. If contrast is used, annotate on screed which view is<br/>being acquired. Body markers are acceptable forms of annotation.</li> </ul> |
| | <ul> <li>Ensure good quality ECG signals are recorded on all images.</li> </ul> |
| | <ul> <li>Distance, time and velocity calibrations must be present on each image. Time, date,<br/>subject ID should be accurately captures on each image.</li> </ul> |
| | <ul> <li>All Image files are to be stored in vendor specific proprietary RAW/NATIVE DICOM<br/>data format (see section 7.3 through 7.5 for system specific downloading instructions).</li> </ul> |
| Echo Views | |
| | High PLAX focusing on Aortic root |
| PLAX | Zoomed view of LVOT and Aortic valve |
| I LAX | Standard 2D PLAX imaging to include LV/LA/AO |
| | Color Doppler of Mitral and Aortic valves |
| | Standard 2D imaging at these levels: |
| PSAX | <ul> <li>1) Aortic Valve; 2) Mitral Valve; 3) Papillary Muscle; 4) Apical</li> </ul> |
| РЭАХ | Color Doppler of the Mitral valve |
| | Color Doppler of Aortic valve at multiple levels, as shown in the image below |


#### Edwards Lifesciences LLC Protocol US IDE Pivotal Trial #2015-08

| | Zoomed view of Aortic valve with and without color Color Doppler of Tricuspid valve and pulmonary valve CW spectral Doppler of Tricuspid regurgitation |
|---|---|
| Apical 4CH | <ul> <li>Standard 2D imaging at increased depth to evaluate atria</li> <li>Standard 2D imaging at decreased depth focusing on LV</li> <li>Views focusing on right ventricle</li> <li>Color Doppler of Mitral valve and Tricuspid valve</li> <li>PW spectral Doppler of Mitral inflow</li> <li>CW spectral Doppler of Mitral flow</li> <li>CW spectral Doppler of Tricuspid regurgitation</li> <li>Tissue Doppler Imaging (TDI) of medial and lateral Mitral annulus</li> </ul> |
| Apical 5CH<br>(BASELINE<br>ONLY) | Tissue Doppler Imaging (TDI) of free-wall tricuspid annulus Zoomed view of LVOT with and without color PW spectral Doppler of LVOT. Place SV 0.5 cm proximal to the Aortic valve. CW spectral Doppler of Aortic valve Color Doppler of Mitral valve Zoomed view of LVOT with and without color |
| Apical 5CH<br>(FOLLOW-UP<br>VISITS ONLY) | <ul> <li>Zoomed view of LVOT with and without color</li> <li>PW spectral Doppler of stent. Place SV just apical to the prosthesis stent.</li> <li>PW spectral Doppler within stent (TAVR only) on the LV side of Aortic valve leaflets</li> <li>CW spectral Doppler of Aortic valve</li> <li>Color Doppler of Mitral valve</li> </ul> |


#### Edwards Lifesciences LLC Protocol US IDE Pivotal Trial #2015-08

| | Standard 2D imaging at increased depth to evaluate atria |
|---|---|
| Apical 3CH | Standard 2D imaging at decreased depth focusing on LV |
| (BASELINE<br>ONLY) | Zoomed view of LVOT with and without color |
| ONET | <ul> <li>PW spectral Doppler of LVOT. Place SV 0.5 cm proximal to the Aortic valve.</li> </ul> |
| | CW spectral Doppler of Aortic valve |
| | Standard 2D imaging at increased depth to evaluate atria |
| | Standard 2D imaging at decreased depth focusing on LV |
| Apical 3CH | Zoomed view of LVOT with and without color |
| (FOLLOW-UP<br>VISITS ONLY) | PW spectral Doppler of stent. Place SV just apical to the prosthesis stent. |
| | PW spectral Doppler within stent (TAVR only) on the LV side of Aortic valve leaflets |
| | CW spectral Doppler of Aortic valve |
| | Color Doppler of Mitral valve |
| | Standard 2D imaging at increased depth to evaluate atria |
| Apical 2CH | Standard 2D imaging at decreased depth focusing on LV |
| | Color Doppler of Mitral valve |
| | Standard 2D imaging |
| Subcostal | Color Doppler of Aortic valve |
| | Color Doppler of Mitral and Tricuspid valves |
| | Diastolic flow reversal of upper abdominal aorta (optional) |
| Right<br>Parasternal<br>(RSB) | CW spectral Doppler of Aortic valve |
| Suprasternal | Standard 2D imaging of aortic arch and descending aorta with and without color |
| Notch (SSN) | PW spectral Doppler with the SV placed in the proximal descending aorta |
| Pedoff CW<br>Spectral | <ul> <li>Acquire highest systolic flow velocity through Aortic valve in the following areas:</li> </ul> |
| Doppler | o 1) Apical, 2) SSN and 3) RSB |


Edwards Lifesciences LLC Protocol US IDE Pivotal Trial #2015-08

.

#### 3.4 Addendum: Specific Comments on Imaging Planes

#### IMAGING TIP 1: PARASTERNAL LONG AXIS VIEW

Parasternal long axis view is recorded with the transducer in the third or fourth intercostals space immediately to the left of the sternum. The transducer should be angled so that aortic valve, mitral valve and left ventricle are in their long axis. It is important that the parasternal long-axis view displays the true long axis of the ventricle with the left ventricle lying horizontally on the image. If it is impossible to obtain a single view which optimally displays the long axis of the aortic valve and aortic root as well as the long axis of the left ventricle, record 2 separate views. It is unacceptable to record an-off-axis view in which the apex "points up" on the screen. If this type of image is obtained try moving the transducer up an interspace or 2 or having the patient take a breath in. Sometimes having the patient move to a more lateral decubitus position will help as well.

#### IMAGING TIP 2: PARASTERNAL LONG AXIS VIEW

Measurement of the left ventricular outflow tract and aortic annulus is a key component of the study. In pre-device imaging, it is important to note that the largest annulus may not be in a plane with valve opening centered in the aorta.

Parasternal short axis view is obtained by angling the probe 90° with respect to the parasternal long axis of the LV. The goal of this view is to obtain information about the aortic valve as well as the LV. This is an essential view post-device to completely assess aortic regurgitation.

#### IMAGING TIP 3: PARASTERNAL SHORT AXIS VIEW

This may be the only view in which post-device medial or lateral aortic regurgitant jets are imaged. Imaging at the level of as well as just below the leaflets may allow you to better image these jets.

Apical four-chamber view provides considerable information including the relative sizes of the right and the left ventricle and the regional function of the LV. The four-chamber view is defined as a view which maximizes the LV long axis and the tricuspid and mitral annular dimensions. In this view, the full excursion of the mitral and tricuspid valves should be seen. The complete endocardial border of the LV will be traced for chamber volume assessment (method of discs) so all aspects including the apex should be visualized. In the


J - 24

Edwards Lifesciences LLC Protocol US IDE Pivotal Trial #2015-08

apical four chamber view, color Doppler of mitral and tricuspid regurgitation should be recorded. The four chamber view should visualize the Lateral, Septal and Apical walls.

Apical two-chamber view should be obtained for the goal of assessment of LV size and function. The complete endocardial border of the LV will be traced for chamber volume assessment (method of discs) so all aspects including the apex should be visualized. The degree of MR by color Doppler will also be assessed. The two chamber should visualize the Anterior, Inferior and apical walls

#### IMAGING TIP 4: APICAL 4 and 2 CHAMBER VIEWS

Because we will measure volumes from the apical views as an important endpoint of the study, please try to avoid apical foreshortening. If the view appears to be foreshortened, please bring the transducer down one interspace and have the patient take a breath in (particularly for the apical two-chamber view). Sometimes this will bring out a better (not foreshortened) view.

Apical 5 chamber and 3 chamber views are obtained to provide detailed information about the aortic valve color, spectral and continuous wave Doppler.

#### IMAGING TIP 5: APICAL 5 and 3 CHAMBER VIEWS

Both these views are essential in imaging post-device aortic regurgitant jets. Because we will be measuring jet vena contracta and jet length, a Res/Zoom view which includes imaging of the entire jet would be helpful. In addition, the 3Ch view may be used in the biplane Simpson's calculation of LV volume when the 2Ch view is inadequate thus careful attention to endocardial definition is important.

MORE IMAGING TIPS: SEE TEACHING PARTNER 3 TRANSTHORACIC ECHO PROTOCOL TEACHING SLIDES


Edwards Lifesciences LLC Protocol US IDE Pivotal Trial #2015-08

#### 4. ECHO SCAN SUBMISSION PROCEDURE

## 4.1 Submitting Echo Images to Imaging Core

- 4.1.1 All images should be uploaded to the image transfer portal at the time of the visit window (or within 2 weeks of image acquisition).
- 4.1.2 The sponsor has provided a check list to be completed by the study qualified sonographer and submitted to the study coordinator for entry in the Electronic Echo Data Transmittal Form (see example 4.1.5) located on the Moving Pictures website <a href="https://mddximage.com">https://mddximage.com</a>.

(Note: the sonographer check list does not need to be submitted and may be retained at the site for personal records.

- 4.1.3 The Study Coordinator is responsible for completely and accurately completing the Electronic Echo Data Transmittal Form. To avoid queries, ensure that no required fields are left blank.
- 4.1.4 If there are questions about completing the Electronic Echo Data Transmittal form, refer to the Moving Pictures "Quick Start Guide", or contact a support team member for assistance (support contact information on Moving Pictures website: <a href="https://mddximage.com">https://mddximage.com</a>).
- 4.1.5 Echo Data Transmittal Form Example




Edwards Lifesciences LLC Protocol US IDE Pivotal Trial #2015-08

#### 4.2 Archival Instructions

- 4.2.1 Complete the Electronic Echo Data Transmittal Form carefully and completely for each echo exam..
- 4.2.2 Archive the Echo study to digital media (DVD) immediately from the ultrasound system that was used to acquire the images (before archiving to Picture Archiving and Communication System [PACS]). Please note: Image files not stored in DICOM format cannot be interpreted.
- 4.2.3 Retain a copy of the DVD on site with study related materials.
- 4.2.4 Follow routine downloading instructions for all ultrasound systems, with the exception of the systems noted below.
- 4.2.5 If there are problems downloading the study to a DVD, Please contact your local ultrasound system application specialist.

# 4.3 GE Vivid 7 System Specific Instructions for Archive Export (RAW Data DICOM data)

- 4.3.1 Archive all studies immediately after image acquisition.
- 4.3.2 Select Archive screen and log in as administrator (ADM). Password should be: ulsadm (all lower case)




Edwards Lifesciences LLC Protocol US IDE Pivotal Trial #2015-08

- 4.3.3 System Setup
  - 1) In Configuration screen select "Connectivity"
  - 2) On the Connectivity screen choose "Dataflow" from top row of options
  - 3) Select CD/DVD Archive from the drop down menu in the "Name" section
  - 4) Highlight Database in the "Selected devices" region, then the Properties button will appear
  - 5) Activate the Properties button



Version 1 - 26 MAY 2016 CONFIDENTIAL

J - 28

Edwards Lifesciences LLC Protocol US IDE Pivotal Trial #2015-08

4.3.4 After activating the Properties button, a new window will appear. Check "Allow Raw Data," and "Allow Multiframe" then change the "Max Framerate" to Full



Version 1 - 26 MAY 2016 CONFIDENTIAL J - 29

Edwards Lifesciences LLC Protocol US IDE Pivotal Trial #2015-08

- 4.3.5 Formatting DVD
  - 1) In Configuration screen select "Connectivity"
  - 2) On the Connectivity screen choose "Tools" from top row of options
  - 3) In the Tools screen the media type should be set to "CD/DVD"
  - 4) Type in label for DVD (4 digit site and 3 digit subject number)
  - 5) Make sure DVD is in drive and select "FORMAT"
- A dialog box will appear to confirm that you wish to format the DVD

  select
  OK.
- Once the DVD is formatted, exit configuration screen




Edwards Lifesciences LLC Protocol US IDE Pivotal Trial #2015-08

- 4.3.6 . Exporting study from Internal Hard Drive to DVD
- Select Archive screen and set "Dataflow" to read "Local Archive Int. HD"
- Select EXPORT from the screen
- The export dialog box will appear. The <u>FROM</u> box should read "Local Archive – Int. HD" and the <u>TO</u> box should read "CD/DVD Archive" from the drop down menus. Select OK.




Edwards Lifesciences LLC Protocol US IDE Pivotal Trial #2015-08

- A screen of patients on the hard drive will appear. Select the patient/subject you wish to export to the DVD and select COPY.
- Once the study has been exported to a DVD, select DONE to finish the copy procedure.
- Select F3 or Alt-E from the keyboard to eject the DVD.



Retain a copy of the DVD on site with study-related materials.

If there are problems downloading the study to a DVD, please contact your local GE application specialist.


Edwards Lifesciences LLC Protocol US IDE Pivotal Trial #2015-08

# 4.4 Philips iE33 System Specific Instructions for Archive Export (NATIVE DICOM data)

- 4.4.1 Archive all studies immediately after image acquisition
- 4.4.2 System set-up
- Select machine "setup" on top row of keyboard to activate set up screen.
- Select "Print/Network" tab on left side of screen (fourth selection down).




Edwards Lifesciences LLC Protocol US IDE Pivotal Trial #2015-08

 On the Print/Network screen select "Device Selection" from the top row of options.



Version 1 - 26 MAY 2016 CONFIDENTIAL J - 34

Edwards Lifesciences LLC Protocol US IDE Pivotal Trial #2015-08

- On the Device selection screen select "Media" from the second row of options.
- Export Compression
- Still Frame Compression: Uncompressed
- Multi-Frame Compression: Compressed
- Monochrome: Send BW as Monochrome, Color as RGB
- Native Data
- Select Export Native Data Compressed
- Check Tissue Doppler Native Data
- Check 2D Native Data
- Check Color Native Data




Edwards Lifesciences LLC Protocol US IDE Pivotal Trial #2015-08

4.4.3 Exporting study from internal hard drive to DVD

- Select "Review" on left side of control panel to activate review screen.
- Select (highlight) subject from exam list.
- On the review screen select "Export To Media"
- Text box will appear

Choose "DVD" and "Export to Media" Select "OK" to process selections



Green Icon at bottom left of screen shows active copying



Retain a copy of the DVD on site with study-related materials.

If there are problems downloading the study to a DVD, please contact your local Philips application specialist.


J - 36

Edwards Lifesciences LLC Protocol US IDE Pivotal Trial #2015-08

#### 5. ECHO QUALITY CONTROL PROCESS

## 5.1 Echo Critique

Echocardiograms will be monitored for adherence to study protocol as well as quality. The Imaging Core Labs will provide feedback in the form of a critique to sites via email for each study subject submitted to the core lab. The critique should be shared with the imaging sonographer to ensure research quality data and to help prevent the possibility of missing data.

## 6. ECHO DATA CLARIFICATION PROCESS (AKA, QUERIES)

#### 6.1 Query Notification

6.1.1 The study coordinator (or designee) and the sponsor will receive an email from MDDX asking for the resolution of any issues that were found during the quality control (QC) process. Prompt response is required from the site designee.

#### 6.2 Echo Data Queries

- 6.2.1 Review the variable name, reported value, and comments/suggestions.
- 6.2.2 Record the corrected, missing, or illegible information in the resolution box.

#### 6.3 Echo Media Queries

- 6.3.1 Review the issue and comments/suggestions
- 6.3.2 Record the corrected information and/or comments of action taken (For Example: sent new images).
- 6.3.3 On the Moving Pictures Electronic Echo Transmittal Form, select that images are being re-submitted.

## 6.4 Echo Query Resolution Form Example


#### Edwards Lifesciences LLC Protocol US IDE Pivotal Trial #2015-08




Edwards Lifesciences LLC Protocol US IDE Pivotal Trial #2015-08

| Written by: Philippe Pibarot | | |
|------------------------------|-------------|----------------|
| Checked by: | Signature: | Date: |
| Checked by: | Signature: | Date: |
| Approved by Director: | Signature: | Date: |
| MOP # P3_001 | Date Issued | Date Effective |


# Appendix K-1 Computed Tomography (CT)

CT Manual of Operations, Appendix K-1

Edwards Lifesciences LLC Protocol US IDE Trial #2015-08

#### Table of Contents

Edwards Lifesciences LLC One Edwards Way Irvine, CA 92614

Document Title: CT Acquisition and Analysis Manual of Operations

Trial Sponsor: Edwards Lifesciences

Protocol Title: A Prospective, Randomized, Controlled, Multi-Center Study to Establish the Safety

and Effectiveness of the SAPIEN 3 Transcatheter Heart Valve in Low Risk Patients Requiring Aortic Valve Replacement who have Severe, Calcific, Symptomatic Aortic

Stenosis

Protocol Identifier: US IDE Trial #2015-08

| 1 | . Acquisition Recommendations for Combined Assessment of the Aortic Root and Aorto-Iliotemoral | |
|---|---|---|
| | Vasculature | 3 |
| | Definition and Identification of the Aortic Annulus and the Annular Plane | 12 |
| | Techniques for Determining the Annular Plane | 13 |
| | Measurements | 17 |
| | Transfemoral Access Analysis | 39 |
| | Bibliography | 43 |
| 2. | Submitting CT Images | 44 |
| 3. | System-Specific CT Acquisition and Reconstruction Techniques | 45 |
| | GE Healthcare CT Scanners | |
| | Philips Hardware | 61 |
| | Siemens Hardware | 77 |
| | Toshiba Hardware | 90 |

PARTNER 3 December 2015, Version 1.0 PARTNER 3 December 2015, Version 1.0

# Acquisition Recommendations for **Combined Assessment** of the Aortic Root and Aorto-Iliofemoral Vasculature

Contrast-enhanced computed tomography (CT) allows for anatomical assessment of the aortic root and the aorto-iliofemoral vasculature within a single examination. Data acquisition strategies and scanning protocols may vary based on scanner system and institutional preferences. The key component of all approaches is an ECG-assisted data acquisition which covers at least the aortic root, while the remainder of the data acquisition may be performed without ECG assistance. If employed properly, ECG assistance allows for artifact-free depiction of the aortic root.

The sequence of patient preparation and data acquisition, and the relevant principles of CT data acquisition will be explained in brief below.

#### ECG-ASSISTED CT DATA ACQUISITION

ECG-assisted data acquisition implies that in parallel to the CT data acquisition, the patient's ECG signal is recorded to do the following:

- · Direct the data acquisition itself
- · Direct the image reconstruction

ECG-assisted data acquisition techniques commonly employed in the clinical environment:

K1-3

- · Retrospective ECG Gating
- · Prospective ECG Triggering
- High-Pitch Helical

PARTNER 3 December 2015, Version 1.0 Currently, there are three different types of



Figure 1 - Retrospective ECG-gated helical data acquisition without dose modulation. The tube current (blue bar) is set at its peak during the entire cardiac cycle. The black boxes indicate the time point of image reconstruction within the cardiac cycle.

#### Retrospective ECG Gating (Spiral/Helical Mode)

- · Helical data acquisition due to continuous movement of the patient through the gantry while the scanner gantry rotates
- · Simultaneously records the ECG signal
- The recorded ECG signal allows for "retrospective" image reconstruction at specific time points of the cardiac cycle (FIGURE 1)
- In general, this technique is available on all scanner platforms capable of cardiac CT
- · Advantage: Allows for dynamic (cine) imaging/ image reconstruction throughout the entire cardiac cycle (early systole - late diastole)
- · Advantage: Greater flexibility in unstable heart rates or rhythms (eq, atrial fibrillation or premature ventricular contractions) - ability to use data from different phases (eg, systole or

PARTNER 3 December 2015, Version 1.0

diastole) and to manually edit the reconstruction (please refer to ECG Editing)

· Disadvantage: Relatively high radiation dose, as full tube current is applied throughout the entire cardiac cycle

#### ECG Editing with Retrospective ECG Gating

- The in-part redundant image data which is acquired using retrospective ECG gating and helical data acquisition allows for manual editing of the ECG signal with adjustment or deletion of certain trigger points (eg, an entire heart beat may be deleted in case of a premature contraction)
- · This technique should be employed in cases of misalignment artifacts due to premature contractions or atrial fibrillation
- . ECG editing has to be performed at the scanner console using the raw data

CAVEAT: Raw data is commonly stored for a limited time only.



Figure 2 - Example of retrospective ECG gating with dose modulation during systole (not recommended). Images reconstructed during systole outside of the window of peak tube current are noisy and uninterpretable.

- · Ideally dose modulation should be switched off to allow for data acquisition with peak tube current throughout the entire cardiac cycle; however, if utilized, it is recommended that dose modulation be used only in diastole set to 20% - 30% peak dose
- in systole CAVEAT: Most automated coronary current during systole.
- due to premature contractions or atrial fibrillation




· ECG editing should be considered to reduce artifacts

K1-5



Figure 3 - Retrospective ECG-gated helical data acquisition with dose modulation. Peak tube current is limited to mid-diastole (not recommended). Image reconstruction at systole (lower row) will likely result in uninterpretable image quality.

#### Dose Modulation in Retrospective ECG Gating:

- · Dose modulation is modulation of the tube current throughout the cardiac cycle with peak tube current (mAs) during a predefined phase of the cardiac cycle and lowered tube current during the remainder of the cardiac cycle (FIGURES 3 & 4)
- Although image reconstruction is still technically feasible throughout the cardiac cycle, images reconstructed outside the preselected phase

will have increased image noise and may not be interpretable

- · For aortic root evaluation, images are usually uninterpretable if tube current is lowered below one third of the peak current
- Due to the pulsatile and conformational changes of the aortic annulus throughout the cardiac cycle with larger dimensions usually found in systole, peak tube current is warranted during systole




Figure 4 - Retrospective ECG-gated helical data acquisition with dose modulation. Peak tube current is limited to systole. Image reconstruction at diastole (middle row) will likely result in uninterpretable image quality.

- · Advantage: Dose reduction
- Disadvantage: Images reconstructed outside of the window of full/peak tube current have increased image noise and may be uninterpretable

PARTNER 3
December 2015, Version 1.0 K1-7



Figure 5 – Prospective ECG-triggered sequential data acquisition. Upper row with diastolic data acquisition (not recommended), lower row with systolic data acquisition.

#### Prospective ECG Triggering (Sequential/Axial Mode)

- Data acquisition is prospectively triggered by the ECG signal (FIGURE 5)
- Data acquisition is performed in a slab-wise (axial, non-helical) fashion while the patient table does not move. The table is moved in between slabs
- Acquisition windows are usually limited to a specific portion of the cardiac cycle (eg, only mid-diastole) with no radiation exposure or image acquisition occurring outside of the acquisition window
- Limitation of the acquisition window often allows for only one single reconstruction, or if the window is slightly broadened ("padding") for slight variation in the reconstruction window
- · Advantage: Lower radiation dose
- Disadvantage: Allows for only limited coverage of the cardiac cycle and almost no correction in case of misregistration or motion artifact


#### Recommendation:

- · If prospective ECG-triggering is employed, the acquisition window should be centered in systole.
- · Due to the limited potential for image correction, this imaging technique should only be employed if radiation dose is a concern.

#### High-Pitch Helical Data Acquisition

- · High-pitch data acquisition is limited to second and third generation dual-source scanners and employs high pitch factors of 3.2-3.4
- Data acquisition can be ECG triggered to aim for systolic or diastolic data acquisition at the level of the aortic root
- This technique allows only for a single reconstruction
- · Advantage: Low radiation exposure
- · Disadvantage: Allows for only a single reconstruction

- table, typically supine, should closely resemble positioning on the cath lab table
- · Placement of ECG electrodes and IV access should follow institutional policies
- Patient instruction on breath-holding prior to scanning may improve compliance with the

#### Note:

Volume scanners with wide z-axis coverage (eq. 256-slice or 320-slice CT scanners) may be capable of covering the entire aortic root with one slab using axial data acquisition and prospective triggering. By extending the acquisition window to cover the entire cardiac cycle, this technique may allow for dynamic imaging, and may then be considered equivalent to retrospective ECG-gating without dose modulation. However, given the prospective nature of the data acquisition, where redundant data is not acquired, ECG editing is not possible.

PARTNER 3 December 2015, Version 1.0 CT Scan - Patient Preparations

- · Positioning of the patient on the scanner
- breath-holding instructions during the scan

K1-9



Figure 6 - Scout views highlighting two different imaging strategies: Left, ECG-assisted data acquisition limited to the aortic root and heart (green box) followed by non-gated CTA of the thorax, abdomen and pelvis (purple box). Right, ECG-assisted data acquisition of the entire thorax (green box) followed by the non-gated CTA of the abdomen and pelvis (purple box).

#### CT Scan - Scan Length and Scan Strategy

In general, there are two different approaches on how to combine the ECG-assisted data acquisition of the aortic root structures and the non-ECG-assisted computed tomography angiography (CTA) of the aorto-iliofemoral vasculature for evaluation of the transfemoral access route (FIGURE 6):

· Cardiac ECG-assisted data acquisition of the heart and aortic root (usually beginning 2 cm below the carina) followed by a non-ECGassisted CTA of the thorax, abdomen, and

pelvis. Although this approach results in repeat data acquisition of the aortic root and cardiac structures, the time-intensive ECG-assisted data acquisition is kept to a minimum.

· ECG-assisted data acquisition of the thorax followed by a non-ECG-assisted CTA of the abdomen and pelvis. The disadvantage of this approach is the relatively long acquisition time required for the entire thorax (may exceed 15 seconds), which increases the risk of breathing artifacts at the level of the cardiac structures.

PARTNER 3

December 2015, Version 1.0

# \mnular Plar

#### In General:

- All studies should be acquired using smallest available scan thickness (\$0.75 mm) based on individual system capabilities: Please refer to your system-specific user manual to determine your detector configuration
- The scan coverage should include the entire aortic arch
- The scan coverage for the non-ECG-assisted CTA of the pelvis should include the femoral heads and extend to shortly above the lesser trochanter
- The data acquisition of the non-ECG-assisted CTA should be performed in the cranial to caudal direction
- Tube voltage, tube current, and pitch should be adapted to institutional CTA protocols

#### Contrast:

- The total dose of contrast varies with scanner, imaging protocol, and body habitus, typically ranging from 60-100 ml.
- Image acquisition timing can be performed using either a timing bolus (test bolus) or bolus tracking. Bolus tracking with a region of interest (eg, in the ascending aorta) is less cumbersome and usually sufficient for imaging of the aortic root.
- Specific contrast protocols should follow institutional policies. A minimum injection rate of approximately 3 to 4 ml/s is usually required to allow for sufficient contrast attenuation of the aortic root.

#### IMAGE RECONSTRUCTION:

ECG-Assisted Image Data of the Aortic Root/Heart

- A small reconstruction field of view should be used to allow for maximum resolution
- The thinnest possible slice thickness should be employed (eg, 0.6 or 0.75 mm)
- If retrospective ECG gating was employed, image reconstructions should cover the entire cardiac cycle (multiphasic data set)
- Reconstruction phases: 0-90% RR at 5 – 10% increments
- Traditional filtered back projection or iterative reconstruction may be used

Non-ECG-Assisted Image Data of the Thorax, Abdomen, and Pelvis

- The slice thickness should be no thicker than 1.5 mm
- Traditional filtered back projection or iterative reconstruction may be used

K1-11


# Definition and Identification of the Aortic Annulus and the Annular Plane

The aortic annulus is not a discrete structure; rather, it is a "virtual" ring formed by the three lowest attachment points of the aortic valve cusps ("hinge points"). Accurately identifying the aortic annular plane is fundamental to proper transcatheter heart valve prosthesis size selection.



Figure 7 – Aortic root anatomy and definition of the annular plane (Image source: Kasel et al. JACC: Cardiovascular Imaging. February 2013)

#### Nomenclature of Viewing Planes

CT images are commonly viewed using multiplanar reformats (MPR). Post-processing platforms provide an axial (transverse), coronal, and sagittal view at the very beginning of processing. Exact orientation of one imaging plane is indicated by the cross hairs in

the two remaining planes. Manipulating the orientation of the cross hairs and the dependent planes results in oblique or double-oblique views, such as a sagittal double-oblique view.


## Techniques for Determining the Annular Plane

There are multiple ways of identifying the correct annular plane using MPRs. Independent of the approach, the final transverse double-oblique view should transect the hinge points of all three cups.

A systematic, step-wise approach has been published by the Society of Cardiovascular Computed Tomography (reproduced with permission):



#### Step 1:

Start out with multiplanar images in axial, sagittal, and coronal orientation.



#### Step 2

Rotate (without moving up and down or left and right) the reference lines in the formerly axial plane in a way so that the line that controls the former sagittal plane crosses the lowest insertion point of the noncoronary cusp, which is located at approximately the 8 o'clock position (note: it is not shown here that this may require to interactively change the level of the formerly axial plane by moving it up and down with the use of the reference line in the formerly coronal image, without rotating it so that the orientation remains unchanged).

K1-13




#### Step 3:

Use the reference line in the coronal image to rotate the former axial plane in a way so that it crudely approximates the plane of the aortic valve.



#### Step 4

In the coronal image, move the reference line that controls the former axial plane up and down to identify the lowest insertion point of the right coronary cusp which is usually located at about the 1 o'clock position. Position the formerly axial plane exactly at the level of that cusp insertion point. Then, move the crosshair in the formerly axial plane exactly onto the right coronary cusp insertion point.



#### Step 5:

The formerly sagittal plane will now show the lowest insertion point both of the right coronary cusp and the noncoronary cusp. In this window, move and rotate the reference line of the former axial plane so that it very exactly crosses both of these insertion points. Once this is achieved, the formerly axial plane will contain 2 of the 3 lowest cusp insertion points.



#### Step 6:

In the former coronal plane, rotate (without moving it) the reference line of the former axial plane until the lowest insertion point of the left coronary cusp just barely appears in the formerly axial window (arrow). Now, the former axial plane is exactly aligned with the lowest cusp insertion points of all 3 aortic cusps and represents both the orientation as well as the level of the "aortic annulus" (image on left). Measurements of aortic annulus dimensions should be performed in this plane.




Figure 8 - Facilitated annular segmentation.

#### Facilitated Annular Segmentation

 Certain post-processing platforms facilitate annular segmentation by manual placement of seeding points at the identified hinge points.
 After placing a seeding point for all three cusps, the plane transecting all three points is automatically displayed.

#### Semi-automated Annular Segmentation

 Certain post-processing platforms perform an automated segmentation of anatomical landmarks, including the basal hinge points, allowing for an automated display of the annular plane

K1-15

#### Note:

Confirmation of the correct identification of the annular plane is warranted for both the facilitated and semiautomated segmentation, ie, by "turning" the cross hairs and verifying the location of the hinge points on the long axis view.

#### PARTNER 3




Figure 9 – Dynamic changes in annular dimensions and configuration throughout the cardiac cycle. Conformational changes occur due to bulging of the aorto-mitral junction (red dashes) towards the left atrium during systole.

#### Importance of Cardiac Phase for Determining Maximum Aortic Annular Dimensions

- The aortic annulus is subject to pulsatile and deformational changes throughout the cardiac cycle
- The annular area may vary greatly between systole and diastole (FIGURE 9). Edwards sizing charts are based on maximum systolic area. Maximum systolic area is determined by evaluating the aortic annulus in 5 10% increments from 25 45% of the R R interval.

#### PARTNER 3


#### Measurements

After proper identification of the annular plane the annulus measurement and ancillary measurements should be performed.

These measurements can be grouped into measurements which depend on the annular plane and measurements which do not depend onto the annular plane.

#### Measurements Depending on Annular Plane

- Annular dimensions
- · Prediction of fluoroscopic angulation
- · Distance to coronary ostia (coronary artery height)
- Sinus height (sinotubular junction height)
- Left Ventricular Outflow Tract (LVOT)
- · Ascending aorta length

#### Measurements Independent of Annular Plane

- Sinus of Valsalva width
- Sinotubular junction (STJ) diameter
- · Ascending aorta diameter

Although several automated tools are commercially available to expedite the valve analysis workflow, it is important to understand the approach for each measurement in order to be capable of performing the assessment manually and to recognize errors which may occur in an automated analysis.

It is recommended to perform the following actions:

- · Identify the annular plane
- · Perform measurements dependent on the annular plane
- · Perform measurements independent of annular plane

K1-17

The annular assessment and measurements are used in conjunction with additional imaging modalities as well as patient characteristics to determine the appropriate prosthesis size.



Figure 10 (A, B, C) - Various descriptors of annular dimensions

#### **Annular Dimensions**

In general, annular dimensions (FIGURE 10) can be expressed in the following terms:

- Area
- Diameter
- Perimeter

It is important to understand that a diameter can be measured using an electronic caliper (simple distance measurement tool) and derived from perimeter or area using a mathematical equation.

Area and perimeter are assessed by utilizing planimetry by manually drawing a contour, a spline (explained below), or semi-automated contour with contrast-edge detection.

The aortic annulus is usually elliptical. A simple distance measurement, such as a long axis or short axis distance, does not integrate the rather complex dimensions of an ellipse.

Alternatively, the maximum or long axis diameter and minimum or short axis diameter can be assessed and then averaged (FIGURE 10B). This represents a more comprehensive assessment of the elliptical anatomy. However, manual caliper measurements are subject to error as a divergence in a single caliper measurement by 2 mm results in a divergence of 1 mm for the averaged value.


Some post-processing platforms provide maximum diameter (long axis) and minimum diameter (short axis) based on annular planimetry. However, these algorithms usually report the most extreme values.

Planimetry is performed by one of the following methods:

- Manual contouring with a region of interest or polygon
- · Manual contouring with a spline
- Semi-automated edge detection

Independent of the approach, planimetry yields an area commonly expressed as mm² or cm². The area measurement can be used to calculate an "effective" area-derived diameter calculated using the formula listed in FIGURE 10A. Some advanced post-processing tools perform this calculation automatically.

A "freehand" contour or region of interest follows the path of the cursor while a polygon is created by placing dots along the annular contour which are automatically connected without interpolation. In contrast a spline tool is similar to an elastic ruler which bends to pass through the manually defined points. Depending on the vendor, these planimetry tools may also yield perimeter. However, a "freehand" contour often results in a irregular line which leads to an artificially increased perimeter. Polygons and splines usually have a smooth contour yielding a more realistic perimeter value. Smoothing algorithms can allow for perimeter assessment using "freehand" contours by correcting the jerky contour.

Edge detection algorithms help to identify the annular contour based on the edge between the contrastattenuated lumen and the non-enhancing mural components. Importantly, automatically drawn contours should be visually validated and if necessary manually corrected.



Figure 11 - Annular assessment in the presence of annular calcifications.

Annular Dimensions in the Presence of Annular Calcifications

Annular calcifications can be classified as:

- · Adherent (crescent)
- Protruding(bulky)

The annular contour should be traced, extrapolating as if the calcification was not present (FIGURE 11).

It is important to also assess the entire anticipated landing zone for the presence of calcifications, for example, at the level of the annulus, sub-annular region (0 to 2 mm below annulus), and the upper LVOT (2 to 6 mm below annulus).

Prosthesis sizing should take into account calcium distribution, location, and size

PARTNER 3 December 2015, Version 1.0 PARTNER 3 December 2015, Version 1.0

K1-19

Prediction of Fluoroscopic Angulation

- · Fluoroscopic angulation required to obtain a coplanar view of the aortic annulus can be obtained prior to the procedure from the CT data set
- This may help to reduce the number of aortograms needed to achieve an acceptable view at the time of the procedure, thus decreasing the amount of contrast material
- Most post-processing platforms report the angulation of each of the three views of the MPR as pairs of degrees [°] RAO/LAO and ° CRA/CAU angulation (FIGURE 12A)
- · These angulations are located on an optimal viewing curve (FIGURE 12B)

Following the annular measurement DO NOT change the angulation or level of the annular plane (transverse double-oblique image) (FIGURE 12A).

By manipulating ("spinning") the cross hairs in the transverse oblique view, the orientation of the coronal doubleoblique view is moved along the optimal viewing curve which is reflected by a change in the displayed values for °RAO/LAO and °CRA/CAU angulation.

- For example, if the implanter prefers a view with 0° CRA/CAU angulation, the coronal view is adjusted to 0° CRA/CAU angulation, and the corresponding LAO angulation is noted
- Common angulation pairs include the following:
- •10° LAO, corresponding CRA/CAU angulation
- CRA/CAU angulation
- •30° LAO, corresponding CRA/CAU angulation

•0° LAO/RAO, corresponding

•0° CRA/CAU, corresponding LAO/RAO angulation






Figure 12 - Required pairs of LAO/RAO and CRA/ CAU angulation to achieve a coplanar view of the aortic annulus are located on the patient-specific optimal viewing curve.

K1-21

#### Coronary Height



Figure 13 - Assessment of coronary artery height.

The distance from the annular plane to the coronary ostia is critical to identify patients with low coronary height. The prosthesis may displace the native leaflets and/or calcium thereby, possibly occluding the ostium.

Following the annular measurement and fluoroscopy angulation assessment do NOT change the angulation or level of the annular plane (transverse double-oblique image).

By spinning the cross hairs on the transverse oblique view, adjust so that the coronal double-oblique view transects the left main ostium.

Measure the vertical height from the annular plane to the inferior aspect of the left coronary ostia. perpendicular to the annular plane, as shown in the image above (FIGURE 13).

Repeat above steps for the right coronary ostia.


# Right coronary cusp

Figure 14 - Assessment of Sinus/STJ Height.

The STJ height is critical in a case of high implantation where the prosthesis may come into contact with the STJ.

#### Step 1:

Do NOT change the angulation or level of the annular plane (transverse double-oblique image).

#### Step 2:

By spinning the cross hairs on the transverse oblique view, adjust so that the coronal double-oblique view transects the center of the left coronary cusp.

# Step 4:

Step 3:

Repeat above steps for the right coronary sinus and noncoronary sinus.

Measure the vertical height from the annular plane

to the STJ, perpendicular to the annular plane, as

shown in the image above (FIGURE 14).


K1-23

#### Left Ventricular Outflow Tract (LVOT)



Figure 15 - Assessment of LVOT area 5 mm below annular plane.

It is important to assess the LVOT for the presence and distribution of calcium. LVOT planimetry informs about LVOT geometry and identifies patients with a septal bulge

#### Step 1:

Do NOT change the angulation or level of the annular plane (transverse double-oblique image)

PARTNER 3


K1-25



Figure 16 - Pronounced septal bulge (white arrow).

#### Step 2:

Change the level of the transverse double-oblique plane 4 to 6 mm into the LVOT without changing its orientation (FIGURE 15)


- Assess the LVOT area by means of planimetry or measure the maximum and minimum diameters
- The LVOT anatomy should be assessed for the presence of a septal bulge (FIGURE 16)

on 1.0

#### Ascending Aorta Length



Figure 17 – Assessment of ascending aortic length.

This measurement is needed for evaluating the feasibility of transaortic access.

#### Step 1

Do NOT change the angulation or level of the annular plane (transverse double-oblique image).

#### Sten 2

Measure the distance from the annular plane to the transection point of the cross hairs and the ascending aortic wall on either coronal oblique or sagittal oblique view (both views result in the same measurement) (FIGURE 16).


K1-27

#### Sinus of Valsalva Width



Figure 18 - Assessment of Sinus Valsalva dimensions.

The sinus width is important to assess for shallow, non-capacious sinuses. Non-capacious sinuses may predispose to coronary occlusion.

#### Step 1:

Change the level of the transverse double-oblique view (annular plane) towards the sinus of Valsalva, usually by scrolling until you reach the widest portion of the sinus of Valsalva.

#### Step 2:

Measure the distance from the left coronary sinus to the opposing commissure using a distance measurement tool (FIGURE 18)

#### PARTNER 3


#### Step 3:

Repeat for the right coronary sinus and the non-coronary sinus, always measuring to the opposing commissure.

#### Step 4:

Average all three values by adding them and dividing by three.

#### Sinotubular Junction (STJ) Diameter



Figure 19 – Assessment of STJ dimensions.

The STJ diameter is critical in a case of high implantation where the prosthesis may come into contact with the STJ.

#### Step 1

Change the level of the transverse double-oblique view towards the STJ; the angulation may have to be changed

#### Step 2:

Identify the STJ and measure the diameter using the distance measurement tool (FIGURE 19)

#### PARTNER 3 December 2015, Version 1.0

K1-29

#### Ascending Aorta Diameter



Figure 20 - Assessment of ascending aortic dimensions.

The ascending aorta diameter is important to evaluate for the presence of an ascending aortic aneurysm, in particular in the setting of transaortic approach.

#### Step 1:

Change the level of the transverse double-oblique view towards the ascending aorta. The angulation has to be changed so that the transverse double-oblique view transects the ascending aorta perpendicular to the long axis (usually resulting in a circular shape of the ascending aorta on the transverse view).

#### Step 2:

Measure the diameter using the distance measurement tool. The measurement should be performed approximately 4 cm above the annular plane (FIGURE 20).

PARTNER 3


## Analysis - Troubleshooting

Good image quality is characterized by sufficient contrast attenuation and images free of artifacts, allowing for proper visualization of the aortic root structures and in particular the aortic annulus, ideally at systole. Artifacts include, but are not limited to, the following:

- Incorrect plane wrong orientation
- · Incorrect plane wrong angulation and too low
- · Incorrect plane too high

- Misalignment artifact
- · Double contours and blurring
- Poor contrast enhancement and image noise

· Breathing artifacts

Importantly, critical measurements such as annular measurements should be documented by means of screen shots (so-called secondary captures) which are ideally archived in, for example in the PACS (Picture Archiving and Communication System).

Screenshots should not only include the view in which the measurement was taken, but also the adjunct views such as the coronal and sagittal double-oblique view in case of an annular measurement on the transverse double-oblique view. These comprehensive screen shots provide valuable information:

- · Positioning of the measurement plane
- · Overall image quality
- Artifacts, which may be subtle or obscured on the measurement plane but more evident on others

PARTNER 3


#### Correct Orientation of the Annular Plane



Figure 23 – Appropriate annular plane segmentation and planimetry.

As discussed earlier, the annular plane transects through the most basal hinge points of all three cusps. Commonly, the center of the cross hairs remains in the center of the annular lumen when obtaining the screenshot (FIGURE 23).




Figure 24 – Appropriate annular plane segmentation and planimetry with cross hairs oriented to show all three hinge points. RC, right coronary cusp; LC, left coronary cusp; NC, non-coronary cusp. Same patient as Figure 23.

The red lines in the oblique coronal and sagittal images indicate the location of the double-oblique transverse image. As the cross hairs actually transect the annular contour four times at 90° intervals, not all of the three hinge points are depicted on the coronal and sagittal oblique views at the same time if the cross hairs remain centered in the annular lumen. Alternatively, the cross hairs can be oriented to transect all three basal hinge points by eccentric orientation of the cross hair center (FIGURE 24).


K1-31

Version 1.0 K1-32

#### Incorrect Plane - Wrong Orientation



Figure 25 – Incorrect plane due to wrong orientation. The plane cuts through the right coronary sinus.

- Incorrect orientation of the annular plane is a common cause of erroneous annular measurements. Frequently, the annular plane transects the basal portion of one sinus as opposed to the most basal hinge point while the two other most basal hinge points are correctly identified.
- In FIGURE 25 the red lines in the oblique coronal and sagittal images indicate the location of the double-oblique axial image.
- Portions of the right coronary cusp can be visualized (white arrow) in the double-oblique transverse view.
- Incorrect angulation commonly results into too large planimetric measurements.

K1-33

#### Incorrect Plane - Wrong Angulation and Too Low



Figure 26 - Wrong angulation and too low. Same angulation as in Figure 24.

 In the setting of wrong angulation (FIGURE 25), a transverse image without sinus tissue can be generated by relocating the level of the transverse double-oblique plane towards the LVOT (FIGURE 26). Although the contour on the transverse double-oblique view appears harmonic, it does not resemble the annular plane. As a consequence, planimetric assessment commonly results in too large measurements.


K1-34

## Incorrect Plane - Too High



Figure 27 – Transverse plane located above the proper annular plane.

 Red lines in the oblique coronal and sagittal images demonstrate the location of the doubleoblique axial image. In the double-oblique axial image, all three coronary cusps are visualized, clearly demonstrating that the plane is too high. This commonly results in overestimation of the annular area. (FIGURE 27)


#### Misalignment Artifact



Figure 28 – Misalignment artifacts (white arrows) truncating the annular contour.

- Irregular heart rhythms such as atrial fibrillation or premature contractions may result in misalignment artifacts due to the variable length of the RR intervals
- Severe misalignment artifact at the annular level (white arrows FIGURE 28) precludes accurate annular assessment
- If the image was acquired using retrospective ECG gating, ECG editing at the CT scanner console can be useful to reduce the artifact burden


K1-35

**Breathing Artifacts** 

#### **Double Contours and Blurring**



Figure 29 – Double contours (white arrows) impairing proper annular assess-

- Cardiac motion and pulsation in addition to irregular heart rhythms such as atrial fibrillation or premature contractions may result in double contours and blurring of the annular contour (white arrows FIGURE 29)
- Severe artifacts preclude accurate annular assessment

#### Poor Contrast Enhancement and Image Noise



Figure 30 – Poor opacification and increased image noise render this data set uninterpretable.

K1-37



Figure 31 – Breathing artifact at the level of the aortic root (white arrow) and evident as a stair-step also involving the sternum (red arrow).

- Breathing artifacts at the annular level can cause artifacts with a similar appearance as misalignment artifacts (white arrows FIGURE 31)
- Breathing artifacts always involve the chest wall, commonly appreciated as a stair-step along the body surface or sternum (red arrow FIGURE 31)
- They usually preclude accurate annular assessment

ARTNER 3 ecember 2015, Version 1.0 PARTNER 3 December 2015, Version 1.0

## Transfemoral Access Analysis

The aorta and iliofemoral vasculature should be evaluated using the acquired CTA data. The aorta can usually be evaluated using axial images and does not necessarily require advanced segmentation. The iliofemoral vasculature should be evaluated using a combination of axial images as well as various post-processing techniques.

#### Aorta

The thoracic and abdominal aorta should assessed for the presence of the following:

- Tortuosity/aneurysm, and in particular partially thrombosed aneurysms
- Non-calcified, exophytic plaque (FIGURE 32)

#### Iliofemoral Vasculature

The iliofemoral arteries should be assessed for the following:

- Vessel diameters
- Vascular calcification
- Tortuosity
- Dissections

A comprehensive analysis includes the following:

- · Review of the vasculature on axial images
- Curved planar reformats (CPRs)
- Volume rendered technique (VRTs)



Figure 32 – Coronal view demonstrating atherosclerotic changes in the aortic arch, including non-calcified plaque (white arrow).

K1-39

#### VascularDimensions

Vascular dimensions should be assessed perpendicular to the long axis of the vessel. On true axial images, only the common femoral arteries are oriented in a perpendicular fashion to the imaging plane. Instead of performing measurements on multiple angulated MPRs, most post-processing platforms allow for semi-automated or automated creation of center lines along the iliofemoral vasculature. The centerlines are then used to create multiple views oriented in a radial fashion in regard to these centerlines.

The required vessel diameters depend on the intended device to be used. Please refer to device-specific IFUs.



Figure 33 – CPRs (two top images) of the right iliofemoral vasculature with short axis views at the level of the common iliac artery and common femoral artery.

PARTNER 3 December 2015, Version 1.0 PARTNER 3 December 2015, Version 1.0

### Vascular Calcification

Vascular calcification can be assessed on axial views, CPRs with short axis views, and VRTs. Calcifications can in general be described and graded with increasing severity using the following terms:

- Spotty
- Confluent
- Horse-shoe and circumferential

In particular horse-shoe and circumferential calcifications are of relevance if vessel dimensions are borderline.

The location and degree of calcifications at the level of the puncture site of the common femoral artery should be assessed. Anteriorly located calcification may interfere with suture systems commonly used for a totally percutaneous, transfemoral approach.



Figure 34 - Nearly circumferential calcification



Figure 35 – Axial image at the level of the common femoral arteries (white arrows). Calcifications are located posteriorly on the right and anteriorly on the left.

K1-41







Figure 36 - Volume rendered imaged in AP (middle), LAO (right) and RAO (left) projection for assessment of iliofemoral tortuosity.

#### Tortuosity

Vascular tortuosity can be best assessed on VRTs given the three-dimensional nature of this technique. Quantification of tortuosity is not standardized. For documentation, AP and oblique views of the iliac vasculature should be obtained.

PARTNER 3 December 2015, Version 1.0 PARTNER 3 December 2015, Version 1.0

# **Bibliography**

Abramson S. The Complete Guide to Cardiac CT. New York: Mc Graw Hill Medical; 2012.

Achenbach S, Delgado V, Hausleiter J, Schoenhagen P, Min J, Leipsic J. SCCT expert consensus document on computed tomography imaging before transcatheter aontic valve implantation (TAVI)/transcatheter aortic valve replacement (TAVR). Journal of Cardiovascular Computed Tomography. 2012; 366-380.

Barbanti M, Yang T-H, Cabau JR, Tamburino C, Wood DA, Jilaihawi H, Leipsic J. (2013). Anatomical and Procedural Features Associated with Aortic Root Rupture During Balloon- Expandable Transcatheter Aortic Valve Replacement. Circulation. 2013; 244-253.

Blanke P, Schoepf UJ, Leipsic JA. CT in Transcatheter Aortic Valve Replacement. Radiology. 2013; 650-669.

Blanke P, Russe M, Leipsic J et al. Conformational pulsatile changes of the aortic annulus: impact on prosthesis sizing by computed tomography for transcatheter aortic valve replacement. JACC Cardiovasc Interv.

September 2012; 5(9):984-94.

Budoff MJ, Shinbane JS. Cardiac CT Imaging. New York: Springer; 2010.

Feuchtner, G. (2013). Imaging of Cardiac Valves by Computed Tomography. Scientifica, 1-13.

Kasel AM, Cassese S, Bleiziff S, Amaki M, Hahn R, Kastrati A, Sengupta P. Standardized imaging for aortic annular sizing: implications for transcatheter valve selection. JACC: Cardiovascular Imaging. 2013 Feb;6(2):249-62. Leipsic J, Gurvitch R, Troy L, Min J, Wood D, Johnson M, Webb J. Multidetector Computed Tomography in Transcatheter Aortic Valve Implantation.

JACC: Cardiovascular Imaging, 2011; 416-429.

Litmanovich DG, Imaging in Transcatheter Aortic Valve Replacement (TAVR): role of the radiologist. *Insights Imaging*. 2014; 123-145.

Mahesh M, Cody D. AAPM/RSNA Physics Tutorial for Residents: Physics of Cardiac Imaging with Multiple-Row Detector CT. RadioGraphics.

2007; 1495-1509. DOI: http://dx.doi. org/10.1148/rg.275075045

Min JK, Berman DS, Leipsic J.

Multimodality Imaging for Transcatheter

Aortic Valve Replacement. Springer; 2013.

Russo M, Tartara P. Trans-Aortic Transcatheter Aortic Valve Replacement with Edwards Sapien- Ascendra 3. 2014, April 10; Retrieved July 1, 2014, from CTSNet: www.ctsnet.org

Schultz CJ, Schoenhagen P, Halliburton SS. Cardiac CT Made Easy: An Introduction to Cardiovascular Multidetector Computed Tomography, Second Edition. CRC Press; 2014.

Wuest W, Anders K, Schuhbaeck A, May MS, Gauss S, Marwan M, Achenbach S. Dual source multidetector CT-angiography before Transcatheter Aortic Valve Implantation (TAVI) using a high-pitch spiral acquisition mode. European Society of Radiology. 2012; 51-58.

#### 2. Submitting CT Images

- 2.1. All images should be uploaded to the image transfer portal (Moving Pictures) at the time of the visit window. Before submitting the CT, ensure the study contains complete systolic and diastolic volume sets and that the Subject ID is available.
- 2.2. The sponsor has provided access to an Electronic Data Transmittal Form (see example 2.4-1) on the Moving Pictures website <a href="https://mddximage.com">https://mddximage.com</a>. This form should be filled out completely and accurately by the study coordinator in order to avoid queries.
- 2.3. If there are questions about completing the Electronic Echo Data Transmittal form, refer to the Moving Pictures "Quick Start Guide", or contact a support team member for assistance (support contact information on Moving Pictures website: <a href="https://mddximage.com">https://mddximage.com</a>).
- 2.4. CT images requiring independent review should be uploaded 72 hours prior to the case being presented.

#### CT Data Transmittal Form Example 2-1



PARTNER 3 December 2015, Version 1.0 PARTNER 3
K1-43 December 2015, Version 1.0

3. System-Specific CT Acquisition and Reconstruction Techniques

# CT Acquisition and Reconstruction Techniques for Transcatheter Aortic Valve Procedure Planning Utilizing GE Healthcare CT Scanners

WRITTEN IN COLLABORATION WITH:



EDITED BY: Philipp Blanke, MD, FSCCT Cardiac Imaging Specialist Center for Heart Valve Innovation St. Paul's Hospital & University of British Columbia Vancouver

Erin Fletcher RN, BSN, RCIS Global Product Training Manager Imaging, Procedure, and Patient Initiatives Edwards Lifesciences

Ann Soderman BS, RT (R)(CT) Global Product Development Leader –Cardiac CT GE Healthcare

Amy Deubig BS, RT (R)(CT) Global Product Marketing Manager – Cardiovascular CT GE Healthcare



PARTNER 3 December 2015, Version 1.0 PARTNER 3

K1-45


This paper is presented as a service to medical personnel by Edwards Lifesciences and GE Healthcare. The information in this white paper has been compiled from available literature. Although every effort has been made to report faithfully the information, the editors and publisher cannot be held responsible for the correctness. This paper is not intended to be, and should not be construed as, medical advice. For any use, the product information guides, inserts, and operation manuals of the various drugs and devices should be consulted. Edwards Lifesciences and the editors disclaim any liability arising directly or indirectly from the use of drugs, devices, techniques, or procedures described in this paper.

WARNING: Any reference to x-ray exposure, intravenous contrast dosage, and other medication is intended as a reference guideline only. The guidelines in this document do not substitute for the judgment of a healthcare provider. Each scan requires medical judgment by the healthcare provider about exposing the patient to ionizing radiation. Use the As Low As Reasonably Achievable (ALARA) radiation dose principle to balance factors such as the patient's condition, size and age; region to be imaged; and diagnostic task.

NOTE: Algorithms/protocols included in this paper are for educational reference only. Edwards does not endorse or support any one specific algorithm/protocol. It is up to each individual clinician and institution to select the treatment that is most appropriate.

Philipp Blanke, MD is a paid consultant to Edwards Lifesciences.


# INTRODUCTION

Transcatheter aortic valve procedures have proven to be an effective alternative in the treatment of aortic stenosis in high risk and inoperable patients. Contrast enhanced computed tomography (CT) has become an integral part of transcatheter aortic valve procedure planning by allowing for anatomical assessment of the aortic root and the aorto-iliofemoral vasculature within a single examination. It is critical that artifact free image data is obtained to allow for reliable anatomical measurements. Data acquisition strategies and scanning protocols may vary depending on scanner manufacturer, system, and institutional preferences. This document provides some recommendations for reliable CT image acquisition for transcatheter aortic valve procedures.

PARTNER 3


K1-47

#### WORK-FLOW RATIONALE

The key component of all approaches is an ECG-assisted data acquisition which covers at least the acrtic root, while the remainder of the data acquisition may be performed without ECG-assistance. If employed properly, ECG-assistance allows for artifactfree depiction of the aortic root. The sequence of patient preparation and the relevant principles of CT data acquisition will be explained in brief below.

#### PATIENT PREPARATION

- · Positioning of the patient on the scanner table, typically supine, should closely resemble positioning on the cath lab table
  - This is important for the prediction of c-arm angulation from the CT dataset.
  - · Placement of ECG-electrodes and IV access should follow institutional policies.
- · Patient instruction on breath-holding prior to scanning may improve compliance with the breath-holding instructions during the scan
  - · Due to the advanced age and frailty of this patient population, additional time may be needed for patient instruction.

Providing time for the patient to practice the breath hold prior to scan acquisition may drastically improve patient compliance and thereby scan quality.

#### CT SCAN - SCAN LENGTH AND SCAN STRATEGY

In general, there are two different approaches on how to combine the ECG-assisted data acquisition of the sortic root structures and the non-ECG assisted computed tomography angiography (CTA) of the aorta-iliofemoral vasculature for evaluation of the transfemoral access route:

1) ECG-assisted data acquisition of the heart and aortic root followed by a non-ECG assisted CTA of the thorax, abdomen and pelvis. Although this approach results in repeat data acquisition of the aortic root and cardiac structures, the time-intensive ECG-assisted data acquisition (in particular when using retrospective ECG-gating) is kept to a minimum which aids in limiting the contrast dose. Furthermore, limiting the ECG-assisted data acquisition also limits the radiation dose intensive component of the examination; although the cardiac scan range is covered twice.

The proposed protocols for all GE scanner Families use this approach. In 40mm detector coverage systems, cardiac data acquisition is performed with retrospective ECG-gating. With the Revolution CT system, with 160mm detector coverage, a one beat, gated whole heart volume scan is performed.

2) ECG-gated data acquisition of the thorax followed by a non-ECG gated CTA of the abdomen and pelvis. The disadvantage of this approach, when using 40 mm detector systems, is the relatively long acquisition time required for the entire thorax (depending on scanner model this will vary but in some cases it may exceed 15 seconds, in particular when using retrospective ECG-gating), which increases the risk of breathing artifacts at the level of the cardiac structures.

#### GEREVOLUTION" CT

#### 1. Scout

#### General

· Lateral and AP scout covering the thorax, abdomen and pelvis including the proximal femoral to the lesser trochanter

#### Data acquisition

- Start: Superior 60 End: Inferior 800
- Tube current 10 mA
- Tube voltage: 120 kV ECG trace: On
- Scout Plane: 90 and 0 degrees
- Auto Voice (Breath hold command): Inspiration

#### Comment

Take note of the iso-center indicator line on the fi scout to ensure that the patient is positioned within 2 cm of isocenter to allow for best image quality. Adjust table height to indicated iso-center location if more than 2 cm off before acquiring the 2nd scout.

2. ECG-gated axial data acquisition of the aortic root/heart (Group 1) followed by non-gated CTA of the thorax, abdomen, and pelvis (Group 2).

#### Smart Prep

#### General

- · Bolus tracking to automatically trigger the diagnostic scan acquisition based on the HU reading in the ROI reaching the prescribed enhancement threshold
- Slice location: approx 2 cm below the carina
- · ROI location: Ascending acrta

#### Data acquisition

Minimum

- Monitoring Delay: 12 sec Monitoring Inter Scan Delay: 1 sec
- Tube voltage: 120 kV
- · Tube current: 100 mA Diagnostic Delay: Auto
- Enhancement Threshold: 200 HU

#### Comment

The effective ('diagnostic') delay between reaching the threshold and the start of the subsequent data acquisition (Group 1) is the combined time comprising the length of the breath hold command (autovoice), the time needed for table movement and the subsequent pre-scan delay (pre-set delay time in Group 1)

#### Group 1 scan parameters - ECG-gated axial data acquisition of the aortic root/heart

#### General

- · ECG-gated axial data acquisition of the aortic root and heart
- · Scan range beginning 2 cm helow the carina to the base of the heart
- Dosemodulation is not recommended to ensure optimal image quality throughout the entire cardiac cycle
- Smart mA automatically sets the tube current to achieve the targeted Noise Index within the range defined by the min and max values

## Data acquisition

- Autovoice (Breath hold command): On (#1 - Suspension)
- Pre-set Delay Time: 2 seconds (Together with the auto voice command and table movement, this results in a diagnostic delay of 4-5sec)
- Scan Type: Cardiac
- Rotation Speed: 0.28 seconds
- SFOV: Cardiac Large DFOV: 25 cm
- Slice thickness: 0.625 mm Collimation: 160 mm (Smart
- Collimation will automatically select the appropriate collimation for the planned scan range
- Tube voltage: 120 kV
- Tube current: Smart mA: Min: 50 mA Max: 600 mA

#### Data reconstruction

- Axial multiphasic reconstruction covering the entire cardiac cycle. 5% or 10% intervals in sinus rhythm
- Slice Thickness: 0.625 mm
- Increment: 0.625 mm
- Iterative Reconstruction ASiR-V: 50%
- Recon: Std
- Use ECG editing if necessary

PARTNER 3 December 2015, Version 1.0 PARTNER 3 December 2015, Version 1.0

K1-50

#### REVOLUTION CT (CONT)

- Repeat acquisition is an additional option which can be used when covering the gated acquisition within a single volume. It may be useful in patients with atrial fibrillation, frequent premature contractions or extremely variable heart rates. See section on ECG Editing to learn how to select the desired heart beat for reconstruction.
- Noise Index: 30 Widenfor SSF: On
- Auto Gating: Off (Dose modulation is not recommended, alternatively ensure max mA during systole
- Targeted Phase reconstruction: 5-95%
- HRVariation Allowance: 4 bpm

#### Group 2 scan parameters - non-gated CTA of the thorax, abdomen, and pelvis

#### General

- · Helical, non-gated acquisition
- Scan range: lung apices to the lesser trochanters of the femoral bone
- · The Prep/Group Delay is needed to allow for the contrast opacified blood to reach the iliofemoral arteries

### Data acquisition

- · Prep/Group Delay 10.0s
- Auto voice (Breath hold command):On (#1-Suspension)
- Scan type: Helical
- · SFOV: Large Body
- Detector coverage: 80 mm
- · Pitch: 0.992
- · Table Speed: 158.75 mm/sec · Rotation Speed: 0.5 seconds
- Slice Thickness: 0.625 mm
- · Tube voltage:
- · 80 kV for BMI < 23 kg/m2 -· 100 kV for BMI 23 - 27 kg/m2
- · 120 kV for BMI >27 kg/m2
- · Tube current: Smart mA: Min: 10 mA Max: 530 mA
- Noise Index:18
- Scan direction: cranio-caudal

#### Data reconstruction

- Slice Thickness: 0.625 mm
- · Increment: 0.625 mm
- Iterative Reconstruction
- ASiR-V: 50% Recon: Std.

#### REVOLUTION CT (CONT)

#### Contrast application protocol

#### General

- Single contrast application for both the ECG-gated axial CTA of the aortic root/heart and the CTA of the thorax/abdomen/pelvis
- · Triphasic administration protocol with pure contrast, followed by a contrast/saline mixture, followed by a saline chaser
- · Placement of IV access per hospital protocol (an 18-guage IV typically provides the highest safety)
- · Automated contrast injection using a dual-cylinder

## Specific

- For normal weighted patients and an iodinated contrast agent with 300 mg/ml apply 30 ml contrast at 3.5 ml/sec, followed by 60 ml of 70% contrast/30% saline at 3.5 ml/sec, followed by 30 ml saline at 3.5 ml/sec; this results in atotalamount of 72 mltotal contrast agent (adjust for contrast agents with differing iodine concentrations)
- For large patients and an iodinated contrast agent with 300 mg/ml apply 40 ml contrast at 4.0 ml/ sec, followed by 80 ml of 70% contrast/30% saline at 4.0 ml/sec, followed by 30 ml saline at 4.0 ml/ sec; this results in a total amount of 96 ml total contrast agent (adjust for contrast agents with differing iodine concentrations)
- Please move this bullet fi bolus monitoring and timing of data acquisition by means of bolus tracking at the level of the ascending aorta with a region of interest placed within the ascending acrta; thresholdset at 200 HU.

PARTNER 3 December 2015, Version 1.0 PARTNER 3 December 2015, Version 1.0

K1-51

REVOLUTION DISCOVERY CT (REVOLUTION HD, REVOLUTION GSI), DISCOVERY CT750 HD, DISCOVERY CT, OPTIMA CT660, REVOLUTION EVO AND LIGHTSPEED VCT SCANNER PLATFORMS:

#### 1. Scout

#### General

 Lateral and AP scout covering the thorax, abdomen and pelvis including the proximal femoral to the lesser trochanter

#### Data acquisition

- Start: Superior 60
- End: Inferior 800 mA: 10 mA
- · ECGtrace:On
- Scout Plane: 90 and 0 degrees
- Auto Voice (Breath hold command): Inspiration

2. Retrospectively ECG-gated data acquisition of the aortic root/heart (Group 1) followed by non-gated CTA of the thorax, abdomen, and pelvis (Group 2).

#### Smart Prep

#### General

- Bolus tracking to automatically trigger the diagnostic scan acquisition based on the HU reading in the ROI reaching the prescribed enhancement threshold.
- Slice location: approximately 2 cm below the carina
- ROI location: Ascending aorta

## Data acquisition

- · Monitoring Delay: 7 sec
- Tubecurrent: 60 mA
- Tube voltage: system sets it to be same as Group 1
- Slice/Collimation: 5 mm
   ISD: 1.4
   Diagnostic Delay: Auto
- Minimum

  Pre-set delay time: 3 seconds
  (this results in a 'diagnostic
  delay' of approximately 5-6sec,
  if rotation time is kept identical
- between both groups, i.e. 0.4sec)
  Enhancement Threshold: 150 HU

#### Comment

The effective ('diagnostic') delay between reaching the threshold and the start of the subsequent data acquisition (Group 1) is the combined time comprising the length of the breath hold command, (auto voice), the time needed for table movement and the subsequent pre-scan delay.

K1-53

REVOLUTION DISCOVERY CT (REVOLUTION HD, REVOLUTION GSI), DISCOVERY CT750 HD, DISCOVERY CT, OPTIMA CT660, REVOLUTION EVO AND LIGHTSPEED VCT SCANNER PLATFORMS: (CONT)

#### Group 1 scan parameters - Retrospectively ECG-gated data acquisition of the aortic root/heart

#### General

- ECG-gated data acquisition of the sortic root and heart
- Scan range: beginning 2 cm below the carina to the base of the heart
- Irregular heartrates (HRs) are frequent within the TAVR population. Using the HR override capability with manually setting the HR to a lower value yields a lower pitch value which results in redundant CT data acquisition and thus provides the greatest fl in image reconstruction (e.g. utilization of SnapShot Segment, SnapShot Burst or SnapShot Burst Plus)



- Keeping as many parameters the same in Group 1 and Group 2 will result in a faster transition between the gated and non-gated groups
- In particular the rotation time needs to be consistent. The non-gated Group 2 is limited to a rotation speed of 0.40 seconds. Thus for heartrates <80 bpm, both groups should employ 0.40 seconds. For heart rates >80 bpm, a rotation speed of 0.35 seconds should be used, however this leads to a longer transition time

#### Data acquisition

- Scan Mode: Cardiac Helical
- Scan Parameter:
- <80 bpm: SnapShot Segment</p>
  >80 bpm: SnapShot Burst
- DFOV: 25 cm
- HR Override: On (manually entermin HR present on the ECG trace)
- · Rotation speed:
- HR < 80 bpm: 0.40 seconds</li>
   HR > 80 bpm: 0.35 seconds
- · Tube voltage:
- · 120 kVp for BMI > 25 kg/m<sup>2</sup>
- 100 kVp for BMI < 25 kg/m²</li>
   Tube current (manual):
   450/600/700 mA for small,
   average and large patients
- ECG Dose modulation is not recommended, alternatively ensure maximum mA in systole (e.g. 25 to 45%, R-peak delay 35%)
- TargetPhase reconstruction:
   5-95%
- Slice/Collimation: 0.625mm
- Scan direction: cranio-caudal
- Pitch: Autopitch (determined by HR)
- Auto voice (Breath hold command): Inspiration only

#### Data reconstruction

- Axial multiphasic reconstruction covering the entire cardiac cycle, 5% or 10% intervals in sinus rhythm
- · Use ECG editing if necessary
- Slice Thickness: 0.625 mm
- Increment: 0.62 mm
- · Recon: Std
- Iterative reconstruction: ASiR (if available) 50%


PARTNER 3


#### Group 2 scan parameter - non-gated CTA of the thorax, abdomen, and pelvis

#### General

- Scan range: Lung apices/upper thoracic inlet to the proximal femoral (lesser trochanter)
- Max mA values will vary between scanner models

#### Data acquisition

- Scan type: Helical
   Pitch: 0.984
- · Table Speed: 39.76 mm
- · Rotation Speed: 0.4 seconds
- Slice Thickness: 1.25 mm
- Collimation: 40 mm
- · Tube Voltage:
  - · 100 kV for BMI < 25 kg/m<sup>2</sup>
  - · 120 kV for BMI > 25 kg/m<sup>2</sup>,
- Tube current: Smart mA Min: 10 mA Max: 700 mA (may vary among scanner systems)
- NoiseIndex:18.4
- · Scan direction: cranio-caudal
- No additional automated breath hold command (no AutoVoice); alternatively mannually instruct patient to slowly exhale

#### Data reconstruction

- · Slice Thickness: 1.25 mm
- · Increment: 0.8 mm
- Recon: Std
- Iterative reconstruction: ASiR (if available) 50%

#### Contrast application protocol

#### General

- Single contrast application for both the retrospectively ECG-gated CTA of the aortic root/ heart and the CTA of the thorax/abdomen/pelvis
- Placement of IV access per hospital protocol (an 18-guage IV typically provides the highest safety)
- Automated contrast injection using a dual-cylinder injector

#### Specific

- Recommended contrast media application: 90 cciodinated contrast medium at 3.5 to 4 cc/sec (300mg/ml iodine contrast agent)
- Contrast bolus monitoring and timing of data acquisition by means of bolus tracking at the level of the ascending aorta with a region of interest placed within the ascending aorta; threshold set at 150 HU.

#### LOW CONTRAST DOSE PROTOCOL FOR 64 SLICE FAMILY OF SCANNERS -

Options for consideration to optimize scan parameters when contrast volumes need to be minimized.

- · Same scanner settings as listed above, except reduce threshold setting for bolus tracking (e.g. 80 HU)
- Reduce scan length of the retrospectively ECG-gated CTA to a minimum to cover only the aortic root as opposed to
  the entire heart, as this is the time-expensive part in regard to data acquisition
- · Reduce total amount of contrast to 50-60 cc
- · Injection rate should be lowered, but should at least be 3.5 cc/sec
- · Threshold to trigger initiation of the retrospective ECG-gated spiral data acquisition can be lowered to 80 HU
- · Use a lower kV such as 80 kV in thin patients
- These alterations should allow for a sufficiently contrast enhanced CT dataset of the aortic root. Contrast attenuation
  of the iliofemoral acquisition may be variable. Lowering EVp may help to maintain adequate opacification of the
  peripheral vessels

#### RECONSTRUCTION OF MULTIPHASIC DATA SET

Multiphase data should be reconstructed to enable evaluation of the aortic valve and aortic root throughout the entire cardiac cycle (e.g. in 10% intervals throughout the cardiac cycle). Although aortic root measurements are recommended in systole multiphase data sets allow for interrogation of other phases if systolic phases have degraded image quality (e.g. motion artifacts). Multiphase reconstruction: From the Prescription (Rx) screen, select the prescription type from the menu. Enter the Start phase/msec, End phase/msec, and Interval to reconstruct.



#### ABSOLUTE RECONSTRUCTIONS

Millisecond prescription for data reconstruction, i.e. reconstruction windows in fixed msec distances from the R-peak, may improve image quality in patients with irregular heart rates. An end-systolic target millisecond reconstruction range is +250 to +300 milliseconds at 25 msec intervals. Hovering the mouse on the ECG trace will indicate phase % and +/-millisecond location.

### REVIEW OF DATA RECONSTRUCTION AND ECG-EDITING

- Image reconstructions of the aortic root and heart should be reviewed immediately after the scan when the raw data is still available
- $\cdot \quad \text{The ECG-gating should be reviewed to ensure that the automated algorithms correctly identifies} \quad \text{the $R$-peaks}$


K1-55


PARTNER 3


#### ECG EDITING ON REVOLUTION CT

It may be helpful to insert, remove, or move a trigger to normalize a heart cycle when a trigger occurs at an incorrect location.

This may occur when abnormal ECG waveform patterns or excessive background noise are present during scan acquisition.

- Open the ECG-gated scan series in the Reconstruction and Image Processing area on the image monitor
- To [insert] a trigger, place the cursor at the intended position on the ECG trace (right-click to "Insert R-peak Trigger"). An additional trigger will display on the ECG trace
- · To [delete] a trigger point on the ECG trace, place the cursor on the trigger and right-click "Delete R-peak Trigger".
- · To [move] a trigger, place the cursor over the trigger and click and drag it to the new location
- To switch to a second heartbeat when repeat acquisition is used; place the cursor in the ECG Editor, right-click and select "Switch Scan". The reconstruction window toggles to the other scan



ECG EDITING ON REVOLUTION DISCOVERY CT (REVOLUTION HD, REVOLUTION GSI),
DISCOVERY CT750 HD, DISCOVERY CT, OPTIMA CT660, REVOLUTION EVO AND LIGHTSPEED
VCT SCANNER PLATFORMS:

Cardiac Helical exams allow for image reconstruction at any point in the RR interval as image data was acquired throughout the entire cardiac cycle using retrospective ECG-gating. The ECG editor provides the ability to move or reposition the reconstruction window.

 $In the ECG \ Editor click the "Rx" icon for the global phase prescription \ method, i.e. the entered phase values are applied to all available heart cycles.$ 

Global phase prescription allows selecting the phases of the cardiac cycle from which images are created. The blue highlighted areas represent the recon windows for each available RR-interval. The example below displays a reconstruction window ranging from 35 to 60% of the RR-interval. Gray areas represents x-ray exposure/available image data within the exam.



ECG-editing. IfR-peaks of the ECG trace were not correctly identified by the trigger points, the trigger points need to be corrected along the ECG trace: Insert, remove, or move a trigger to normalize a heart cycle when a trigger occurs at an undesirable location.



- To [insert] a trigger, place the cursor at the intended location along the ECG trace (right-click "Insert Trigger"). An
  additional trigger point (red line) appears on the ECG trace
- Following insertion of a trigger point, a recon window needs to be added (right-click "Add Recon Window").
   Confirm that the recon window is in the desired location before confirming image reconstruction
- · To[delete] a trigger point on the ECG trace, place the cursor on the trigger (red line), right-click "Delete Trigger"
- · To [move] a trigger, place the cursor over the trigger and click and drag it to the desired location

K1-57


Deleting a trigger affects the position of reconstruction windows in adjacent RR-intervals, when relative reconstructions (%) are employed. In contrast "Delete Image Recon Window" retains the trigger point while image data following the selected trigger point does not contribute to image reconstruction, thus not affecting adjacent RR-intervals. This approach may be employed to improve image quality, e.g. in cases of premature contractions or atrial fi extremely variable heart rates.

· Place the cursor in the blue image reconstruction window in the ECG editor, right click "Delete Image Recon Window"





· An orange (relaxed phase) or red (ungated) area appears on the trace if reconstruction window removal results in insufficient z-axis overlap to create gated images in order to compensate for the removed recon window. Relaxed phase reconstruction windows indicate where relaxed phase reconstruction images will be created. The images are reconstructed as close to the requested phase as possible, with a maximum of a 20% phase offset

In contrast to the global phase prescription across all RR-intervals, reconstruction windows can also be moved manually. Manually move or adjust recon window of one or more heart cycles, e.g. in setting of varying heart rates. Always review the images created from the edit ECG Trace process. Editing the trace changes the reconstruction using the original scan data.

- Achenbach S, Delgado V, Hausleiter J, et al. SCCT expert consensus document on computed tomography imaging before transcatheter acrtic valve implantation (TAVI)/transcatheter acrtic valve replacement (TAVI). J Cardiovasc Comput Tomogr 2012;6(6)566-380.
- Blanke P, Bulla S, Baumann T, et al. Thoracic Aorta: Prospective Electrocardiographically Triggered CT Angiography with Dual-Source CT-Feasibility, Image Quality, and Dose Reduction. Radiology 2010;255(1):207-217.
- 3. Blanke P, Russe M, Leipsic J, et al. Conformational Pulsatile Changes of the Aortic Annulus. JACC Cardiovasc Imaging 2012;5(9):984-994
- 4. Blanke P, Schoepf UJ, Leipsic J. CT in Transcatheter Acrtic Valve Replacement. Radiology 2013-269(3):650-669.
- Gurvitch B, Wood DA, Leipzic J, et al. Multislice Computed Tomography for Prediction of Optimal Angiographic Deployment Projections: During Transcatheter Acrtic Valve Implantation. JACC Cardiovasc Imaging 2010;3(11):1167-1165.
- 6. Leipsic J, Gurvitch R, LaBounty TM, et al. Multidetector Computed Tomography in Transcatheter Acrtic Valve Implantation. JACC Cardiovasc Imaging 2011;4(4):416-429.
- 7. Litmanovich DE, Ghersin E, Burke DA, et al. Imaging in Transcatheter Aortic Valve Replacement (TAVR): role of the radiologist. Insights Imaging

Edwards, Edwards Lifesciences, and the stylized E logo are trademarks of Edwards Lifesciences Corporation. All other trademarks are the property of their respective owners.

© 2015 Edwards Lifesciences Corporation. All rights reserved. PP-US-0168 v1.0 E5667/6-15/THV

© GE Healthcare, 2015

#### Edwards Lifesciences | edwards.com

One Edwards Way | Irvine, California 92614 USA Switzerland | Japan | China | Brazii | Australia | India



PARTNER 3


K1-60


K1-59


# CT Acquisition and Reconstruction Techniques for Transcatheter Aortic Valve Procedure Planning Utilizing Philips Hardware

WRITTEN IN COLLABORATION WITH:

# **PHILIPS**

EDITED BY:
Philipp Blanke, MD, FSCCT
Cardiac Imaging Specialist
Center for Heart Valve Innovation
St. Paul's Hospital & University of British Columbia
Vancouver

Erin Fletcher RN, BSN, RCIS Global Product Training Manager Imaging, Procedure, and Patient Initiatives Edwards Lifesciences

Philips Personnel Ronda Bruce Thomas Ivanc Thomas Naypauer Rolf Raijimakers

PARTNER 3




This paper is presented as a service to medical personnel by Edwards Lifesciences and Philips. The information in this white paper has been compiled from available literature. Although every effort has been made to report faithfully the information, the editors and publisher cannot be held responsible for the correctness. This paper is not intended to be, and should not be construed as, medical advice. For any use, the product information guides, inserts, and operation manuals of the various drugs and devices should be consulted. Edwards Lifesciences and the editors disclaim any liability arising directly or indirectly from the use of drugs, devices, techniques, or procedures described in this paper.

WARNING: Any reference to x-ray exposure, intravenous contrast dosage, and other medication is intended as a reference guideline only. The guidelines in this document do not substitute for the judgment of a healthcare provider. Each scan requires medical judgment by the healthcare provider about exposing the patient to ionizing radiation. Use the As Low As Reasonably Achievable (ALARA) radiation dose principle to balance factors such as the patient's condition, size and age; region to be imaged; and diagnostic task.

NOTE: Algorithms/protocols included in this paper are for educational reference only. Edwards does not endorse or support any one specific algorithm/protocol. It is up to each individual clinician and institution to select the treatment that is most appropriate.

Philipp Blanke, MD is a paid consultant to Edwards Lifesciences.


## INTRODUCTION

Transcatheter aortic valve procedures have proven to be an effective alternative in the treatment of aortic stenosis in high risk and inoperable patients. Contrast enhanced computed tomography (CT) has become an integral part of transcatheter aortic valve procedure planning by allowing for anatomical assessment of the aortic root and the aorto-iliofemoral vasculature within a single examination.

It is critical that artifact free image data is obtained to allow for reliable anatomical measurements. Data acquisition strategies and scanning protocols may vary depending on scanner manufacturer, system, and institutional preferences. This document provides some recommendations for reliable CT image acquisition for transcatheter aortic valve procedures.

#### WORK-FLOW RATIONALE

The key component of all approaches is an ECG-assisted data acquisition which covers at least the aortic root, while the remainder of the data acquisition may be performed without ECG assistance. If employed properly, ECG assistance allows for artifact-free depiction of the aortic root. The sequence of patient preparation and the relevant principles of CT data acquisition will be explained in brief below.

#### PATIENT PREPARATION

- Positioning of the patient on the scanner table, typically supine, should closely resemble positioning on the cath lab table.
  - · This is important for the prediction of c-arm angulation from the CT dataset.
  - Placement of ECG-electrodes and IV access should follow institutional policies.
- Patient instruction on breath-holding prior to scanning may improve compliance with the breath-holding instructions during the scan.
  - Due to the advanced age and frailty of this patient population, additional time may be needed for patient instruction.

Providing time for the patient to practice the breath hold prior to scan acquisition may drastically improve patient compliance and thereby scan quality.

#### CT SCAN - SCAN LENGTH AND SCAN STRATEGY

In general, there are two different approaches on how to combine the ECG-assisted data acquisition of the acrtic root structures and the non-ECG assisted computed tomography angiography (CTA) of the acrtofilio/femoral vasculature for evaluation of the transfemoral access route:

- 1) Cardiac ECG-assisted data acquisition of the heart and aortic root (usually beginning 2cm below the carina) followed by a non-ECG assisted CTA of the thorax, abdomen and pelvis. Although this approach results in repeat data acquisition of the aortic root and cardiac structures, the time-intensive ECG-assisted data acquisition is kept to a minimum which aids in limiting the contrast dose. Furthermore, limiting the ECG-assisted data acquisition also limits the radiation dose intensive component of the examination; although the cardiac scan range is covered twice. The proposed protocols below all use this approach.
- 2) ECG-assisted data acquisition of the thorax followed by a non-ECG assisted CTA of the abdomen and pelvis. The disadvantage of this approach is the relatively long acquisition time required for the entire thorax (may exceed 15 seconds), which increases the risk of breathing artifacts at the level of the cardiac structures.

NOTE: The following protocols are fully editable by the user (in particular tube current and tube voltage settings may be changed). Customized protocols can be saved as alternate protocols.


K1-63


#### PHILIPS BRILLIANCE ICT, INGENUITY, IQon, BRILLIANCE 64

| 1. Surview (Topogram/Scout) | | |
|---|---|---|
| General AP topogram/scout covering the thorax, abdomen and pelvis including the proximal femoral to the lesser trochanter | Data acquisition (manufacturers' default settings) - Length: 750 mm - Tubevoltage: 120 kV - Tubecurrent: 30 mA - Field of View: 500 mm | |
| 2. Non-enhanced scan (optional) | | |
| General Can be used for quantification of annular calcification Can be used for planning of subsequent contrast-enhanced data acquisition | Data acquisition Acquisition mode: Prospective ECG-gating, axial Pulsing window: 75% of RR-interval Tubevoltage: 120 kV Tubecurrent: 55 mAs Anatomical dose modulation: No Slice/Collimation: AUTO Scan direction cranio-caudal Rotation time: 0.4 sec | Data reconstruction Axial reconstruction within the pulsing window: 75% phase Field of View limited to the heart: 220 mm Slice thickness (thin): 2.5 mm Increment (thin): 2.5 mm Filter: CB |
| 3. Locator | | |
| General Planlocation of Locator on Surview: 2 cm below carina Place region of interest (ROI) within the ascending acrta | Data acquisition (manufacturers' default settings) Delay: None Tube current: Automatically populated and is set to 30 mAs Tube voltage: Automatically populated and is set to 120 kVp Slice/Collimation: Automatically populated and is set to 16 x 0.625 mm | |
| 4. Bolus Tracking | | |
| General Same location as #3 Threshold: change/difference of 110 HU in the ROI within the ascending actta to trigger cardiac contrast enhanced data acquisition (#5) | Data acquisition (manufacturers' default settings) Delay: Variable (use minimum delay possible) Tube current: Automatically populated and is set to 30 m.As Tube voltage: Automatically populated and is set to 120 kVp Slice/Collimation: Automatically populated and is set to 16 x 0.625 mm | |

PHILIPS BRILLIANCE iCT, INGENUTTY, IQon, BRILLIANCE 64 (CONT)

## $5. \,Retrospectively\,ECG-gated\,cardiac\,data\,acquisition-Contrast\,enhanced$

#### General

- · Retrospectively ECG-gated data acquisition of the aortic root and heart
- · Plan data acquisition on Surview: Scan range beginning 2 cm below the carina to the base of the heart
- Use unenhanced CaSc CT data for planning if available

#### Data acquisition

- Delay after monitoring has reached threshold: 5 sec
- Breath hold command: Inspiration only Tube voltage: 120 kV Tube current: 800 mAs (1000
- mAs for large patients) Anatomical dose modulation: NO
  - Dose modulation throughout the cardiac cycle: full exposure throughout is preferred, alternatively dose modulation with peak dose in systole
  - Slice/Collimation: AUTO
  - · Scan direction cranio-caudal
  - Pitch: Auto Pitch Rotation time: 0.4 sec

#### Data reconstruction · Axial multiphasic

- reconstruction covering the entire cardiac cycle, 5% or 10% intervals in sinus rhythm
- Use ECG editing if necessary Field of View limited to the heart: 220 mm
- Slice thickness: 0.9 mm Increment: 0.45 mm
- Filter: XCB
- Iterative reconstruction: iDose4 or IMR

#### 6. CTA of the thorax/abdomen/pelvis - Contrast enhanced

#### General

· Scan range: Upper thoracic aperture to the proximal femoral (lesser trochanter)

## Data acquisition

- Delay: Variable (use minimum delay possible)
- No additional automated breath hold command; alternatively manual instruction to slowly exhale
- Tube voltage: 120 kV
- Tube current: 251 mAs
- Anatomical dose modulation: Z-Modulation; 3-D Modulation
- · Slice/Collimation: AUTO
- Scan direction: cranio-caudal
- · DoseRight: YES
- · DoseRight Index: 26
- · Pitch: MAX per DRI
- · Rotation time: MIN per DRI · FOV: 350 mm

## Data reconstruction

- Axial reconstructions
- Slice thickness thin: 1.5mm Increment: Contiguous or
- Filter: B for ST Recon, YB for Lung Recon
- Iterative reconstruction: iDose4 or IMR


PARTNER 3 K1-65 December 2015, Version 1.0


#### PHILIPS INGENUITY CT SP/CORE/ELITE

NOTE: SP and Core, 64 row detector; collimation 64 x 0.625 mm; 40 mm z-axis coverage; Elite, 128 slice, 64 x 0.625 mm detector row system with dual focal spot positions to double the number of slices within the 40 mm z-axis gantry coverage.

#### 1. Surview (Topogram/Scout) General Data acquisition (manufacturers' default settings) · AP topogram/scout covering the thorax, abdomen and pelvis · Length: 750 mm including the proximal femoral Tube voltage: 120 kV to the lesser trochanter Tubecurrent:30mA · Field of View: 500 mm 2. Non-enhanced scan (optional) Data reconstruction General Data acquisition · Can be used for quantification Acquisition mode: Prospective Axial reconstruction within the pulsing window: 75% phase of annular calcification ECG-gating, axial Can be used for planning of Pulsing window: 75% of RR-Field of View limited to the heart: 220 mm subsequent contrast-enhanced interval Tube voltage: 120 kV Slice thickness (thin): 2.5 mm data acquisition Tube current: 55mAs · Increment (thin): 2.5 mm Anatomical dose modulation: No Filter: CB Slice/Collimation: AUTO Scan direction cranio-caudal Rotation time: Core/Elite: 0.4 sec SP: 0.33 sec 3. Locator General Data acquisition Plan location of Locator on (manufacturers' default settings) Surview: 2 cm below carina Delay: None Placeregion of interest (ROI) Tube current: Automatically within the ascending aorta populated and is set to 30 mAs Tube voltage: Automatically populated and is set to 120 kVp Slice/Collimation: Automatically populated and is set to 16 x 0.625 mm

#### 4. Bolus tracking

General

- · Samelocation as#3
- Threshold; change difference of 110 HU in the ROI within the ascending aorta to trigger cardiaccontrast enhanced data acquisition (#5)

## Data acquisition

- (manufacturers' default settings)
  Delay: Variable (use minimum
- delay possible)
  Tubecurrent: Automatically
- populated and is set to 30 mAs
- · Tube voltage: Automatically
- populated and is set to 120 kVp Slice/Collimation: Automatically populated and is set to 16 x 0.625 mm

#### 5. Retrospectively ECG-gated cardiac data acquisition - Contrast enhanced

#### Genera

- ECG-assisted data acquisition of the sortic root and heart
- Plan data acquisition on Surview: Scan range beginning 2 cm below the carina to the base of the heart
- Use unenhanced CaSc CT data for planning if available

#### Data acquisition

- Delay after monitoring has reached threshold: 5 seconds
- Breath hold command: Inspiration only
- Tube voltage: 120 kV
   Tube current: 800 m As (1000 m
- Tubecurrent: 800 mAs (1000 mAs for large patients)
- Anatomical dose modulation: No
   Dose modulation throughout the cardiac cycle: full exposure throughout is preferred, alternatively dose modulation
- with peak dose in systole
  Slice/Collimation: AUTO
- Scan direction: cranio-caudal
   Pitch (if helical): AutoPitch
- (based on heart rate)
  Rotation time:
  Core/Elite: 0.3 sec
  SP: 0.27 sec

#### Data reconstruction

- Axial multiphasic reconstruction covering the entire cardiac cycle, 5% or 10% intervals in sinus rhythm
- Use ECG editing if necessary
- Field of View limited to the heart: 220 mm
- Slice thickness: 0.9 mm
- · Increment: 0.45 mm · Filter: XCB
- Iterative reconstruction: iDose'

### 6. CTA of the thorax/abdomen/pelvis - Contrast enhanced

### General

Scan range: Upper thoracic aperture to the proximal femoral (lesser trochanter)

# Data acquisition Delay: Variable (use minimum

- delay possible)
  No additional automated breath
- hold command; alternatively manualinstruction to slowly exhale
- Tube voltage: 120 kV
   Tubecurrent: 251 mAs
- Anatomical dose modulation
   Z-Modulation, 3-D Modulation
- Slice/Collimation: AUTO
   Scan direction: cranio-caudal
- · Pitch: MAX per DRI
- Rotation time: MIN per DRI
- FOV: 350 mm

### Data reconstruction

- Axial reconstructions
- Slice thickness thin: 3 mm
- Increment: 3 mm
- Filter: B for ST Recon, YB for Lung Recon
- Iterative reconstruction: iDose<sup>4</sup>
   or IMR

PARTNER 3 December 2015, Version 1.0 PARTNER 3 December 2

K1-67


#### PHILIPS BRILLIANCE ICT ELITE

| 1. Surview (Topogram/Scout) | | |
|---|---|---|
| General • AP topogram/scout covering the thorax, abdomen and pelvis including the proximal femoral to the lesser trochanter | Data acquisition<br>(manufacturers' default settings)<br>• Length: 750 mm<br>• Tube voltage: 120 kV<br>• Tube current: 30 mA<br>• Field of View: 500 mm | |
| 2. Non-enhanced scan (optional) | | |
| General Can be used for quantification of annular calcification Can be used for planning of subsequent contrast-enhanced data acquisition | Data acquisition Acquisition mode: Prospective ECG-gating, axial Pulsing window: 75% of RR-interval Tube voltage: 120 kV Tubecurrent: 55 mAs Anatomical dose modulation: NO Slice/Collimation: AUTO) Scan direction cranio-caudal Rotation time: 400 msec Scan time: 16 sec Scan length: 14 cm | Data reconstruction Axial reconstruction within the pullsing window: 75% phase Field of View limited to the heart: 220 mm Slice thickness (thin): 2.5 mm Increment (thin): 2.5 mm Filter: CB |
| 3. Locator | | |
| General Plan location of Locator on Surview: 2 cm below carina Place region of interest (ROI) within the ascending aorta | Data acquisition (manufacturers' default settings) Delay: None Tubecurrent: Automatically populated and is set to 30 mAs Tube voltage: Automatically populated and is set to 120 kVp Slice/Collimation: Cycle time: Automatically populated and is set to 16 x 0.625 mm | |

#### 4. Bolus tracking

#### General

- Samelocationas#3
- Threshold; change/difference of 150 HU to trigger cardiac contrastenhanced data acquisition (#5)

## Data acquisition

- (manufacturers' default settings)
  Delay: Variable (use minimum delay possible)
- Tube current: Automatically populated and is set to 30 mAs
   Tube voltage: Automatically
- populated and is set to 120 kVp · Slice/Collimation: Automatically populated and is set to 16 x 0.625 mm

## 5. Retrospectively ECG-gated cardiac data acquisition - Contrast enhanced

#### General

- ECG-assisted data acquisition of the aortic root and heart
- Plan data acquisition on
   Surview: Scanrange beginning
   2 cm below the carina to the
   base of the heart
- Use unenhanced CaSc CT data for planning if available

#### Data acquisition

- Delay after monitoring has reached threshold: 5 seconds
- Breath hold command: Inspiration only
- Tube voltage: 120 kV
   Tubecurrent: 800 mAs (1000 for large patients)
- Anatomical dose modulation: No
   Dose modulation throughout the cardiac cycle: full exposure throughout is preferred, alternatively dose modulation
- with peak dose in systole
  Slice/Collimation: AUTO
- Scan direction cranio-caudal
   Pitch (if helical): Autopitch
- Rotation time: 0.27 sec

## Data reconstruction

- Axial multiphasic
  reconstruction covering the
  entire cardiac cycle, 5% or
  10% intervals in sinus rhythm
- Use ECG editing if necessary
   Field of View limited to the heart: 220 mm
- · Slice thickness: 0.9 mm
- · Increment: 0.45 mm
- Filter:XCB
- Iterative reconstruction: iDose<sup>4</sup> or IMR


K1-69


#### 6. CTA of the thorax/abdomen/pelvis - Contrast enhanced General Data acquisition Data reconstruction · Scan range: Upper thoracic · Delay: Variable (use minimum Axial reconstructions delay possible) Slice thickness thin: 3 mm aperture to the proximal femoral (lesser trochanter) · No additional automated · Increment: 3 mm breath hold command; Filter: Bfor ST Recon, alternatively manual YB for Lung instruction to slowly exhale Iterative reconstruction: iDose4 Tube voltage: 120 kV · Tubecurrent: 251 mAs · Anatomical dose modulation: Z-Modulation, 3-D Modulation · Slice/Collimation: AUTO · Scan direction: cranio-caudal · DoseRight: YES · DoseRight Index: 26 · Pitch: MAX per DRI · Rotation time: MIN per DRI • FOV: 350 mm

#### PHILIPS IQon SPECTRAL CT

| 1. Surview (Topogram/Scout) | | |
|---|---|---|
| General AP topogram/scout covering the thorax, abdomen and pelvis including the proximal femoral to the lesser trochanter | Data acquisition<br>(manufacturers' default settings)<br>• Length: 750 mm<br>• Tube voltage: 120 kV<br>• Tube current: 30 mA<br>• Field of View: 500 mm | |
| 2. Non-enhanced scan (optional) | | |
| General Can be used for quantification of annular calcification Can be used for planning of subsequent contrast-enhanced data acquisition | Data acquisition Acquisition mode: Prospective ECG-gating, axial Pulsing window: 75% of RR-interval Tube voltage: 120 kV Tube current: 42 mAs Anatomical dose modulation: NO Slice/Collimation: AUTO Scan direction: cranio-caudal Rotation time: 0.33 sec | Data reconstruction Axial reconstruction within the pullsing window: 75% Field of View limited to the heart: 220 mm Slice thickness (thin): 2.5 mm Increment (thin): 2.5 mm Filter: CB |
| 3. Locator | | |
| General Plan location of Locator on Surview: 2 cm below carina Placeregion of interest (ROI) within the ascending aorta | Data acquisition (manufacturers' default settings) Delay: None Tube current: Automatically populated and its set to 30 mAs Tube voltage: Automatically populated and its set to 120 kVp Slice/Collimation: Automatically populated and is set to 16 x 0.625 mm | |
| 4. Bolus tracking | | |
| General Same location as #3 Threshold, change/difference of 110 HU to trigger cardiac contrast enhanced data acquisition (#5) | Data acquisition (manufacturers' default settings) Delay: Variable (use minimum delay possible) Tube current: Automatically populated and is set to 30 mAs Tube voltage: Automatically populated and is set to 120 kVp Slice/Collimation: Automatically populated and is set to 16 x 0.625 mm | |


PARTNER

K1-71


### 5. Retrospectively ECG-gated cardiac data acquisition - Contrast enhanced

#### General

- ECG-assisted data acquisition of the aortic root and heart
- Plan data acquisition on Surview: Scan range beginning 2 cm below the carina to the base of the heart
- · Use unenhanced CaSc CT data for planning if available

#### Data acquisition

- Delay after monitoring has reached threshold: 5 seconds
- Breath hold command: Inspiration only
- Tubevoltage: 120 kV
- Tubecurrent: 620 mAs (775 mAs for large patients)
- Anatomical dose modulation:
- Dose modulation throughout the cardiac cycle: full exposure throughout is preferred, alternatively dose modulation with peak dose in systole Slice/Collimation: AUTO
- · Scan direction cranio-caudal
- · Pitch (if helical); AutoPitch

## Rotation time: 0.27 sec

#### Data reconstruction

- · Axial multiphasic reconstruction covering the entire cardiac cycle, 5% or 10% intervals in sinus rhythm
- Use ECG editing if necessary
- Field of View limited to the
- heart: 220 mm Slice thickness: 0.9 mm
- · Increment: 0.45 mm
- · Filter: XCB
- · Iterative reconstruction: iDose or IMR
- Conventional and Spectral results

## 6. CTA of the thorax/abdomen/pelvis - Contrast enhanced

· Scan range: Upper thoracic aperture to the proximal femoral (lesser trochanter)

#### Data acquisition

- Delay: Variable (use minimum delay possible)
- No additional automated breath hold command: alternatively manual instruction to slowly exhale
- Tubevoltage: 120 kV
- · Tubecurrent: 193 mAs · Anatomical dose modulation:
- Z-Modulation, 3-D Modulation · Slice/Collimation: AUTO
- · Scan direction: cranio-caudal
- · DoseRight: YES
- DoseRight Index: 26
- · Pitch: MAX per DRI
- · Rotation time: MIN per DRI
- · FOV: 350 mm

#### Data reconstruction

- Axial reconstructions
- Slice thickness thin: 3 mm
- · Increment: 3 mm
- Filter: Bfor ST Recon YB for Lung
- Iterative reconstruction: iDose or IMR
- Conventional or Spectral results

## Contrast application protocol

#### General

- · Single contrast application for both the retrospectively ECG-gated CTA of the aortic root/ heart and the CTA of the thorax/abdomen/pelvis
- Placement of IV access per hospital protocol (an 18-guage IV typically provides the highest safety)
- Automated contrast injection using a dual-cylinder

#### Specific

- Recommended contrast media application: Site specific and scan protocol driven
- Contrast bolus monitoring and timing of data acquisition by means of bolus tracking at the level of the ascending aorta with a region of interest placed within the ascending aorta; threshold set at 110 HU above baseline, delay to start of data acquisition after reaching threshold 5 sec

#### LOW-CONTRAST DOSE PROTOCOL - RATIONAL FOR ALL SCANNER TYPES

- Reduce scan length of the retrospectively ECG-gated CTA to a minimum to cover only the acrtic root as opposed to the entire heart, as this is the time-intensive part in regard to data acquisition
- · Injection rate and total amount of contrast may be lowered
- · Threshold to trigger initiation of the retrospective ECG-gated spiral data acquisition can be lowered to 80 HU
- · Reduce tube voltage to increase contrast attenuation

These alterations should allow for a sufficiently contrast enhanced CT dataset of the aortic root. Contrast attenuation of the iliofemoral acquisition may be variable.

#### RECONSTRUCTION OF MULTIPHASIC DATA SET

The image data of the acrtic root and heart should be reconstructed as multiphasic data set throughout the entire cardiac cycle in 5% or 10% intervals, allowing for cine review of the anatomy.

#### REVIEW OF DATA RECONSTRUCTION AND ECG-EDITING

- · Image reconstructions of the aortic root and heart should be reviewed immediately after the scan when raw data is
- · The ECG-gating should be reviewed to ensure that the automated algorithms correctly identifies the R-peaks
- · If any R points were not correctly identified, manual correction should be performed. This can enhance the quality of cardiac images in the presence of heart rate irregularities
- · To activate the editing tools, click the pencil icon. If the icon is grayed out, editing has been disabled



K1-74

PARTNER 3



· Right-click on an arrhythmia to Accept or Reject



- · Double-click on the wave to add a new R point
- · Move an existing R point by drag and drop
- · Double click on a R point to delete it



· Movephase points by drag and drop



· Additional options are available in the right-click menu



· The undo option functions with the editing tools. Click this to delete your edit



#### References

- Achenbach S, Delgado V, Hausleiter J, et al. SCCT expert consensus document on computed tomography imaging before transcatheter aortic valve implantation (TAVI)/transcatheter aortic valve replacement (TAVIS). J Cardiovasc Comput Tomogr 2012:6(s)566-350.
- Blanke P, Bulla S, Baumann T, et al. Thoracic Austa: Prospective Eletrocardiographically Triggered CT Angiography with Dual-Source CT-Feanibity, Image Quality, and Dose Rechartion. Radiology 2010;255(1):207-217.
- 3. Blanke P, Russe M, Leipsic J, et al. Conformational Pulsatile Changes of the Aortic Annulus. JACC Cardiovasc Imaging 2012;5(9):984-994
- 4. Blanke P, Schoepf UJ, Leipeic J. CT in Transcatheter Acrtic Valve Replacement. Radiology 2013;269(3):650-669.
- Gurvitch R, Wood DA, Leipnic J, et al. Multiplice Computed Tomography for Prediction of Optimal Angiographic Deployment Projections During Transcatheter Acrtic Valve Implantation. JACC Cardiovasc Imaging 2010;3(11):1157-1165.
- $6. \ \ Leipsic J, Gurvitch R, LaBounty TM, et al. \ Multidetector \ Computed Tomography in Transcatheter Acretic Valve Implantation. \\ JACC \ Cardiovasc Imaging 2011:4(4):416-429.$
- Litmanovich DE, Ghersin E, Burke DA, et al. Imaging in Transcatheter Aortic Valve Replacement (TAVR): role of the radiologist. Insights Imaging 2014; 5:123-145.

Edwards, Edwards Lifesciences, and the stylized E logo are trademarks of Edwards Lifesciences Corporation. All other trademarks are the property of their respective owners.

© 2015 Edwards Lifesciences Corporation. All rights reserved. PP-US-0069 v1.0 E5668/6-15/THV

© Philips, 2015

Edwards Lifesciences | edwards.com

One Edwards Way | Irvine, California 92614 USA Switzerland | Japan | China | Brazii | Australia | India



# CT Acquisition and Reconstruction Techniques for Transcatheter Aortic Valve Procedure Planning Utilizing Siemens Hardware

# WRITTEN IN COLLABORATION WITH: SIEMENS Healthcare

EDITED BY:
Philipp Blanke, MD
Cardiac Imaging Specialist
Center for Heart Valve Innovation
St. Paul's Hospital & University of British Columbia
Vancouver

Erin Fletcher RN, BSN, RCIS Global Product Training Manager Imaging, Procedure, and Patient Initiatives Edwards Lifesciences

Ricarda Grund
Application Specialist & Product Manager
User Services – Computed Tomography
Siemens Healthcare GmbH
Customer Solutions




K1-78

PARTNER 3


This paper is provided as an educational resource to medical personnel by Edwards Lifesciences and Siemens. The information in this white paper has been compiled from available literature. Although every effort has been made to faithfully report the information, the editors and publisher cannot be held responsible for the correctness. This paper is not intended to be, and should not be construed as, medical advice. For any use, the product information guides, inserts, and operation manuals of the various drugs and devices should be consulted. Edwards Lifesciences, Siemens and the editors disclaim any liability arising directly or indirectly from the use of drugs, devices, techniques, or procedures described in the reference guide.

WARNING: Any reference to X-ray exposure, intravenous contrast dosage, and other medication is intended as a reference guideline only. The guidelines in this document do not substitute for the judgment of a health care provider. Each scan requires medical judgment by the health care provider about exposing the patient to ionizing radiation. Use the As Low As Reasonably Achievable (ALARA) radiation dose principle to balance factors such as the patient's condition, size, and age; region to be imaged; and diagnostic task.

NOTE: Algorithms/protocols included in this book are for educational reference only. Edwards does not endorse or support any one specific algorithm/ protocol. It is up to each individual clinician and institution to select the treatment that is most appropriate.

Philipp Blanke, MD is a paid consultant to Edwards Lifesciences.

#### INTRODUCTION

Transcatheter aortic valve procedures have proven to be an effective alternative in the treatment of aortic stenosis in high risk and inoperable patients. Contrast enhanced computed tomography (CT) has become an integral part of transcatheter aortic valve procedure planning by allowing for anatomical assessment of the aortic root and the aorto-iliofemoral vasculature within a single examination. It is critical that artifact free image data is obtained to allow for reliable anatomical measurements. Data acquisition strategies and scanning protocols may vary depending on scanner manufacturer, system, and institutional preferences. This document provides

and institutional preferences. This document provides recommendations for reliable CT image acquisition for transcatheter aortic valve procedures.


PARTNER 3

K1-79


#### WORK-FLOW RATIONALE

The key component of all approaches is an ECG-assisted data acquisition that covers at least the acrtic root, while the remainder of the data acquisition may be performed without ECG assistance. If employed properly, ECG assistance allows for artifact-free depiction of the acrtic root. The sequence of patient preparation and the relevant principles of CT data acquisition will be explained in brief below.

#### PATIENT PREPARATION

- Position the patient, typically supine, on the scanner table to closely resemble cath
  lab table positioning. This is important for the prediction of C-arm angulation from
  the CT dataset.
- · Place ECG-electrodes and IV access in accordance with institutional policies.
- Provide time for the patient to practice the breath hold prior to scan acquisition to improve patient compliance and thereby scan quality.
- Allow additional scanning and instruction time as needed due to the advanced age and frailty of this patient population.

#### CT SCAN - SCAN LENGTH AND SCAN STRATEGY

In general, two different approaches are used to combine the ECG-assisted data acquisition of the sortic root structures and the non-ECG-assisted computed tomography angiography (CTA) of the acrto/ilio/femoral vasculature for evaluation of the transfemoral access route:

- 1) Cardiac ECG-assisted data acquisition of the heart and aortic root (usually beginning 2cm below the carrina) followed by a non-ECG-assisted CTA of the thorax, abdomen, and pelvis. Although this approach results in repeat data acquisition of the aortic root and cardiac structures, the time-intensive ECG-assisted data acquisition is kept to a minimum that aids in limiting the contrast dose. Furthermore, by limiting the ECG-assisted data acquisition this decreased the radiation dose-intensive portion of the examination, although the cardiac scan range is covered twice. The proposed protocols for all Siemens scanner families use this approach.
- 2) ECG-assisted data acquisition of the thorax followed by a non-ECG-assisted CTA of the abdomen and pelvis. The disadvantage of this approach is the relatively long acquisition time required for the entire thorax (may exceed 15 seconds), which increases the risk of breathing artifacts at the level of the cardiac structures.

#### SIEMENS SOMATOM DEFINITION FLASH AND SOMATOM FORCE

Siemens SOMATOM Flash and Siemens SOMATOM Force systems are dual-source CT systems allowing for a heart rate independent temporal resolution of 75 msec and 66 msec, respectively, when rotation times of 285 msec and 250 msec are employed.

| 1. Topogram | | |
|---|---|---|
| General AP topogram covering the thorax, abdomen, and pelvis including the proximal femoral to the lesser trochanter | Data acquisition • Manufacturers' default setting | |
| 2. CaSc (optional) | | |
| General Can be used for visualization of annular calcification Can be used for planning of subsequent contrast-enhanced data acquisition | Data acquisition Prospective ECG-triggering CARE KV: Off Ref. kVp: 120 kVp CARE dose 4D: On Ref. mAs: 80 mAs/rot Default trigger in end-systole Slice/Collimation: 2 x 128 x 0.6 mm (Flash) 2 x 192 x 0.6 mm (Force) Scan direction cranio-caudal Rotation time: 285 msec (Flash) 250 msec (Force) | Data reconstruction Axial reconstruction within the pulsing window, commonly Best Diast Field of view limited to the heart Slice thickness: 0.75 mm Increment: 0.5 mm Convolution kernel: Heart View medium CaSc B36f (Flash) Qr36 (Force) |
| 3. Premonitoring for Bolus tracking | (CARE Bolus) | |
| General Plan location of pre-monitoring on topogram: 2 cm below carina Alternatively plan pre-monitoring using the CaSC CT data Pre-monitoring using the bold transect through ascending aorta Placeregion of interest (ROI) within the ascending aorta | Data acquisition (manufacturers' default settings) Delay: 2s Effective (eff.) mAs: 120 mAs Effective (eff.) kVp: 120 kVp Slice/Collimation: Acq. 1 x 10.0 mm Cycle time: 1.57s | |
| 4. Monitoring for Bolus tracking (C. | ARE Bolus) | |
| General Same location as pre-monitoring Threshold: Change of 100HU to trigger retrospective ECG-gated spiral data acquisition (#5) | Data acquisition (manufacturers' default settings) Delay: 2s Effective (eff.) mAs: 20 mAs Effective (eff.) kVp: 120 kVp Slice/Collimation: Acq.lx10.0mm Cycle time: 1.57s | |


December 2013, Ver

K1-82

## SIEMENS SOMATOM DEFINITION FLASH AND SOMATOM FORCE (CONT)

#### 5. Retrospective ECG-gated spiral data acquisition - Contrast enhanced

#### General

- ECG-gated dual source data acquisition of the aortic root and heart
- Plan data acquisition on topogram: Scan range beginning 2 cm below the carina to the apex of the heart
- Use unenhanced CaSc CT data for planning if available

#### Data acquisition

- Delay after monitoring has reached threshold: 4 seconds
- Breath hold command: Inspiration only
- CARE KV: On (Dose saving optimized for "vasculature")
- Ref. kVp: 120 kVp
- Reference tube current: 250 mAs/rot
- Anatomical dose modulation: CARE Dose 4D on
- · Pulsing (dose modulation
- throughout cardiac cycle): Off Slice/Collimation: 2 x 128 x 0.6 mm (Flash) 2 x 192 x 0.6 mm (Force)
- Scan direction: Cranio-caudal
- Pitch: automatic (adaption to heart rate)
- Rotation time: 285 msec (Flash) 250 msec (Force)

#### Data reconstruction

- Axial multiphasic reconstruction covering the entire cardiac cycle, 5 or 10% intervals in sinus rhythm, 50 msec intervals in atrial fibrillation
- Use ECG editing if necessary
- Field of view limited to the heart
- Slice thickness: 0.75 mm
- Increment: 0.5 mm
- Medium smooth convolution kernel with either filtered back projection B26f (Flash) Bv40 (Force) or iterative reconstruction (e.g SAFIRE, strength 3, 126f)

#### 6. High-pitch CTA of the thorax, abdomen, pelvis - Contrast enhanced

#### General

- High-pitch ("Flash") dual source data acquisition of the thorax, abdomen, and pelvis
- Scan range: Upper thoracic aperture to the proximal femoral (lesser trochanter)

## Data acquisition

- Delay 5s (minimum delay; needed for repositioning the patient table and adjusting the tube-detector system)
- No additional automated breath hold command; alternatively manual instruction to slowly exhale.
- CARE KV: On (Dose saving optimized for "vasculature")
- Ref. kVp: 100 kVp
- Reference tube current: 200 mAs/rot
- Anatomical dose modulation: CARE Dose 4D on
- · Slice/Collimation: 2 x 128 x 0.6 mm (Flash) 2 x 192 x 0.6 mm (Force)
- · Pitch:
- 3.4 (Flash) 3.2 (Force)
- Rotation time: 285 msec (Flash) 250 msec (Force)

#### Data reconstruction

- Axial reconstructions
- Slice thickness: 0.75 mm
- · Increment: 0.5 mm
- Medium smooth convolution kernel with either filtered back projection B26f (Flash) Bv40 (Force) or iterative reconstruction (e.g SAFIRE/ ADMIRE, strength 3, 126f)

K1-83

#### Contrast application protocol

#### General

- Single contrast application for both the retrospectively ECG-gated CTA of the aortic root/ heart and the CTA of the thorax/abdomen/pelvis
- Placement of an IV access in an antecubital vein (an 18-guage IV typically provides the highest safety)
- Automated contrast injection using a dual-cylinder injector

## Specific

- Contrast bolus monitoring and timing of data acquisition by means of bolus tracking at the level of the ascending acrts with an ROI placed within the ascending acrts; threshold set at 100 HU above baseline, delay to start of data acquisition after reaching threshold 6 sec
- The proposed delay can be considered a default setting and may be increased in patients with por ejection fraction. This may help prevent the highpitch spiral acquisition from outrunning the bolus.


K1-84 Page 204

#### SIEMENS SOMATOM DEFINITION AS64 AND AS+

Siemens SOMATOM Definition AS64 and AS+ are dual-source CT systems for a heart rate independent temporal resolution of 150 msec and 142 msec, respectively, when rotation times of 300 msec and 285 msec are employed.

| 1. Topogram | | |
|---|---|---|
| General • AP topogram view covering the thorax, abdomen, and pelvis including the proximal femoral to the lesser trochanter | Data acquisition • Manufacturers' default setting | |
| 2. CaSc (optional) | | |
| General Can be used for visualization of annular calcification Can be used for planning of subsequent contrast-enhanced data acquisition | Data acquisition Prospective ECG-triggering CARE KV: Off Ref. kVp: 120 kVp CARE dose 4D: On Ref. mAs: 80 mAs/rot Default trigger in end-systole Slice/Collimation: 64 x 0.6 mm (AS64) 128 x 0.6 mm (AS+) Scan direction: Cranio-caudal Rotation time: 300 msec (AS64) 285 msec (AS6+) | Data reconstruction Axial reconstruction within the pulsing window, commonly Best Diast Field of view limited to the heart Slice thickness: 0.75 mm Increment: 0.5 mm Convolution kernel: B35f Heart View medium CaSc |
| 3. Pre-monitoring for Bolus tracking | (CARE Bolus) | |
| General Plan location of pre-monitoring on topogram: 2 cm below carina Alternatively plan pre-monitoring using the CaSc CT data. Pre-monitoring should transect through assending aorta. Place ROI within the ascending aorta | Data acquisition (manufacturers' default settings) Delay: 2s Effective (eff.) mAs: 20 mAs Effective (eff.) kVp: 120 kVp Slice/Collimation: Acq. 1 x 10.0 mm Cycle time: 1.16s | |
| 4. Monitoring for Bolus tracking (CA | AREBolus) | |
| General Same location as pre-monitoring Threshold: Change of 100HU to trigger retrospective ECG-gated spiral data acquisition (#5) | Data acquisition (manufacturers' default settings) Delay: 10s Effective (eff.) mAs: 20 mAs Effective (eff.) kVp: 120 kVp Slice/Collimation: Acq. 1 x 10.0 mm Cycle time: 1.16s | |

#### 5. Retrospective ECG-gated spiral data acquisition - Contrast enhanced

#### General

- · ECG-gated data acquisition of
- the aortic root and heart · Plan data acquisition on topogram: Scan range beginning 2 cm below the carina to the apex of the heart
- Use unenhanced CaSc CT data for planning if available

## Data acquisition

- · Delay after monitoring has
- reached threshold: 7 seconds Breath hold command:
- Inspiration only CARE KV: On (Dose saving optimized for "vasculature")
- Ref. kVp: 120 kVp
  - Reference tube current: 250 mAs/rot
  - Anatomical dose modulation: CARE Dose 4D on
  - Pulsing (dose modulation throughout cardiac cycle): Off
  - Slice/Collimation: 64 x 0.6 mm (AS64) 128 x 0.6 mm (AS+)
  - Scan direction: Cranio-caudal
- · Pitch: Automatic (adaption to heart rate)
- Rotation time: 300 msec (AS64) 280 msec (AS+)

#### Data reconstruction

- Axial multiphasic reconstruction covering the entire cardiac cycle, 5 or 10% intervals in sinus rhythm, 50 msec intervals in atrial fibrillation
- Use ECG editing if necessary
- Field of view limited to the heart
- Slice thickness: 0.75 mm
- Increment: 0.5 mm
- Medium smooth convolution kernel with either filtered back projection (B26f) or iterative reconstruction (e.g SAFIRE, strength 3, I26f)

## 6. CTA of the thorax/abdomen/pelvis - Contrast enhanced

### General

· Scan range: Upper thoracic aperture to the proximal femoral (lesser trochanter)

## Data acquisition

- (manufacturers' default settings) Delay 5s (minimum delay; needed for repositioning of the patient table and adjusting the tube-detector system)
- No additional automated breath hold command; alternatively manual instruction
- to slowly exhale.
  CARE KV: On (Dose saving optimized for "vasculature")
- Ref. kVp: 100 kVp · Reference tube current: 200 mAs/rot
- · Anatomical dose modulation:
- CARE Dose 4D on · Slice/Collimation:
- 64 x 0.6 mm (AS64) 128 x 0.6 mm (AS+) · Scan direction: Cranio-caudal
- · Pitch: 1.45
- Rotation time: 300 msec (AS64) 285 msec (AS+)

#### Data reconstruction

- Axial reconstructions
- Slice thickness: 0.75 mm Increment: 0.5 mm
- Medium smooth convolution kernel with either filtered back projection (B26f) or iterative reconstruction (e.g SAFIRE, strength 3, I26f)

PARTNER 3


K1-85


#### Contrast application protocol

#### General

- Single contrast application for both the retrospectively ECG-gated CTA of the aortic root/ heart and the CTA of the thorax/abdomen/pelvis
- Placement of IV access in an antecubital vein (an 18-guage IV typically provides the highest safety)
- Automated contrast injection using a dual-cylinder injector

## Specific

Contrast bolus monitoring and timing of data acquisition by means of bolus tracking at the level of the ascending a orta with a ROI placed within the ascending acut; threshold set at 100 HU above baseline, delay to start of data acquisition after reaching threshold? see

#### LOW-CONTRAST DOSE PROTOCOL - RATIONALE FOR ALL SCANNER TYPES

- · Same scanner settings as listed above, except the threshold setting for bolus tracking
- Reduce scan length of the retrospectively ECG-gated CTA(#5) to a minimum to cover
  only the aortic root as opposed to the entire heart, as this is the time-intensive partin
  recard to data acquisition
- Injection rate might be lowered
- Threshold to trigger initiation of the retrospective ECG-gated spiral data acquisition can be lowered to 80 HU
- Systems with the capability of low kV data acquisition (70kV-90kV, Force) may allow for reduced iodine delivery rates as low kV data acquisition increases iodine attenuation; CARE KV settings need to be adjusted (setting 4-7).

These alterations should allow for a sufficiently contrast-enhanced CT dataset of the aortic root. Contrast attenuation of the iliofemoral acquisition may be variable.

# DOSE MODULATION FOR RETROSPECTIVE ECG-GATED SPIRAL DATA ACQUISITION

The protocols listed above do not employ dose modulation for the retrospective ECG-gated spiral data acquisition, allowing for image reconstructions throughout the entire cardiac cycle at a constant image noise level. This allows for identifying the reconstruction phase with largest annular dimensions and optimal image quality. If dose modulation is employed, peak dose should be applied during systole with a pulsing window set to 5–35%. MinDOSE should not be used, as this renders images non-interpretable outside of the pulsing window.

#### RECONSTRUCTION OF MULTIPHASIC DATA SET

Multiphasic ("dynamic", "cine") data sets can be reconstructed using a relative approach (percentage intervals [%] between two R-peaks) or an absolute approach (fixed distance of the reconstruction window from the R-peak, reported as [msec]).

The relative approach (e.g. 5 or 10% intervals) performs well in regular sinus rhythm. In case of increased heart rate variability, atrial fibrillation, or ectopic beats, absolute reconstruction should be employed (e.g. 50 msec) in combination with ECG-editing if necessary.

CAVEAT: "Best Diastole" and "Best Systole" are algorithms which aim at automated identification of optimal reconstruction phases with the least coronary artery motion in Diastole or Systole. However, these algorithms are intended for coronary CTA and not aortic root imaging.

#### REVIEW OF DATA RECONSTRUCTION AND ECG-EDITING

- Image reconstructions of the aortic root and heart should be reviewed immediately
  after the scan when raw data is still available
- The ECG-gating should be reviewed to ensure that the automated algorithms correctly identified the R-peaks (dots, also known as "Syncs" should be aligned with R-peaks)
- If R-peaks were not correctly identified, manual correction should be performed (e.g. "Insert Sync" if an R-peak was not identified, or "Delete Sync" if a Sync was placed on anything other than the R-peak; alternatively Syncs can also be shifted manually)
- In case of ectopic contractions, absolute reconstruction should be used and the Sync of the ectopic beat should be deleted



If mis-registration or stair-step artifacts are present, ECG-editing should be
employed with either modification of trigger-points (if they were initially incorrectly
identified by the algorithm) or deletion of trigger-points (in premature contraction
or attrial fibrillation).


K1-87


## Written in collaboration with:

# SIEMENS

#### References

- Achenbach S, Delgado V, Hausleiter J, et al. SCOT expert consensus document on computed tomography imaging before transcatheter acrtic valve implantation (TAVI)/transcatheter acrtic valve replacement (TAVR). J Cardiovasc Comput Tomogr 2012:6(6)866-380.
- Blanke P, Bulla S, Baumann T, et al. Thoracic Aneta-Prospective Electrocardiographically Triggered OT Angiography with Dual-Source OT-Feasibility, Image Quality, and Dose Reduction. Radiology 2010;255(1):207-217.
- 3. Blanke P, Russe M, Leipsic J, et al. Conformational Pulsatile Changes of the Aortic Annulus. JACC Cardiovasc Imaging 2012;5(9):984-994.
- 4. Blanke P, Schoepf UJ, Leipsic J. CT in Transcatheter Aortic Valve Replacement. Radiology 2013:269(3):650-669.
- Gurvitch B. Wood DA, Leipzic J, et al. Multiclice Computed Tomography for Prediction of Optimal Angiographic Deployment Projections During Transcatheter Acrtic Valve Implantation. JACC Cardiovacc Imaging 2010;3(11):1187-1185.
- 6. Leipsic J, Gurvitch B, LaBounty TM, et al. Multidetector Computed Tomography in Transcatheter Acrtic Valve Implantation. JACC Cardiovasc Imaging 2011:4(4):416-429.
- Litmanovich DE, Ghersin E, Burke DA, et al. Imaging in Transcatheter Aortic Valve Replacement (TAVR): role of the radiologist. Insights Imaging 2014; S:123-145.

Edwards, Edwards Lifesciences, and the stylized E logo are trademarks of Edwards Lifesciences Corporation. All other trademarks are the property of their respective owners.

© 2015 Edwards Lifesciences Corporation. All rights reserved. PP-ALL-0018 v3.0 E5665/6-15/THV

© Siemens Healthcare GmbH, 2015

## Edwards Lifesciences | edwards.com

One Edwards Way | Irvine, California 92614 USA Switzerland | Japan | China | Brazil | Australia | India



# CT Acquisition and Reconstruction Techniques for Transcatheter Aortic Valve Procedure Planning Utilizing Toshiba Hardware

#### WRITTEN IN COLLABORATION WITH:

## TOSHIBA

Leading Innovation >>>

#### EDITED BY:

Philipp Blanke, MD, FSCCT Cardiac Imaging Specialist Center for Heart Valve Innovation St. Paul's Hospital & University of British Columbia Vancouver

Erin Fletcher RN, BSN, RCIS Global Product Training Manager Imaging, Procedure, and Patient Initiatives Edwards Lifesciences, THV – Global

Matt Fernandes R.T. (R)(CT) Marketing Clinical Support Specialist, CT Toshiba America Medical Systems




K1-89


This paper is provided as an educational resource to medical personnel by Edwards Lifesciences and Toshiba. The information in this white paper has been compiled from available literature. Although every effort has been made to fauthfully report the information, the editors and publisher cannot be held responsible for the correctness. This paper is not intended to be and should not be construed as medical advice. For any use, the product information guides, inserts, and operation manuals of the various drugs and devices should be consulted. Edwards Lifesciences, Toshiba, and the editors disclaim any liability arising directly or indirectly from the use of drugs, devices, techniques, or procedures described in this paper.

WARNING: Any reference to X-ray exposure, intravenous contrast dosage, and other medication is intended as a reference guideline only. The guidelines in this document do not substitute for the judgment of a health care provider. Each scan requires medical judgment by the health care provider about exposing the patient to ionizing radiation. Use the As Low As Reasonably Achievable (ALARA) radiation dose principle to balance factors such as the patient's condition, size, and age; region to be imaged; and diagnostic task.

NOTE: Algorithms/protocols included in this paper are for educational reference only. Edwards does not endorse or support any one specific algorithm/protocol. It is up to each individual clinician and institution to select the treatment that is most appropriate.

Philipp Blanke, MD is a paid consultant for Edwards Lifesciences.


## INTRODUCTION

Transcatheter aortic valve procedures have proven to be an effective alternative in the treatment of aortic stenosis in high risk and inoperable patients. Contrast enhanced computed tomography (CT) has become an integral part of transcatheter aortic valve procedure planning by allowing for anatomical assessment of the aortic root and the aorto-iliofemoral vasculature within a single examination. It is critical that artifact free image data is obtained to allow for reliable anatomical measurements. Data acquisition strategies and scanning protocols may vary depending on scanner manufacturer, system, and institutional preferences. This document provides recommendations for reliable CT image acquisition for transcatheter aortic valve procedures.

K1-91 PARTNER 3

#### WORK-FLOW RATIONALE

The key component of all approaches is an ECG-assisted data acquisition that covers at least the aortic root, while the remainder of the data acquisition may be performed without ECG assistance. If employed properly, ECG assistance allows for artifact-free depiction of the aortic root. The sequence of patient preparation and the relevant principles of CT data acquisition will be explained in brief below.

#### PATIENT PREPARATION

- Position the patient, typically supine, on the scanner table to closely resemble catheterization table positioning. This is important for the prediction of C-arm angulation from the CT dataset.
- · Place ECG-electrodes and IV access in accordance with institutional policies.
- Provide time for the patient to practice the breath hold prior to scan acquisition, as it
  may significantly improve patient compliance and thereby scan quality.
- Plan additional scanning and instruction time as needed, due to the advanced age and frailty of this patient population.

#### CT SCAN - SCAN LENGTH AND SCAN STRATEGY

In general, two different approaches are used to combine the ECG-assisted data acquisition of the sortic root structures and the non-ECG-assisted computed tomography angiography (CTA) of the sorto/ilio/femoral vasculature for evaluation of the transfemoral access route:

- 1) Cardiac ECG-assisted data acquisition of the heart and aortic root (usually beginning 2 cm below the carina) followed by a non-ECG-assisted CTA of the thorax, abdomen, and pelvis. Although this approach results in repeat data acquisition of the aortic root and cardiac structures, the time-intensive ECG-assisted data acquisition is kept to a minimum that aids in limiting the contrast dose. Furthermore, limiting the ECG-assisted data acquisition also limits the radiation dose intensive component of the examination, although the cardiac scan range is covered twice. The proposed protocols for the Aquilion ONE Family and the Aquilion PRIME and Aquilion 64/VeloCT 128 Families without variable helical pitch (VHP) use this approach.
- 2) ECG-assisted data acquisition of the thorax followed by a non-ECG assisted CTA of the abdomen and pelvis. The disadvantage of this approach is the relatively long acquisition time required for the entire thorax (may exceed 15 seconds), increases the risk of breathing artifacts at the level of the cardiac structures. The proposed protocols for the Aquilion PRIME Family and Aquilion 64/VeloCT 128 Family utilities with (was this approach.

TOSHIBA - AQUILION ONE 640/AQUILION ONE VISION

#### 1. Scanogram General Data acquisition · AP/LAT Scanogram covering · AP Scanogram: the thorax, abdomen, and 120 kVp/50 mA pelvis including the proximal LAT Scanogram: femoral to the lesser trochanter 120 kVp/100 mA 2. Non-enhanced scan (optional) - Calcium Score Data acquisition Data reconstruction General · Can be used for quantification Acquisition mode: Ca Score Field of View limited to the of annular calcification Volume Mode heart (220 mm) · Can be used for planning of · Tube voltage: 120 kVp Slice thickness 0.5 mm subsequent contrast-enhanced Tube current: SURE Exposure Increment 0.25 mm R-R Scanning Window: data acquisition SUREIQ: Ca Score (FC 12) HR<71 bpm (75%); HR>71 · Volume data can be acquired as a single-beat/one rotation bpm (40%) (determined by scanner) Slice/Collimation: 0.5/240 (120 mm)Rotation time Aquilion ONE 640: 350 msec Aquilion ONE ViSION: 275 msec 3. S&V Scan and View General Data acquisition Plan location of SURE Start (manufacturers' default settings) on AP Scanogram view: Delay: 0 seconds · Tube current: 50 mA Center of volume Placeregion of interest (ROI) · Tube voltage: 120 kVp within the descending aorta Slice/Collimation: 0.5 mm x4 · Rotation Time: Aquilion ONE 640: 350 msec Aquilion ONE ViSION: 275 msec 4. Bolus tracking - SUREStart General Data acquisition (manufacturers' default settings) Same location as #3 Threshold: 300 HU · Delay: 10 seconds · Tubecurrent:50mA · Tube voltage: 100 kVp Slice/Collimation: 0.5 mm x4 · Rotation Time: Aquilion ONE 640: 350 msec Aguilion ONE ViSION: 275 msec Cycle time/repetition: 2 second intermittent interval Voicetiming: 14 seconds PARTNER 3


K1-94

#### TOSHIBA - AQUILION ONE 640/AQUILION ONE VISION (CONT)

#### 5. ECG-assisted cardiac data acquisition - Contrast enhanced

#### General

- · ECG-assisted data acquisition of the aortic root and heart as a single beat/one rotation scan
- Plan volume acquisition on scanogram view: Scan range beginning 1 cm below the carina to the apex of the heart
- Use unenhanced CaSc CT data for planning if available
- Set medium FOV (320 mm) -Must match helical CTA

#### Data acquisition

- No delay after monitoring has reached threshold (system starts immediately with data acquisition)
- Breath hold command: Inspiration only (Breath command set in SUREStart at 14 seconds after beginning of contrast injection)
- Tubevoltage: 100 kVp
- Tube current: SURE Exposure (automatically selects the tube current based on the patient size)
- Target mode set to 50% and exposure window set to 1000 msec will ensure full R-R scan. The exposure time can be adjusted based upon HR. This is a single beat/one rotation scan
- Slice/Collimation: Configured based upon desired scanlength (0.5x240/0.5x280/0.5x320)
- Rotation time: Aguilion ONE 640: 350 msec Aguilion ONE VISION: 275 msec

- Axial multiphasic reconstruction covering the entire cardiac cycle in 5% or 10% intervals
- Use ECG editing if necessary Field of View limited to the heart (220 mm)
- Slice thickness: 0.5 mm

Data reconstruction

- Increment: 0.25 mm SUREIQ: Cardiac CTA (FC 03)
- Iterative reconstruction: ATDR 3D

## 6. CTA of the thorax/abdomen/pelvis - Contrast enhanced

## General

- · Scan range: Upper thoracic aperture to the proximal femoral (lesser trochanter)
- Set medium FOV (320 mm) -Must match volume scan

## Data acquisition

- Delay: 6 seconds (minimum delay needed to reposition scanner and continue with non-gated acquisition)
- No additional automated breath hold command; alternatively manual instruction to slowly exhale
- Tubevoltage: 100 kVp Tube current: SURE Exposure (automatically selects the tube
- current based on the patient size) Slice/Collimation: 0.5 mmx80
- Scan direction: Cranio-caudal
- Pitch: Fast
- Rotation time: AquilionONE 640:350 msec Aguilion ONE VISION: 275 тес

#### Data reconstruction

- · Slice thickness: 1.0 mm
- · Increment: 0.8 mm
- SUREIQ: CTA Body FC 08
- Iterative reconstruction: AIDR 3D

## Contrast application protocol

#### General

- · Single contrast application for both the ECGassisted as a single beat/one rotation scan of the aortic root/heart and the CTA of the thorax/ abdomen/pelvis
- · Placement of IV access per institutional protocol (an 18-guage IV typically provides the highest safety)
- Automated contrast injection using a dual-cylinder injector

#### Specific

- Recommended contrast media application: 50-90 cciodinated contrast medium at
- Contrast bolus monitoring and timing of data acquisition by means of bolus tracking at the level of the descending acrts with an ROI placed within the descending aorta; threshold set at 250 HU

#### RECOMMENDATIONS FOR A LOW-CONTRAST PROTOCOL

- Use lower range of total amount of contrast (50 cc)
- · Place ROI for bolus tracking (SURSStart) in ascending acrts as this decreases the delay between contrast administration/arrival to the start of the data acquisition
- Athreshold of 250 HU ensures a contrast attenuation of at least 250 HU in the aortic root, however with 50 cc of contrast, attenuation of the non-gated scan may be variable

#### TOSHIBA - AQUILION PRIME WITH VARIABLE HELICAL PITCH (vHP OPTIONAL)

#### 1. Scanogram General Data acquisition · APScanogram: AP/LAT Scanogram covering the thorax, abdomen, and 120 kVp/50 mA pelvis including the proximal LAT Scanogram: femoral to the lesser trochanter 120 kVp/100 mA

## 2. Non-enhanced scan (optional) - Calcium Score

## General

- · Can be used for quantification of annular calcification
- · Can be used for planning of subsequent contrast-enhanced data acquisition

## Data acquisition

- Tube voltage: 120 kVp

## Acquisition mode:

- Scan & Scan (sequential mode)
- R-R Scanning Window:
- Sequential scan using step and shoot mode
- Tube current: SURE Exposure
- HR<71 bpm (75%): HR>71 bpm (40%)
- Slice/Collimation: 3.0 mmx4
- Rotation time: 350 msec

## Data reconstruction

- Field of View limited to the heart(220mm) Slice thickness: 0.5 mm
- Increment: 0.25 mm
- SUREIQ: Ca Score (FC 12)

## 3. S&V Scan and View

## General

- · Plan location of SUREStart on APScanogram view: 1cm below carina
- · Place region of interest (ROI) within the descending acrts

## Data acquisition (manufacturers' default settings)

- Delay: 0 seconds Tubecurrent: 50 mA
- · Tube voltage: 120 kVp
- Slice: 0.5 mmx4
- Rotation Time: 350 msec

#### PARTNER 3


#### TOSHIBA - AQUILION PRIME WITH VARIABLE HELICAL PITCH (vHP, OPTIONAL) (CONT)

#### 4. Bolus tracking - SUREStart General Data acquisition · Same location as #3 (manufacturers' default settings) · Threshold: 180 HU · Delay: 10 seconds Tubecurrent: 50 mA Tube voltage: 100 kVp Slice/Collimation: 0.5 mmx4 Rotation Time: 350 msec · Cycle time/repetition: 2 second intermittent interval 5. ECG-gated thoracic data acquisition and non-gated data acquisition of the abdomen and pelvis-Contrast enhanced General Thoracic Data acquisition Data reconstruction · Utilize vHP (optional scan · Delay after monitoring has Axial multiphasic mode on Aquilion PRIME reached threshold: 5 seconds reconstruction covering the family of CT scanners) Breath hold command: entire cardiac cycle in 5% or · Allows for one helical scan/ Inspiration only 10% intervals one breath hold combining Tube voltage: 100 kVp Use ECG editing if necessary gated thoracic and non-· Tube current and anatomical FieldofViewlimitedtothe gated abdominal/pelvic data dose modulation: SURE Exposure heart (220 mm) XYZModulation Slice thickness: 0.5 mm acquisition Plan helical scan from above Helical retrospectively ECG · Increment: 0.25 mm apices of the proximal femoral gated mode using vHP SUREIQ: Cardiac CTA (FC 03) to the lesser trochanter Slice/Collimation: 0.5 mmx80 Iterative reconstruction: The retrospectively ECG-gated Rotation time: 350 msec AIDR 3D helical acquisition should be Pitch: Cardiac (automatically set to start above lung apices to set by SURE Cardio) below apex of the heart Abdominal/Pelvic Data acquisition Data reconstruction · Tube voltage: 100 kVp Slice thickness: 1.0 mm · Tube current and anatomical · Increment: 0.8mm SURBIQ: CTA Body (FC 08) dose modulation: SURE Exposure XYZ Modulation Iterative reconstruction: Slice/Collimation: 0.5 mmx80 AIDR 3D Scan direction: Cranio-caudal Pitch: Standard · Rotation time: 350 msec Contrast application protocol

## General

- Single contrast application for both the retrospectively ECG-gated CTA of the acrtic root/ heart and the CTA of the thorax/abdomen/pelvis
- Placement of IV access per institutional protocol (an 18-guage IV typically provides the highest safety)
- Automated contrast injection using a dual-cylinder injector

## Specific

- Recommended contrast media application: 90 cc iodinated contrast medium at 4 cc/sec
- Contrast bolus monitoring and timing of data acquisition by means of bolus tracking at the level of the descending aorta with an ROI placed within the descending aorta; threshold set at 180 HU

K1-97

#### TOSHIBA - AQUILION PRIME WITHOUT VARIABLE HELICAL PITCH (vHP)

| General | Data acquisition | |
|---|---|---|
| AP/LAT Scanogram covering | · AP Scanogram: | |
| the thorax, abdomen, and | 120 kVp/50 mA | |
| pelvis including the proximal | · LAT Scanogram: | |
| femoral to the lesser trochanter | 120 kVp/100 mA | |
| 2. Non-enhanced scan (optional) – C | Calcium Score | |
| General Can be used for quantification of annular calcification Can be used for planning of subsequent contrast-enhanced data acquisition | Data acquisition Acquisition mode: Scan & Scan (sequential mode) Tube voltage: 120 kVp Tube current: SURRE Exposure R.R. Scanning Window: HR<71 bpm (75%); HR>71 bpm (40%) Slice/Collimation: 3.0 mmx4 Rotation time: 350 mass. | Data reconstruction Field of View limited to the heart (220 mm) Slice thickness: 0.5 mm Increment: 0.25 mm substitute: 0.25 mm Substitute: 0.25 mm |
| | Notation time: 350 msec | |
| 3. S&V Scan and View | · Rotation time: 350 msec | |
| 3. S&V Scan and View General | Data acquisition | |
| General Plan location of SURES tart on AP Scanogram view: 1cm | Data acquisition (manufacturers' default settings) • Delay: 0 seconds | |
| General Plan location of SUREStart on AP Scanogram view: 1cm below carina | Data acquisition (manufacturers' default settings) Delay: 0 seconds Tubecurrent: 50 mA | |
| General Plan location of MRES Start on AP Scanogram view: 1cm below carina Place ROI within the | Data acquisition (manufacturers' default settings) • Delay: 0 seconds • Tube current: 50 mA • Tube voltage: 120 kVp | |
| General Plan location of SUREStart on AP Scanogram view: 1cm below carina | Data acquisition (manufacturers' default settings) • Delay: 0 seconds • Tube current: 50 mA • Tube voltage: 120 kVp • Slice/Collimation: 0.5 mmx4 | |
| General Plan location of MRES Start on AP Scanogram view: 1cm below carina Place ROI within the | Data acquisition (manufacturers' default settings) • Delay: 0 seconds • Tube current: 50 mA • Tube voltage: 120 kVp | |
| General Plan location of MURSS start on AP Scanogram view: 1cm below carina Place ROI within the descending acrta | Data acquisition (manufacturers' default settings) • Delay: 0 seconds • Tube current: 50 mA • Tube voltage: 120 kVp • Slice/Collimation: 0.5 mmx4 | |
| General Plan location of SURESStart on AP Scanogram view: 1cm below carina Place ROI within the descending aorta 4. Bolus tracking - SUREStart General | Data acquisition (manufacturers' default settings) Delay: 0 seconds Tube current: 50 mA Tube voltage: 120 kVp Slice/Collimation: 0.5 mmx4 Rotation Time: 350 msec | |
| General Plan location of SURES Start on AP Scanogram view: 1cm below carina Place ROI within the descending aorta Bolus tracking - SURES Start General Same location as #3 | Data acquisition (manufacturers' default settings) Delay: 0 seconds Tube current: 50 mA Tube voltage: 120 kVp Slice/Collimation: 0.5 mmx4 Rotation Time: 350 msec | |
| General Plan location of SURESStart on AP Scanogram view: 1cm below carina Place ROI within the descending aorta 4. Bolus tracking - SUREStart General | Data acquisition (manufacturers' default settings) Delay: 0 seconds Tube current: 50 mA Tube voltage: 120 kVp Slice/Collimation: 0.5 mmx4 Rotation Time: 350 msec Data acquisition (manufacturers' default settings) Delay: 10 seconds | |
| General Plan location of SURES Start on AP Scanogram view: 1cm below carina Place ROI within the descending aorta Bolus tracking - SURES Start General Same location as #3 | Data acquisition (manufacturers' default settings) Delay: 0 seconds Tube current: 50 mA Tube voltage: 120 kVp Slice/Collimation: 0.5 mmx4 Rotation Time: 350 msec Data acquisition (manufacturers' default settings) Delay: 10 seconds Tube current: 50 mA | |
| General Plan location of SURES Start on AP Scanogram view: 1cm below carina Place ROI within the descending aorta Bolus tracking - SURES Start General Same location as #3 | Data acquisition (manufacturers' default settings) Delay: 0 seconds Tube voltrage: 120 kVp Slice/Collimation: 0.5 mmx4 Rotation Time: 350 msec Data acquisition (manufacturers' default settings) Delay: 10 seconds Tube current: 50 mA Tube voltrage: 100 kVp | |
| General Plan location of SURES Start on AP Scanogram view: 1cm below carina Place ROI within the descending aorta Bolus tracking - SURES Start General Same location as #3 | Data acquisition (manufacturers' default settings) Delay: 0 seconds Tube current: 50 mA Tube voltage: 120 kVp Slice/Collimation: 0.5 mmx4 Rotation Time: 350 msec Data acquisition (manufacturers' default settings) Delay: 10 seconds Tube current: 50 mA Tube voltage: 100 kVp Slice/Collimation: 0.5 mmx4 | |
| General Plan location of SURES Start on AP Scanogram view: 1cm below carina Place ROI within the descending aorta Bolus tracking - SURES Start General Same location as #3 | Data acquisition (manufacturers' default settings) Delay: 0 seconds Tube voltrage: 120 kVp Slice/Collimation: 0.5 mmx4 Rotation Time: 350 msec Data acquisition (manufacturers' default settings) Delay: 10 seconds Tube current: 50 mA Tube voltrage: 100 kVp | |


TOSHIBA - AQUILION PRIME WITHOUT VARIABLE HELICAL PITCH (vHP) (CONT)

#### 5. ECG-gated data acquisition of the aortic root/heart

#### General

· Retrospectively ECG-gated helical acquisition of the aortic root and heart.

#### ECG-gated Data acquisition of the aortic root and heart

- Delay after monitoring has reached threshold: 5 seconds
- Breath hold command: Inspiration only
- Tube voltage: 100 kVp
- Tube current and anatomical dose modulation: SURE Exposure XYZModulation
- Helical retrospective ECG Gated mode
- Slice/Collimation: 0.5 mmx80
- · Rotation time: 350 msec
- · Pitch: Cardiac (set by SURE Cardio)

## Data reconstruction

- Axial multiphasic reconstruction covering the entire cardiac cycle, 5% or 10% intervals in sinus rhythm
- · Use ECG editing if necessary Field of View limited to the
- heart (220 mm) Slice thickness: 0.5 mm
- · Increment: 0.25 mm
- · surs IQ: Cardiac CTA (FC 03)
- Iterative reconstruction:
- AIDR 3D

### 6. CTA of the thorax/abdomen/pelvis - Contrast enhanced

· Non-gated data acquisition of the thorax, abdomen, and pelvis immediately following the prior data acquisition

#### Thorax/Abdominal/Pelvic Data acquisition

- Delay prior to scan scans: 7 seconds (minimum delay needed to reposition scanner and continue with non-gated acquisition)
- No additional automated breath hold command; alternatively manual instruction to slowly exhale
- Tube voltage: 100 kVp
- · Tube current and Anatomical dose modulation: SURE Exposure XYZModulation
- Slice/Collimation: 0.5 mmx80
- · Scan direction: Cranio-caudal
- · Pitch: Standard
- · Rotation time: 350 msec

## Data reconstruction

- Slice thickness: 1.0mm Increment: 0.8 mm
- SURE IQ: CTA Body (FC 08)
- Iterative reconstruction: AIDR 3D

Contrast application protocol

- · Single contrast application for both the retrospectively ECG-gated CTA of the aortic root/ heart and the CTA of the thorax/abdomen/pelvis
- · Placement of IV access per institutional protocol (an 18-guage IV typically provides the highest safety)
- Automated contrast injection using a dual-cylinder injector

- Recommended contrast media application: 80 100 cc iodinated contrast medium at 4 cc/sec
- Contrast bolus monitoring and timing of data acquisition by means of bolus tracking at the level of the descending acrts with an ROI placed within the descending aorta; threshold set at 180 HU

TOSHIBA - AQUILION 64 AND AQUILION VELOCT 128 WITH vHP

## 1. Scanogram

#### General

· AP/LAT Scanogram covering the thorax, abdomen, and pelvis including the proximal femoral to the lesser trochanter

#### Data acquisition APScanogram:

- 120 kVp/50 mA LAT Scanogram:
- 120 kVp/100 mA

#### 2. Non-enhanced scan (optional) - Calcium Score

#### General

- · Can be used for quantification of annular calcification
- · Canbe used for planning of subsequent contrast-enhanced data acquisition

#### Data acquisition

- Acquisition mode Scan & Scan (sequential mode)
  - Tube voltage: 120kVp
- Tube current: 300mA (Aquilion 64), SURE Exposure (Velo CT 128)
- R-R Scanning Window: HR<71 bpm (75%); HR>71 bpm (40%)
- Slice/Collimation: 3.0 mmx4
- Rotation time: 400 msec, 350 msec (optional)

## Data reconstruction

- Field of View limited to the heart (220mm)
- Slice thickness: 0.5mm
- Increment: 0.25mm
- · SUREIQ: Ca Score (FC12)

#### 3. S&V Scan and View

#### General

- Plan location of SURE Start on AP Scanogram view: 1 cm below carina
- Placeregion of interest (ROI) within the descending aorta

#### Data acquisition (manufacturers' default settings)

- Delay: 0 seconds
- Tube current: 50 mA
- Tube voltage: 120 kVp
- Slice/Collimation: 0.5 mm x4
- Rotation time: 400 msec (350 msec optional)

## 4. Bolus tracking - SUREStart

#### General

- Same location as #3
- · Threshold: 180 HU

## Data acquisition (manufacturers' default settings)

- Delay: 10 seconds
- · Tube current: 50 mA
- · Tube voltage: 100 kVp
- Slice/Collimation: 0.5 mmx4
- Rotation time: 400 msec (350 msecoptional)
- Cycletime/repetition: 2 second intermittent interval


K1-99


K1-100 Page 212

TOSHIBA - AQUILION 64 AND AQUILION VELOCT 128 WITH vHP (CONT)

#### 5. ECG-gated thoracic data acquisition and non-gated data acquisition of the abdomen and pelvis-Contrast enhanced

## General

- Utilize Variable Helical Pitch (vHP)vHPisanoptional scan mode on Aquillion 64 and Aquilion VeloCT 128 CT scanners
- Allows for one helical scan/one breath hold combining gated/ non-gated data acquisition.
- Plan helical scan from above apices to below ischium. The retrospectively ECG-gated helical acquisition should be set to start above lung apices to below apex of the heart

## Thoracic Data acquisition

- Delay after monitoring has reached threshold: 5 seconds. Breath hold command:
- Inspiration only Tube voltage 100 kVp
- Tube current: fixed tube current adjusted to BMI. e.g. 400mA (Aquilion 64), SURE Exposure XYZ Modulation (Velo CT 128)
- Helical retrospective ECG Gated mode using vHP
- Slice/Collimation: 0.5x64 Rotation time: 400 msec.
- 350msec (optional) Pitch: Cardiac (Set by SURE Cardio)

## Abdominal/Pelvic Data acquisition

- Tube voltage 100 kVp
- · Tube current and Anatomical dose modulation: SURE Exposure XYZModulation
- Slice/Collimation: 0.5x64 Scan direction: cranio-caudal
- Pitch: Standard
- Rotation time: 350 msec

## Data reconstruction

- Axial multiphasic reconstruction covering the entire cardiac cycle, 5% or 10% intervals in sinus rhythm
- Use ECG editing if necessary Field of View limited to the heart
- Slice thickness- 0.5 mm
- Increment = 0.25 mm <sup>SURE</sup>IQ: Cardiac CTA FC 03 (Velo CT 128), FC 43 (Aquilion 64)
- Quantum De-noising Software (QDS +) (Aquilion 64)
- Boost 3D (Aquilion 64)
- Iterative reconstruction -
- AIDR 3D (Velo CT 128)

### Data reconstruction

- Axial reconstructions 3mmx3mm
- Slice thickness thin 1.0mm · Increment - 0.8mm
- SUREIQ: CTA Body FC 08
- Quantum De-noising Software
- (QDS +) (Aquilion 64)
- Boost 3D (Aquilion 64)
- Iterative reconstruction -AIDR 3D (Velo CT 128)

#### Contrast application protocol

· Non-gated data acquisition

of the thorax, abdomen, and

General

pelvis.

- · Single contrast application for both the retrospectively ECG-gated CTA of the aortic root/ heart and the CTA of the thorax/abdomen/pelvis
- placement of IV access per hospital protocol (an 18-guage IV typically provides the highest safety)
- automated contrast injection using a dual-cylinder injector

#### Specific

- Recommended contrast media application: 90 cc iodinated contrast medium at 4 cc/sec
- Contrast bolus monitoring and timing of data acquisition by means of bolus tracking at the level of the descending acrts with a region of interest placed within the descending acrts; threshold set at 180 HU.

#### TOSHIBA - AQUILION 64 AND AQUILION VELOCT 128 WITHOUT vHP

#### 1. Scanogram

#### General

· AP/LAT Scanogram covering the thorax, abdomen, and pelvis including the proximal femoral to the lesser trochanter

## Data acquisition

- AP Scanogram:
- 120 kVp/50 mA LAT Scanogram: 120 kVp/100 mA

#### 2. Non-enhanced scan (optional) - Calcium Score

#### General

- · Can be used for quantification of annular calcification
- · Canbe used for planning of subsequent contrast-enhanced data acquisition

#### Data acquisition

- Acquisition mode Scan & Scan (sequential mode)
- Tube voltage: 120 kVp
- Tube current: 300mA (Aquilion 64), SURE Exposure (Velo CT 128)
- R-R Scanning Window: HR<71 bpm (75%); HR>71 bpm (40%)
- Slice/Collimation: 3.0 mm x4
- Rotation time: 400 msec (350 msec optional)

## Data reconstruction

- Field of View limited to the heart(220mm)
- Slice thickness 0.5 mm
- Increment 0.25 mm
- · SUREIQ: Ca Score (FC 12)

## 3. S&V Scan and View

#### General

- Plan location of SURE Start on AP Scanogram view: 1 cm below carina
- · Place ROI within the descending aorta

## Data acquisition (manufacturers' default settings)

- Delay: 0 seconds
- Tube current: 50 mA
- Tube voltage: 120 kVp
- Slice/Collimation: 0.5 mm x4
- Rotation time: 400 msec
- (350 msec optional)

## 4. Bolus tracking - SUREStart

#### General

 Same location as #3 · Threshold: 180 HU

## Data acquisition (manufacturers' default settings)

- Delay: 10 seconds
- · Tube current: 50 mA
- · Tube voltage: 100 kVp
- Slice/Collimation: 0.5 mm x4
- Rotation time: 400 msec (350 msecoptional)


K1-101

#### TOSHIBA - AQUILION 64 AND AQUILION VELOCT 128 WITHOUT vHP (CONT)

#### 5. ECG-gated data acquisition of the aortic root/heart - Contrast enhanced

#### General

 Retrospectively ECG-gated helical acquisition of the aortic root and heart

#### Thoracic Data acquisition

- Delay after monitoring has reached threshold: 5 seconds
- Breath hold command: Inspiration only
- Tube voltage 100 kVp
- Tube current: fixed tube current adjusted to BMI, e.g. 400 mA (Aquilion 64), SURE Exposure XYZ Modulation (Velo CT 128)
- Helical retrospective ECG Gated mode
- · Slice/Collimation: 0.5 mm x64
- Rotation time: 400 msec (350 msec optional)
- · Pitch: Cardiac (set by SURE Cardio)

#### Data reconstruction

- Axial multiphasic reconstruction covering the entire cardiac cycle, 5% or
- 10% intervals in sinus rhythm Use ECG editing if necessary
- Field of View limited to the
- Slice thickness: 0.5 mm Increment: 0.5 mm SUREIQ: Cardiac CTA FC 43 (Aquilion 64), FC 03 (VeloCT 128)
- Quantum De-Noising Software (QDS +) (VeloCT 128)
- Boost 3D (VeloCT 128)
- Iterative reconstruction -AIDR 3D (VeloCT 128)

#### 6. Contrast enhanced ECG-assisted cardiac data acquisition

#### General

· Non-gated data acquisition of the thorax, abdomen, and pelvis.

#### Abdominal/Pelvic Data acquisition

- Delay between scans: 7 seconds Tube voltage 100 kVp
- · Tube current and Anatomical dose modulation: SUREExposure XYZModulation
- Slice/Collimation: 0.5 mm x64
- Scan direction: Cranio-caudal
- · Pitch: Standard Rotation time: 400 msec (350 msec optional)

#### Data reconstruction

- Increment: 0.8mm
- SUREIQ: CTA Body FC 08

- Axial reconstructions: 3 mm x
- Slice thickness: 1.0mm
- Quantum De-Noising Software (QDS +)

K1-103

- Boost 3D
- Iterative reconstruction -AIDR 3D (VeloCT 128)

#### Contrast application protocol

- · Single contrast application for both the retrospectively ECG-gated CTA of the aortic root/ heart and the CTA of the thorax/abdomen/pelvis
- · Placement of IV access per institutional protocol (an 18-guage IV typically provides the highest safety)
- Automated contrast injection using a dual-cylinder injector

- Recommended contrast media application: 80 100 cc iodinated contrast medium at 4 cc/sec
- Contrast bolus monitoring and timing of data acquisition by means of bolus tracking at the level of the descending acrts with an ROI placed within the descending aorta; threshold set at 180 HU

#### RECOMMENDATIONSFOR A LOW-CONTRAST PROTOCOL

- Use reduced amount of contrast material (e.g. 50 60 cc)
- Place ROI for bolus tracking (SUREStart) in ascending acrts as this decreases the delay between contrast administration/arrival to the start of the data acquisition
- · Reducethresholdforbolustrackingto160HU
- · Limit the Z-axis coverage of the ECG-gated data acquisition to the acrtic root, as this is the Time-intensive part of the examination (due to the low pitch value for ECG-gated data acquisition)
- This approach should allow for sufficient contrast attenuation of the acrtic root, however contrast attenuation of the non-gated scan may be variable

#### RECONSTRUCTION OF MULTIPHASIC DATA SET

Multiphasic ('dynamic', 'cine') data sets can be reconstructed using a relative approach (percentage intervals [%] between two R-peaks) or an absolute approach (fixed distance of the reconstruction window form the R-peak, reported as [msec]).



Relative Reconstruction settings in 5% intervals

For retrospectively ECG-gated CT data, the relative approach (e.g. 5% or 10% intervals) performs well in regular sinus rhythm. In case of increased heart rate variability, atrial fibrillation, or ectopic beats, absolute reconstruction should be employed in combination with ECG-editing if necessary.



Absolute Reconstruction settings in 50 ms intervals

#### REVIEW OF DATA RECONSTRUCTION AND ECG-EDITING

- · Image reconstructions of the aortic root and heart should be reviewed immediately after the scan when raw data is still available
- The ECG-gating should be reviewed to ensure that the automated algorithms correctly identifi the R-peaks
- If R-peaks were not correctly identified, manual correction should be performed (e.g. add an R-peakifan R-peakwas not identified or delete an R-peakifan R-peakwas placed on anything other than the R-peak; alternatively R-peaks can be shifted manually)
- In case of ectopic contractions, absolute reconstruction should be used and the R-peak of the ectopic beat should be deleted



ECG-editing screen showing correctly identified R-peaks.


- Achenbach S, Delgado V, Hausleiter J, et al. SCCT expert consensus document on computed tomography imaging before transcatheter acrtic valve implantation (TAVI)/transcatheter acrtic valve replacement (TAVI). J Cardiovasc Comput Tomogr 2012;6(6)566-350.
- Blanke P, Bulla S, Baumann T, et al. Thoracic Aorta: Prospective Eletrocardiographically Triggered CT Angiography with Dual Source CT-Feanblity, Image Quality, and Dose Reduction. Radiology 2010;255(1):207-217.
- 3. Blanke P, Russe M, Leipsic J, et al. Conformational Pulsatile Changes of the Aortic Annulus. JACC Cardiovasc Imaging 2012;5(9):984-994.
- 4. Blanke P, Schoepf UJ, Leipzic J. CT in Transcatheter Aortic Valve Replacement. Radiology 2013;269(3):650-669.
- Gurvitch B. Wood DA. Leipsic J. et al. Multitide: Computed Tomography for Prediction of Optimal Angiographic Deployment Projections During Transcatheter Aortic Valve Implantation. JACC Cardiovasc Imaging 2010;3(11):1157-1155.
   Leipsic J, Gurvitch B, LaBounty TM, et al. Multidetector Computed Tomography in Transcatheter Aortic Valve Implantation. JACC Cardiovasc Imaging 2011;4(4):416-429.
- Litmanovich DE, Ghersin E, Burke DA, et al. Imaging in Transcatheter Aortic Valve Replacement (TAVR): role of the radiologist. Insights Imaging 2014; 5:125-146.

Edwards, Edwards Lifesciences, and the stylized E logo are trademarks of Edwards Lifesciences Corporation. All other trademarks are the property of their respective owners.

© 2015 Edwards Lifesciences Corporation. All rights reserved. PP-US-0167 v1.0 E5666/6-15/THV

@Toshiba Medical Systems Corporation 2015. All rights reserved. Design and specifications are subject to change without notice.

Edwards Lifesciences | edwards.com

One Edwards Way I Irvine, California 92614 USA Switzerland | Japan | China | Brazii | Australia | India



PARTNER 3

# Appendix K-2 Sub-Study CT

CT Substudy Manual of Operations

Edwards Lifesciences LLC Protocol US IDE Trial #2015-08

Edwards Lifesciences LLC

One Edwards Way

Irvine, CA 92614

Document Title: CT Substudy Manual of Operations

Trial Sponsor: Edwards Lifesciences

Protocol Title: A Prospective, Randomized, Controlled, Multi-Center Study to Establish

the Safety and Effectiveness of the SAPIEN 3 Transcatheter Heart Valve in Low Risk Patients who have Severe, Calcific, Aortic Stenosis Requiring

Aortic Valve Replacement.

Protocol Identifier: US IDE Trial #2015-08

Edwards Lifesciences LLC Protocol US IDE Trial #2015-08

Document Approval: St. Paul's Cardiac CT Core Lab, Edwards Lifesciences, LLC

Document title: CT Procedure Manual

Document version: Version 3.0; Nov 2017

Study number: 2015-08

| Name/Title | Signature/Date |
|---|---|
| Jonathon Leipsic, MD<br>Director, CT Core Lab<br>University British Columbia | |
| Philipp Blanke, MD<br>Director, CT Core Lab<br>University British Columbia | |
| Vinny Podichetty, MD<br>Director, PARTNER 3 Trial<br>Edwards Lifesciences | |
| Kyle Bilhorn, MPH<br>Sr. Manager, Clinical Core Labs<br>Edwards Lifesciences | |

#### Edwards Lifesciences LLC Protocol US IDE Trial #2015-08

# Contents\_Toc498693158

| 1. | Site-preparation | E |
|----|-------------------------|----|
| 2. | Site Validation | 6 |
| | CT Data Acquisition | |
| 4. | CT Data Reconstructions | 12 |
| 5 | Submitting CT Images | 18 |

Edwards Lifesciences LLC Protocol US IDE Trial #2015-08

## DOCUMENT REVISION HISTORY

Document Revision History begins with the first revision after the initial approved version

| Section updated in version | Changes resulting in version | Reason for |
|---|---|---|
| FINAL_v 2.0,_May 2016 | FINAL_v 3.0, Nov 2017 | change |
| Headers and throughout document | Headers | Removed the "- |
| Sub-study | Substudy | " to align with |
| | | the protocol |
| | | and other trial |
| | | resources |
| Section 2 | Section 2 | Updating with |
| a. All sites will be required to submit | b. All sites will be required to submit to | new url and |
| to the Imaging Core Lab, a de- | the Imaging Core Lab, a de-identified | image vendor |
| identified sample of a CT | sample of a CT performed per section | name. |
| performed per section 3 via | 3 via Bioclinica Smart Submit at | |
| Moving Pictures WebSend at | https://smartsubmit.bioclinica.com. | |
| https://www.mddximage.com | | |
| Section 3 | Section 3 | Per the CT core |
| Single-source 64-row scanners are | Single-source 64-row scanners are | lab, adequate |
| not sufficient | sufficient if heart rate is adequately | imaging may |
| | controlled | be obtained in |
| | | 64-slice |
| | | scanners when |
| | | the heart rate |
| | | is appropriately |
| Section 2 Heart Date Centre! | Costion 2 Heart Bate Control | Controlled |
| Section 3, Heart Rate Control | Section 3, Heart Rate Control | Adding upper |
| | Heart rate for single-source 64-slice | parameter for |
| | scanners must be <80 bpm to ensure | appropriate |
| | adequate image quality. | heart rate |
| | | control in |
| | | single-source |
| | | 64-slice |
| | | scanners |

#### Edwards Lifesciences LLC Protocol US IDE Trial #2015-08

| Section update<br>FINAL_v 2.0,_ | | Changes resulting in version<br>FINAL_v 3.0, Nov 2017 | | Reason for<br>change |
|---|---|---|---|---|
| Table 2 | | Table 2 | | Adding |
| Scanner Single-source | Acquisition<br>mode<br>ECG-gated, | Scanner Single-source volume scanner with extended z-axis | Acquisition mode<br>ECG-gated, 'one-<br>beat, one-slab'<br>volume acquisition | acquisition<br>modes for<br>additional |
| volume scanner GE Revolution (16cm coverage) Philips iCT 256 (8cm coverage) Toshiba Aquilion One/Vision or Aquilion Premium (16cm coverage) | 'one-beat, one-<br>slab' volume<br>acquisition | GE Revolution (16cm coverage) Toshiba Aquilion One/Vision or Aquilion Premium (16cm coverage) Philips iCT 256 (8cm coverage) | | scanners to be<br>used in the<br>substudy |
| Dual-Source scanner • Siemens Somatom Definition, Flash, Force | Helical/spiral<br>acquisition with<br>retrospective<br>ECG-gating (do<br>not use high-<br>helical pitch<br>acquisition or<br>step-and shoot<br>mode) | Sing-Source scanner with limited z-axis coverage and Dual- Source scanner • All GE systems except for GE Revolution • All Philips systems systems <sup>2</sup> • All Toshiba systems except for Aquilion | Helical/spiral<br>acquisition with<br>retrospective ECG-<br>gating | |
| Table 2 footnote<br>Note – For Dual-Source<br>use of high-pitch helica<br>should be avoided. | • | One/Vision Table 2 footnote Note – <sup>1</sup> Philips iCT 256 ceither ECG-gated, 'one-bevolume acquisition or He acquisition with retrospe For Dual-Source CT scann pitch helical data acquisitiavoided. | eat, one-slab'<br>lical/spiral<br>ctive ECG-gating; <sup>2</sup><br>eer, the use of high- | |

Edwards Lifesciences LLC Protocol US IDE Trial #2015-08

#### 1. Site-preparation

In order to reach the highest rate of diagnostic scans possible, and to salvage potentially non-diagnostic data by means of ECG-editing etc., all sites participating in the CT substudy will be responsible for completing all required training and ensuring their institution's scanner and protocols are compatible with the scanning protocol outlined in section 3 of this document.

#### 2. Site Validation

The purpose of the Site CT Qualification Process is to ensure adherence to the imaging protocol as well as ensure compatibility between site CT acquisition, upload process and the Core Lab analysis tools.

Site will be validated upon successful completion of the following items:

- 1. Completing and returning a follow-up survey (will be sent to site by Edwards Lifesciences).
- 2. The first submission of a CT of an enrolled substudy patient to the Imaging Core Lab.
  - c. All sites will be required to submit to the Imaging Core Lab, a de-identified sample of a CT performed per section 3 via Bioclinica Smart Submit at <a href="https://smartsubmit.bioclinica.com">https://smartsubmit.bioclinica.com</a>.
  - A critique of the CT qualification scan will be emailed or faxed to the site and study sponsor as notification of the qualification status
  - If the site does not qualify with the first submission, the Imaging Core Lab will use the critique to recommend changes for resubmission of another CT study.

#### 3. CT Data Acquisition

Contrast-enhanced computed tomography (CT) allows for assessment of the Transcatheter Heart Valve (THV) in regard to positioning, expansion, and leaflet morphology and function. Similarly, it allows evaluation of Surgical Aortic Valves (SAVs) and their leaflets. However, image interpretation, particularly in regard to leaflet assessment, can be significantly limited by motion and mis-registration artifacts as well as beam-hardening artifact or poor contrast attenuation.

This section provides recommendations and requirements for scanner selection and data acquisition techniques. Adherence to these guidelines is essential to provide sufficient image data sampling while minimizing potential artifacts; thereby optimizing the diagnostic yield.

Data acquisition strategies and scanning protocols vary based on scanner systems. For the purpose of this substudy, an <a href="ECG-assisted">ECG-assisted</a> data acquisition which covers at least the aortic root throughout the entire cardiac cycle is required.

The relevant principles of CT data acquisition will be explained in brief below.

V3.0 Nov 2017 CONFIDENTIAL

K-2 - 6

Edwards Lifesciences LLC Protocol US IDE Trial #2015-08

NOTE: Only cardiac CT imaging is required for the post-TAVR CT scan at 30 days and at one year for the purpose of the substudy. A CTA of the thorax, abdomen and pelvis is NOT required at 30 days and one year.

#### Scanner selection

It is required that post-TAVR CT scans are performed with either

- Dual-source systems or
- Single-source volume scanners.

Single-source 64-row scanners are sufficient if heart rate is adequately controlled.

Note: The scanner employed ideally shall remain the same for the 30 day and one year CT examination.

#### Heart rate control

CT data acquisition at lower heart rates is preferred as this minimizes motion artifacts. Administration of heart rate controlling medications (e.g. beta blockers) should be considered in patients with accelerated heart rates (e.g., >65 bpm), in particular when using single-source volume scanners. Heart rate for single-source 64-slice scanners must be <80 bpm to ensure adequate image quality.

Note: Administration should follow institutional protocols such as those commonly used for coronary CTA. Contraindications for Beta-Blockers need to be considered

#### Contrast enhancement

Contrast administration protocols should be adopted from institutional protocols for coronary CTA. For recommendations see Table 1.

Table 1: Recommendations for contrast administration:

| Parameter | Recommendation |
|---|---|
| Iodine concentration | Iodinated contrast agent as per institutional standards |
| Flow rate | 4-6ml/sec |
| Volume | As per institutional standard for routine coronary cardiac CT, commonly 50-80cc |
| IV-access | Antecubital vein is recommended |
| Timing | Bolus tracking to allow for peak contrast in the ascending aorta |

Edwards Lifesciences LLC Protocol US IDE Trial #2015-08

#### Data Acquisition Mode

The ECG-assisted, contrast enhanced image acquisition of the aortic root constitutes the main and most important part of the post-TAVR CT scan at 30 days and one year. To allow for evaluation of potential leaflet restriction, and to ensure abundant image data in case of artifacts, it is required that the entire cardiac cycle is covered, independent of the acquisition mode employed. Table 2 provides and overview of acquisition modes stratified by scanner type to meet imaging requirements.

Table 2: Required acquisition modes stratified by CT system

| Scanner | Acquisition mode |
|---|---|
| Single-source volume scanner with extended | ECG-gated, 'one-beat, one-slab' volume acquisition |
| z-axis coverage | |
| GE Revolution (16cm coverage) Toshiba Aquilion One/Vision or Aquilion Premium (16cm coverage) Philips iCT 256 (8cm coverage) | |
| Sing-Source scanner with limited z-axis coverage and Dual-Source scanner All GE systems except for GE Revolution All Philips systems <sup>1</sup> All Siemens systems <sup>2</sup> All Toshiba systems except for Aquilion One/Vision | Helical/spiral acquisition with retrospective ECG-<br>gating |

Note – <sup>1</sup> Philips iCT 256 can be operated with either ECG-gated, 'one-beat, one-slab' volume acquisition or Helical/spiral acquisition with retrospective ECG-gating; <sup>2</sup> For Dual-Source CT scanner, the use of high-pitch helical data acquisition should be avoided.

Edwards Lifesciences LLC Protocol US IDE Trial #2015-08

#### Dose modulation

In order to achieve constant, diagnostic image quality throughout the cardiac cycle, we recommend maintaining peak tube current throughout the cardiac cycle and to avoid dose modulation (Figure 1 and 2).



Figure 1 — Retrospective ECG-gated helical data acquisition without dose modulation. The tube current (blue bar) is set at its peak during the entire cardiac cycle. The black boxes indicate the time point of image reconstruction within the cardiac cycle.

Edwards Lifesciences LLC Protocol US IDE Trial #2015-08



Figure 2 - ECG-gated, 'one-beat, one-slab' volume acquisition without dose modulation. The tube current (blue bar) is set at its peak during the entire cardiac cycle. The black boxes indicate the time point of image reconstruction within the cardiac cycle.

Edwards Lifesciences LLC Protocol US IDE Trial #2015-08

#### Scan coverage

The ECG-assisted data acquisition has to at least cover the entire SAV/THV (Figure 3). Scan coverage can be extended to include the entire heart, however this will increase the radiation burden to the patient.

CAVEAT: Please consider that the aortic root changes position during the cardiac cycle, with the potential of only partially covering the SAV/THV during certain parts of the cardiac cycle. Ensure that the anticipated scan range covers the SAV/THV throughout the entire cardiac and accommodates for changes in position.



Figure 3 – Scout views. Scan coverage can be limited to the THV/SAV as opposed to the entire heart, but should include the entire THV/SAV.

#### Scan settings

- Peak tube current: Scan settings should follow the institutional standard. Lower tube current can be
  used if anticipated increase in image noise is compensated by iterative image reconstruction.
- Tube voltage: Data acquisition with low tube voltage (e.g. 70-100kVp) should be avoided, as this
  increases beam hardening and streak artifacts of the metal components of the SAVs and THVs.
  Instead, data acquisition should be performed at 120kVp, alternatively at 140kVp. The latter however
  can significantly reduce the attenuation of the iodinated contrast media. Scan settings should be
  reviewed and care should be taken to avoid use of automated tube voltage selection algorithms in
  favour of manual selection of tube voltage.

Dose modulation should be avoided. If however dose-modulation is used, tube current should only be lowered to a level to still allow for diagnostic image quality.

Edwards Lifesciences LLC Protocol US IDE Trial #2015-08

Note - When using Siemens scanners (Siemens Healthcare, Forchheim, Germany), the use of MinDOSE (algorithm to lower tube current to 4% of peak current) should be avoided.

Table 3: Recommendations for scan parameters

| Parameter | Recommendation |
|---|---|
| Tube current | Absolute or reference tube current settings similar to institutional settings for routine coronary cardiac CT |
| Dose modulation | Dose modulation is not recommended in order to allow for images of equal, diagnostic image quality throughout the entire cardiac cycle |
| Tube voltage | 120kVp, alternatively 140kVp to reduce beam hardening artifacts of stent frame (in particular with volume-scanners); use of 100kVp or 80kVp is not recommended; automated algorithms for tube voltage selection may need to be overridden |
| Collimation | Thinnest possible, e.g. 0.625 with GE and Philips hardware, 0.6mm with Siemens Hardware, 0.5mm/0.25mm with Toshiba hardware |

#### 4. CT Data Reconstructions

#### Raw data protection

In order to allow for further image reconstruction if primary reconstructions are artifact impaired or insufficient, raw data should be protected from automated deletion on the scanner console. Raw data protection should occur immediately after data acquisition.

# **Data Reconstructions**

Image data should be reconstructed as follows:

- · Thin sliced axial reconstructions
- These should cover the entire cardiac cycle as multiphase/multiphasic reconstructions (AKA 4D-CT, cine)
- Reconstruction field of view should be limited to the heart, using a 512 x 512 matrix.
- Thin sliced reconstruction can be reconstructed in an overlapping fashion (increment < slice thickness)</li>

Multiphasic reconstructions are typically reconstructed in an interval fashion, either using a relative (percentage) approach, or an absolute approach (msec).

Edwards Lifesciences LLC Protocol US IDE Trial #2015-08

- For Single-Source Volume scanner (GE Revolution, Philips iCT256, Toshiba Aquilion One/Vision):
  - 5% or 10% increments
- 2. For Dual-Source systems (Siemens Somatom Definition, Flash, Force):
  - . 5% or 10% increments (relative reconstruction)
  - or 50ms increments (absolute reconstruction)

As opposed to relative reconstruction, absolute reconstruction is less susceptible to stair-step and double contour artifacts in the setting of atrial fibrillation or premature contractions. In absolute reconstruction, the distance of the reconstruction window to the preceding R-peak remains constant independent of the length of the RR-interval. When using retrospective ECG-gating, absolute reconstructions are favorable in particular for systolic/end-systolic image reconstruction.

Table 4: Recommendations for image reconstruction parameters

| Parameter | Recommendation |
|---|---|
| Reconstruction<br>Technique | Either filtered back projection or iterative reconstruction are acceptable. If iterative reconstruction is used, the strength/weighting should be intermediate (e.g. ADMIRE/SAPHIRE/IRIS strength 3, ASIR 40%) |
| Slice thickness | Thinnest possible, e.g. 0.625 with GE and Philips hardware, 0.6mm with<br>Siemens Hardware, 0.5mm/0.25mm with Toshiba hardware |
| Slice overlap | Slice overlap is recommended to improve MPR quality; e.g. 0.4 mm increment with 0.6 mm slice thickness when using Siemens equipment |
| Reconstruction field of view and matrix | Small field of view (FOV) limited to the heart; 512 x 512 matrix |
| Reconstruction<br>kernel | Same kernel as used for coronary CTA per institutional standard; alternatively use edge-pronounced kernel ('stent' kernel, e.g. 146f) in particular with pronounced blooming, |
| Multiphasic | Coverage of the entire cardiac cycle: |
| reconstruction | Volume scanner (GE Revolution, Philips iCT256, Toshiba Aquilion One/Vision): • 5% or 10% increments |
| | Other scanner: |

Edwards Lifesciences LLC Protocol US IDE Trial #2015-08

#### R-peak recognition

Prior to image reconstruction, the ECG-stripe should be reviewed to ensure that the scanner correctly sensed the R-peaks for timing of image reconstructions. Commonly, if R-peak recognition was incorrect, such as in the case of weak ECG-signal or artifacts, R-peak recognition and thus image synchronization can be manually corrected. This applies for both ECG-gated, 'one-beat, one-slab' volume acquisition as well as helical acquisition with retrospective ECG-gating.

#### ECG-editing with retrospective ECG-gating

Due to low pitch values, and thus redundant image data sampling, helical acquisition with retrospective ECG-gating allows for ECG-editing to improve the quality of image reconstructions. ECG-editing is particularly useful in the setting of

- Atrial fibrillation
- Premature atrial and ventricular contractions (PACs and PVCs)

Atrial fibrillation and ectopic heart beats result in RR-intervals of significantly different length, leading to stair-step and double-contour artifacts.

In case of premature contractions, ECG-editing aims at avoiding image reconstruction which uses image data from RR-intervals which are affected by the premature contractions. Importantly, these may differ in regard to diastolic or systolic image reconstruction. It is important to understand how and which RR-intervals are affected by premature contractions.

- Preceding RR-Interval which is terminated by PVC/PAC: Shortening of diastole of the preceding RR-interval (e.g. missing mid/end-diastolic image data in case of diastolic image reconstruction)
- RR-Interval beginning with PVC/PAC: Relative shift of cardiac phases within the ectopic RR-interval due to reduced LV loading within the shortened preceding RR-interval.
- Subsequent RR-Interval (only with PVC): Due to increased LV filling during compensatory pause,
   LV ejection increases in the subsequent RR-interval.

In particular, in coronary CTA, end-systole has been proven to be the cardiac phase yielding most reliable image quality, in particular when using high temporal resolution systems such as dual-source scanners. This is because end-systole can be considered the most stable phase within the cardiac cycle in regard to impact of increased heart rate variability with varying length of the RR-intervals. While the position of end-systole in the cardiac cycle is directly related to the length of the LV ejection time, it remains fairly constant with regard the absolute distance from the R-peak in msec.

The length of the preceding RR-interval determines the LV filling state, and thus the length of the LV ejection time and position of end-systole (Figure 4).

Edwards Lifesciences LLC Protocol US IDE Trial #2015-08

- If the preceding RR-interval is shorter, LV filling is reduced and the subsequent LV ejection time is shorter, i.e. end-systole is closer to the R-peak.
- If the preceding RR-interval is longer, LV filling is increased and the LV ejection time is longer, i.e. end-systole is closer to the R-peak.



Figure 4 — Dependency of the position of end-systole on the length of the preceding RR-interval. The length of the preceding RR-interval determines the LV filling state, and thus the length of the LV ejection time and position of end-systole.

The above stated relationship is important to understand its influence on end-systole timing in premature contractions and atrial fibrillation. Importantly, there are differences between PACs and PVCs with regard to the subsequent RR-interval following the RR-interval beginning with the PAC/PVC (Figure 5).

# Premature atrial contraction:

- 1. The RR-interval prior to the PAC is shortened, often missing mid-/end-diastole.
- 2. The RR-interval beginning with the PAC, end-systole shifts towards the R-peak.
- 3. The subsequent RR-interval is not affected.

Edwards Lifesciences LLC Protocol US IDE Trial #2015-08

#### Premature ventricular contraction:

- 1. The RR-interval prior to the PVC is shortened, often missing mid-/end-diastole.
- 2. The RR-interval beginning with the PVC, end-systole shifts towards the R-peak.
- The subsequent RR-interval is affected, as the RR-interval beginning with the PVC is elongated due to the compensatory pause, leading to increased LV filling and shift of end-systole in the subsequent RR-interval.



Figure 5 - Influence of PACs/PVCs on the position of end-systole.

Helical acquisition with retrospective ECG-gating and its inherent low pitch values with redundant image data sampling, allows for ECG editing to help eliminate the negative impact of premature ventricular contractions. This is performed by manually deselecting specific RR-intervals that contain extra-systoles.

Edwards Lifesciences LLC Protocol US IDE Trial #2015-08

In the setting of PACs or PVCs, the following approach is recommended when performing end-systolic image reconstruction using an absolute [msec] reconstruction technique (Figure 6):

- Keep reconstruction window in shortened RR-interval which is terminated by PAC/PVC, as position of end-systole is not affected.
- Eliminate reconstruction window in RR-interval beginning with PAC/PVC, as position of endsystole is altered, being closer to the R-peak.
- Only in PVCs the subsequent RR-interval is affected, given the compensatory pause with increased LV filling. If possible without resulting in a data gap, the reconstruction window in the subsequent should be deleted/deactivated.



Figure 6 - Approach to end-systolic data reconstruction in PACs/PVCs using ECG-editing and absolute (msec) reconstruction.

Edwards Lifesciences LLC Protocol US IDE Trial #2015-08

The situation is very different, when diastolic images are being reconstructed. In the setting of PACs or PVCs, the following approach is recommended when performing diastolic image reconstructions (commonly with relative [%] reconstruction) (Figure 7):

- Eliminate reconstruction window in the RR-interval which is terminated by the PAC/PVC, if this RR-interval is shortened (most commonly). Note: Shortening of the RR-interval impacts the absolute position of the reconstruction window when using a percentage/relative reconstruction. Furthermore, lack of mid-/late-diastolic data would also interfere with absolute reconstruction.
- 2. If possible, also eliminate reconstruction window in RR-interval beginning with PAC/PVC.
- 3. In PVC, the subsequent RR-interval may be affected, but data gap may not allow for deletion.



Figure 7 - - Approach to diastolic data reconstruction in PACs/PVCs using ECG-editing and relative (%) reconstruction.

## 5. Submitting CT Images

Refer to Appendix K-1 for CT submission instructions.

# Appendix L Histopathology

# 1.0 Purpose

The purpose of the following protocol is to provide the Investigator (clinical site) with procedures for handling and assessing the study valve after explantation. The assessment should include gross examination, identification of the primary failure mode and contributory factors leading to the explant (if possible), photographs and other documentation, and preparation of the explanted valve for shipment to the Sponsor or designated Histopathology Laboratory for further analysis. Also, included is an overview of the procedures to be followed by the Sponsor and/or designated Histopathology Laboratory for gross analysis, as well as macro and micro histopathology analysis. Investigational valves that are removed at any time an allegation of device malfunction should be returned to the Sponsor for evaluation. All other explants (those not with an allegation of device malfunction) should be sent to the Histopathology Core Lab. Refer to section 6.0 for tissue shipment information.

# 2.0 Valve Explanation Procedure

Upon autopsy (only), prior to removal of the valve from the heart, obtain *in situ* photographs of the inflow and outflow tracts, valve leaflets, and conduit tissue. Using care, the valve should be excised in a fashion so as to keep the valve and surrounding structure as intact as possible.

For all explants (those obtained at autopsy as described above or through valve replacement surgery following standard surgical practice), once removed the valve should be rinsed of all residual blood by gently agitating in sterile Lactated Ringers solution.

Prior to shipment of the valve to the Sponsor or designated Histopathology Laboratory for further dissection and pathologic analysis, grossly examine the explanted tissue *in toto* and record observations on the explanted valve CRF. Gross photographs will be taken of both inflow and outflow tracks. Observations of stent frame apposition and neointimal incorporation will be documented.

Swab cultures of possibly infected areas should be taken, sent to the appropriate laboratory and documented in the pathology report. If no infection is obvious, then no culture swab is necessary.

#### 3.0 Tissue Dissection Procedure

Once the valve has been explanted, grossly examined, and photographed, the tissue should be sent to the Sponsor or designated Histopathology Laboratory for histological analysis. Place the sample into a specimen cup or equivalent container. The specimen cup should contain 10% buffered formalin solution. On the outside of the container, label the study patient number, valve serial number, site number, and date of explant. The tissues will be examined at the Sponsor or designated histopathology laboratory to determine the morphology of the tissue/valve, as well as to assess leaflet calcification, and general histopathology. The valve tissues will be stained with H&E, Von Kossa, or other relevant stains and will be reviewed by a certified pathologist.

#### 4.0 Fixation

Explanted study valve samples shall be submitted in 10% formalin.

#### 5.0 Documentation

Please provide the following supporting documents to enable complete explant assessment. The documents should enable the Sponsor to determine explant date, duration of implant, surgical pathology, mediating study patient history, reason for reoperation, gross description, and pathology notes. The documents may be returned with the shipped tissue.

- Operative report dictated at the explant
- Sponsor Case Report Forms
- Pathology report (once available)
- Blood study results (once available)
- Preoperative Echocardiographic Report (Just Prior to Explant)

# 6.0 Tissue Shipment

Investigational valves that are removed at any time with an allegation of device malfunction should be returned to the Sponsor for evaluation. Contact your sponsor representative for assistance with the return which will include a Compliant Report (completed by the Sponsor) and biohazard packaging.

# Shipping Address:

Edwards Lifesciences LLC 1212 Alton Pkwy Irvine, CA 92606 Attention: Returned Goods CER/RGA#:

Investigational valves that are removed for any reason other than an allegation of device malfunction should be sent to the Histopathology Laboratory. Place the specimen container within two, separately sealed biohazard plastic bags. Place the sealed sample in a small non-crushable box. Ship the tissue to the Sponsor's designated Histopathology Laboratory by Federal Express PRIORITY (Sponsor billing number 0900-2768-9) or equivalent shipping service:

Histology Core Laboratory: Renu Virmani, MD

CV Path Institute. Inc. 19 Firstfield Road Gaithersburg, MD 20878 Phone: 301-208-3745 Ext. 105

# 7.0 Procedure for Evaluation at Sponsor or Designated Histopathology Laboratory

Gross Examination and Photographs:

If possible, photographs should be taken at each stage of dissection to better document observations. Assessment of the valve leaflets and commissures will include presence of leaflet fenestrations, tears, thrombus formations and calcified nodules. Photographs will be taken of all suspected abnormalities. The gross examination should include macroscopic assessment of the following:

Mobility and shape of leaflets; Calcification (leaflet and conduit);

Host tissue overgrowth; Evidence of infection;
Leaflet wear or degeneration; Aneurysm formation;
Leaflet thickness; Valve thrombosis;
Leaflet fenestrations; Tissue rejection;
Fibrosis sheathing; Inflammation.

# 8.0 Radiographic Analysis

Additionally, X-rays will be taken of all valve/devices to assess placement and apposition of the stent frame to the host vessel and to identify leaflet calcification. X-rays will be in both transverse and longitudinal planes.

# 9.0 Dissection and Sampling

A portion of each valve assembly, to include one commissure and one half of each adjacent valve leaflet, will be removed from the assembly and submitted for scanning electron microscopic examination. The portion will be removed by making two longitudinal cuts through the length of the host vessel and metal stent frame. The remaining valve leaflets will be excised away at the point of attachment to the assembly.

# Scanning Electron Microscopy

Scanning electron microscopy will be employed to assess degree of intimal incorporation of the metal stent frame, endothelial coverage of the host vessel neointima and valve leaflets. Leaflet surface topology will be assessed and any defects in the surface identified.

# 10.0 Histopathology Evaluation

#### Paraffin:

Valve leaflets will be inked on the outflow surfaces to maintain orientation. Serial slices of the leaflets will be made from base to free edge and flat embedded for cross-sectional examination. Hematoxylin and eosin, trichrome, Movat pentachrome, Von Kossa calcium, and Phosphotungstic acid-hematoxylin stains will be performed on all sections.

#### Plastic:

The remaining valve assembly (minus the portion removed for SEM) will be processed and embedded in methylmethacrylate plastic. Transverse sections will be sawed and ground from the area of the superior tip of the first stent strut (proximal end), from the mid portion near the proximal end of the short bar assembly (not to include PET skirt) and from the distal end through the short bar assembly and commissures.

# Transmission electron microscopy (TEM)

One half of each valve leaflet from the mid-portion will be reserved for transmission electron microscopy. The section will be of full leaflet thickness, flat embedded in epoxy resin and cross-sectioned. TEM will be employed to assess collagen integrity and calcium deposition.

# **Explant Shipping Form**

Please enter the following information and fax the form to CV Path at (301) 208-3745 24 hours prior to shipment.

Ship to: TBD

| Protocol #: SAPIE | N 3 Expanded Indication | Subject ID: | |
|---|---|---|---|
| Sponsor: <u>Edwa</u> | rds Lifesciences | Device Type: <u>SAPI</u> | EN 3 ™ THV |
| Study Site: | | Site Principal Investigate | or: |

| Item Shipped (Serial Number) | Sender:<br>Print Name / Signature | Date<br>Harvested<br>(If available) | Shipping Tracking Number | Date Sent |
|---|---|---|---|---|

| Comments: |
|-----------|

Please keep a copy of this form in the subject study file. If possible, please include a copy of this form in the package

# Appendix M EQ-5D-5L



Health Questionnaire

English version for the UK

UK (English) © 2009 EuroQol Group EQ-5D™ is a trade mark of the EuroQol Group

| Under each heading, please tick the ONE box that best descr | ribes your health TO |
|---|---|
| MOBILITY | |
| I have no problems in walking about | |
| I have slight problems in walking about | |
| I have moderate problems in walking about | _ |
| I have severe problems in walking about | _ |
| I am unable to walk about | _ |
| SELF-CARE | |
| I have no problems washing or dressing myself | |
| I have slight problems washing or dressing myself | |
| I have moderate problems washing or dressing myself | |
| I have severe problems washing or dressing myself | |
| I am unable to wash or dress myself | |
| USUAL ACTIVITIES (e.g. work, study, housework, family or leisure activities) | |
| I have no problems doing my usual activities | |
| I have slight problems doing my usual activities | |
| I have moderate problems doing my usual activities | |
| I have severe problems doing my usual activities | |
| I am unable to do my usual activities | |
| PAIN / DISCOMFORT | |
| I have no pain or discomfort | |
| I have slight pain or discomfort | _ |
| I have moderate pain or discomfort | _ |
| I have severe pain or discomfort | _ |
| I have extreme pain or discomfort | _ |
| ANXIETY / DEPRESSION | |
| I am not anxious or depressed | |
| I am slightly anxious or depressed | |
| I am moderately anxious or depressed | |
| I am severely anxious or depressed | |
| I am extremely anxious or depressed | П |

2

UK (English) © 2009 EuroQol Group EQ-5D™ is a trade mark of the EuroQol Group

The best health

- · We would like to know how good or bad your health is TODAY.
- This scale is numbered from 0 to 100.
- 100 means the <u>best</u> health you can imagine.
   0 means the <u>worst</u> health you can imagine.
- Mark an X on the scale to indicate how your health is TODAY.
- Now, please write the number you marked on the scale in the box below.

YOUR HEALTH TODAY =

3

UK (English) © 2009 EuroQol Group EQ-5D™ is a trade mark of the EuroQol Group

# Appendix N Kansas City Cardiomyopathy Questionnaire (KCCQ)

# The KC Cardiomyopathy Questionnaire

The following questions refer to your heart failure and how it may affect your life. Please read and complete the following questions. There are no right or wrong answers. Please mark the answer that best applies to you.

Heart failure affects different people in different ways. Some feel shortness of breath while
others feel fatigue. Please indicate how much you are limited by heart failure (shortness of
breath or fatigue) in your ability to do the following activities over the past 2 weeks.

## Place an X in one box on each line

| Activity | Extremely<br>Limited | Quite a bit<br>Limited | Moderately<br>Limited | Not at all<br>Limited | Limited for<br>other reasons or<br>did not do the<br>activity |
|---|---|---|---|---|---|
| Dressing yourself | | | | | |
| Showering/Bathing | | | | | |
| Walking 1 block on<br>level ground | | | | | |
| Doing yardwork,<br>housework or<br>carrying groceries | | | | | 0 |
| Climbing a flight of<br>stairs without<br>stopping | | | | | |
| Hurrying or jogging (as if to catch a bus) | | | | | |
| 2. Compared with 2 weeks ago, have your symptoms of heart failure (shortness of breath, fatigue, or ankle swelling) changed? My symptoms of heart failure have become Much Slightly Not changed Slightly Much I've had no symptoms worse worse better better over the last 2 weeks | | | | | |

PARTNER 3 Trial. Version 5.0 DEC 2018

Copyright @1992 -2005 John Spertus, MD, MPH

Original US English

| when you woke up | | nines did you nave | swelling in | your reet, ankles t | or legs |
|---|---|---|---|---|---|
| Every morning | 3 or more times<br>a week, but not<br>every day | 1-2 times a week | Less than o week | nce a Never or<br>past 2 v | · |
| Over the past 2 It has been | | has swelling in you | ır feet, ankles | s or legs bothered | you? |
| Extremely bothersome | Quite a bit<br>bothersome | Moderately bothersome | Slightly<br>bothersome | Not at all<br>bothersome | I've had n<br>swelling<br>□ |
| 5. Over the past 2<br>what you was | | e, how many times h | nas <b>fatigue</b> lis | mited your ability | to do |
| All of the Seve<br>time times pe | ral At least<br>er day once a day | 3 or more times<br>per week but not<br>every day | 1-2 times<br>per week | Less than once<br>a week | Never over<br>the past 2<br>weeks |
| | ] [ | | | | |
| 6. Over the past 2 | 2 weeks, how much | ı has your <b>fatigue</b> b | othered you? | | |
| Extremely bothersome | Quite a bit<br>bothersome | • | Slightly<br>othersome | Not at all<br>bothersome | I've had<br>no fatigue<br>□ |
| | weeks, on average<br>nat you wanted? | e, how many times h | as s <b>hortne</b> ss | of breath limited | d your |
| All of the Seve time times pe | | 3 or more times per week but not every day | 1-2 times<br>per week | Less than once<br>a week | Never over<br>the past 2<br>weeks |
| Copyright ⊗1992 -2005 Jo | ohn Spertus, MD, MPH | | | Original | US English |

| 8. Over the past 2 weeks. how much has your shortness of breath bothered you? | | | | | |
|---|---|---|---|---|---|
| | | | • | | had no<br>s of breath |
| 9. Over the <u>past 2 weeks</u> , on average, how many times have you been forced to sleep sitting up in a chair or with at least 3 pillows to prop you up because of shortness of breath? | | | | | |
| Every night W | 3 or more times a reek, but not every | | Less than of a week | | |
| | | sen for a number o<br>, if your heart failu | | | rou |
| Not at all sure | Not very sure | Somewhat sure | Mostly sure | Completely | sure |
| | | at things you are ab<br>or example, weighin | | | |
| Do not understand<br>at all | Do not understa<br>very well | and Somewhat<br>understand | Mostly<br>understa | • | • |
| 12. Over the past | 2 weeks, how mucl | n has your heart fai | lure limited yo | ur enjoyment of lif | e? |
| It has extremely<br>limited my<br>enjoyment of life | It has limited my<br>enjoyment of life<br>quite a bit | | It has sligh<br>limited m<br>enjoyment o | ny enjoym | ent of |
| 13. If you had to s<br>would you feel | | ur life with your he | art failure the | way it is <u>right now</u> | , how |
| Not at<br>satisfi | all Mostly<br>ied dissatisfie | Somewhat<br>d satisfied | Mostly<br>satisfied<br>□ | Completely satisfied | |
| Copyright ©1992 -2005 Jo | hn Spertus, MD, MPH | | | Original US Er | nglish |

| your heart failure? | | | | | | |
|---|---|---|---|---|---|---|
| I felt that way I fe<br>all of the time most<br>□ | | | ccasionally l<br>t that way | I rarely felt that<br>way | I never felt<br>way | that |
| | 15. How much does your heart failure affect your lifestyle? Please indicate how your heart failure may have limited your participation in the following activities over the past 2 weeks. | | | | | |
| | Plea | se place an X | in one box | on each line | | |
| Activity | Severely<br>limited | Limited quite a bit | Moderately<br>limited | Slightly<br>limited | Did not<br>limit at all | Does not<br>apply or did<br>not do for<br>other reasons |
| Hobbies, | | | | | | |
| recreational activities | | | | | | |
| Working or<br>doing household<br>chores | | | | | | |
| Visiting family<br>or friends out of<br>your home | | | | | | |
| Intimate<br>relationships<br>with loved ones | | | | | | |

Copyright @1992 -2005 John Spertus. MD. MPH

Original US English

Appendix O

SF-36

# Your Health and Well-Being

This survey asks for your views about your health. This information will help keep track of how you feel and how well you are able to do your usual activities. Thank you for completing this survey!

For each of the following questions, please mark an  $\boxtimes$  in the one box that best describes your answer.

1. In general, would you say your health is:



2. Compared to one year ago, how would you rate your health in general now?



3. The following questions are about activities you might do during a typical day. Does your health now limit you in these activities? If so, how much?

| | | Yes,<br>limited<br>a lot | Yes,<br>limited<br>a little | No, not<br>limited<br>at all |
|---|---|---|---|---|
| a | Vigorous activities, such as running, lifting heavy objects, participating in strenuous sports | | 2 | 3 |
| ь | Moderate activities, such as moving a table, pushing a vacuum cleaner, bowling, or playing golf | 🗆 1 | 2 | 3 |
| e | Lifting or carrying groceries | 1 | 2 | 3 |
| d | Climbing several flights of stairs | 1 | 2 | 3 |
| e | Climbing one flight of stairs | 1 | 2 | 3 |
| ſ | Bending, kneeling, or stooping | 1 | 2 | 3 |
| 8 | Walking more than a mile | 🗆 1 | 2 | 3 |
| h | Walking several hundred yards | 🗌 1 | 2 | 3 |
| i | Walking one hundred yards | 🗆 1 | 2 | 3 |
| j | Bathing or dressing yourself | | 2 | 3 |

| 4. | During the past 4 weeks, how much of the time have you had any of the |
|---|---|
| | following problems with your work or other regular daily activities as a |
| | result of your physical health? |

| | | All of<br>the time | Most of<br>the time | Some of<br>the time | A little of<br>the time | None of<br>the time |
|---|---|---|---|---|---|---|
| | ' | lacksquare | lacksquare | lacksquare | lacksquare | lacksquare |
| a | Cut down on the <u>amount of</u><br>time you spent on work or<br>other activities | 🔲 1 | 2 | 3 | 🗆 4 | 5 |
| b | Accomplished less than you would like | 1 | 2 | 3 | 4 | 5 |
| c | Were limited in the <u>kind</u> of work or other activities | 1 | 2 | 3 | 🗆 4 | 5 |
| d | Had <u>difficulty</u> performing the work or other activities (for example, it took extra effort) | | 2 | 3 | 4 | 5 |

5. During the <u>past 4 weeks</u>, how much of the time have you had any of the following problems with your work or other regular daily activities <u>as a result of any emotional problems</u> (such as feeling depressed or anxious)?

| | | All of<br>the time | Most of<br>the time | Some of the time | A little of<br>the time | None of<br>the time |
|---|---|---|---|---|---|---|
| | Cut down on the <u>amount of</u><br>time you spent on work or<br>other activities | | 2 | 3 | 4 | 5 |
| , | Accomplished less than you would like | | 2 | 3 | 4 | 5 |
| : | Did work or other activities less carefully than usual | | 2 | 3 | 4 | 5 |

6. During the <u>past 4 weeks</u>, to what extent has your physical health or emotional problems interfered with your normal social activities with family, friends, neighbors, or groups?

| Not at all | Slightly | Moderately | Quite a bit | Extremely |
|------------|----------|------------|-------------|-----------|
| _ ı | _ 2 | 3 | _ 4 | 5 |

7. How much bodily pain have you had during the past 4 weeks?

| None | Very mild | Mild | Moderate | Severe | Very severe |
|------|-----------|------|----------|--------|-------------|
| 1 | 2 | 3 | _ 4 | 5 | 6 |

8. During the <u>past 4 weeks</u>, how much did <u>pain</u> interfere with your normal work (including both work outside the home and housework)?

| Not at all | A little bit | Moderately | Quite a bit | Extremely |
|------------|--------------|------------|-------------|-----------|
| | 2 | 3 | □ 4 | 5 |

9. These questions are about how you feel and how things have been with you during the past 4 weeks. For each question, please give the one answer that comes closest to the way you have been feeling. How much of the time during the past 4 weeks...

| | | _ | All of<br>e time | Most of<br>the time | Some of the time | A little of the time | None of the time |
|---|---|---|---|---|---|---|---|
| , Did | l you feel full of life? | | 1 | 2 | 3 | | 5 |
| ь На | ve you been very nerv | ous? | . 1 | 2 | 3 | | 5 |
| dur | ve you felt so down in<br>nps that nothing could<br>er you up? | 1 | 1 | 2 | 3 | | 5 |
| d Hav | ve you felt calm and<br>ceful? | | 1 | 2 | 3 | | 5 |
| . Did | l you have a lot of ene | rgy? | . 1 | 2 | 3 | 4 | 5 |
| r Hav | ve you felt downheart<br>l depressed? | ed | | 2 | 3 | | 5 |
| 8 Did | l you feel worn out? | | | 2 | 3 | 4 | 5 |
| h Ha | ve you been happy? | | . 1 | 2 | 3 | 4 | 5 |
| , Did | l you feel tired? | | | 2 | 3 | 4 | 5 |
| em | | interfere<br>:.)?<br>Most of | d with y | our social | activities<br>little of | (like visiting | |
| | the time t | he time | the ti | me th | e time | the time | |
| | <b>▼</b> | ▼<br>□ 2 | <b>▼</b> | 3 | <b>▼</b> | <b>▼</b> | |

# 11. How TRUE or FALSE is each of the following statements for you?

| | | Definitely<br>true | Mostly<br>true | Don't<br>know | Mostly<br>false | Definitely false |
|---|---|---|---|---|---|---|
| | | $\blacksquare$ | lacksquare | lacksquare | lacksquare | lacksquare |
| â | I seem to get sick a little easier than other people | 🗆 1 | 2 | 3 | | 5 |
| ь | I am as healthy as<br>anybody I know | 🗌 1 | 2 | 3 | 4 | 5 |
| c | I expect my health to get worse | 🗆 1 | 2 | 3 | 4 | 5 |
| A | My health is excellent | | Π, | | | |

# Thank you for completing these questions!

# Appendix P References

- Bonow, R.O., et al., ACC/AHA 2006 guidelines for the management of patients with valvular heart disease: a report of the American College of Cardiology/American Heart Association Task Force on Practice Guidelines (writing Committee to Revise the 1998 guidelines for the management of patients with valvular heart disease) developed in collaboration with the Society of Cardiovascular Anesthesiologists endorsed by the Society for Cardiovascular Angiography and Interventions and the Society of Thoracic Surgeons. J Am Coll Cardiol, 2006. 48(3): p. e1-148.
- 2. Siu SC, Silversides CK. Bicuspid aortic valve disease. J Am Coll Cardiol. 2010; 55(25):2789-2800. DOI: 10.1016/j.jacc.2009.12.068.
- 3. Michelena HI, Desjardins VA, Avierinos JF, et al. Natural history of asymptomatic patients with normally functioning or minimally dysfunctional bicuspid aortic valve in the community. Circulation. 2008; 117(21):2776-2784. DOI: 10.1161/circulationaha.107.740878.
- 4. Roberts WC, Ko JM. Frequency by decades of unicuspid, bicuspid, and tricuspid aortic valves in adults having isolated aortic valve replacement for aortic stenosis, with or without associated aortic regurgitation. Circulation. 2005; 111(7):920-925. DOI: 10.1161/01.cir.0000155623.48408.c5.
- 5. Frank, S., A. Johnson, and J. Ross, Jr., Natural history of valvular aortic stenosis. Br Heart J, 1973. 35(1): p. 41-6.
- 6. Gardin, J.M., et al., Aortic stenosis: can severity be reliably estimated noninvasively? Chest, 1980. 77(2): p. 130-1.
- 7. Murakami, T., et al., Changes in patterns of left ventricular hypertrophy after aortic valve replacement for aortic stenosis and regurgitation with St. Jude Medical cardiac valves. Artif Organs, 2000. 24(12): p. 953-8.
- 8. Rankin, J.S., et al., Determinants of operative mortality in valvular heart surgery. J Thorac Cardiovasc Surg, 2006. 131(3): p. 547-57.
- 9. Chiappini, B., et al., Outcome after aortic valve replacement in octogenarians. Ann Thorac Surg, 2004. 78(1): p. 85-9.
- 10. Thourani, V.H., et al., Outcomes of surgical aortic valve replacement in high-risk patients: a multiinstitutional study. Ann Thorac Surg, 2011. 91(1): p. 49-55; discussion 55-6.
- 11. Connolly, H.M., et al., Severe aortic stenosis with low transvalvular gradient and severe left ventricular dysfunction: result of aortic valve replacement in 52 patients. Circulation, 2000. 101(16): p. 1940-6.
- 12. Bouma, B.J.v.D.B., R. B.; van Der Meulen, J. H.; Verheul, H. A.; Cheriex, E. C.; Hamer, H. P.; Dekker, E.; Lie, K. I.; Tijssen, J. G., To operate or not on elderly patients with aortic stenosis: the decision and its consequences. Heart, 1999. 82(2): p. 143-8.
- 13. Brown, J.M., et al., Isolated aortic valve replacement in North America comprising 108,687

- patients in 10 years: changes in risks, valve types, and outcomes in the Society of Thoracic Surgeons National Database. J Thorac Cardiovasc Surg, 2009. 137(1): p. 82-90.
- 14. Thourani, V.H., et al., Long-term outcomes after isolated aortic valve replacement in octogenarians: a modern perspective. Ann Thorac Surg, 2008. 86(5): p. 1458-64; discussion 1464-5.
- 15. Cribier, A., et al., Percutaneous transcatheter implantation of an aortic valve prosthesis for calcific aortic stenosis: first human case description. Circulation, 2002. 106(24): p. 3006-8.
- 16. Thomas, M. and O. Wendler, Transcatheter aortic valve implantation (TAVI): how to interpret the data and what data is required? EuroIntervention, 2009. 5(1): p. 25-7.
- 17. Grube, E., et al., Percutaneous aortic valve replacement for severe aortic stenosis in high-risk patients using the second- and current third-generation self-expanding CoreValve prosthesis: device success and 30-day clinical outcome. J Am Coll Cardiol, 2007. 50(1): p. 69-76.
- 18. Walther, T., et al., One-year interim follow-up results of the TRAVERCE trial: the initial feasibility study for trans-apical aortic-valve implantation. Eur J Cardiothorac Surg, 2011. 39(4): p. 532-7.
- 19. Svensson, L.G., et al., United States feasibility study of transcatheter insertion of a stented aortic valve by the left ventricular apex. Ann Thorac Surg, 2008. 86(1): p. 46-54; discussion 54-5.
- 20. Thomas, M., et al., One-Year Outcomes of Cohort 1 in the Edwards SAPIEN Aortic Bioprosthesis European Outcome (SOURCE) Registry: The European Registry of Transcatheter Aortic Valve Implantation Using the Edwards SAPIEN Valve. Circulation, 2011. 124(4): p. 425-33.
- 21. Thomas, M. Balloon-Expandable Edwards SAPIEN: The Expanding (including Cohort 2) SOURCE Registry: 30 Day Outcomes from 2,300 Edwards TAVI Patients and Predictors of Mortality. in TCT. 2010. Washington, DC.
- 22. Thomas, M. Updates from the SOURCE Registry: Echo Data, Subset Analyses, and Impact of EuroSCORE on Clinical Outcomes. in TCT. 2009. San Francisco, CA.
- 23. Wendler, O. Transapical Aortic Valve Implantation Early Results from the SOURCE Registry. in EACTS. 2009. Vienna, Austria.
- 24. Lefevre, T., et al., One year follow-up of the multi-centre European PARTNER transcatheter heart valve study. Eur Heart J, 2011. 32(2): p. 148-57.
- Kodali, S. Pooled Analysis with Extended Follow-Up from the REVIVE II and REVIVAL II Transfemoral Feasibility Registries. in TCT. 2008. Washington, DC.
- 26. Finsterer, J. and C. Stollberger, Strategies for primary and secondary stroke prevention in atrial fibrillation. Neth J Med, 2008. 66(8): p. 327-33.

- 27. Thoracic Aorta: Prospective Electrocardiographically Triggered CT Angiography with Dual-Source CT—Feasibility, Image Quality, and Dose Reduction. Blanke P, Bulla S, Baumann T, et al. Radiology 2010:255;207-217.
- 28. Freitag G. Methods for assessing noninferiority with censored data. Biometrical journal. Biometrische Zeitschrift. 2005; 47(1):88-98; discussion 99-107.
- 29. Makkar RR, Fontana G, Jilaihawi H, et al. Possible Subclinical Leaflet Thrombosis in Bioprosthetic Aortic Valves. The New England journal of medicine. 2015; 373(21):2015- 2024.
- 30. Pache G, Schoechlin S, Blanke P, et al. Early hypo-attenuated leaflet thickening in balloon-expandable transcatheter aortic heart valves. European heart journal. 2015.
- 31. O'Brien, S.M., et al., The Society of Thoracic Surgeons 2008 cardiac surgery risk models: part 2--isolated valve surgery. Ann Thorac Surg, 2009. 88(1 Suppl): p. S23-42.
- 32. Comparison of 12 risk stratification schemes to predict stroke in patients with nonvalvular atrial fibrillation. Stroke, 2008. 39(6): p. 1901-10.
- 33. Independent predictors of stroke in patients with atrial fibrillation: a systematic review. Neurology, 2007. 69(6): p. 546-54.
- 34. Gottesman, R.F., et al., Delirium after coronary artery bypass graft surgery and late mortality. Ann Neurol, 2010. 67(3): p. 338-44.
- 35. Durack, D.T., A.S. Lukes, and D.K. Bright, New criteria for diagnosis of infective endocarditis: utilization of specific echocardiographic findings. Duke Endocarditis Service. Am J Med, 1994. 96(3): p. 200-9.
- 36. Fried, L.P., et al., Frailty in older adults: evidence for a phenotype. J Gerontol A Biol Sci Med Sci, 2001. 56(3): p. M146-56.
- 37. Stolerman, Ian. Encyclopedia of Psycho-pharmacology. London UK: Springer; 2010.
- 38. Perlman GY, Blanke P, Dvir D, et al. Bicuspid Aortic Valve Stenosis: Favorable Early Outcomes With a Next-Generation Transcatheter Heart Valve in a Multicenter Study. JACC. Cardiovascular interventions. 2016;9(8):817-824. DOI: 10.1016/j.jcin.2016.01.002. No Epub.

# Appendix Q Actigraphy/QOL Sub-Study QOL measures [Enrollment Closed]

# Visual Analogue Scale (VAS) 1

A Visual Analogue Scale (VAS) is a measurement instrument that tries to measure a characteristic or attitude that is believed to range across a continuum of values and cannot easily be directly measured. For example, the amount of pain that a patient feels ranges across a continuum from none to an extreme amount of pain. From the patient's perspective this spectrum appears continuous ± their pain does not take discrete jumps, as a categorization of none, mild, moderate and severe would suggest. It was to capture this idea of an underlying continuum that the VAS was devised.

Operationally a VAS is usually a horizontal line, 100 mm in length, anchored by word descriptors at each end, as illustrated in Fig. 1. The patient marks on the line the point that they feel represents their perception of their current state. The VAS score is determined by measuring in millimeters from the left hand end of the line to the point that the patient marks. There are many other ways in which VAS have been presented, including vertical lines and lines with extra descriptors. As such an assessment is clearly highly subjective, these scales are of most value when looking at change within individuals.

# Figure 1 VAS example

| How severe is your pain today? Place a vertical mark on the line below to in | dicate |
|---|---|
| how bad you feel your pain is today. | |
| No pain | Very severe pair |

# PF-10 Health Survey<sup>2</sup>

The Optum<sup>™</sup> PF-10 Health Survey is a Health Survey that uses just 10 questions to measure physical health and well-being from the patient's point of view. Taking only two to three minutes to complete, the PF-10 is a practical, reliable and valid measure of physical health and is particularly useful in large population health surveys or for applications that combine a generic and disease-specific health survey. As the survey uses norm-based scoring, comparisons can be made among the other generic health surveys (SF-36v2<sup>®</sup> and SF-8<sup>™</sup>). It is a widely used tool for monitoring population health, comparing and analyzing disease burden and predicting medical

The PF-10 is available in multiple modes of administration and in both standard four-week and acute one-week recall periods.

# KCCQ-123

expenses.

| The Kansas City Cardiomyopathy Ques | tionnaire (KCCQ) | is a 23-item | ı, self- |
|---|---|---|---|
| administered instrument that quantifies | physical function, | symptoms ( | frequency, |

severity and recent change), social function, self-efficacy and knowledge, and quality of life.

In the KCCQ, an overall summary score can be derived from the physical function, symptom (frequency and severity), and social function and quality of life domains. For each domain, the validity, reproducibility, responsiveness and interpretability have been independently established. Scores are transformed to a range of 0-100, in which higher scores reflect better health status.

The KCCQ-12 reduces the KCCQ's 23 items to 12. This short version significantly increase the speed and ease of questionnaire administration while preserving the sensitivity, specificity, and reliability of the original instruments.

<sup>&</sup>lt;sup>1</sup> VAS source: <a href="http://buderimosteopathy.com.au/wp-content/uploads/2012/02/VAS.pdf">http://buderimosteopathy.com.au/wp-content/uploads/2012/02/VAS.pdf</a>

<sup>&</sup>lt;sup>1</sup> https://www.optum.com/optum-outcomes/what-we-do/health-surveys/sf-12v2-health-survey.html

<sup>&</sup>lt;sup>1</sup> http://cvoutcomes.org/pages/3214